## Nitto BioPharma Inc.

Statistical Analysis Plan

NBF-006-001: A Phase I/lb Open-Label, Multi-Center, Dose-Escalation Study to Investigate the Safety, Pharmacokinetics and Preliminary Efficacy of Intravenous NBF-006 in Patients with Non-Small Cell Lung, Pancreatic, or Colorectal Cancer Followed by a Dose Expansion Study in Patients with KRAS-Mutated Non-Small Cell Lung Cancer

**Investigational Product: NBF-006** 

NCT03819387

14 March 2023





# Statistical Analysis Plan Final Version 2.0; March 14, 2023

#### Protocol No. NBF-006-001

IND Number: 139860

A Phase I/Ib Open-Label, Multi-Center, Dose-Escalation Study to Investigate the Safety, Pharmacokinetics and Preliminary Efficacy of Intravenous NBF-006 in Patients with Non-Small Cell Lung, Pancreatic, or Colorectal Cancer Followed by a Dose Expansion Study in Patients with KRAS-Mutated Non-Small Cell Lung Cancer

| Prepared by: | Dailan Danforth | Electronically signed by: Dallan<br>7 Danforth<br>Re-ason: author<br>Date: Mar 16: 2023 10:28 EDT | Date: | 16-Mar-2023 |
|---|---|---|---|---|
| | Dailan Danforth, MP | H, MS | | |
| | Associate Director, E | Biostatistics | | |
| | Theradex Oncology | | | |
| Reviewed by: | Judy DeChamplas | Electronically signed by: Judy<br>DisChamplain<br>Reason, approval<br>Date: Mer 16, 2023 11:02 EDT | Date: | 16-Mar-2023 |
| | Judy DeChamplain, I | MS, PMP | -COMMON CO. | |
| | Global Head of Open | | | |
| | Theradex Oncology | | | |
| | Jose Mejias | Electronically signed by: Jose Majias<br>Reason: approval<br>Date: Mar 16, 2023 11:08 EDT | Date: | 16-Mar-2023 |
| | Jose Mejias, B.S. | | | |
| | Director, Statistical F | | | |
| | Theradex Oncology | тодганины | | |
| | 0 | Electronically signed by: Zachary<br>Albaugh<br>Reason: approval<br>Date: Mar 16, 2023 10 22 EDT | Date: | 16-Mar-2023 |
| | Zachary Albaugh | | | |
| | Senior Clinical Proje | ct Manager | | |
| | Theradex Oncology | | | |
| | Joachim Gullbo | Electronically signed by Joachim<br>Gullbo<br>Reason: approval<br>Date: Mar 17, 2023 08:53 EDT | Date: | 17-Mar-2023 |
| | Joachim Gullbo, MD | PhD | | ======================================= |
| | Medical Monitor | | | |
| | Theradex Oncology | | | |
| Approved by: | Sonya Zabludoff | Electronically signed by Sonya<br>Zabbudoff<br>Reason: approval<br>Date: Mar 20, 2023 12:14 PIDT | Date: | 20-Mar-2023 |
| Approved by. | Sonya Zabludoff, Ph | D<br>cal Operations (GCP Clin | | |



## Statistical Analysis Plan Final Version 2.0; March 14, 2023

#### Protocol No. NBF-006-001

IND Number: 139860

A Phase I/Ib Open-Label, Multi-Center, Dose-Escalation Study to Investigate the Safety, Pharmacokinetics and Preliminary Efficacy of Intravenous NBF-006 in Patients with Non-Small Cell Lung, Pancreatic, or Colorectal Cancer Followed by a Dose Expansion Study in Patients with KRAS-Mutated Non-Small Cell Lung Cancer

Sponsor: Nitto BioPharma, Inc.

10618 Science Center Drive, San Diego, California, 92121

USA

CRO: Theradex Oncology

4365 Route 1 South

Suite 101

Princeton, New Jersey 08540

USA



# **TABLE OF CONTENTS**

| | | | | Page No. |
|---|---|---|---|---|
| 1.0 | Introdu | ction | | 7 |
| | 1.1 | Stud | y Documents Used in the Preparation of this Docu | ıment8 |
| 2.0 | Objectiv | es and E | indpoints | 9 |
| 3.0 | Study D | esign | | 10 |
| | 3.1 | Over | rall Study Design | 10 |
| | 3.2 | Bline | ding and Unblinding | 13 |
| | 3.3 | Rano | domization and Stratification | 13 |
| | 3.4 | Sam | ple Size | 13 |
| 4.0 | Manage | ment of | Analysis Data | 14 |
| | 4.1 | Data | Handling | 14 |
| | 4.2 | Miss | ing Data | 14 |
| | 4.3 | Codi | ng Conventions for Events and Medications | 14 |
| 5.0 | Statistic | | ods | |
| | 5.1 | Gene | eral | 14 |
| | | 5.1.1 | Definitions | 15 |
| | | 5.1.2 | Visit Window | 15 |
| | 5.2 | Stati | istical Analysis Populations | 15 |
| | | 5.2.1 | Intent-to-Treat (ITT) | 15 |
| | | 5.2.2 | Safety Evaluable | 15 |
| | | 5.2.3 | Efficacy Evaluable | 15 |
| | | 5.2.4 | Pharmacokinetic Evaluable | |
| | 5.3 | Stud | y Population Characteristics | 16 |
| | | 531 | Study Enrollment | |



| | 5.3.2 | Patient Disposition16 |
|---|---|---|
| | 5.3.3 | Protocol Deviations16 |
| | 5.3.4 | Demographics |
| | 5.3.5 | Baseline Disease Characteristics17 |
| | 5.3.6 | Prior Cancer Therapy18 |
| | 5.3.7 | Prior Medical History18 |
| 5.4 | Effica | ncy Analyses18 |
| | 5.4.1 | Best Overall Tumor Response per RECIST 1.119 |
| | 5.4.2 | Duration of Overall Response23 |
| | 5.4.3 | Duration of Stable Disease per RECIST 1.124 |
| 5.5 | Safet | y and Tolerability Analysis24 |
| | 5.5.1 | Study Drug Exposure and Compliance24 |
| | 5.5.2 | Dose Limiting Toxicity24 |
| | 5.5.3 | Adverse Events25 |
| | 5.5.4 | Laboratory Data26 |
| | 5.5.5 | Electrocardiogram Data27 |
| | 5.5.6 | Other Safety Parameters27 |
| | 5.5.7 | Concomitant Measures27 |
| | 5.5.8 | Pharmacokinetic Analyses27 |
| | | 5.9 Estimation of population pharmacokinetic<br>ters using population pharmacokinetic (PopPK) modeling<br>approach 29 |
| | 5.5.10 | Biomarker Related Analyses30 |
| Changes | to Plann | ned Analyses30 |
| Referen | ces | 30 |
| Index of | Tables a | nd Figures37 |
| | Changes | 5.3.3 5.3.4 5.3.5 5.3.6 5.3.7 5.4 Effica 5.4.1 5.4.2 5.4.3 5.5 Safet 5.5.1 5.5.2 5.5.3 5.5.4 5.5.5 5.5.6 5.5.7 5.5.8 5.parame 5.5.10 Changes to Plant References |



| | 8.1 | Tables | 37 |
|---|---|---|---|
| | 8.2 | Figures | 39 |
| 9.0 Inde | ex of A | Appendix Listings | 40 |
| Figure 1 | Part | A and B Study Design Schematic | 10 |
| Figure 2 | Dose | Escalation Study Design (3+ 3 Schema) | 11 |
| Table 1 | Obje | ctives and Related Endpoints | 9 |
| Table 2 | | A NBF-006 Dose Levels | |
| Table 3 | Part | B NBF-006 Dose Levels | 13 |
| Table 4 | | onse: Patients with target (+/- non-target) disease | |
| Table 5 | | onse: Patients with non-target disease only | |
| Table 6 | Best | overall response when CR and PR confirmation required | 22 |
| Table 7 | | ST 1.1 Event /Censored Date used in DOR | |
| Table 8 | Dose | Limiting Toxicity | 25 |
| Table 9 | | cal Laboratory Parameters Collection | |
| Table 10 | PK P | arameters | 28 |
| Table 7-1 | Stud | y Calendar Part A (Protocol Amendment 4.0 Table 3) | 31 |
| Table 7-2 | Stud | y Calendar Part B (Protocol Amendment 4.0 Table 4) | 34 |



# **Abbreviations**

| AE(s) | Adverse Event(s) |
|---|---|
| ALP | Alkaline Phosphatase |
| ALT | Alanine Transaminase |
| API | Active Pharmaceutical Ingredient |
| AST | Aspartate Transaminase |
| BOR | Best Overall (Tumor) Response |
| Cls | Confidence Intervals |
| CR | Complete Response |
| CRO | Contract Research Organization |
| CT | Computerized Tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DLT | Dose-Limiting Toxicity |
| DOR | Duration of Overall Response |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group Performance Status |
| eCRF | Electronic Case Report Form |
| EOI | End of Infusion |
| GCP | Good Clinical Practice |
| GGT | Gamma Glutamyl Transferase |
| GSTT1 | Glutathione S-Transferase theta class |
| ICF | Informed Consent Form |
| IMP | Investigational Medicinal Products |
| ITT | Intent to Treat |
| KRAS | Gene in the Ras Family of Oncogenes (Kirsten Ras Oncogene Homolog) |
| MedDRA | Medical Dictionary for Regulatory Activities |
| ms | Millisecond |
| MTD | Maximum Tolerated Dose |
| N | Number |
| NCI | National Cancer Institute |
| NSCLC | Non-Small Cell Lung Cancer |
| ORR | Overall Response Rate |
| 05 | Overall Survival |
| PD | Progressive Disease |
| PK | Pharmacokinetic |
| PR | Partial Response |
| PR | PR Segment Duration in ECG |
| PT | Preferred Term |
| QT | OT Interval in ECG |
| QTcF | Fridericia Corrected QT Interval in ECG |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SAE | Serious Adverse Event(s) |
| SAP | Statistical Analysis Plan |
| SD | Stable Disease |
| siRNA | Small Interfering Ribonucleic Acid |
| SOC | MedDRA System Organ Class |
| SOI | Start of Infusion |
| TEAEs | Treatment-Emergent Adverse Events(s) |
| UCR | - I THE TOTAL OF THE TAXABLE PROPERTY OF TAXABLE PROPERTY OF T |
| | Unconfirmed Complete Response |
| ULN | Unconfirmed Partial Response Upper Limit of Normal |
| NAME OF TAXABLE PARTY. | White Blood Cell Count |
| WHO-DD | World Health Organization Drug Dictionary |



## 1.0 Introduction

This Statistical Analysis Plan (SAP) describes analyses and data presentations for Nitto BioPharma, Inc. Protocol NBF-006-001. It provides details of the analysis populations, derived variables, and statistical methods to be used in the analyses and reporting of safety and efficacy data.

The purpose of the SAP is to ensure the credibility of the study findings by specifying the statistical approaches to study data analyses prospectively. The SAP final 1.0 was used for the interim analysis of Part A of the study. Based on this interim analysis, specification of potential additional analyses to be included in the final analysis of data derived from Part B of the study may be incorporated in an amended version of the protocol and SAP, which is finalized prior to database lock for Part B of the study. Such additional analyses may, for example, entail assessments of efficacy in specific biomarker-defined subsets of study subjects of potential relevance based on exploratory analysis of the interim (Part A) biomarker data. All statistical analyses detailed in this SAP are conducted using SAS statistical software (version 9.4 or higher).

The Theradex Medical Monitor, supported by the Nitto BioPharma, Inc. GCP Clinical Lead as required in the setting of serious adverse events (SAEs), will be responsible for the assessment of ongoing safety data for the study. This will include a review of all adverse events (AEs) (serious and non-serious AEs) as they are reported, and laboratory and ECG results. Safety data will be reviewed periodically by a safety review committee consisting of Theradex Oncology Medical Monitor, Nitto BioPharma, Inc., and Investigators. Details are provided in the Safety Management Plan and/or the Communication Plan. Nitto BioPharma, Inc. will make decisions on dose modifications, cohort dose escalation, and transition to dose expansion phase (Part B) based on recommendations by the core safety committee comprised of the Theradex Medical Monitor, Investigators, and the Nitto BioPharma, Inc. GCP Clinical Lead.



# 1.1 Study Documents Used in the Preparation of this Document

The following documents were used in preparation of this SAP:

# **List of Study Documents**

| Study Document | Approval Date | |
|------------------------|---------------|-----|
| Protocol Amendment 4.0 | 06 June 2022 | 433 |
| 1165 Annotated CRF | 18 May 2021 | |



#### **Objectives and Endpoints** 2.0

#### Table 1 **Objectives and Related Endpoints**

| Objective | Endpoint |
|---|---|
| Primary (Part A Dose Escalation) | |
| To determine the safety profile, maximum tolerated dose (MTD), and recommended doses for Part B of NBF-006 in patients with advanced (NSCLC), pancreatic, or colorectal cancer for dose levels 1-4 (0.15, 0.3, 0.6, and 1.2 mg/kg) and in patients with KRAS-mutated NSCLC for dose level 5 (1.6 mg/kg). | Number of patients with DLTs and AEs. |
| Secondary (Part A Dose Escalation) | |
| To evaluate preliminary efficacy of NBF-006 in patients with advanced NSCLC, pancreatic, or colorectal cancer for dose levels 1-4 (0.15, 0.3, 0.6, and 1.2 mg/kg) and in patients with KRAS-mutated NSCLC for dose level 5 (1.6 mg/kg). To investigate the pharmacokinetics (PK) of NBF-006. | Best overall response (CR, PR, SD) per RECIST 1.1 and PK parameters (C <sub>max</sub> , clearance [CL], volume of distribution [V <sub>ss</sub> ], terminal elimination half-life [T <sub>1/2</sub> ], area under the curve [AUC] <sub>0-t</sub> ) of siRNA, duration of overall response, duration of stable disease. |
| Exploratory (Part A Dose Escalation) | |
| To evaluate correlation between biomarkers and clinical outcome. To evaluate correlation between KRAS mutations and clinical outcome. | Biomarkers may include, but<br>are not necessarily limited to,<br>GSTP or related proteins of<br>the GST family. |
| Primary (Part B Dose Expansion) | |
| To evaluate preliminary efficacy and safety profile of NBF-006 in patients with KRAS-mutated NSCLC. | Best overall response (CR, PR,<br>SD) per RECIST 1.1 and safety<br>(DLT, AEs), duration of overall<br>response, duration of stable<br>disease. |
| Secondary (Part B Dose Expansion) | |
| To investigate the PK of NBF-006 | PK parameters (C <sub>max</sub> , CL, V <sub>ss</sub> , T <sub>1/2</sub> , AUC <sub>0-t</sub> , AUC <sub>0-m</sub> ) of siRNA. |
| Exploratory (Part B Dose Expansion) | |
| To evaluate correlation between glutathione S-<br>transferase pi (GSTP) messenger ribonucleic acid<br>(mRNA) knockdown (KD) in surrogate tissue<br>(peripheral blood mononuclear cells [PBMCs]),<br>biomarkers, and clinical outcome. | Biomarkers may include, but<br>are not necessarily limited to,<br>GSTP or related proteins of<br>the GST family |



## 3.0 Study Design

## 3.1 Overall Study Design

This is an open-label, non-placebo-controlled study conducted in two parts - Part A (dose escalation) followed by Part B (dose expansion).

Figure 1 Part A and B Study Design Schematic



The end of study is defined as the last patient last visit date in the trial.

#### Part A Dose Escalation Phase

Patients in Part A will have previously treated progressive or metastatic NSCLC, pancreatic, or colorectal cancer, with or without KRAS mutation status.

In both parts, NBF-006 will be administered via intravenous (IV) infusion over 70 minutes once a week for 4 weeks followed by a 2-week rest period. The length of each cycle is 6 weeks.

The first dose level (0.15 mg/kg) will be a single patient cohort. If any grade 2 or greater drug-related event occurs during the first cycle of treatment, the cohort will be expanded up to 3 patients. If a dose-limiting toxicity (DLT) occurs during the first cycle, the cohort will be expanded up to 6 patients before proceeding with dose escalation.

Subsequent cohorts in the dose escalation phase will enroll patients following the standard 3+3 design. If 1 out of 3 patients experience a DLT during the first cycle of treatment, the dose cohort will be expanded up to 6 patients. If no DLT is observed in the first three patients enrolled at the



highest dose, this cohort will be expanded to 6 patients. If 2 or more out of 6 patients experience DLTs, the MTD has been exceeded, and dose escalation will cease. Up to 3 additional patients will be enrolled at a lower dose if only 3 patients were treated at that dose level, to confirm safety of that dose. To collect clinically important information in the target population, and prepare for Part B, the 6-patient cohort(s) must each include at least 3 patients with histologically or cytologically confirmed progressive or metastatic NSCLC, up to dose level 4 (1.2 mg/kg) in Part A. In dose level 5 (1.6 mg/kg) in Part A and all patients in Part B, only patients with previously treated NSCLC with KRAS mutation will be included. Once safety has been confirmed in Part A at 1.6 mg/kg (i.e., 0-1 DLT in 6 patients), an additional 4 patients with KRAS-mutated NSCLC will be enrolled in Part B of the study at this dose level. Stratification for GSTT1-null genotype patients will not occur in Part A.

One dose de-escalation is permitted.

Enroll 3 patients at a dose level

1 DLT
2-3 DLT

Escalate to next dose

1 of 6 DLT

Stop

MTD=Previous dose

MTD=Previous dose

Figure 2 Dose Escalation Study Design (3+ 3 Schema)



Note that if a dose level is not tolerated, the protocol implies that three additional subjects should be enrolled at the next lowest dose level to confirm that it is the MTD (defined as dose at which 0-1 subjects experience DLTs).

Table 2 Part A NBF-006 Dose Levels

| Dose Level | NBF-006 Dose | Number of Patients# |
|------------|--------------|---------------------|
| 1 | 0.15 mg/kg | 1-6* |
| 2 | 0.3 mg/kg | 3-6 |
| 3 | 0.6 mg/kg | 3-6 |
| 4 | 1.2 mg/kg | 3-6 |
| 5 | 1.6 mg/kg | 3-6 |

<sup>\*</sup>Two patients were dosed at 0.15 mg/kg; however, the first patient did not complete Cycle 1 due to disease progression and was replaced with another patient.

The definition of MTD will be based on review of safety data and DLTs corresponding to the first cycle of therapy in at least 6 evaluable patients. MTD will be defined as the highest dose where 0 or 1 out of 6 patients have DLTs.

## Part B Dose Expansion Phase

After MTD is confirmed in Part A for up to dose level 4 or 5 (1.2 or 1.6 mg/kg), enrollment in Part B may commence. Part B will enroll patients with previously treated progressive or metastatic NSCLC with confirmed KRAS mutation.

Two doses levels that will be explored further in Part B are 0.6 mg/kg and 1.2 mg/kg. Approximately twenty patients will be enrolled in Part B, with 10 patients enrolled in each of the two cohorts. Both cohorts will be stratified for GSTT1-null genotype patients. Once dose level 5 (1.6 mg/kg) has been confirmed to be safe in Part A, an additional 4 patients will then be enrolled at 1.6 mg/kg, for a planned total of 24 patients in Part B. The proportion of GSTT1-null patients treated at the highest dose level (1.6 mg/kg) will be balanced with the previous two expansion cohorts as much as possible by applying stratification rules in Part B (depending on the distribution of patients enrolled in Part A, unstratified).

<sup>\*</sup>The 6-patient cohort(s) must each include at least 3 patients with histologically or cytologically confirmed progressive or metastatic NSCLC.



Part B NRF-006 Dose Levels Table 3

| | TEL GOO DOSC ECTEIS | |
|------------|---------------------|--------------------|
| Dose Level | NBF-006 Dose | Number of Patients |
| 3 | 0.6 mg/kg | 10 |
| 4 | 1.2 mg/kg | 10 |
| 5 | 1.6 mg/kg | 4* |

<sup>\*</sup>Dose level 5 pending confirmation of safety in Part A

For both phases, NBF-006 will be administered via intravenous (IV) infusion over 70 minutes once a week for 4 weeks followed by a 2-week rest period. The length of each cycle is 6 weeks.

# Duration of Therapy

Upon completion of Cycle 1, in the absence of disease progression or unacceptable toxicity, patients may continue to be treated with NBF-006 at the same dose and schedule until disease progression, death, withdrawal of consent, investigator decision to remove patient, or intolerable toxicity, whichever occurs first. A patient may continue on study (even if one or more criterion meets Disease Progression per RECIST 1.1) at the Investigator's discretion if deemed that the drug is well-tolerated and that the patient may continue to receive benefit from continuing treatment.

## 3.2 Blinding and Unblinding

This is an open-label study; blinding techniques are not required.

### 3.3 Randomization and Stratification

This is an open-label, non-placebo-controlled study. Randomization is only implemented in IWRS for Part B at 0.6 and 1.2 mg/kg. Patients enrolled in Part B will be stratified for GSTT1-null genotype to ensure equal allocation to the cohorts with different doses. Patients treated at the highest dose level in Part B will be balanced for GSTT1-null genotype to match the distribution of patients at the other (stratified) dose levels as much as possible but may depend on the first 6 patients treated at this dose in Part A (not stratified). Stratification for GSTT1-null genotype patients will not occur in Part A.

## 3.4 Sample Size

This is an exploratory trial and therefore no sample size calculations have been performed. The number of patients in Part A (up to 20) is based on



the planned number of dose escalation cohorts required to identify the MTD. The planned number of patients in Part B is approximately 20-24. Unless the reason was toxicity (i.e., a DLT), any patient who discontinues after receiving less than 4 doses during Cycle 1 will be replaced.

#### 4.0 Management of Analysis Data

The data from all study centers will be pooled together for analyses.

## Data Handling

Unscheduled laboratory results will not be analyzed for the visit summary of continuous values but will be included in the laboratory shift tables.

# 4.2 Missing Data

All partial date value(s) will be presented in the patient listing, as they are recorded on the eCRF. Unless otherwise specified, no imputation of values for missing data will be performed. The missing values will not be reported as a "0" numerical value in the database, and the missing values will not be included in the overall dataset.

If the start date/time of an AE is partially or completely missing, the AE will be assumed as Treatment-Emergent AE (TEAE). If the timing of a given concomitant medication cannot be determined, it will be included in the listings/summaries as concomitant.

4.3 Coding Conventions for Events and Medications

| Event/Medication | Coding/Mapping Conventio |
|-----------------------------------|--------------------------|
| AE, Medical History Coding | MedDRA version 21.1 |
| Lab Test Grade | NCI CTCAE version 5.0 |
| Prior and Concomitant Medications | WHO-DDE version 2018 |

#### 5.0 Statistical Methods

#### 5.1 General

Demographic and baseline characteristics, efficacy assessments, and safety data will be summarized by Dose Cohort and Overall for Part A; by dose level 0.6 mg/kg, 1.2 mg/kg, and 1.6 mg/kg (if dose level deemed safe), and Overall for Part B. Results from Part A and Part B will be presented separately for safety and baseline data, but for efficacy data, include all the 10 patients at 1.6 mg/kg, so can be compared to other expansion cohorts.



Continuous data will be presented as n, mean, standard deviation, median, minimum, and maximum. Categorical data will be presented as frequency counts and percentages. All raw data collected will be listed.

#### 5.1.1 Definitions

Baseline: The last measurements taken prior to first exposure to study drug, including Day 1 measurements taken pre-dosing. If patients have no value as defined above for a particular parameter, the baseline value will be missing.

## 5.1.2 Visit Window

In order to summarize longitudinal data per timepoint, assessment will be allocated to visits using pre-defined time windows. Unless otherwise specified, the schedule of event and windowing in protocol will be used. The deviations from visit windows will be captured by protocol deviations.

## 5.2 Statistical Analysis Populations

## 5.2.1 Intent-to-Treat (ITT)

All participants who were enrolled (signed consent) into the study, irrespective of whether study medication was administered or not. Demographic and baseline data are based on ITT population.

### 5.2.2 Safety Evaluable

All patients who received any component of study treatment. Safety data and study drug exposure are based on Safety Evaluable population.

## 5.2.3 Efficacy Evaluable

Patients with measurable disease by RECIST 1.1 who had a baseline assessment and at least one post-baseline assessment. Efficacy Evaluable is the population for efficacy analyses.

#### 5.2.4 Pharmacokinetic Evaluable

Patients who receive at least 1 dose of study treatment and have blood samples collected for at least 6 hours after the end of infusion. Patients who do not complete the study treatment infusion will be excluded from the pharmacokinetic analysis.



## 5.3 Study Population Characteristics

## 5.3.1 Study Enrollment

Patient enrollment, eligibility, and study populations are summarized by frequency and percentage of patients.

## 5.3.2 Patient Disposition

The disposition of patients, based on the reasons reported for study withdrawal, is summarized by frequency and percentage of patients.

### 5.3.3 Protocol Deviations

A classified list of protocol deviations can be found in the Project Management Plan, Appendix E. Protocol deviations are categorized by Theradex Oncology and Nitto BioPharma, Inc. as:

#### Minor:

Where evidence exists that departure(s) from the protocol requirements, ICH-GCP or local requirements has occurred with evidence that:

- Does not have a significant impact on the research participant's rights, safety or welfare; the integrity of the data; nor substantially alter risks to subjects.
- Isolated/infrequent procedure-related deviations (e.g., ECOG not performed, missed lab tests, PK time point deviations).
- Failure to follow ICH-GCP procedures for significant study processes (example: IMP accountability logs, patient identification code list) that can be retrospectively or prospectively corrected.

## Major:

Where evidence exists that significant and unjustified departure(s) from the protocol requirements, ICH-GCP or local requirements has occurred with evidence that:

- The safety or well-being of trial subjects have the significant potential to be jeopardized.
- There are a significant number of Minor non-compliances within a single area of responsibility, indicating a systemic quality assurance failure.
- Impact significantly upon secondary study endpoints
- Variance from a protocol specified procedure results in questionable data.



#### Critical:

Where evidence exists that significant and unjustified departure(s) from the protocol requirements, ICH-GCP or local requirements has occurred with evidence that:

- The safety or well-being of trial subjects have been jeopardized.
- The scientific value of the trial has been jeopardized.
- The clinical trial data are unreliable.
- There are a number of Major non-compliances across areas of responsibility, indicating a systemic quality assurance failure.
- Impacts significantly upon primary study endpoints.
- There has been clinical research misconduct or fraudulent activity.

## 5.3.4 Demographics

Demographics, including age categories (18 to 64, 65+), sex, race, ethnicity, and ECOG performance status, are summarized by frequency and percentage of patients within each category.

Age is summarized using descriptive statistics (n, mean, standard deviation, median, minimum, and maximum). The exact age is calculated in years without decimal places as follows:

Age (years) = (Year of First Dose – Year of Birth) – Correction, Where: Correction = 1, if Birth Month > First Dose Month or Birth Month = First Dose Month and Birth Day > First Dose Day; Else: Correction = 0 (First Dose is first study drug administration).

### 5.3.5 Baseline Disease Characteristics

Primary site, disease stage, KRAS genotype mutation are summarized by frequency and percentage of patients. Duration of disease is calculated from the date of initial diagnosis to the date of first study drug administration for NSCLC (with or without KRAS mutation), pancreatic cancer, and colorectal cancer tumor types for each dose levels in Part A and B, respectively. EGFR Mutation, ALK/ROSI gene fusion will be summarized for the 14 early enrolled patients in Part A. Smoking history will be summarized for NSCLC patients in Part A and NSCLC patients in Part B in the category of never, former, current for NSCLC patients and the duration



of tobacco consumption. GSTT1 genotype will be summarized in the category of null and wild type.

## 5.3.6 Prior Cancer Therapy

Prior cancer therapies, including chemotherapy, hormone therapy, immunotherapy, and other prior therapies for NSCLC (with or without KRAS mutation), pancreatic cancer, and colorectal cancer tumor types for each dose levels in Part A and Part B, respectively, prior cancer radiation, and prior surgeries are summarized by frequency and percentage of patients within each category. Number of patients with prior cancer therapies of 1 regimen, 2, 3, 4, 5, >=6 regimens and best response will be summarized by frequency and percentage of patients by dose level. Prior medications will be listed.

## 5.3.7 Prior Medical History

Medical History will be coded using MedDRA version 21.1 and summarized by system organ class (SOC) and preferred term (PT) by dose level.

## 5.4 Efficacy Analyses

Patients with measurable disease will be assessed at baseline and reevaluated at the end of even numbered cycles for dose levels 1-4 in Part A and at baseline and at the end of every cycle for dose level 5 in Part A and all patients in Part B of the study. The patients could be assessed outside these protocol-specified windows at the investigator's discretion. Efficacy Evaluable population is used for efficacy analyses. Statistical comparisons will not be made among the dose levels.

The primary measure of tumor response is the overall response (CR+PR) reported and confirmed. An initial response of complete response (CR) or partial response (PR) based on RECIST 1.1 should be confirmed by a second imaging evaluation. The efficacy endpoints include best overall response (BOR), overall response rate (ORR = rate of PR + CR), disease control rate (DCR= rate of SD+PR+CR), duration of overall response (DOR), duration of CR, and duration of stable disease (SD).

BOR summary table in number (%) is provided. Duration of overall response, complete response, and stable disease life table estimates will be summarized. All efficacy tables and figures will be presented by dose



level at 0.15, 0.3, 0.6, 1.2 mg/kg and overall for Part A; by dose level 0.6, 1.2, 1.6 mg/kg (including the 1.6 mg/kg from Part A) and overall for Part B.

## 5.4.1 Best Overall Tumor Response per RECIST 1.1

Tumor responses and progression will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. All measurable lesions up to a maximum of two lesions per organ and five lesions in total, representative of all involved organs, should be identified as target lesions and measured at baseline. Target lesions should be selected based on their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the baseline sum diameters, which will be used as reference by which to characterize the objective tumor response.

All other lesions (or sites of disease) including pathological lymph nodes should be identified as non-target lesions and should be also recorded at baseline. Measurements of these lesions are not required, and these lesions should be followed as "present," "absent," or in rare cases "unequivocal progression".

BOR is defined as the best response assessment depending on the findings of target, non-target lesion and new lesions from the start of study treatment until disease progression or recurrence. Valid response assessments (ranked from best to worst) are CR, PR, SD, and PD. CR or PR with only one evaluation will also be presented as unconfirmed PR (uPR) or unconfirmed CR (uCR). BOR for a patient without any valid assessments is not evaluable (NE). Symptomatic deterioration is not considered PD. The primary evaluation of efficacy will focus on PR and CR but analyses incorporating uPR and uCR will also be performed.

BOR is based on the overall response captured on the eCRF off-study summary. All available valid tumor assessments will be used, invalid assessments (not evaluable due to incomplete assessment, not assessed, or missing) will be ignored.

Response Assessment after Palliative Radiotherapy



Palliative radiotherapy, which was implemented in Protocol Amendment 4 (dated 06-Jun-2022), is allowed as medically indicated after completion of the first treatment cycle, and after discussion with medical monitor. Lesions assigned as targets at baseline should preferably not be included in the radiotherapy field, as it would preclude further response assessment per RECIST. Following palliative radiotherapy of RECIST target lesions, the irradiated lesion(s) and overall response assessment should be NA/Not evaluated, but remaining target and non-target lesions should continue to be monitored (an individualized schedule for radiology assessment is acceptable).

BOR is summarized as the number (%) of patients in each response category (CR, PR, SD, PD, and NE) for NSCLC (with or without KRAS mutation), pancreatic cancer, and colorectal cancer tumor types in Part A and Part B, respectively. Patients are counted once in each of the response categories based on their best response assessment.

- PR and CR must be confirmed by a repeat assessment.
- A confirmed CR is a CR which is followed by another CR without any intervening assessments of PD.
- A confirmed PR is a PR preceded or followed by a CR or another PR, allowing for one interim assessment of SD.
- All other assessments of CR or PR are considered unconfirmed responses uCR or uPR.
- For SD, follow-up measurements must meet the SD criteria at least 5 weeks (35 days) after study entry.
- If the first two scheduled assessments are not evaluable and followed by PD or death, BOR is NE.

ORR is defined as the proportion of patients with a BOR of confirmed CR or confirmed PR. ORR<sub>2</sub> will also be provided for all CR (including uCR) and all PR (including uPR). DCR is defined as the proportion of patients with a BOR of CR or PR or SD. DCR<sub>2</sub> will also be provided for all CR (including uCR), all PR (including uPR), and SD. The two-sided 95% Clopper-Pearson [1] Cls is calculated for ORR, ORR<sub>2</sub>, DCR, DCR<sub>2</sub>using the following SAS code:

LowerCL = 1-betainv (1-alpha/2, N-x+1, x)

UpperCL = betainv (1-alpha/2, x+1, N-x)

where: N=sample size, X=number of responders, alpha=0.05 for a 95% confidence interval.



Best percent changes from baseline in target tumor size based on RECIST 1.1 (waterfall plots) and percent change from baseline in tumor response overtime (spider plot) will be provided for NSCLC, pancreatic cancer, and colorectal cancer patients respectively.

Table 4 provides a summary of the overall response status calculation at each time point for patients who have measurable disease at baseline. When patients have non-measurable disease, Table 5Table 5Table 5Table 5 should be used.

CR and PR must be confirmed by a repeat assessment at least 4 weeks but no later than 5 weeks for patients in dose levels 1-4 (0.15, 0.3, 0.6, and 1.2 mg/kg) in Part A after the criteria for response are first met. Response will be confirmed at 4 weeks or at the next scheduled scan (at Week 6 of the following cycle) for patients in dose level 5 (1.6 mg/kg) in Part A and all patients in Part B. If a confirmative scan is done after 4 weeks, the next scheduled scan (at Week 6 of the following cycle) may be omitted.

Follow-up measurements for SD must meet the SD criteria at least 5 weeks after study entry. In this circumstance, the best overall response can be interpreted as in Table 6Table 6Table 6Table 6Table 6Table 5Table 5Table 5.Table 5

Table 4 Response: Patients with target (+/- non-target) disease

| <b>Target Lesions</b> | Non-target Lesions | <b>New Lesions</b> | Overall Response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR / non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | NE |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |



PD=progressive disease, NE=not evaluable

Table 5 Response: Patients with non-target disease only

| Non-target Lesions | <b>New Lesions</b> | Overall Response |
|--------------------|--------------------|------------------|
| CR | No | CR |
| Non-CR / non-PD | No | Non-CR / non-PD* |
| Not all evaluated | No | NE |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

CR=complete response; PD=progressive disease; NE=not evaluable \* Non-CR/non-PD is preferred over SD for non-target disease

Table 6 Best overall response when CR and PR confirmation required

| Overall<br>response<br>First time<br>point | Overall response<br>Subsequent time<br>point | BEST overall response |
|---|---|---|
| CR | CR | CR |
| CR | PR | SD, PD or PR* |
| CR | SD | SD provided minimum criteria for SD duration met, otherwise PD |
| CR | PD | SD provided minimum criteria for SD duration met, otherwise PD |
| CR | NE | SD provided minimum criteria for SD duration met, otherwise NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | SD provided minimum criteria for SD duration met, otherwise PD |
| PR | NE | SD provided minimum criteria for SD duration met, otherwise NE |
| NE | NE | NE |

CR=complete response; PR=partial response; SD=stable disease; PD=progressive disease; NE=nonevaluable

\* If CR is truly met at first time point, then any disease seen at a subsequent time point, even disease meeting PR criteria relative to baseline, makes the disease PD at that point (since disease must have reappeared after CR). Best response would depend on whether minimum duration for SD was met. However, sometimes 'CR' may be claimed



when subsequent scans suggest small lesions were likely still present and in fact the patient had PR, not CR, at the first time point. Under these circumstances, the original CR should be changed to PR and the best response is PR.

## 5.4.2 Duration of Overall Response

DOR is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started). Only patients with a confirmed CR or PR are included in the analysis. For a patient without evidence of PD, DOR censoring details are listed in Table 7.

The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.

Cls for the median duration times are calculated using Brookmeyer and Crowley method [2]. Cls for point estimates of the survival distribution are calculated using the method by Kalbfleisch and Prentice [3].

Duration of treatment per dose level with patient's response overtime (swimmer plot) will be presented for Part A and Part B, respectively.

Table 7 RECIST 1.1 Event /Censored Date used in DOR

| Scer | nario | Outcome | Date |
|---|---|---|---|
| A | No baseline assessment | Censored* | Date of first dose |
| В | Progression at or before next scheduled assessment | Progressed | Date of progression |
| C1 | Progression after one missing assessment | Progressed | Date of progression |
| C2 | Progression after two or more missing assessments | Censored* | Date of last<br>evaluable<br>assessment |
| D | No progression | Censored* | Date of last<br>evaluable<br>assessment |
| E | Discontinued treatment due to toxicity, withdrew consent without progressive disease (PD) | Censored* | Date of last<br>evaluable<br>assessment |
| F | No evaluable tumor assessments or drop out before first follow-<br>up period | Censored* | Date of enrollment |
| G | New anticancer therapy given (including localized therapy to<br>target lesions such as radiotherapy or surgery, after which<br>RECIST response will be NA). | Censored* | Date of last<br>evaluable<br>assessment |



\*Censored = without progressive disease at that time

## 5.4.3 Duration of Stable Disease per RECIST 1.1

Stable Disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started. Duration of stable disease will be analyzed in a similar method as DOR.

## 5.5 Safety and Tolerability Analysis

Safety analyses are based on Safety Evaluable population. Descriptive statistics are used to summarize the safety parameters. Safety data include AEs, laboratory parameters, vital signs, electrocardiogram (ECG) parameters, and ECOG performance status. Protocol schedule of events and windowing will be used for the applicable safety table assessments.

## 5.5.1 Study Drug Exposure and Compliance

NBF-006 exposure and compliance are summarized for cycle 1 and all treatment cycles using descriptive statistics. Number of subjects to whom NBF-006 is administered will be summarized. Duration of Exposure is defined as the duration between the first and last dose of study drug (last dose date - first dose date+1) during the treatment period. Total Dose is defined as the sum of all study drug administered over the entire course of the study. Total intended dose is defined as the sum of intended doses during the duration of exposure, based on no modifications to the protocol-specified dose and schedule.

Percent Compliance is defined as the total dose divided by total intended dose multiplied by 100% for each patient. The frequency and percentage of patient receiving <100%, 100%, and >100% of their intended dose will be summarized.

The number of patients with dose delayed and interrupted will be each summarized using frequency counts and percentages, along with the reasons for patients receiving NBF-006.

## 5.5.2 Dose Limiting Toxicity



DLT is defined as any treatment-related toxicity during the first cycle (42) days) that meets any of the following criteria based on CTCAE version 5.0 for all patients enrolled in the study, regardless of their replacement.

#### Table 8 Dose Limiting Toxicity

#### A DLT will be defined as

- (1) Treatment-related hematological toxicities including Grade 4 neutropenia, any grade neutropenic fever, ≥ Grade 3 thrombocytopenia lasting longer than 3 consecutive days, ≥ Grade 3 thrombocytopenia with bleeding, any other confirmed hematological toxicity ≥ Grade 4
- (2) Treatment-related non-hematological toxicity ≥ Grade 3 including Electrolyte abnormalities that do not resolve within 48 hours of intervention, ≥ Grade 3 infusion-related reactions, Grade 3 cytokine release syndrome, any hepatic toxicity meeting Hy's Law criteria, Grade 3 nausea/vomiting or diarrhea or other self-limited or medically controllable toxicities that last > 72 hours regardless of medical intervention
- (3) Any other treatment-related toxicity, i.e., greater than at baseline, is clinically significant and/or unacceptable, does not respond to supportive care and results in a disruption of the dosing schedule of more than 14 days
- (4) Any death not clearly due to the underlying disease or extraneous causes DLT excludes: Alopecia of any grade

#### 5.5.3 Adverse Events

TEAEs are defined as adverse events that occurred on or after the first dose date of study drug up to 30 days post the last dose date. If an AE occurs before the first dose of study drug, it will be considered as non-treatment emergent.

TEAEs are summarized by frequency and percentage of patients and tabulated by MedDRA system organ class (SOC) and preferred term (PT), by maximum NCI-CTCAE version 5.0 grade and by unrelated, unlikely, possible, probable and definite relationships to NBF-006. Serious adverse events (SAEs), TEAEs leading to treatment discontinuation and death are summarized. Drug-related TEAEs by CTCAE grade, and drug-related grade 3 or greater TEAEs are summarized. Patients with multiple instances of a specific TEAE or AE are counted once within a summary category-SOC, PT, maximum grade, or closest relationship to treatment. Infusion-related reactions (IRR) by severity grade will be summarized by dose. Number of



IRR per patient per dose level will be summarized as well. All AEs, DLTs, and IRRs will be listed respectively.

# 5.5.4 Laboratory Data

Laboratory data will be summarized by laboratory tests for the treatment period, defined as the time from first dose up to 30 days post last dose of study drug. Laboratory data will be converted to SI units prior to summarization. All laboratory tests will be provided in patient listings. The listings indicate the normal ranges for each parameter. Each value, if appropriate, is classified as falling above (H), below (L), or within normal range and graded using the CTCAE criteria.

The observed data and change from baseline will be summarized at each of the laboratory timepoints, using descriptive statistics, for hematology, chemistry and urinalysis laboratory tests, as specified below in Table 9.

The changes from baseline to maximum CTCAE grade during treatment will be summarized by frequency and percentage of patients using shift tables for every gradable hematology and chemistry test. Maximum CTCAE Grade is defined as the highest CTCAE version 5.0 grade reported for a patient after first dose and up to 30 days post last dose.

Table 9 Clinical Laboratory Parameters Collection

| Hematology | Serum Chemistry | Urinalysis |
|---|---|---|
| Hemoglobin | Sodium | Glucose |
| Hematocrit | Potassium | Protein |
| WBC and | BUN | Ketones |
| differential | Calcium<br>SGOT/ALT | Nitrite |
| Platelet | SGPT/AST | Leukocyte esterase |
| | Alkaline phosphatase | Specific gravity |
| | Total protein | pH |
| | Total bilirubin | Microscopic analysis WBC, RBC, bacteria, epithelia |
| | Albumin | cells, casts, mucous, crystals |
| | Creatinine | The Control of the Co |
| | Glucose | |

A listing of patients with grade 3 or 4 laboratory values during treatment period from first dose up to 30 days post last dose study drug will also be provided.



## 5.5.5 Electrocardiogram Data

ECG parameters including heart rate, PR, QT, and QTcF observed data and change from baseline will be summarized by visit. The average of the triplicate ECG measurements performed pre-infusion on or before Day 1 will serve as baseline. The number and percentage of QT and QTcF in categories of interval ≤440, >440, >480, >500 ms, and increase from baseline >30 ms or >60 ms will be summarized. Patient listings of QT/QTcF maximum change from baseline >50 ms or increase to 500 ms will be provided.

## 5.5.6 Other Safety Parameters

Vital signs including blood pressure, heart rate, respiration rate, and temperature, as well as weight will be summarized using descriptive statistics. Change from baseline to maximum ECOG scores will be summarized by frequency and percentage of patients using shift tables. Pain Assessment will be listed.

#### 5.5.7 Concomitant Measures

Concomitant measures will be coded using the World Health Organization Drug Dictionary (WHO-DD version 2018), tabulated by drug class and term, and summarized by frequency and percentage of patients. Patients are counted only once in each summary category (e.g., drug class or term). All concomitant medications that were ongoing at Day 1 of treatment or taken on Day 1 of treatment or thereafter up to the last dose of study drug will be summarized within each category and listed. Palliative radiotherapy is allowed upon implementation of Protocol Amendment 4 (dated 06-Jun-2022) as medically indicated after completion of the first treatment cycle, and after discussion with medical monitor and will be listed separately.

## 5.5.8 Pharmacokinetic Analyses

## 5.5.8.1 Summary of PK Concentration Data

Mean and individual NDT-05-1040 plasma concentration-time curves on Day 1 and Day 22 of Cycle 1 will be expressed graphically using both linear and semi-logarithmic scale. PK concentration data will be summarized using descriptive statistics: number of patients, arithmetic mean (Mean), standard deviation (SD), %coefficient variance (CV%), minimum (Min), median (Med), and maximum (Max). Individual data will be reported using



the actual collection time points whereas mean summary data will be reported using nominal time points.

5.5.8.2 Estimation of Individual Pharmacokinetic Parameters Using Non-Compartmental Analysis (NCA)

Individual PK parameters will be calculated from plasma concentrationtime profiles of NDT-05-1040 using non-compartmental analysis (NCA) method on Day 1 and Day 22 of Cycle 1. NCA will be conducted) to obtain estimation of individual PK parameters in Phoenix WinNonlin 64, version 8.3.4.

## Calculation of PK Parameters

For the calculation of PK parameters, actual times and dose will be used in PK parameter calculations. All plasma concentrations that are below limit of quantification (BLQ) will be set as zero. The following parameters will be calculated and reported:

Table 10 PK Parameters

| PK parameter | Definition |
|---|---|
| Cmax | maximum plasma concentration observed |
| T <sub>max</sub> | time to maximum plasma concentration, or first maximum plasma concentration if this occurs at more than 1 time point |
| Cmin | minimum plasma concentration observed |
| AUC <sub>0-t</sub> | area under the plasma concentration-time curve from time 0 to the last quantifiable concentration, calculated by the linear up/log down trapezoidal rule |
| AUC <sub>0-72</sub> | area under the plasma concentration-time curve from time 0 to 72 hours, calculated by the linear up/log down trapezoidal rule |
| AUC <sub>0</sub> | area under the plasma concentration-time curve extrapolated to infinity, calculated as $AUC_{0-t}+C_{last}/\lambda_z$ |
| Vz | volume of distribution during terminal elimination phase following intravenous administration $V_z = \left(\frac{Dose}{\lambda_Z*AUC_{0-\infty}}\right)$ |
| V <sub>55</sub> | Volume of distribution at equilibrium following intravenous administration, Vss = (MRTINF + CL) |
| CL | total body clearance following intravenous administration $CL = \left(\frac{Dose}{AUC_{0-\infty}}\right)$ |



| PK parameter | Definition |
|---|---|
| T <sub>1/2</sub> | first-order terminal elimination half-life, calculated as $ln(2)/\lambda_z$ |

The minimum requirement for CL,  $V_z$ ,  $V_{ss}$  and  $T_{1/2}$  calculation will be the inclusion of at least 3 consecutive plasma concentrations above the lower limit of quantification (LLOQ) with at least one of these concentrations following  $C_{max}$ .  $R^2$  adjustment of the terminal elimination phase regression line must be greater than or equal to 0.80. To have a meaningful reportable  $AUC_{0-\infty}$ , CL,  $V_z$ ,  $V_{ss}$ ,  $T_{1/2}$ ,  $\% AUC_{0-\infty}$  (percent extrapolated) will not exceed 30%.

## Descriptive Analysis and Presentation of PK Parameters

PK parameters will be summarized by dose level using descriptive statistics including number of patients, arithmetic mean (Mean), %coefficient of variation (CV%), standard deviation (SD), median (Median), minimum (Min) and maximum (Max) values.

Additional analysis will be performed on calculated PK parameters to assess dose proportionality for the  $C_{max}$ ,  $AUC_{0-72}$  and  $AUC_{0-\infty}$  at Cycle 1 Day1 and Day22 and to estimate accumulation ratio ( $R_{acc}$ ) for the  $C_{max}$ ,  $AUC_{0-72}$ ,  $AUC_{0-\infty}$  at Cycle 1.

# 5.5.9 Estimation of population pharmacokinetic parameters using population pharmacokinetic (PopPK) modeling approach

To quantify the typical disposition characteristics and sources of PK variability (such as between-subject, within-subject, and inter-occasion variability), population pharmacokinetic (PopPK) analyses will be performed by an outside vendor Ann Arbor Pharmacometrics Group, Inc. (A2PG) and will be included in the final Clinical Study Report. In addition, PopPK analysis will be used to quantitatively identify the impact of covariates (such as age, sex, race, body weight, concomitant medications, disease state) on systemic drug exposures and assess their potential implications on dosing regimen.

A population PK model will be developed using the nonlinear mixed-effects modeling approach. The data will be analyzed in NONMEM (version 7.3.0 whereas R (version 3.6.1 (2019-07-05) and RStudio (v1.3.959-1) will be used for pre- and post-processing of data. Detailed PopPK analysis will be



described in a separate stand-alone modeling plan and a specific report will be produced to reflect the entire PopPK analysis work performed by Amador.

Final pharmacokinetics analyses will be performed by an outside vendor and will be included in the final Clinical Study Report.

## 5.5.10 Biomarker Related Analyses

The actual value, change from baseline for cytokines (TNF-α, IL-1β, IL-6, and IFN-y) and complements (CH50, Bb, C3a, and C5a) will be listed. Spaghetti plots overtime will be provided for each patient for cytokines and complements. The actual value for complements assessment, ADA assay, and exploratory biomarkers will be listed. Other biomarkers related analyses will be provided in separate reports.

Listing to show mRNA level for GST family (GSTP1, GSTT1, MGST3 and GSTM3) will be provided. Spaghetti plots overtime will be provided for each patient for GSTP1 will be provided.

#### 6.0 Changes to Planned Analyses

Not applicable.

#### 7.0 References

- [1] Clopper CJ, Pearson ES The use of confidence or fiducial limits illustrated in the case of the binomial. Biometrika 1934; 26(4):404-13.
- [2] Brookmeyer R Crowley J. A confidence interval for the median survival time, Biometrics 1982;38:29-41.
- [3] Kalbfleisch JD, Prentise RL. The Statistical Analysis of Failure Time Data. New York: John Wiley & Sons, Inc. 1980.



#### Study Calendar Part A (Protocol Amendment 4.0 Table 3) Table 7-1

| | 4 | Cycle 1 | | | | | | | | Cyc | le 2 | | | C | ycle 3 & | beyone | 1 | EOT | 30-day |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Part A<br>Evaluations | Pre-<br>treat-<br>ment* | Wk<br>1<br>D1 | Wk 2<br>D8<br>±3 | Wk 3<br>D15<br>±3 | Wk 4<br>D22<br>±3 | Wk 5<br>D29-35 | Wk 6<br>D36-42 | Wk 1<br>D1 | Wk 2<br>D8<br>±3 | Wk 3<br>D15<br>±3 | Wk 4<br>D22<br>±3 | Wk 5<br>D29-35 | Wk 6<br>D36-42 | Wk 1<br>D1 | Wk 2<br>Wk 3<br>Wk 4 | Wk<br>5 | Wk<br>6 | | safety<br>FU visi<br>(±3) |
| Informed consent (incl. optional biopsy consent) | × | | | | | | | | | | | | | | | .,. | | | |
| Medical history | × | | | | | | | | | | | | | | | | | | |
| Physical exam | X | Xp | | | | . 9 | - S | X | | | | 0 | | × | | 4 | | X | × |
| Weight | х | Xe | | | | 9 | | × | | | | | | × | | | | X | × |
| Vital signs* | × | Xp | X | X | × | | | × | × | X | × | | | X | | | | X | |
| ECG' | X | Xp | | | х | 4 3 | | | | | | | | | | | | X | |
| ECOG performance status | × | Xp | | | | | | × | | | | | | × | | | | × | × |
| Tumor measurement <sup>6</sup><br>(tumor markers, if<br>applicable) | x | | | | | | x | | | | | | × | | | | x | × | |
| Hematology <sup>b</sup> | × | X <sub>p</sub> | X | х | х | | | × | х | × | X | | | X | - 8 | | | X | × |
| Blood chemistry | x | Χp | X | х | х | | | X | х | X | × | | | x | 7. | | | X | × |
| Urinalysis | X | Χp | | | | 8 8 | 1 0 | X | | | | 0 | | X | 1 0 | | | X | X |
| Blood sample for<br>immune activation<br>biomarkers | | × | | | | | | | | | | | | | | | | | |
| Pregnancy test | X* | | | | | 0 3 | - 0 | X | | | | | | X | 1 0 | 67 | | X | 7.0 |
| Blood sample for ADA assay <sup>c</sup> | | × | | х | | | | × | | | | | | × | | | | × | × |
| PK blood sampling <sup>d</sup> | | × | × | | × | 2 3 | | × | | | | | | | | | | | |
| Blood sample for<br>exploratory biomarkers | х | | | | | | | | | | | | | | | | | | |
| Blood sample for GSTP<br>KD <sup>a</sup> | | × | х | | | | | | | | | | | | | | | | |

NBF-006-001 Statistical / Copyright® 2016 by Theradex Oncology, Princeton NJ All rights reserved Statistical Analysis Plan Final Version 2.0; March 14, 2023

31



| You | х | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| GSTT1 genotyping <sup>p</sup> | х | | | | | | | | | - P | | | |
| Optional biopsy | × | | 1777.77 | | × | | | | | | | | |
| NBF-006 administration " | | × | × | × | × | × | × | × | × | × | × | | |
| Concomitant medications | × | | < throughout study > | | | | | | | | | | |
| Adverse events | | | throughout study> | | | | | | | | | × | × |

a: Screening assessments may be performed within 28 days of study to treatment initiation, unless specified.

b: For Cycle 1 Day 1, these tests may be performed within 3 days prior to Cycle 1 Day 1. Physical exam and pre-treatment tests done within 3 days of Cycle 1 Day 1 do not need to be repeated for Wk1D1 unless clinically indicated.

- C ADA assay timepoints:
  - Cycle 1, Day 1: pre-dose
  - Cycle 1, Day 15: pre-dose
  - Cycle 2, Cycle 4, Cycle 6, Cycle 8, etc. (i.e., every even numbered cycle), up to one year. Day 1 pre-dose
  - Year 2 and beyond: every 6 months
  - EOT
  - 30-day safety follow up visit
- d: PK timepoints:
  - Cycle 1, Day 1:
    - Before start of infusion (SOI),
    - During the infusion: 20 m (±5min) after the start of the last infusion step implemented at 6 mL/min rate
  - End of Infusion (EOI); after EOI: 0.5 hr (±5min), 2 hr (±10min), 6 hr (±15min), 24 hr (±1hr), 48 hr (±2hr), 72 hr (±3hr)
  - Cycle 1, Day 8: pre-dose
  - Cycle 1, Day 22:
    - Before SOI
    - During the infusion; 20 min (±5min) after the start of the last infusion step implemented at 6 mL/min rate
    - End of Infusion (EOI); after EOI: 0.5 hr (±5min), 2 hr (±10min), 6 hr (±15min), 24 hr (±1hr), 48 hr (±2hr), 72 hr (±3hr)
  - Cycle 2, Day 1: pre-dose
- e: Wtal signs, including blood pressure, heart rate, respiration rate, and temperature. During Cycle 1: Before SOI, EDI; after EDI: 1hr (±5min), 2hr (±10min), Other days; only before SOI and EOI.
- f. Standard 12-lead ECG (in triplicate) while patient is in semi-recumbent position. Perform at screening. Cycle 1 First and fourth doses: within 15 minutes prior to SOI, then 15 min (±5min). 30 min (±10min), 1 hr (±10min) (at EOI)

NBF-006-001 Statistical Analysis Plan Copyright® 2016 by Theradex Oncology, Princeton NJ

Final Version 2.0; March 14, 2023

All rights reserved

32



- g: Tumor measurement by RECIST version 1.1 and tumor markers will be collected at baseline and at the end of every even numbered cycle in Part A, dose levels 1-4 (0.15 mg/kg, 0.3 mg/kg, 0.6 mg/kg, 1.2 mg/kg) and at the end of every cycle for dose level 5 (1.6 mg/kg), if applicable; the same method used at baseline for a patient should be used consistently for all evaluations throughout the study. To be assigned a status of PR or CR, changes in tumor measurements must be confirmed by repeat assessments that should be performed at 4 weeks but no later than 5 weeks for patients in dose levels 1-4 (0.15 mg/kg, 0.3 mg/kg, 0.6 mg/kg, and 1.2 mg/kg) in Part A after the criteria for response are first met. Response will be confirmed at 4 weeks or at the next scheduled scan (at Week 6 of the following cycle) for patients in dose level 5 (1.6 mg/kg) in Part A. If a confirmative scan is done after 4 weeks, the next scheduled scan at Week 6 of the following cycle may be omitted. In the case of SD, follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 5 weeks.
- h: Hematology, including hemoglobin, white blood cell with differential, and platelet count.
- E Blood chemistry, including sodium, potassium, blood urea nitrogen, glucose, SGOT/SGPT (ALT/AST), alkaline phosphatase, total protein, total bilirubin, albumin, creatinine, and calcium.
- Blood samples collected during Cycle 1 (Week 1) for all patients treated in Part A of the study for determination of complement (CH50, Bb, C3a, C5a) and cytokines (IFN-y, IL-1β, IL-6, TNF-α):
  - Pre-dose
  - 10 ± 3 minutes after 50f
  - 60 ± 10 minutes after EOI
  - 6 hr ± 15 minutes after EOI
  - 24 hr ± 1 hr after EOI
- k: Pregnancy test; for women of childbearing potential, a negative pregnancy test (urine or serium) must be done within 7 days prior to study treatment initiation and documented.
- It. Confirmation of KRAS mutation: optional for Part A dose levels 1-4 and mandatory for Part A dose level 5 (1.6 mg/kg). Obtain archive sample if available; otherwise, a fresh biogsy (low or minimal risk only) is required. If such type of biopsy is needed but cannot feasibly be collected, the Sponsor and Medical Monitor should be consulted. Genomic tumor profile report is acceptable in lieu of a biopsy. Note: if at any time during the trial a biopsy is performed as part of routine medical care, we may request a sample.
- m: NBF-006 is administered IV QC (minimum 4 days apart) preferably on a Monday or Tuesday (to accommodate the PK schedule) during Cycle 1.
- n: GSTP KD time points collected in the 6 patients from Part A at dose level 5 (1.6 mg/kg):
  - · Cycle 1, Day 1:
    - Before SOI
    - After EOI: 6 hr (±15min), 24 hr (±1hr)
  - Cycle 1, Day 8: before 5OI

o: Optional biopsy collected during screening and 24(±3) hours after the 4th dose in cycle 1. Only for patients signing the optional biopsy consent, and when the biopsy can be safely obtained. p: In Part A of the study, patients will not be stratified for the GSTT1- null genotype, but whole blood samples will still be collected during the screening visit and batch-analyzed at a central laboratory.

Note: Each patient must remain in clinic for a 6-hour safety observation period after each NBF-006 infusion, until the safety review committee has reviewed a 3-patient cohort and recommended a reduced observation time at that dose level. Please see Protocol Amendment Section 8.1.2.8 for details.

NBF-006-001 Statistical Analysis Plan Copyright© 2016 by Theradex Oncology, Princeton NJ All rights reserved 33 Final Version 2.0; March 14, 2023



# Table 7-2 Study Calendar Part B (Protocol Amendment 4.0 Table 4)

| Part B Evaluations | | Cycle 1 | | | | | | | | Cyc | le 2 | | | C | ycle 3 & | beyon | d | EOT | 30-day |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-<br>treat-<br>ment <sup>4</sup> | Wk 1<br>D1 | Wk 2<br>D8<br>±3 | Wk 3<br>D15<br>±3 | Wk 4<br>D22<br>±3 | Wk 5<br>D29-35 | Wk 6<br>D36-42 | Wk 1<br>D1 | Wk 2<br>D8<br>±3 | Wk 3<br>D15<br>±3 | Wk 4<br>D22<br>±3 | Wk 5<br>D29-35 | Wk 6<br>D36-42 | Wk 1<br>D1 | Wk2<br>Wk3<br>Wk4 | Wk<br>5 | Wk<br>6 | | safety<br>FU visit<br>(±3) |
| Informed consent (incl. optional biopsy consent) | х | | | | | | | | | | | | | | | | | | |
| Medical history | х | | | | | | | | | | | | | | | | | | |
| Physical exam | X | ΧÞ | | | | 1 6 | | х | | | | | 8 0 | X | | | S | X | X |
| Weight | x | Xp | | | | | | × | | | | | | × | | | | X | X |
| Vital signs* | X | Xt | X | X | X | | | X | × | × | × | | | × | | | | X | |
| ECG' | х | Xp | | | Х | 2 0 | | | | | | 6 | | | | | | X | |
| ECOG performance status | × | Xt | | | | | | X | | | | | | × | | | | × | × |
| Tumor measurement <sup>6</sup><br>(tumor markers, if<br>applicable) | × | | | | | | х | | | | | | × | | | | × | x | |
| Hematology <sup>b</sup> | х | Χp | x | х | X | | | х | × | × | × | | | х | | | | X | X |
| Blood chemistry | × | Xe | × | X | х | 7 | | × | X | × | × | 0 | | × | | | | X | X |
| Urinalysis | X | Xp | | | | | | X | | | | | | х | | | | × | X |
| Blood sample for<br>immune activation<br>biomarkers | | х | | | | | | | | | | | | | | | | | |
| Pregnancy test | X <sub>s</sub> | | | | | | | × | | | | | | × | | | | X | 2.77 |
| Blood sample for ADA assay <sup>c</sup> | | х | | X | | | | х | | | | | | х | | | | х | х |
| PK blood sampling d | | × | X | | х | 3 | | X | | | | | | | | | | | |
| Blood sample for<br>exploratory biomarkers | × | | | | | | | | | | | | | | | | | | |
| Blood sample for GSTP<br>KD <sup>o</sup> | | х | × | | | | | | | | | | | | | | | | |

NBF-006-001 Statistical Analysis Plan Copyright® 2016 by Theradex Oncology, Princeton NJ All rights reserved 34


Final Version 2.0; March 14, 2023



| Adverse events | | | | nagara a monaga | < | th | roughou | it study | | ·····> | | X | × |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Concomitant medications | х | | < | | | | | | | | | x | |
| NBF-006 administration<br>m | | × | X | × | x | × | × | х | × | × | X | | |
| Optional biopsy <sup>o</sup> | х | | | - 3 | х | | | | | | | | |
| GSTT1 genotyping <sup>2</sup> | х | | | | | | | | | | | | |
| Confirmation of KRAS<br>mutation '<br>(Part B mandatory) | х | | | | | | | | | | | | |

- a: Screening assessments may be performed within 28 days of study to treatment initiation, unless specified.
- b: For Cycle 1 Day 1, these tests may be performed within 3 days prior to Cycle 1 Day 1, Physical exam and pre-treatment tests done within 3 days of Cycle 1 Day 1 do not need to be repeated for Wk1D1 unless clinically indicated.
- C ADA assay timepoints:
  - Cycle 1, Day 1: pre-dose
  - Cycle 1, Day 15: pre-dose
  - Cycle 2, Cycle 4, Cycle 6, Cycle 8, etc. (i.e., every even numbered cycle), up to one year: Day 1 pre-dose
  - Year 2 and beyond: every 6 months
  - **EOTs**
  - 30-day safety follow up visit
- d: PK timepoints:
  - Cycle 1, Day 1:
    - Before start of infusion (SOI),
    - During the infusion; 20 m (±5min) after the start of the last infusion step implemented at 6 mL/min rate
  - End of Infusion (EOI); after EOI: 0.5 hr (±Smin), 2 hr (±10min), 6 hr (±15min), 24 hr (±1hr)
  - Cycle 1, Day 8: pre-dose
  - Cycle 1, Day 22:
    - Before SOI
    - During the infusion: 20 m (±5min) after the start of the last infusion step implemented at 6 mL/min rate
    - End of Infusion (EOI); after EOI: 0.5 hr (±5min), 2 hr (±10min), 6 hr (±15min), 24 hr (±1hr)
  - Cycle 2, Day 1: pre-dose
- e: Vital signs, including blood pressure, heart rate, respiration rate, and temperature. During Cycle 1: Before SOI, EOI; after EOI: 1hr (±5min), 2hr (±10min), Other days: only before SOI and EOL.
- ft. Standard 12-lead ECG (in triplicate) while patient is in semi-recumbent position. Perform at screening, Cycle 1 First and fourth doses: within 15 minutes prior to SOI, then 15 min (±5min), 30 min (±10min), 1 hr (±10min) (at EOI)

NBF-006-001 Statistical Analysis Plan Copyright® 2016 by Theradex Oncology, Princeton NJ

Final Version 2.0; March 14, 2023

All rights reserved

35


- g: Tumor measurement by RECIST version 1.1 and tumor markers will be measured at baseline and at the end every cycle, if applicable; the same method used at baseline for a patient should be used consistently for all evaluations throughout the study. To be assigned a status of PR or CR, changes in tumor measurements must be confirmed at 4 weeks or at the next scheduled scan (at Week 6 of the following cycle). If a confirmative scan is done after 4 weeks, the next scheduled scan at Week 6 of the following cycle may be omitted. In the case of SD, follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 5 weeks.
- h: Hematology, Including hemoglobin, white blood cell with differential, and platelet count.
- E Blood chemistry, including sodium, potassium, blood urea nitrogen, glucose, SGOT/SGPT (ALT/AST), alkaline phosphatase, total protein, total billrubin, albumin, creatinine, and caldium.
- j. Blood samples collected during Cycle 1 (Week 1) for all patients treated in Part B of the study for determination of complement (CH50, Bb, C3a, C5a):
  - Pre-dose
  - 10 ± 3 minutes after SOI
  - 60 ± 10 minutes after EOI
  - 6 hr ± 15 minutes after EOI
  - 24 hr ± 1 hr after EOI

Dose levels 3 (0.6 mg/kg) and 4 (1.2 mg/kg) did not result in immune activation in Part A and therefore, cytokine activity will not be monitored at those two dose levels in Part B. However if a patient, during or after any infusion of NBF-006, develops IRR symptoms (e.g. backache, fever, nausea, headache, rash, rapid heartbeat, low blood pressure, or trouble breathing), best attempts should be made to collect cytokines as described for Part A with the exception of 10 ± 3 minutes after SDI, which should be collected as close as feasible to the IRR. If there is no meaningful cytokine induction in the 6-patient dose level 5 (1.6 mg/kg) during Part A, then cytokine testing will also not be needed in the remaining 4 patients at that same dose level (1.6 mg/kg), unless there are symptoms of IRR. However, complement samples will continue to be collected for all patients.

- k: Pregnancy test: for women of childbearing potential, a negative pregnancy test (urine or serum) must be done within 7 days prior to study treatment initiation and documented.
- It: Confirmation of KRAS mutation required for Part B. Obtain archive sample if available; otherwise, a fresh biopsy (low or minimal risk only) is required. If such type of biopsy is needed but cannot feasibly be collected, the sponsor and Medical Monitor should be consulted. Genomic tumor profile report is acceptable in lieu of a biopsy. Note: if at any time during the trial a biopsy is performed as part of routine medical care, we may request a sample.
- m: NBF-006 is administered IV QC (minimum 4 days apart) preferably on a Monday or Tuesday (to accommodate the PK schedule) during Cycle 1.
- n: GSTP mRNA KD time points:
  - Cycle 1, Day 1:
    - Before SOI
    - After EOt: 6 hr (±15min), 24 hr (±1hr)
  - Cycle 1, Day 8: before 5OI
- Optional biopsy collected during screening and 24 (±3) hours after the 4th dose in cycle 1. Only for patients signing the optional biopsy consent, and when the biopsy can be safely obtained.
   In Part B of the study, patients will be stratified for the GSTT1- null genotype. Analysis will be done at a central lab from blood samples collected during the screening visit. Initial patients may be enrolled before the GSTT1 status is known.

Note: Each patient must remain in clinic for a 6-hour safety observation period after the first diose, 2 hours after EOI for remaining doses in Cycle 1. The observation period may be further reduced to 30 minutes starting Cycle 2, after Medical Monitor and Investigator safety review. Please see Protocol Amendment Section 8.1.2.8 for details.

NBF-006-001 Statistical Analysis Plan Copyright© 2016 by Theradex Oncology, Princeton NJ All rights reserved 36 Final Version 2.0; March 14, 2023




#### 8.0 Index of Tables and Figures

#### 8.1 Tables

```
Table 14.1.1.1 Study Populations (Dose Escalation Part A)
Table 14.1.1.2 Patient Disposition (Dose Escalation Part A) 15
Table 14.1.2 Demographics (Dose Escalation Part A) 16
Table 14.1.3.1 Baseline Disease Characteristics for NSCLC (Dose Escalation Part A) 18
Table 14.1.3.1 Baseline Disease Characteristics for NSCLC (Dose Expansion Part B) 21
Table 14.1.3.2 Baseline Disease Characteristics for Pancreatic Cancer (Dose Escalation
Part A) 23
Table 14.1.3.3 Baseline Disease Characteristics for Colorectal Cancer (Dose Escalation
Part A) 23
Table 14.1.4 Summary of Medical History (Dose Escalation Part A)
Table 14.1.5.1 Prior Cancer Therapy for NSCLC (Dose Escalation Part A)
Table 14.1.5.2 Prior Cancer Therapy for Pancreatic Cancer (Dose Escalation Part A) 28 Table 14.1.5.3 Prior Cancer Therapy for Colorectal Cancer (Dose Escalation Part A) 28
Table 14.2.1.1 Best Overall Response Summary based for NSCLC (Dose Escalation Part A
and Dose Expansion Part B)
                              30
Table 14.2.1.2 Best Overall Response Summary based for Pancreatic Cancer (Dose
Escalation Part A)
                      32
Table 14.2.1.3 Best Overall Response Summary based for Colorectal Cancer (Dose
                      32
Escalation Part A)
Table 14.2.2.1 Life Table Summary of Duration of Overall Response (Dose Escalation
Part A) 36
Table 14.2.2.2 Life Table Summary of Duration of Overall Response (Dose Expansion Part
B)
       38
Table 14.2.3.1 Life Table Analysis of Duration of Overall Response: Confidence
Intervals for Point Estimates (Dose Escalation Part A)
Table 14.2.3.2 Life Table Analysis of Duration of Overall Response: Confidence
Intervals for Point Estimates (Dose Expansion Part B)
                                                             47
Table 14.2.4 Patient Listing for Duration of Overall Response
Table 14.2.5.1 Life Table Summary of Duration of Stable Disease (Dose Escalation Part
A)
       50
Table 14.2.5.2 Life Table Summary of Duration of Stable Disease (Dose Expansion Part
B)
       51
Table 14.2.6.1 Life Table Analysis of Duration of Stable Disease: Confidence Intervals
for Point Estimates (Dose Escalation Part A) 53
Table 14.2.6.2 Life Table Analysis of Duration of Stable Disease: Confidence Intervals
for Point Estimates (Dose Expansion Part B)
                                             55
Table 14.2.7 Patient Listing of Duration of Stable Disease 57
Table 14.3.1.1 Overall Summary of Treatment-Emergent Adverse Events (Dose Escalation
Part A) 59
Table 14.3.1.2 Summary of Treatment-Emergent Adverse Events by System Organ Class and
Preferred Term (Dose Escalation Part A)
                                            60
Table 14.3.1.3 Summary of Treatment-Emergent Adverse Events by System Organ Class
(Dose Escalation Part A)
                             61
Table 14.3.1.4 Summary of Drug-Related, Treatment-Emergent Adverse Events by System
Organ Class and Preferred Term (Dose Escalation Part A)
                                                             63
Table 14.3.1.5 Summary of Grade 3 or Greater, Treatment-Emergent Adverse Events by
System Organ Class and Preferred Term (Dose Escalation Part A)
                                                                     64
Table 14.3.1.6 Summary of Grade 3 or Greater, Drug-Related, TEAE by System Organ Class
and Preferred Term (Dose Escalation Part A) 65
Table 14.3.1.7 Summary of TEAE by Maximum Severity Grade, System Organ Class and
Preferred Term (Dose Escalation Part A)
                                              66
Table 14.3.1.8 Summary of Drug-Related, TEAE by Maximum Severity Grade, System Organ
Class and Preferred Term (Dose Escalation Part A)
                                                     67
Table 14.3.1.9 Summary of Serious Adverse Events by System Organ Class and Preferred
Term (Dose Escalation Part A) 68
Table 14.3.1.10 Summary of Death On-Study or within 30 Days Post Last Dose (Dose
Escalation Part A) 69
Table 14.3.2.1 Patient Listing of Treatment-Emergent Adverse Events Leading to Death
       71
Table 14.3.2.2 Patient Listing of Serious Adverse Events
Table 14.3.2.3 Patient Listing of Treatment-Emergent Adverse Events Leading to Drug
Withdrawn
```



```
Table 14.3.2.4 Patient Listing of Dose Limiting Toxicities 74
Table 14.3.3.1 Summary of Dose Limiting Toxicities by System Organ Class and Preferred
Term During Cycle One 76
Table 14.3.3.2 Summary of Infusion Related Reaction by Maximum Severity Grade, System
Organ Class and Preferred Term (Dose Escalation Part A)
Table 14.3.4 Patient Listing of Grade 3 and 4 Abnormal Laboratory Values During
              79
Treatment
Table 14.3.5.1.1 Summary of NBF-006 Administration and Compliance for Cycle One (Dose
Escalation Part A)
                     81
Table 14.3.5.1.2 Summary of NBF-006 Administration and Compliance for All Treatment
Cycles (Dose Escalation Part A)
                                    83
Table 14.3.5.1.3 Summary of NBF-006 Dose Delayed/Interrupted/Withdrawn (Dose
                     85
Escalation Part A)
Table 14.3.5.1.4 Summary of Concomitant Measures (Dose Escalation Part A) 86
Table 14.3.5.2.1 Summary of Change from Baseline during Treatment Period for
Hematology Tests (Dose Escalation Part A)
                                            87
Table 14.3.5.2.1 Summary of Change from Baseline during Treatment Period for
Hematology Tests (Dose Expansion Part B)
                                            88
Table 14.3.5.2.2 Summary of Change from Baseline during Treatment Period for Blood
Chemistry Tests (Dose Escalation Part A)
                                            89
Table 14.3.5.2.2 Summary of Change from Baseline during Treatment Period for Blood
                                            90
Chemistry Tests (Dose Expansion Part B)
Table 14.3.5.2.3 Summary of Change from Baseline during Treatment Period for
Urinalysis Tests (Dose Escalation Part A)
                                            91
Table 14.3.5.2.3 Summary of Change from Baseline during Treatment Period for
Urinalysis Tests (Dose Expansion Part B)
                                            92
Table 14.3.5.3.1 Summary of Shift from Baseline to Maximum CTCAE Grade during
Treatment Period for Hematology Tests (Dose Escalation Part A)
Table 14.3.5.3.2 Summary of Shift from Baseline to Maximum CTCAE Grade during
Treatment Period for Blood Chemistry Tests (Dose Escalation Part A) 94
Table 14.3.5.3.3 Summary of Shift from Baseline to Maximum CTCAE Grade during
Treatment Period for Urinalysis Tests (Dose Escalation Part A)
Table 14.3.5.5.1 Summary of ECG Data and Change from Baseline by Visit (Dose
Escalation Part A)
                     98
Table 14.3.5.6.1 Summary of ECG Parameter QT and QTcF Data by Visit (Dose Escalation
Part A) 100
Table 14.3.5.7.1 Summary of Shift from Baseline to Maximum ECOG Score (Dose Escalation
Part A) 101
Table 14.3.5.7.2 Summary of Shift from Baseline to Maximum ECOG Score (Dose Expansion
Part B) 102
Table 14.4.1.1 Summary of Mean Change from Baseline in TNF-α Overtime (Dose Escalation
Part A) 104
Table 14.4.1.2 Summary of Mean Change from Baseline in TNF-α Overtime (Dose Expansion
Part B) 105
Table 14.4.2.1 Summary of Mean Change from Baseline in IL-lβ Overtime (Dose Escalation
Part A) 106
Table 14.4.2.2 Summary of Mean Change from Baseline in IL-1β Overtime (Dose Expansion
Part B) 106
Table 14.4.3.1 Summary of Mean Change from Baseline in IL-6 Overtime (Dose Escalation
Part A) 106
Table 14.4.3.2 Summary of Mean Change from Baseline in IL-6 Overtime (Dose Expansion
Part B) 106
Table 14.4.4.1 Summary of Mean Change from Baseline in IFN-y Overtime (Dose
Escalation Part A)
                    107
Table 14.4.4.2 Summary of Mean Change from Baseline in IFN-V Overtime (Dose Expansion
Part B) 107
Table 14.4.5.1 Summary of Mean Change from Baseline in Complement-CH50 Overtime (Dose
Escalation Part A)
                    107
Table 14.4.5.2 Summary of Mean Change from Baseline in Complement-CH50 Overtime (Dose
Expansion Part B)
                     107
Table 14.4.6.1 Summary of Mean Change from Baseline in Complement-Eb Overtime (Dose
Escalation Part A) 107
Table 14.4.6.2 Summary of Mean Change from Baseline in Complement-Bb Overtime for
Dose Expansion (Part B)
                             108
Table 14.4.7.1 Summary of Mean Change from Baseline in Complement-C3a Overtime (Dose
Escalation Part A)
                     108
Table 14.4.7.2 Summary of Mean Change from Baseline in Complement-C3a Overtime (Dose
Expansion Part B)
                     108
```



Table 14.4.8.1 Summary of Mean Change from Baseline in Complement-C5a Overtime (Dose Escalation Part A) 108
Table 14.4.8.2 Summary of Mean Change from Baseline in Complement-C5a Overtime (Dose Expansion Part B) 108

#### 8.2 Figures

```
Figure 14.2.1.1: Best Change from Baseline in Tumor Measurements for NSCLC (Waterfall
Plot) for Dose Escalation (Part A) and Dose Expansion (Part B)
                                                                   33
Figure 14.2.1.2: Best Change from Baseline in Tumor Measurements for Pancreatic Cancer
(Waterfall Plot) (Dose Escalation Part A) 33
Figure 14.2.1.3: Best Change from Baseline in Tumor Measurements for Colorectal Cancer
(Waterfall Plot) (Dose Escalation Part A)
                                             33
Figure 14.2.1.4.1: Percent Change from Baseline in Tumor Response for NSCLC (Spider
Plot) (Dose Escalation Part A)
                                     34
Figure 14.2.1.4.2: Percent Change from Baseline in Tumor Response for NSCLC (Spider
Plot) (Dose Expansion Part B) 35
Figure 14.2.1.5: Percent Change from Baseline in Tumor Response for Pancreatic Cancer
(Spider Plot) (Dose Escalation Part A)
                                             35
Figure 14.2.1.6: Percent Change from Baseline in Tumor Response for Colorectal Cancer
(Spider Plot) (Dose Escalation Part A)
                                             35
Figure 14.2.2.1: Duration of Overall Response (Kaplan-Meier) (Dose Escalation Part A)
       40
Figure 14.2.2.2: Duration of Overall Response (Kaplan-Meier) (Dose Expansion Part B)
Figure 14.2.2.3: Duration of Overall Complete Response (Kaplan-Meier) (Dose Escalation
Part A) 42
Figure 14.2.2.4: Duration of Overall Complete Response (Kaplan-Meier) (Dose Expansion
Part B) 43
Figure 14.2.2.5: Duration of Treatment per Dose Level with Patient's Response Overtime
(Swimmer Plot) (Dose Escalation Part A)
                                             44
Figure 14.2.2.6: Duration of Treatment per Expansion Cohort with Patient's Response
Overtime (Swimmer Plot) (Dose Expansion Part B)
                                                    44
Figure 14.2.5.1: Duration of Stable Disease (Kaplan-Meier) (Dose Escalation Part A)
       52
Figure 14.2.5.2: Duration of Stable Disease (Kaplan-Meier) (Dose Expansion Part B) 52
Figure 14.4.1.1: Spaghetti Plot for Individual Change from Baseline in TNF-\alpha Overtime
                             109
(Dose Escalation Part A)
Figure 14.4.1.2: Spaghetti Plot for Individual Change from Baseline in TNF-α Overtime
(Dose Escalation Part B)
                             109
Figure 14.4.2.1: Spaghetti Plot for Individual Change from Baseline in IL-1β Overtime
(Dose Escalation Part A)
                             110
Figure 14.4.2.2: Spaghetti Plot for Individual Change from Baseline in IL-1β Overtime
(Dose Escalation Part B)
                             110
Figure 14.4.3.1: Spaghetti Plot for Individual Change from Baseline in IL-6 Overtime
(Dose Escalation Part A)
                             110
Figure 14.4.3.2: Spaghetti Plot for Individual Change from Baseline in IL-6 Overtime
(Dose Escalation Part B)
                             110
Figure 14.4.4.1: Spaghetti Plot for Individual Change from Baseline in IFN-y Overtime
(Dose Escalation Part A)
                            111
Figure 14.4.4.2: Spaghetti Plot for Individual Change from Baseline in IFN-y Overtime
(Dose Escalation Part B)
                             111
Figure 14.4.5.1: Spaghetti Plot for Individual Change from Baseline in Complement-CH50
                                     111
Overtime (Dose Escalation Part A)
Figure 14.4.5.2: Spaghetti Plot for Individual Change from Baseline in Complement-CH50
Overtime (Dose Escalation Part B)
                                     111
Figure 14.4.6.1: Spaghetti Plot for Individual Change from Baseline in Complement-Bb
Overtime (Dose Escalation Part A)
                                     111
Figure 14.4.6.2: Spaghetti Plot for Individual Change from Baseline in Complement-Bb
Overtime (Dose Escalation Part B)
                                     112
Figure 14.4.7.1: Spaghetti Plot for Individual Change from Baseline in Complement-C3a
Overtime (Dose Escalation Part A)
Figure 14.4.7.2: Spaghetti Plot for Individual Change from Baseline in Complement-C3a
Overtime (Dose Escalation Part B)
                                     112
Figure 14.4.8.1: Spaghetti Plot for Individual Change from Baseline in Complement-C5a
Overtime (Dose Escalation Part A)
                                     112
```



Figure 14.4.8.2: Spaghetti Plot for Individual Change from Baseline in Complement-C5a Overtime (Dose Escalation Part B) 112

Figure 14.4.9.1: Spaghetti Plot for Individual Change from Baseline in GSTP1 mPNA Level Overtime (Dose Escalation Part A) 113

Figure 14.4.9.2: Spaghetti Plot for Individual Change from Baseline in GSTP1 mPNA Level Overtime (Dose Escalation Part B) 113

#### 9.0 Index of Appendix Listings

```
Listing 16.2.1.1 Patient Disposition 116
Listing 16.2.2.1 Inclusion/Exclusion Criteria
                                                      117
Listing 16.2.4.1 Demographics 118
Listing 16.2.4.2.1 Disease Related Characteristics 119
Listing 16.2.4.2.2 Baseline KRAS Mutation Assessment 120
Listing 16.2.4.3 Medical History
Listing 16.2.4.4 Prior Cancer Therapy 122
Listing 16.2.4.5 Prior Medications
                                      123
Listing 16.2.4.6 Prior Cancer Radiation
                                              124
Listing 16.2.4.7 Prior Cancer Surgeries
                                              125
Listing 16.2.4.8 Pregnancy Test
                                      126
Listing 16.2.5.1 NBF-006 Administration
                                              127
Listing 16.2.6.1 Extent of Disease: Target and Non-Target Lesions 128
Listing 16.2.6.2 Cycle Response Assessment 130
Listing 16.2.7.1 Adverse Events
                                      131
Listing 16.2.7.2.1 Treatment-Emergent Adverse Events Leading to Dose Interrupted 132
Listing 16.2.7.2.2 Treatment-Emergent Adverse Events Leading to Dose Delayed
                                                                                      133
Listing 16.2.7.2.3 Treatment-Emergent Adverse Events Leading to Drug Withdrawn
                                                                                     134
Listing 16.2.7.3 Serious Adverse Events
                                              135
Listing 16.2.7.4 Patients with Incomplete Adverse Event Information Excluded from
Summary Tables 136
Listing 16.2.7.5 Death Summary
                                      137
Listing 16.2.8.1 Clinical Laboratory Tests Hematology
                                                              138
                                              Blood Chemistry
Listing 16.2.8.2 Clinical Laboratory Tests
                                                                      139
Listing 16.2.8.3 Clinical Laboratory Tests - Urinalysis
Listing 16.2.9.1 Vital Signs 141
Listing 16.2.9.2 Physical Examination 142
Listing 16.2.9.3 Electrocardiogram 143
Listing 16.2.9.4 ECOG Performance Status
Listing 16.2.9.5 Infusion-Related Reactions 146
Listing 16.2.9.6 Pain Assessment
                                     147
Listing 16.2.9.7 Immune Activation Markers - Cytokines Assessment 148
Listing 16.2.9.8 Immune Activation Markers - Complement Assessment 149
Listing 16.2.9.9 Anti-Drug Antibody (ADA) Assay
                                                      150
Listing 16.2.9.10 KRAS Mutation Assessment
Listing 16.2.9.11 GSTT1 Genotyping 152
Listing 16.2.9.12 Exploratory Tumor Biopsy
Listing 16.2.9.13 GSTP mRNA KD Sample 154
Listing 16.2.9.14 GST Family - GSTP1 mRNA Level
Listing 16.2.9.15 GST Family - GSTT1 mRNA Level
                                                      155
                                                      156
Listing 16.2.9.16 GST Family - MGST3 mPNA Level
Listing 16.2.9.17 GST Family - GSTM3 mPNA Level
                                                      157
                                                      158
Listing 16.2.9.18 Pharmacokinetics Data Collection
Listing 16.2.10.1 Concomitant Measures
                                              160
Listing 16.2.10.2 Concomitant Measures - Palliative Radiotherapy
```

# Nitto NBF-006-001\_SAP Part A & B Final 2.0\_clean\_14Mar2023

Final Audit Report 2023-03-20

Created: 2023-03-16

By: Zachary Albaugh (ZAlbaugh@theradex.com)

Status: Signed

Transaction ID: CBJCHBCAABAApU4pC5ZcgruuCFu1BE5rmWpFcnwWObKyP

## "Nitto NBF-006-001\_SAP Part A & B Final 2.0\_clean\_14Mar202 3" History

- Document created by Zachary Albaugh (ZAlbaugh@theradex.com) 2023-03-16 - 2:18:10 PM GMT-IP address: 65.128.24.19
- Document emailed to Dailan Danforth (DDanforth@theradex.com) for signature 2023-03-16 - 2:21-40 PM GMT
- Document emailed to Judy DeChamplain (jdechamplain@theradex.com) for signature 2023-03-16 2:21:40 PM GMT
- Document emailed to Jose Mejias (jmejias@theradex.com) for signature 2023-03-16 - 2:21:40 PM GMT
- Document emailed to Zachary Albaugh (ZAlbaugh@theradex.com) for signature 2023-03-16 - 2:21:40 PM GMT
- Document emailed to Joachim Gullbo (jgullbo@theradex.com) for signature 2023-03-16- 2:21:40 PM GMT
- Document emailed to sonya.zabludoff@nitto.com for signature 2023-03-16 - 2:21:41 PM GMT
- Zachary Albaugh (ZAlbaugh@theradex.com) authenticated with Adobe Acrobat Sign. 2023-03-16 - 2:22:03 PM GMT
- Document e-signed by Zachary Albaugh (ZAlbaugh@theradex.com)
  Signing reason: approval
  Signature Date: 2023-03-16 2:22:03 PM GMT Time Source; server- IP address: 65.128.24.19



Email viewed by Dailan Danforth (DDanforth@theradex.com) 2023-03-16 - 2:26:56 PM GMT-IP address: 104.47.58.254

Dailan Danforth (DDanforth@theradex.com) authenticated with Adobe Acrobat Sign. 2023-03-16 - 2:28:01 PM GMT

6 Document e-signed by Dailan Danforth (DDanforth@theradex.com)

Signing reason: author

Signature Date: 2023-03-16 - 2:28:01 PM GMT - Time Source: server- IP address: 24.2:241.195

Email viewed by Judy DeChamplain (jdechamplain@theradex.com) 2023-03-18 - 3:01:11 PM GMT- IP address: 104.47.59.254

Judy DeChamplain (jdechamplain@theradex.com) authenticated with Adobe Acrobat Sign. 2023-03-16 - 3:02:05 PM GMT

Document e-signed by Judy DeChamplain (jdechamplain@theradex.com)

Signing reason: approval

Signature Date: 2023-03-16 - 3:02:05 PM GMT - Time Source: server- IP address: 72.94.90.100

Email viewed by Jose Mejias (jmejias@theradex.com)
2023-03-18 - 3:06:11 PM GMT-IP address: 104.47.58.254

Jose Mejias (jmejias@theradex.com) authenticated with Adobe Acrobat Sign.

2023-03-16 - 3:08:20 PM GMT

Document e-signed by Jose Mejias (jmejias@theradex.com)

Signing reason: approval

Signature Date: 2023-03-16 - 3:08:20 PM GMT - Time Source: server- IP address: 73:226 136:254

Email viewed by Joachim Gullbo (jgullbo@theradex.com)

2023-03-17 - 12:53:26 PM GMT- IP address: 104.47.56.254

Joachim Gullbo (jgullbo@theradex.com) authenticated with Adobe Acrobat Sign. 2023-03-17 - 12:53:48 PM GMT

Document e-signed by Joachim Gullbo (jgullbo@theradex.com)

Signing reason: approval

Signature Date: 2023-03-17 - 12:53:48 PM GMT - Time Source: server- IP address: 73:255:180:248

nitto.com

2023-03-20 - 7:14:09 PM GMT- IP address: 104.47.23.126

Signer sonya.zabludoff@nitto.com entered name at signing as Sonya Zabludoff 2023-03-20 - 7:14:37 PM GMT- IP address; 138.226.67.6 Sonya Zabludoff (sonya.zabludoff@nitto.com) authenticated with Adobe Acrobat Sign. 2023-03-20 - 7:14:39 PM GMT

Signature Date: 2023-03-20 - 7:14:39 PM GMT - Time Source; server- IP address: 136:226:67.8

- Signing reason: approval
  Sonya Zabludoff (sonya.zabludoff@nitto.com)
- Agreement completed.

2023-03-20 - 7:14:39 PM GMT

Names and email addresses are entered into the Acrobat Sign service by Acrobat Sign users and are unverified unless otherwise noted,





#### Table Shells, Listings and Figures for Statistical Analysis Plan

Signature Page Final Version 2.0; March 14, 2023 Protocol No. NBF-006-001 IND Number: 139860

A Phase I/Ib Open-Label, Multi-Center, Dose-Escalation Study to Investigate the Safety, Pharmacokinetics and Preliminary Efficacy of Intravenous NBF-006 in Patients with Non-Small Cell Lung, Pancreatic, or Colorectal Cancer Followed by a Dose Expansion Study in Patients with KRAS-Mutated Non-Small Cell Lung Cancer

| repared by: | Dailan Danforth | Electronically signed by: Dailan<br>Danforth<br>Reason: author<br>Date: Mar 16, 2023-10-29 EDT | Date: | 16-Mar-2023 |
|---|---|---|---|---|
| | Dailan Danforth, MF | | | |
| | Associate Director, E | Biostatistics | | |
| | Theradex Oncology | | | |
| Reviewed by: | Judy DeChamplai | Electronically signed by Judy<br>y DeChampian<br>Reason: approval<br>Data: Mar 16: 2023 11:03 EDT | Date: | 16-Mar-2023 |
| | Judy DeChamplain, I | MS. PMP | of the sale | |
| | Global Head of Ope | | | |
| | Theradex Oncology | | | |
| | Jose Mejias | Electronically signed by Jose Mejias<br>Reason: approval<br>Date: Mar 21, 2023 08:58 EDT | Date: | 21-Mar-2023 |
| | Jose Mejias, B.S. | | | |
| | Director, Statistical I | | | |
| | Theradex Oncology | | | |
| | ر<br>ا | Electronically signed by Zachary<br>Albuigh<br>Reason approval<br>Date: Mar 16: 2023 10:25 EDT | Date: | 16-Mar-2023 |
| | Zachary Albaugh | | | |
| | Senior Clinical Proje | ct Manager | | |
| | Theradex Oncoloy | | | |
| | Joackim Gullbo | Electronically signed by Joachim<br>Gullbo<br>Reason approval<br>Date Mar 17, 2023 08:54 EDT | Date: | 17-Mar-2023 |
| | Joachim Gullbo, MD | PhD | | |
| | Medical Monitor | | | |
| | Theradex Oncoloy | | | |
| Approved by: | Sonya Zabludoff | Electronically signed by: Sonya<br>, Zabludotf<br>Reason approval<br>Date: Mwi 20: 2023 12:13 PDT | Date: | 20-Mar-2023 |
| | Sonya Zabludoff, Ph | | | |
| | 그리다 시장 하다는 것이 없어요. 그리는 사이지를 받는 것이다. | cal Operations (GCP Clini | cal Dir | ector & Project |
| | Nitto BioPharma, Inc | 일 10분이 150 10분이 보고 있다. 그렇게 하는 다른 보이라면 ! | | |



### Table Shells, Listings and Figures for Statistical Analysis Plan

Signature Page Final Version 2.0; March 14, 2023

> Protocol No. NBF-006-001 IND Number: 139860

A Phase I/Ib Open-Label, Multi-Center, Dose-Escalation Study to Investigate the Safety, Pharmacokinetics and Preliminary Efficacy of Intravenous NBF-006 in Patients with Non-Small Cell Lung, Pancreatic, or Colorectal Cancer Followed by a Dose Expansion Study in Patients with KRAS-Mutated Non-Small Cell Lung Cancer

Sponsor: Nitto BioPharma, Inc.

10618 Science Center Drive, San Diego, California, 92121

USA

CRO: Theradex Oncology, Inc.

4365 Route 1 South

Suite 101

Princeton, New Jersey 08540

USA

2



#### 1.0 Table of Contents

| | | | Page No. |
|---|---|---|---|
| 1.0 | Tabl | le of Contents | 3 |
| 2.0 | Prog | gramming Considerations | 4 |
| 2.1 | 1 TLF | Outputs | 4 |
| 2.2 | 2 Data | a Conventions and Rules | 4 |
| 2.3 | 3 NBF | -006 Starting Dose and Dose Levels | 5 |
| 2.4 | 4 Out | put Presentation Rules | 5 |
| 3.0 | Inde | ex of Tables and Figures | 6 |
| 14 | <b>i.</b> 1 | Demographic and Baseline Data Summary Tables | 13 |
| 14 | 1.2 | Efficacy Data Summary Tables and Figures | 29 |
| 14 | l.3 | Safety Data Summary Tables | 58 |
| | 14.3.1 | Display of Adverse Events | 58 |
| | 14.3.2 | Listings of Death, Other Serious and Significant Adverse Events. | 70 |
| | 14.3.3 | Adverse Events of Special Interest | 75 |
| | 14.3.4 | Abnormal Laboratory Value Listing | 78 |
| | 14.3.5 | Other Safety Data Summary Tables | 80 |
| 14 | 1.4 | Biomarker Data Summary Tables | 103 |
| 4.0 | Inde | ex of Listing | 114 |



#### 2.0 Programming Considerations

All tables, data listings, figures (TLFs), and statistical analyses will be generated using SAS® Version 9.4.

#### 2.1 TLF Outputs

Unless otherwise noted, the estimated mean and median for a set of values are printed out to one more significant digit than the original values; Standard Deviations are printed out to 2 more significant digits than the original values. The minimum and maximum will be reported the same significant digits as the original values. For example, for age:

| N | XX |
|--------------------|------|
| Mean | XX.X |
| Standard Deviation | X.XX |
| Median | XX.X |
| Minimum | XX |
| Maximum | XX |

Percentage values will be printed with one digit to the right of the decimal point in parentheses 1 space after the count (e.g., 7 (12.8%), 13 (5.4%).

#### 2.2 Data Conventions and Rules

This section provided rules for calculations and definitions for naming conventions that are common to all applicable tables.

The baseline value of a variable is defined as the last value obtained on or before the administration date and time of the first study drug dose.

For any variable where percent change from baseline is evaluated at Visit X: Percent Change from Baseline value = [(Visit X value - Baseline value)/Baseline value] x100

For any variable where absolute change from Baseline is evaluated at Visit X: Absolute Change from Baseline value = Visit X value - Baseline value

Concomitant drugs missing both start and stop dates or having a start date prior to the last dose of study drug and missing the stop date or having a stop date after the start of study drug and missing the start date, are counted as concomitant.



<u>Relative Study Day</u>: The first day of treatment is Day 1. A minus (-) sign indicated days prior to the start of treatment (e.g., Day -3 represented 3 days before start of therapy; there is no Day 0). The relative study day for a specific visit (day of study relative to start of treatment) is calculated as Visit Date - Date of First Dose +1 (for post-treatment visits) and Visit Date - Date of First Dose (for Screening visits).

#### 2.3 NBF-006 Starting Dose and Dose Levels

The pre-planned doses of NBF-006 will be

Dose Level 1: 0.15 mg/kg

Dose Level 2: 0.3 mg/kg

Dose Level 3: 0.6 mg/kg

Dose Level 4: 1.2 mg/kg

Dose Level 5: 1.6 mg/kg

#### 2.4 Output Presentation Rules

Tables and figures will be presented separately for Part A and Part B, adjust titles as below:

Title (Dose Escalation Part A)

Title (Dose Expansion Part B)

For Baseline and Safety tables and figures, present Part A dose escalation at dose levels 0.15, 0.3, 0.6, 1.2, 1.6 mg/kg (6 patients), and overall; present Part B expansion cohorts at 3 Dose Level 0.6, 1.2, 1.6 mg/kg (4 patients), and overall.

For Efficacy data, present Part A dose escalation at dose level 0.15, 0.3, 0.6, 1.2 mg/kg, and overall; present Part B expansion cohorts at 3 Dose Level 0.6, 1.2, 1.6 mg/kg (4 patients, also include the 6 patients from Part A at 1.6 mg/kg), and overall.



Page No.

#### 3.0 Index of Tables and Figures Table 14.1.1.2 Patient Disposition (Dose Escalation Part A)....... 15 Table 14.1.3.1 Baseline Disease Characteristics for NSCLC (Dose Escalation Table 14.1.3.1 Baseline Disease Characteristics for NSCLC (Dose Expansion Table 14.1.3.2 Baseline Disease Characteristics for Pancreatic Cancer (Dose Table 14.1.3.3 Baseline Disease Characteristics for Colorectal Cancer (Dose Table 14.1.4 Summary of Medical History (Dose Escalation Part A) ...... 24 Table 14.1.5.1 Prior Cancer Therapy for NSCLC (Dose Escalation Part A)............... 25 Table 14.1.5.2 Prior Cancer Therapy for Pancreatic Cancer (Dose Escalation Table 14.1.5.3 Prior Cancer Therapy for Colorectal Cancer (Dose Escalation Table 14.2.1.1 Best Overall Response Summary based for NSCLC (Dose Table 14.2.1.2 Best Overall Response Summary based for Pancreatic Cancer Table 14.2.1.3 Best Overall Response Summary based for Colorectal Cancer Table 14.2.2.1 Life Table Summary of Duration of Overall Response (Dose Table 14.2.2.2 Life Table Summary of Duration of Overall Response (Dose Table 14.2.3.1 Life Table Analysis of Duration of Overall Response: Confidence Intervals for Point Estimates (Dose Escalation Part A)...... 45



| Table | 14.2.3.2 Life Table Analysis of Duration of Overall Response: Confidence Intervals for Point Estimates (Dose Expansion Part B) | 47 |
|---|---|---|
| Table | 14.2.4 Patient Listing for Duration of Overall Response | |
| | 14.2.5.1 Life Table Summary of Duration of Stable Disease (Dose Escalation Part A) | |
| Table | 14.2.5.2 Life Table Summary of Duration of Stable Disease (Dose Expansion Part B) | 51 |
| Table | 14.2.6.1 Life Table Analysis of Duration of Stable Disease: Confidence Intervals for Point Estimates (Dose Escalation Part A) | 53 |
| Table | 14.2.6.2 Life Table Analysis of Duration of Stable Disease: Confidence Intervals for Point Estimates (Dose Expansion Part B) | 55 |
| Table | 14.2.7 Patient Listing of Duration of Stable Disease | 57 |
| Table | 14.3.1.1 Overall Summary of Treatment-Emergent Adverse Events (Dose Escalation Part A) | 59 |
| Table | 14.3.1.2 Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Dose Escalation Part A) | 60 |
| Table | 14.3.1.3 Summary of Treatment-Emergent Adverse Events by System Organ Class (Dose Escalation Part A) | 61 |
| Table | 14.3.1.4 Summary of Drug-Related, Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Dose Escalation Part A) | 63 |
| Table | 14.3.1.5 Summary of Grade 3 or Greater, Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Dose Escalation Part A) | 64 |
| Table | 14.3.1.6 Summary of Grade 3 or Greater, Drug-Related, TEAE by System Organ Class and Preferred Term (Dose Escalation Part A) | 65 |
| Table | 14.3.1.7 Summary of TEAE by Maximum Severity Grade, System Organ Class and Preferred Term (Dose Escalation Part A) | 66 |
| Table | 14.3.1.8 Summary of Drug-Related, TEAE by Maximum Severity Grade, System Organ Class and Preferred Term (Dose Escalation Part A) | 67 |
| Table | 14.3.1.9 Summary of Serious Adverse Events by System Organ Class and Preferred Term (Dose Escalation Part A) | 68 |



| Table | 14.3.1.10 Summary of Death On-Study or within 30 Days Post Last Dose (Dose Escalation Part A) | 69 |
|---|---|---|
| Table | 14.3.2.1 Patient Listing of Treatment-Emergent Adverse Events Leading to Death | 71 |
| Table | 14.3.2.2 Patient Listing of Serious Adverse Events | 72 |
| Table | 14.3.2.3 Patient Listing of Treatment-Emergent Adverse Events Leading to Drug Withdrawn | 73 |
| Table | 14.3.2.4 Patient Listing of Dose Limiting Toxicities | 74 |
| Table | 14.3.3.1 Summary of Dose Limiting Toxicities by System Organ Class and Preferred Term During Cycle One | 76 |
| Table | 14.3.3.2 Summary of Infusion-Related Reaction by Maximum Severity<br>Grade, System Organ Class and Preferred Term (Dose Escalation Part<br>A) | 77 |
| Table | 14.3.4 Patient Listing of Grade 3 and 4 Abnormal Laboratory Values During Treatment | 79 |
| Table | 14.3.5.1.1 Summary of NBF-006 Administration and Compliance for Cycle One (Dose Escalation Part A) | 81 |
| Table | 14.3.5.1.2 Summary of NBF-006 Administration and Compliance for All Treatment Cycles (Dose Escalation Part A) | 83 |
| Table | 14.3.5.1.3 Summary of NBF-006 Dose Delayed/Interrupted/Withdrawn (Dose Escalation Part A) | 85 |
| Table | 14.3.5.1.4 Summary of Concomitant Measures (Dose Escalation Part A) | 86 |
| Table | 14.3.5.2.1 Summary of Change from Baseline during Treatment Period for Hematology Tests (Dose Escalation Part A) | 87 |
| Table | 14.3.5.2.1 Summary of Change from Baseline during Treatment Period for Hematology Tests (Dose Expansion Part B) | 88 |
| Table | 14.3.5.2.2 Summary of Change from Baseline during Treatment Period for Blood Chemistry Tests (Dose Escalation Part A) | 89 |
| Table | 14.3.5.2.2 Summary of Change from Baseline during Treatment Period for Blood Chemistry Tests (Dose Expansion Part B) | 90 |
| Table | 14.3.5.2.3 Summary of Change from Baseline during Treatment | |



| | Period for Urinalysis Tests (Dose Escalation Part A) | 91 |
|---|---|---|
| Table | 14.3.5.2.3 Summary of Change from Baseline during Treatment Period for Urinalysis Tests (Dose Expansion Part B) | 92 |
| Table | 14.3.5.3.1 Summary of Shift from Baseline to Maximum CTCAE Grade during Treatment Period for Hematology Tests (Dose Escalation Part A) | 93 |
| Table | 14.3.5.3.2 Summary of Shift from Baseline to Maximum CTCAE Grade during Treatment Period for Blood Chemistry Tests (Dose Escalation Part A) | 94 |
| Table | 14.3.5.3.3 Summary of Shift from Baseline to Maximum CTCAE Grade during Treatment Period for Urinalysis Tests (Dose Escalation Part A) | 95 |
| Table | 14.3.5.5.1 Summary of ECG Data and Change from Baseline by Visit (Dose Escalation Part A) | 98 |
| Table | 14.3.5.6.1 Summary of ECG Parameter QT and QTcF Data by Visit (Dose Escalation Part A)1 | 00 |
| Table | 14.3.5.7.1 Summary of Shift from Baseline to Maximum ECOG Score (Dose Escalation Part A) | 01 |
| Table | 14.3.5.7.2 Summary of Shift from Baseline to Maximum ECOG Score (Dose Expansion Part B) | 02 |
| Table | 14.4.1.1 Summary of Mean Change from Baseline in TNF-α Overtime (Dose Escalation Part A)1 | 04 |
| Table | 14.4.1.2 Summary of Mean Change from Baseline in TNF-α Overtime (Dose Expansion Part B) | 05 |
| Table | 14.4.2.1 Summary of Mean Change from Baseline in IL-1β Overtime (Dose Escalation Part A) | 06 |
| Table | 14.4.2.2 Summary of Mean Change from Baseline in IL-1β Overtime (Dose Expansion Part B)1 | 06 |
| Table | 14.4.3.1 Summary of Mean Change from Baseline in IL-6 Overtime (Dose Escalation Part A) | 06 |
| Table | 14.4.3.2 Summary of Mean Change from Baseline in IL-6 Overtime (Dose Expansion Part B) | 06 |
| Table | 14.4.4.1 Summary of Mean Change from Baseline in IFN-γ Overtime (Dose Escalation Part A)1 | 07 |



| Table 14.4.4.2 Summary of Mean Change from Baseline in IFN-y Overtime (Dose Expansion Part B) | )7 |
|---|---|
| Table 14.4.5.1 Summary of Mean Change from Baseline in Complement-<br>CH50 Overtime (Dose Escalation Part A)10 | )7 |
| Table 14.4.5.2 Summary of Mean Change from Baseline in Complement-<br>CH50 Overtime (Dose Expansion Part B) | )7 |
| Table 14.4.6.1 Summary of Mean Change from Baseline in Complement-Bb Overtime (Dose Escalation Part A) | )7 |
| Table 14.4.6.2 Summary of Mean Change from Baseline in Complement-Bb Overtime for Dose Expansion (Part B)10 | )8 |
| Table 14.4.7.1 Summary of Mean Change from Baseline in Complement-<br>C3a Overtime (Dose Escalation Part A)10 | )8 |
| Table 14.4.7.2 Summary of Mean Change from Baseline in Complement-<br>C3a Overtime (Dose Expansion Part B) | )8 |
| Table 14.4.8.1 Summary of Mean Change from Baseline in Complement-<br>C5a Overtime (Dose Escalation Part A) | )8 |
| Table 14.4.8.2 Summary of Mean Change from Baseline in Complement-<br>C5a Overtime (Dose Expansion Part B) | )8 |
| Figure 14.2.1.1: Best Change from Baseline in Tumor Measurements for NSCLC (Waterfall Plot) for Dose Escalation (Part A) and Dose Expansion (Part B) | 33 |
| Figure 14.2.1.2: Best Change from Baseline in Tumor Measurements for Pancreatic Cancer (Waterfall Plot) (Dose Escalation Part A) | 33 |
| Figure 14.2.1.3: Best Change from Baseline in Tumor Measurements for Colorectal Cancer (Waterfall Plot) (Dose Escalation Part A) | 33 |
| Figure 14.2.1.4.1: Percent Change from Baseline in Tumor Response for NSCLC (Spider Plot) (Dose Escalation Part A) | 34 |
| Figure 14.2.1.4.2: Percent Change from Baseline in Tumor Response for NSCLC (Spider Plot) (Dose Expansion Part B) | 35 |
| Figure 14.2.1.5: Percent Change from Baseline in Tumor Response for Pancreatic Cancer (Spider Plot) (Dose Escalation Part A) | 35 |
| Figure 14.2.1.6: Percent Change from Baseline in Tumor Response for Colorectal Cancer (Spider Plot) (Dose Escalation Part A) | |
| Figure 14.2.2.1: Duration of Overall Response (Kaplan-Meier) (Dose Escalation Part A)4 Figure 14.2.2.2: Duration of Overall Response (Kaplan-Meier) (Dose Expansion Part B)4 | |
| Figure 14.2.2.3: Duration of Overall Complete Response (Kaplan-Meier) (Dose Escalation Part A) | |



| Figure 14.2.2.4: Duration of Overall Complete Response (Kaplan-Meier) (Dose |
|---|
| Expansion Part B)43 |
| Figure 14.2.2.5: Duration of Treatment per Dose Level with Patient's Response |
| Overtime (Swimmer Plot) (Dose Escalation Part A)44 |
| Figure 14.2.2.6: Duration of Treatment per Expansion Cohort with Patient's Response |
| Overtime (Swimmer Plot) (Dose Expansion Part B)44 |
| Figure 14.2.5.1: Duration of Stable Disease (Kaplan-Meier) (Dose Escalation Part A)52 |
| Figure 14.2.5.2: Duration of Stable Disease (Kaplan-Meier) (Dose Expansion Part B)52 |
| Figure 14.4.1.1: Spaghetti Plot for Individual Change from Baseline in TNF-α Overtime |
| (Dose Escalation Part A)109 |
| Figure 14.4.1.2: Spaghetti Plot for Individual Change from Baseline in TNF-α Overtime |
| (Dose Escalation Part B)109 |
| Figure 14.4.2.1: Spaghetti Plot for Individual Change from Baseline in IL-1β Overtime |
| (Dose Escalation Part A)110 |
| Figure 14.4.2.2: Spaghetti Plot for Individual Change from Baseline in IL-1β Overtime |
| (Dose Escalation Part B)110 |
| Figure 14.4.3.1: Spaghetti Plot for Individual Change from Baseline in IL-6 Overtime |
| (Dose Escalation Part A)110 |
| Figure 14.4.3.2: Spaghetti Plot for Individual Change from Baseline in IL-6 Overtime |
| (Dose Escalation Part B)110 |
| Figure 14.4.4.1: Spaghetti Plot for Individual Change from Baseline in IFN-γ Overtime |
| (Dose Escalation Part A)111 |
| Figure 14.4.4.2: Spaghetti Plot for Individual Change from Baseline in IFN-γ Overtime |
| (Dose Escalation Part B)111 |
| Figure 14.4.5.1: Spaghetti Plot for Individual Change from Baseline in Complement- |
| CH50 Overtime (Dose Escalation Part A)111 |
| Figure 14.4.5.2: Spaghetti Plot for Individual Change from Baseline in Complement- |
| CH50 Overtime (Dose Escalation Part B)111 |
| Figure 14.4.6.1: Spaghetti Plot for Individual Change from Baseline in Complement-Bb |
| Overtime (Dose Escalation Part A)111 |
| Figure 14.4.6.2: Spaghetti Plot for Individual Change from Baseline in Complement-Bb |
| Overtime (Dose Escalation Part B)112 |
| Figure 14.4.7.1: Spaghetti Plot for Individual Change from Baseline in Complement-C3a |
| Overtime (Dose Escalation Part A)112 |
| Figure 14.4.7.2: Spaghetti Plot for Individual Change from Baseline in Complement-C3a |
| Overtime (Dose Escalation Part B)112 |
| Figure 14.4.8.1: Spaghetti Plot for Individual Change from Baseline in Complement-C5a |
| Overtime (Dose Escalation Part A)112 |
| Figure 14.4.8.2: Spaghetti Plot for Individual Change from Baseline in Complement-C5a |
| Overtime (Dose Escalation Part B)112 |
| Figure 14.4.9.1: Spaghetti Plot for Individual Change from Baseline in GSTP1 mRNA |
| Level Overtime (Dose Escalation Part A)113 |



| Figure 14.4.9.2: Spaghetti | Plot for Individual Char | nge from Baseline in ( | GSTP1 mRNA |
|---|---|---|---|
| Level Overtime | (Dose Escalation Part B) | ) | 113 |



| 14.1 | Demograph | ic and l | Baseline | Data ! | Summary | Tables |
|------|-----------|----------|----------|--------|---------|--------|
|------|-----------|----------|----------|--------|---------|--------|



#### DIRECTORY/FILE.SAS


#### Table 14.1,1,1 Study Populations (Dose Escalation Part A) All Enrolled (N=n)

| | NBF-006 Dose Level (mg/kg) for Escalation (Part A) | | | NBF-006 Dose Expansion (mg/kg) (Part B) | | | | |
|---|---|---|---|---|---|---|---|---|
| Study Population | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | nnn | nnn | nnn | nnn | nna | nnn | nnn |
| Patients Enrolled [1] | mm(xx,x96) | nn(xx,x%) | nn(xxx%) | rm(xx.x96) | пп(хосх%) | nn(xx.x%) | nn(xxx4) | rm(xx.x%) |
| Met All Eligibility Criteria | m(xx.x%) | nn(xx,x%) | mn(xx.x96) | rin(xx.x96) | mm(xxxx95) | nn(xx.x%) | mn(xxxx4b) | rm(xx.x96) |
| Did Not Meet All Eligibility Criteria | rrrr(xx,x96) | nn(xx,x%) | mm(xxxx96) | rim(xxx.x96) | rim(xxxx94) | nn(xx.x%) | mn(xxxxX) | nn(xx.x94) |
| Waiver | mm(xx.x96) | mn(xx.x%) | nn(xxxx9t) | rin(xx.x96) | rm(xxxx96) | nn(xx.x96) | nn(xxxxii) | mn(xx.x96) |
| Intent-to-Treat [1] | nn(xx.x96) | nn(xx.xl6) | mn(xxxx46) | nn(xx.x%) | mm(xxxx96); | nn(xx.x96) | nn(xxxxXI) | nn(xx.x%) |
| Safety Evaluable [2] | nn(xx.x96) | nn(xx.x%) | (discording | nin(xx.x96) | rin(xxxx94) | nn(xx.x96) | nrr(xxxxx96) | nn(xx.x96) |
| Efficacy Evaluable [3] | nn(xx,x%) | mn(xx,x46) | nn(xx,x/lib) | nn(xx,x%) | nn(xxxx96) | nn(xx,x%) | mn(xxxx46) | nn(xx,x96) |

<sup>[1]</sup> intent-to-Treat (ITT) includes all participants who were enrolled (signed consent) into the study, irrespective of whether study medication was administrated or not.

Present Part A and Part B output separately, adjust title for Part B accordingly.

<sup>[2]</sup> Safety Evaluable include all patients who received any component of study treatment.

<sup>[3]</sup> Efficacy Evaluable include patients with measurable disease by RECIST 1.1 who had a baseline assessment and at least one post-baseline assessment. Cross-References; Listing 16.2.1.1, 16.2.2.1

FROGRAMMERS NOTES:



#### DIRECTORY/FILE.SAS


#### Table 14.1,1.2 Patient Disposition (Close Escalation Part A) Intent-to-Treat (N=n)

| | NBF-006 Dose Level (mg/kg) for Escalation (Part A) | | | NBF-006 Dose Expansion (mg/kg) (Part B) | | | Part B) | |
|---|---|---|---|---|---|---|---|---|
| Patient Disposition | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patient | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Patients Off-Study [1] | mm(xx.x96) | nn(xx,x%) | rm(xxxx%) | rm(xx.x96) | mm(xxxx96) | nn(xx.x%) | nn(xxx4) | nn(xx.x% |
| Reasons for Off-Study [2] | | | | | | | | |
| Off-Study Reason | mm(xx,x96) | nn(xx,x46) | nn(xxxx46) | rm(xx,x96) | mm(xxxx94) | nn(xxx96) | nn(xxxxXI) | nn(xx.x% |
| Off-Study Reason | mm(xxx.x96) | mn(xx,xHi) | nntxxxx4b). | rin(xx.x96) | rim(xxxx94) | nn(xx.x96) | nn(xxxxiii) | rin(xx.x96 |
| Off-Study Reason | nn(xx.x96) | mn(xx,x46) | nn(xxx9b) | nn(xx,x96) | nn(xxxx96) | nn(xx,x%) | mn(xxxx/6) | nn(xx,x96 |
| Off-Study Reason | mm(xx,x96) | nn(xx.x46) | nn(xxxx46) | nn(xx.x96) | mm(xxxx94) | nn(xx.x96) | mn(xxxx46) | nn(xx.x94 |
| Off-Study Reason | mm(xx,x96) | nn(xx,x%) | mn(xxxxqun | nmbxx,x96) | rin(xxxx96) | nn(xx,x%) | nn(xxxxiii) | nn(xx.x96) |

<sup>[1]</sup> Number of Patients used as denominator to calculate percentages.
[2] Patients Off-Study used as denominator to calculate percentages.
Cross-References: Listing 16.2.1.1

PROGRAMMER'S NOTES:

Only present Off-Study reason categories that are used in the database from the "Off-Study" CRF.

Sort "Reasons for Off-Study" in descending order of "Overal" frequency.
Present Part A and Part B output separately, adjust title for Part B accordingly.

15



DIRECTORY/FILE.SAS

FINAL – ddmmmyythh:mm Page 1 of x

## Table 14.1.2 Demographics (Dose Escalation Part A) Intent-to-Treat (N=n)

| | NBF-00 | 6 Dose Level (m; | g/kg) for Escalat | ion (Part A) | NBF-006 Dose Expansion (mg/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|---|
| Demographics | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patient | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Age (years) | | | | | | | | |
| N | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean | xx.x | XX.X | XX.X | XX.X | xx.x | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| Median | xx.x | XX.X | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x |
| Minimum | XX | xx | XX | XX | xx | XX | XX | xx |
| Maximum | xx | XX | XX | xx | xx | XX | xx | xx |
| Age Group (years) [1] | | | | | | | | |
| 18 to 64 | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| 65 + | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Sex [1] | | | | | | | | |
| Male | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Female | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Race [1] | | | | | | | | |
| White | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Asian | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Black or African American | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Native Hawaiian or Pacific Islander | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| American Indian or Alaska native | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Not Reported | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Other | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Ethnicity [1] | | | | | | | | |
| Hispanic or Latino | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Not Hispanic or Latino | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 16 Final Version 2.0, March 14, 2023




| feight (kg)<br>N | nnn | nnn | nnn | nnn | non | nnn | nnn | nnn |
|---|---|---|---|---|---|---|---|---|
| Mean | XXXX | xx.x | xx.x | xx.x | XX.X | XX.X | XXX | XX,X |
| Standard Deviation | X.XX | X.XX. | N.XX | X.XX | K.XX | X.XX | X.XX | XXX |
| Median | XX.X | XX,X | XX.X | XX.X | XXXX | XX.X | XX.X | XX.X |
| Minimum | 300 | ×× | xx | XX | XX | XX | XX | XX |
| Maximum | XX | xx<br>xx | xx<br>xx | xx | xx<br>xx | xx<br>xx | XX | XX<br>XX |
| WI: | | | | | | | | |
| N | ппп | nnn | nnn | nnn | ann | nnn | nnn | nnn |
| Mean | 300,0 | XX.X | xxx | xx.x | XX.X | XXXX | XX.X | XX.X |
| Standard Deviation | X,XX | x.xx | x,xx | X,XX | 36.30X | XXX | XXX. | %.XX |
| Median | 300,00 | xx.x | XX.X | xx.x | XX.X | xx.x | XX.X | XX.X |
| Minimum | 300 | XX | xx | XX | XX | XX | XX | XX |
| Maximum | XX | XX | xx | kx. | XX | XX | XX | 300 |

<sup>[1]</sup> Number of Patients used as denominator to calculate percentages.

Cross-References: Listing 16.2.4.1, 16.2.9.1

PROGRAMMER'S NOTES:

Sort Age categories as shown in table.

If age is missing, the exact age was calculated in years without decimal places as follows:

Age (years) = (Year of On-Study - Year of Birth) - Correction

Where: Correction = 1, if Birth Month > On-Study Month or Birth Month = On-Study Month and Birth Day > On-Study Day Else: Correction = 0

17

Sort Age categories as shown in table.

Sort Sex categories in descending order of "Overal" frequency.
Sort Ethnicity Origin categories in descending order of "Overall" frequency.
Present Part A and Part B output separately, adjust title for Part B accordingly.



DIRECTORY/FILE.SAS

FINAL – ddmmmyy:hh:mm Page 1 of x

#### Table 14.1.3.1 Baseline Disease Characteristics for NSCLC (Dose Escalation Part A) Intent-to-Treat (N=n)

| | | NBF-006 Dose Leve | (mg/kg) for Escalation | (Part A) |
|---|---|---|---|---|
| Baseline Disease Characteristics | 0.15 | 0.3 | onwards | Overall |
| Number of Patient | nnn | nnn | nnn | nnn |
| Primary Site [1] | | | | |
| Primary Site | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Primary Site | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Primary Site | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Disease Stage [1] | | | | |
| Stage | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Stage | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Stage | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| ECOG Performance Status [1] | | | | |
| 0 | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| 1 | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| 2 | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| EGFR Mutation [1] | | | | |
| Yes | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| No | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Unknown | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| ALK/ROSI Gene Fusion [1] | | | | |
| Yes | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| No | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Unknown | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| KRAS Genotype Mutated [1] | | | | |
| Yes | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| No | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Unknown | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Duration of Disease (month) [2] | | | | |
| BF-006-001 | Statistical Analysis Plan | Final Version 2.0, | March 14, 2023 | |
| opyright© 2016 by Theradex Oncology®, Princetor<br>Il rights reserved | 1 NJ<br>18 | Confident | al – Entire Page | |



| N | nnn | nnn | nnn | nnn |
|---|---|---|---|---|
| Mean | xx.x | XX.X | XX.X | xx.x |
| Standard Deviation | x.xx | X_XX | x.xx | x.xx |
| Median | xx.x | xx.x | xx.x | xx.x |
| Minimum | xx | xx | xx | xx |
| Maximum | XX | xx | xx | xx |
| Smoking History [3] | | | | |
| Never | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Former | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Duration of Tobacco Use (month) | | | | |
| N | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | X_XX | x.xx | x.xx |
| Median | xx.x | xx.x | xx.x | xx.x |
| Minimum | xx | XX | XX | XX |
| Maximum | xx | xx | xx | xx |
| Current | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Duration of Tobacco Use (month) | | | | |
| N | nnn | nnn | nnn | nnn |
| Mean | xx.x | XX.X | XX.X | XX.X |
| Standard Deviation | x.xx | X_XX | x.xx | x.xx |
| Median | xx.x | xx.x | XX.X | XX.X |
| Minimum | xx | xx | XX | XX |
| Maximum | XX | xx | xx | xx |
| GSTT1 Genotype [1][4] | | | | |
| Null | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Wild Type | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Unknown | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 19

Final Version 2.0, March 14, 2023


NSCLC= Non-Small Cell Lung Cancer; GSTT1= Glutathione S-Transferase theta class
[1] Number of Patients used as denominator to calculate percentages.
[2] Duration of disease is calculated from the date of initial diagnosis to the date of first study drug administration.
[3] Number of NSCLC patients used as denominator to calculate percentages.

<sup>[4]</sup> This genotype only determined for the 1.6 mg/kg dose level. Cross-References: Listing 16.2.4.2.1, 16.2.4.2.2



PROGRAMMER'S NOTES:

PROGRAMMER'S NOTES:
Calculated in Months: (Date of Initial Diagnosis - Date of First Dosel/ (365.25/12).
Sort categories in descending order of "Overail" frequency.
Note: "01jan" used when day and month missing from date of diagnosis. "01" used when only day missing from date of diagnosis.
Remove "Primary Site" if there is only one site input in data for NSCLC.
Sort ECOC Performance Status categories as shown in table.
Present Part A and Part B output separately, adjust title for Part B accordingly.
Present GSTT1 only if result data is available. GSTT1 data is also available for 1.6 mg/kg in Part A.



DIRECTORY/FILE.SAS

FINAL – ddmmmyy:hh:mm Page 1 of x

## $Table\ 14.1.3.1$ Baseline Disease Characteristics for NSCLC (Dose Expansion Part B) Intent-to-Treat (N=n)

| | | NBF-006 Dose E | xpansion (mg/kg) (Par | t B) |
|---|---|---|---|---|
| Baseline Disease Characteristics | 0.6 | 1.2 | 1.6 | Overall |
| N. J. CD. C. | | | | |
| Number of Patient | nnn | nnn | nnn | nnn |
| Primary Site [1] | | | | |
| Primary Site | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Primary Site | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Primary Site | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Disease Stage [1] | | | | |
| Stage | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Stage | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Stage | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| KRAS Genotype Mutated [1][2] | | | | |
| Yes | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| No | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Unknown | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Duration of Disease (month) [3] | | | | |
| N | nnn | nnn | nnn | Nnn |
| Mean | xx.x | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx |
| Median | xx.x | xx.x | XX.X | xx.x |
| Minimum | xx | XX | XX | xx |
| Maximum | xx | xx | xx | XX |
| Smoking History [4] | | | | |
| Never | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Former | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Duration of Tobacco Use (month) | | | | |
| N | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx |
| NEE OOF OO4 | Caratination Annal India Disc. | Fi11/i | | |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 21 Final Version 2.0, March 14, 2023




| Median | xx.x | 300.00 | xx.x | XXXX |
|---|---|---|---|---|
| Minimum | xx | XX | XX | 306 |
| Maximum | ×× | 100 | xx | 300 |
| Current | nn(xx,x\$6) | rm(xxxx96) | nn(xx,x56) | nn(xxx96) |
| Duration of Tobacco Use (month) | | | | |
| N | nnn | nnn | nnn | Non |
| Mean | xx.x | XX.X | XX.X | XXXX |
| Standard Deviation | x.xx | W.XX | N.100 | XXX |
| Median | xx.x | 300.00 | xx.x | XXX |
| Minimum | ×× | XX | ×× | XX |
| Maximum | xx | XX | xx | XX |
| GSTT1 Genotype [1] | | | | |
| Null | nn(xx,x%) | rm(xxxx96) | nn(xx,x96) | rin(xxxx%) |
| Wild Type | rm(xx.x%) | mn(xxxx96) | rin(xx.x56) | (46x,30x)mn |
| Linknown | ryn(xx.x96) | rm(xxxx94) | rint(xx.x96) | mm(xxx,x%) |

NSCLC= Non-Small Cell Lung Cancer; GSTT1= Glutathione S-Transferase theta class

#### PROGRAMMERS NOTES:

Calculated in Months: (Date of Initial Diagnosis - Date of First Dose)/ (365,25/12). Sort categories in descending order of "Overal" frequency.

Note: '01jan' used when day and month missing from date of diagnosis. '01' used when only day missing from date of diagnosis.

22

Remove "Primary Site" if there is only one site input in data for NSCLC.

Present Part A and Part B output separately, adjust title for Part B accordingly.

Present GSTT1 only if result data is available.

<sup>[1]</sup> Number of Patients used as denominator to calculate percentages.

<sup>[2]</sup> In dose expansion for NSC, C, all patients must have KRAS Genotype Mutated but, not have EGFR and ALK/ROSI Gene mutation.

<sup>[3]</sup> Duration of disease is calculated from the date of initial diagnosis to the date of first study drug administration.

<sup>[4]</sup> Number of NSCLC patients used as denominator to calculate percentages.

Cross-References: Listing 16.2.4.2.1, 16.2.4.2.2



#### <Use the above table as template for tables as below>

#### Table 14.1.3.2

Baseline Disease Characteristics for Pancreatic Cancer (Dose Escalation Part A) Intent-to-Treat (N=n)

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg

[1] Number of Patients used as denominator to calculate percentages.

[2] Duration of disease is calculated from the date of initial diagnosis to the date of first study drug administration.

Cross-References: Listing 16.2.4.2.1, 16.2.4.2.2 PROGRAMMER'S NOTES:

Calculated in Months: (Date of Initial Diagnosis - Date of First Dosey (365.25/12).

Sort categories in descending order of "Overail" frequency.

Note: '01jan' used when day and month missing from date of diagnosis. '01' used when only day missing from date of diagnosis.

Remove "Primary Site" if there is only one site input in data for Pancreatic Cancer

This table is only for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg, not for Part A (1.6 mg/kg).

Remove Smoking History, EGFR Mutation, ALK/ROSI Gene Fusion, which are only for NSCLC patients.

#### Table 14.1.3.3

Baseline Disease Characteristics for Colorectal Cancer (Dose Escalation Part A) Intent-to-Treat (N=n)

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg.

[1] Number of Patients used as denominator to calculate percentages.

[2] Duration of disease is calculated from the date of initial diagnosis to the date of first study drug administration,

Cross-References: Listing 16.2.4.2.1, 16.2.4.2.2

PROGRAMMER'S NOTES:

Calculated in Months: (Date of Initial Diagnosis - Date of First Dose) (365.25/12).

Sort categories in descending order of "Overall" frequency.

Note: '01]an' used when day and month missing from date of diagnosis. '01' used when only day missing from date of diagnosis.

Remove "Primary Site" if there is only one site input in data for Colorectal Cancer

This table is only for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg, not for Part A (1.6 mg/kg).

Remove Smoking History, EGFR Mutation, ALK/ROSI Gene Fusion, which are only for NSCLC patients.

NBF-005-001

Copyright© 2016 by Therades Oncology®, Princeton NJ

All rights reserved

Statistical Analysis Plan

23




DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b


#### Table 14.1,4 Summary of Medical History (Dose Escalation Part A) Intent-to-Treat (N=n)

| MedDRA System Organ Class | NBF-00 | 6 Dose Level (m | g/kg) for Escalat | ion (Part A) | NBF-006 Dose Expansion (mg/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|---|
| MedORA Preferred Term [1][2] | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patient | nnn | nnn | nnn | nnn | nnn | nna | nnn | nnn |
| Number of Patients with Any<br>Medical History | nn(xx.x%) | nn(xx.x%) | nn(xxxXII) | rm(xx.x96) | nn(xxx%) | nn(xx.x%) | nn(xxxXI) | nn(xx.x%) |
| MedDRA System Organ Class | mn(xx,x%) | nn(xx.x16) | nn(xxx46) | nm(kx.x96) | nn(xxx96) | nn(xxx96) | nn(xxxxW) | nn(xx.x%) |
| MedDRA Preferred Term | nn(xx.x96) | mn(xx,x%) | nntxxxx4b). | rin(xx.x96) | rim(xxxx94) | nn(xx,x96) | nn(xxxx46) | mn(xx.x96) |
| MedDRA Preferred Term | nn(xx.x96) | nn(xx,x46) | nn(xxx9b) | nn(xx,x96) | nn(xxxx96) | nn(xx,x%) | rin(xxx16) | rin(xx,x96) |
| MedDRA Preferred Term | nn(xx,x96) | nn(xx.x%) | mm(xxxx36) | nn(xx.x96) | rin(xxxx94) | nn(xx.x96) | mm(xxxx46) | nn¢xx.x94 |
| MedDRA Preferred Term | nn(xx.x96) | nn(xx.x%) | mn(xxxx94) | nm(xx.x96) | rin(xxxx94) | nn(xx.x96) | nn(xxxxiii) | nn(xx.x96 |
| MedDRA System Organ Class | nn(xx,x%) | nn(xx.xl6) | nn(xxx46) | nn(xx.x96) | rin(xxxx96) | nn(xxx96) | mm(xxxxx46) | mn(xx.x90 |
| MedDRA Preferred Term | nn(xx,x96) | nn(xx.x%) | (dPx_xx)nn | rinčxx.x96) | nn(xxxx96) | nn(xx,x56) | nn(xxxxXii) | mn(xx.x96) |
| MedDRA Preferred Term | nn(xx,x%) | nn(xx,xi6) | mn(xx.x96) | nn(xx.x%) | nn(xxx96) | nn(xx,x%) | mm(xxxx46) | nn(xx.x% |
| MedDRA Preferred Term | mm(xx.x96) | nn(xx.x%) | mm(xx,x%) | rim(xx,x%) | rin(xxxx/6) | nn(xx,x96) | пп(хосжін) | nn(xx.x96 |

[1] MedDRA version 21.1

[2] Number of Patients is used as denominator to calculate percentages.

[3] Patients with multiple Medical History Events were only counted once within a summary category; system organ class and preferred term. Patients with events in more than one category were counted once within each category.

Cross-References: Usting 16.2.4.3
PROGRAMMERS NOTES:

Include all "Therapeutic Class" categories found in the database,
Sort "Therapeutic Class" column in descending order based on "Overal" column frequency count.

Present Part A and Part B output separately, adjust title for Part B accordingly.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan

24




mm:rl/tymmmbb - JAVI3 ZAZ.3JRYY9DTD39IQ zAZ.3JRY78DTD30IQ df\tau basef q f\0.0-000-000 Phase 1/1b

## Table 14.1.5.1 Prior Cancer Therapy for NSCLC (Dose Escalation Part A) Intent-to-Treat (N=n)

| opvrieht© 2016 by Theradex Oncologe | | 9 sizylenA leoitzi | ueli | Final Version 2.0 | , March 14, 2023 | | | |
|---|---|---|---|---|---|---|---|---|
| Unknown | (%x-xx)uu | (%x.xx)nn | (%x-xx)uu | (%x·xx)uu | (%x·xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Not Applicable | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x.xx)nn |
| Progressive Disease | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Stable Disease | (%x-xx)uu | (%x·xx)uu | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Partial Response | (%x-xx)uu | (%x·xx)uu | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Complete Response | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Best Response | | | | | | | | |
| <br>Яедітепз | (%x-xx)uu | (%x.xx)nn | (%x*xx)uu | (%x-xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| гиәші <b>З</b> әң 7 | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| 1 Regimen | (%x-xx)uu | (%x.xx)nn | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Ио Regimen | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x·xx)uu |
| Prior Immunotherapy | | | | | | | | |
| Пиклоwn | (%x-xx)uu | (%x-xx)uu | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu |
| Not Applicable | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Progressive Disease | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Stable Disease | (%x-xx)uu | (%x.xx)nn | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu |
| Partial Response | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x·xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Complete Response | (%x·xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x*xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Best Response | | | | | | | | |
| <br>snəmigəA ə=< | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x.xx)nn |
| Z Regimens | (%x-xx)uu | (%x·xx)uu | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu |
| 1 Regimen | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x*xx)uu | (%x·xx)uu | (%x·xx)uu | (%x.xx)nn |
| No Regimen | (%x-xx)uu | (%x.xx)nn | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu |
| Prior Chemotherapy | | | | | | | | |
| Vumber of Patient | uuu | uuu | uuu | uuu | uuu | uuu | uuu | uuu |
| Prior Cancer Therapy [1][2] | 21.0 | 6.0 | ouwards | Overall | 9.0 | 2.1 | 9.1 | Overall |
| | NBE-0 | n) ləvəl əsoO ə0 | ng/kg) for Escalat | (A hsq) noi: | NBL | -006 Dose Exps | l) (g/kg) (noizni | (8 the |

Sonfidential - Entire Page

Copyright© 2016 by Theradex Oncology®, Princeton M All rights reserved

57



| Il rights reserved | | 97 | | Confider | age4 əntire Page | | | |
|---|---|---|---|---|---|---|---|---|
| opyright© 2016 by Theradex Oncolog<br>SPF-006-001 | | 3 sizylenA lesitzi | uel | Final Version 2.0 | ), March 14, 2023 | | | |
| Stable Disease | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x·xx)uu | (%x·xx)uu |
| Partial Response | (%x-xx)uu | (%x·xx)uu | (%x*xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Complete Response | (%x-xx)uu | (%x·xx)uu | (%xxx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Best Response | | | | | | | | |
| девітепз<br>Яевітепз | (%x-xx)uu | (%x-xx)uu | (%x*xx)uu | (%x-xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Z Regimens | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x·xx)uu |
| 1 Regimen | (%x-xx)uu | (%x·xx)uu | (%x <sup>-</sup> xx)uu | (%x-xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu |
| Мо Regimen | (%x-xx)uu | (%x·xx)uu | (%x*xx)uu | (%x·xx)uu | (%x-xx)u u | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| All lines of Therapies | | | | | | | | |
| Unknown | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x·xx)uu | (%x·xx)uu |
| 9lds⊃ilqqA foN | (%x-xx)uu | (%x.xx)nn | (%xxx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x·xx)uu | (%x·xx)uu |
| Progressive Disease | (%x-xx)uu | (%x.xx)nn | (%xxx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x·xx)uu | (%x.xx)nn |
| Stable Disease | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x*xx)uu | (%x·xx)uu | (%x·xx)uu | (%x.xx)nn |
| Partial Response | (%x-xx)uu | (%x·xx)uu | (%x*xx)uu | (%x·xx)uu | (%x*xx)uu | (%x·xx)uu | (%x·xx)uu | (%x·xx)uu |
| Best Response<br>Complete Response | (%x·xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu | (%x.xx)nn |
| <br>э=6 Regimens | (%x-xx)uu | (%x.xx)nn | (%x-xx)uu | (%x-xx)uu | (%x·xx)uu | (%x·xx)uu | (%x-xx)uu | (%x.xx)nn |
| Z Regimens | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x·xx)uu |
| 1 Regimen | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| иэті <b>д</b> эя оN | (%x-xx)uu | (%x.xx)nn | (%x:xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x·xx)uu | (%x·xx)uu |
| Other Prior Therapies | | | | | | | | |
| Unknown | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x·xx)uu |
| 9ldspilgqA foU | (%x-xx)uu | (%x·xx)uu | (%xxx)uu | (%x·xx)uu | (%x-xx)u u | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Progressive Disease | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x·xx)uu | (%x.xx)nn |
| Stable Disease | (%x-xx)uu | (%x·xx)uu | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x-xx)u u | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| 92noq29A leit169 | (%x-xx)uu | (%x·xx)uu | (%xxx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu |
| Complete Response | (%x-xx)uu | (%x.xx)nn | (%x*xx)uu | (%x·xx)uu | (%x-xx)uu | (%x·xx)uu | (%x-xx)uu | (%x.xx)nn |
| Best Response | | | | | | | | |
| Regimens | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x.xx)nn |
| z Regimens | (%x-xx)uu | (%x.xx)nn | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x·xx)uu | (%x·xx)uu | (%x.xx)nn |
| nəmigəA f | (%x-xx)uu | (%x.xx)nn | (%x <sup>-</sup> xx)uu | (%x·xx)uu | (%x·xx)uu | (%x·xx)uu | (%x·xx)uu | (%x.xx)nn |
| No Regimen | (%x-xx)uu | (%x·xx)uu | (%x*xx)uu | (%x·xx)uu | (%x-xx)uu | (%x-xx)uu | (%x-xx)uu | (%x·xx)uu |
| Prior Hormone Therapy | | | | | | | | |



| Progressive Disease | nn(xxxx%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x46) | nn(xx.x%) | nn(xx.x%) | nn(xx.x16) | nn(xx.x%) |
|---|---|---|---|---|---|---|---|---|
| Not Applicable | nn(xxxx%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x46) | nn(xx.x%) | nn(xx.x%) | nn(xx.x16) | nn(xx.x%) |
| Unknown | nn(xxxx%) | nn(xx,x%) | nn(xx.x%) | nn(xx.x46) | nn(xx.x%) | nn(xx.x%) | nn(xx.x16) | nn(xx.x%) |
| Prior Cancer Radiation [2] | nn(xxx,x%) | nn(xx.x%) | nn(xx.x%) | nn(xx,x16) | nn(xx.x/6) | nn(xx.x96) | nn(xx;x%) | nn(xx.x%) |
| Prior Cancer Surgeries [2] | | nn(xx,x%) | nn(xx.x%) | nn(xx,x16) | nn(xx.x/6) | nn(xx.x96) | nn(xx;x%) | nn(xx.x%) |

Present Part A and Part B output separately, adjust title for Part B accordingly.

NSCLC= Non-Small Cell Lung Cancer
[1] Number of Patients used as denominator to calculate percentages.
[2] Patients may be counted in inore than one prior therapy categories.
Cross-References: Listing 16.2.4.4, 16.2.4.5, 16.2.4.6, 16.2.4.7
PROGRAMMERS NOTES:



#### <Use the above as template repeat for>

#### Table 14,1,5,2 Prior Cancer Therapy for Pancreatic Cancer (Dose Escalation Part A) Intent-to-Treat (N=n)

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg,

- [1] Number of Patients used as denominator to calculate percentages.
- [2] Patients may be counted in more than one prior therapy categories. Cross-References; Listing 16.2.4.4, 16.2.4.5, 16.2.4.6, 16.2.4.7 PROGRAMMERS NOTES;

This table is only for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg, not for Part A (1.6 mg/kg)

#### Table 14.1.5.3 Prior Cancer Therapy for Colorectal Cancer (Dose Escalation Part A) Intent-to-Treat (N=n)

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg.

- [1] Number of Patients used as denominator to calculate percentages.
- [2] Patients may be counted in more than one prior therapy categories.

Cross-References: Listing 16.2.4.4, 16.2.4.5, 16.2.4.6, 16.2.4.7

PROGRAMMER'S NOTES:

This table is only for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg, not for Part A (1.6 mg/kg).

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 28




# 14.2 Efficacy Data Summary Tables and Figures

Statistical Analysis Plan

29



DIRECTORY/FILE.SAS

FINAL – ddmmmyythhtmm Page 1 of x

Table 14.2.1.1

Best Overall Response Summary based for NSCLC (Dose Escalation Part A and Dose Expansion Part B)

Efficacy Evaluable (N=n)

| | NBF-006 D | ose Level (mg | /kg) for Escala | ation (Part A) | NBF-006 Dose Expansion (mg/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|---|
| Best Overall Response | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patient | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Best Overall Response [1] | | | | | | | | |
| Complete Response (CR) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| CR Unconfirmed (uCR) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Partial Response (PR) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| PR Unconfirmed (uPR) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Stable Disease (SD) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Progressive Disease (PD) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Not Evaluable (NE) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Missing | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Overall Response (CR or PR) [2][3] | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Lower 95% Confidence Limit | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx_x% | xx.x% |
| Upper 95% Confidence Limit | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% |
| Overall Response 2 (CR or uCR or PR or uPR) [3][4] | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Lower 95% Confidence Limit | xx.x% | xx.x% | xx_x% | xx.x% | xx.x% | xx.x% | xx_x% | xx.x% |
| Upper 95% Confidence Limit | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% |
| Disease Control Rate (CR or PR or SD) [3][5] | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Lower 95% Confidence Limit | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% |
| Upper 95% Confidence Limit | xx.x% | xx.x% | xx_x% | xx.x% | xx.x% | xx.x% | xx_x% | xx.x% |
| Disease Control Rate 2 (CR or uCR or PR or uPR or SD) [3][6] | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Lower 95% Confidence Limit | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% |
| Upper 95% Confidence Limit | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% |
| Complete Response (CR) [3] | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Lower 95% Confidence Limit | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx_x% | xx.x% |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 30 Final Version 2.0, March 14, 2023



| Upper 95% Confidence Limit | xx.x46 | xx.x96 | xx.x46 | xx.x96 | ****** | хх.х% | жжж | xx.x96 |
|---|---|---|---|---|---|---|---|---|
| Complete Response 2 (CR or uCR) [3][7] | mn(xxxx/H) | nn(xx,x95) | nn(xx,x56) | nn(xx,x%) | nn(xx,x%) | nn(xxx%) | mn(xx.x%) | nn(xx,x96) |
| Lower 95% Confidence Limit | xxxx/H | xx,x95 | xx,x56 | xx,x% | xx,x% | xxx% | xx.x% | xx,x96 |
| Upper 95% Confidence Limit | xxxx/H | xx,x95 | xx,x56 | xx,x% | xx,x% | xxx% | xx.x% | xx,x96 |

# NSCLC= Non-Small Cell Lung Cancer

Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg except Part A 1.6 mg/kg, Part B at 0.6, 1.2 & 1.6 mg/kg including the 1.6 mg/kg from Part A.

- [1] Number of Patients is used as denominator to calculate percentages.
- [2] Overall Response is based on patients with either a Complete Response (CR) or Partial Response (PR).
- [3] Clopper-Pearson method is used for the calculation of the 95% confidence interval.
- [4] Overall Response 2 is based on patients with CR or uCR or PR or uPR.
- [5] Disease Control Rate is based on patients with CR or PR or SD.
- [6] Disease Control Rate 2 is based on patients with CR or uCR or PR or uPR or SD.
- [7] Complete Response 2 is based on patients with CR or uCR.
- Cross-References: Figure 14.2.1.1, Listing 16.2.6.2

#### PROGRAMMER'S NOTES:

Assumptions: Assessments of SD before Study week 5 (35 days) were treated as missing. Confirmatory scans for CR and PR must have been at least 4 weeks following initial documentation of a valid overall response.

The two-sided 95% Clopper-Pearson confidence interval was calculated for the overall response rates using the following SAS® code.

EdwerCL = 1-betainv (1-alpha/2, N-x=1, x)

UpperCl. = betainv (1-alpha/2, x+1, N-x)

where: N=sample size, X=number of responders, alpha=0.05 for a 95% confidence interval.

Derive uCR and uPR per SAP, they are not collected on CRF.

Remove missing if no missing value.

Present Part A and Part B output in same table.

Present Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg except Part A 1.6 mg/kg. Present Part B at 0.6, 1.2 & 1.6 mg/kg including the 1.6 mg/kg from Part A.



<Use the above as template repeat for>

## Table 14.2.1.2

Best Overall Response Summary based for Pancreatic Cancer (Dose Escalation Part A)

Efficacy Evaluable (N=n)

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg Cross-References; Figure 14.2.1.2, Listing 16.2.6.2

PROGRAMMERS NOTES:

This table is only for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg, not for Part A 1.6 mg/kg.

Table 14.2.1.3 Best Overall Response Summary based for Colorectal Cancer (Dose Escalation Part A) Efficacy Evaluable (N=n)

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg Cross-References; Figure 14.2.1.3, Listing 16.2.6.2 PROGRAMMER'S NOTES;

This table is only for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg, not for Part A 1.6 mg/kg.

32



Figure 14.2.1.1; Best Change from Baseline in Tumor Measurements for NSCLC (Waterfall Plot) for Dose Escalation (Part A) and Dose Expansion (Part B) Efficacy Evaluable (N=n)



Horizontal reference ranges using definitions for progression (+20) and partial response (+30)
Y-axis scale should always be -100 to 100 to avoid presenting extreme values. Values that are capped as a result of this restriction to the scale are marked with \*
Cross-References: Table 14.2.1.1. Listings 16.2.6.2

PROGRAMMER'S NOTES:

Horizontal reference ranges use (+20) for progression and (-30) for partial response.

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use colors and/or patterns, and legend to present different dose levels.

Add patient number with best response.

Present Part A and Part & output in same figure.

<Use the above as template repeat for>

Figure 24.2.1.2: Best Change from Baseline in Tumor Measurements for Pancreatic Cancer (Waterfall Plot) (Dose Escalation Part A)

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg

Cross-References: Table 14.2.1.2. Listings 16.2.6.2

PROGRAMMERS NOTE: This is for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg.

Figure 34.2.1.3: Sest Change from Baseline in Tumor Measurements for Colorectal Cancer (Waterfall Plot) (Oose Escalation Part A)

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg Cross-References: Table 14.2,1.3, Listings 16.2.6.2

PROGRAMMER'S NOTE: This is for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg.

| N8F-006-001 | Statistical Analysis Plan | Final Version 2.0, March 14, 2023 |
|---|---|---|
| Copyright© 2016 by Theradex Occology®, Pri | nceton NJ | |



Figure 44.2.1.4.1: Percent Change from Baseline in Turnor Response for NSCLC (Spider Plot) (Dose Escalation Part A) Efficacy Evaluable (N=r)



For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg except Part A 1.6 mg/kg.

Y-axis scale should always be -100 to 100 to avoid presenting extreme values, Values that are capped as a result of this restriction to the scale are marked with \* Cross-References: Table 14.2.1.1. Listings 16.2.6.2

PROGRAMMERS NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Add patient number and responses.

Use colors and/or patienns, and legend to present different dose levels.

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg except Part A 1.6 mg/kg.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan

34




# <Use the above as template repeat for>

Figure 54.2.1.4.2: Percent Change from Baseline in Tumor Response for NSCLC (Spider Plot) (Dose Expansion Part 8) Efficacy Evaluable (N=n)

For Part 8 at 0.6, 1.2.8 1.6 mg/kg including the 1.6 mg/kg from Part A.
Y-axis scale should always be -100 to 100 to avoid presenting extreme values. Values that are capped as a result of this restriction to the scale are marked with \*
Cross-References: Table 14.2.1.1. Listings 16.2.6.2

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Add patient number and responses

Use colors and/or patterns, and legend to present different dose levels. Present Part 8 at 0.6, 1.2 & 1.6 mg/kg including the 1.6 mg/kg from Part A.

## <Use the above as template repeat for>

Figure 64.2.1.5: Percent Change from Baseline in Tumor Response for Pancreatic Cancer (Spider Plot) (Dose Escalation Part A) Efficacy Evaluable (N=n)

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg. Cross-References: Table 14.2.1.2, Listings 16.2.6.2

PROGRAMMERS NOTE:

This is for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/sg. Use colors and/or patterns, and legend to present different dose levels.

Figure 74.2.1.6: Percent Change from Baseline in Tumor Response for Colorectal Cancer (Spider Plot) (Dose Escalation Part A) Efficacy Evaluable (N=n)

For Part A dose level at 0.15, 0.3, 0,6, 1.2 mg/kg.

Cross-References: Table 14.2.1.3, Listings 16.2.6.2

PROGRAMMER'S NOTE:

This is for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg.
Use colors and/or patterns, and legend to present different dose levels.

Statistical Analysis Plan

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved


35



DIRECTORY/FILE.SAS FINAL – ddmmmyy:hh:mm NBF-006-001 Phase 1/1b Page 1 of x

#### Table 14.2.2.1 Life Table Summary of Duration of Overall Response (Dose Escalation Part A) Efficacy Evaluable (N=n)

| | | NBF-006 Dose | e Level (mg/kg) for | Escalation (Part A) | |
|---|---|---|---|---|---|
| Duration of Overall Response | 0.15 | 0.3 | 0.6 | 1.2 | Overall |
| Number of Patients | xx | xx | XX | XX | xx |
| Number of Fatients Number of Events | xx<br>xx (xx.x%) | xx<br>xx (xx.x%) | xx (xx.x%) | xx<br>xx (xx.x%) | xx<br>xx (xx.x%) |
| | • , | • ' | • / | , , | • / |
| Number of Censored [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Duration of Overall Response [1][3] | | | | | |
| 75% Progression-free | xxx days | xxx days | xxx days | xxx days | xxx days |
| Median | xxx days | xxx days | xxx days | xxx days | xxx days |
| Lower 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days | xxx days |
| Upper 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days | xxx days |
| 25% Progression-free | xxx days | xxx days | xxx days | xxx days | xxx days |
| Last Observation | xxx days | xxx days | xxx days | xxx days | xxx days |
| Duration of Overall CR [21[3] | | | | | |
| 75% Progression-free | xxx days | xxx days | xxx days | xxx days | xxx days |
| Median | xxx days | xxx days | xxx days | xxx days | xxx days |
| Lower 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days | xxx days |
| Upper 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days | xxx days |
| 25% Progression-free | xxx days | xxx days | xxx days | xxx days | xxx days |
| Last Observation | xxx days | xxx days | xxx days | xxx days | xxx days |
| Progression-Free Rate | | | | | |
| Baseline | 100.0% | 100.0% | 100.0% | 100.0% | 100.0% |
| 2 cycles (84 days) | xx.x % | xx.x % | xx.x % | xx.x % | xx.x % |
| 4 cycles (168 days) | xx.x % | xx.x % | xx.x % | xx.x % | xx.x % |
| 6 cycles (252 days) | xx.x % | xx.x % | xx.x % | xx.x % | xx.x % |
| 8 cycles (336 days) | xx.x % | xx.x % | xx.x % | xx.x % | xx.x % |
| Last Event (xxx days) | xx.x % | xx.x % | xx.x % | xx.x % | xx.x % |

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg except Part A 1.6 mg/kg.

NBF-006-001 Statistical Analysis Plan Final Version 2.0, March 14, 2023 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved 36

<sup>[1]</sup> Duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Only



patients with a confirmed CR or PR are included in the analysis. Symptomatic deterioration is not considered PD. For a patient without evidence of disease progression, duration of overall response will be consored at the date of last evaluable tumor assessment.

[2] Duration of overall complete response is measured from the time measurement interia are first met for CR until the first date that recurrent disease is objectively documented. Only patients with a confirmed CR are included in the analysis. Symptomatic deterioration is not considered PD. For a patient without evidence of disease progression, duration of overall CR will be censored at the date of last evaluable turnor assessment.

[3] Life Table estimates are calculated using Kaplan-Meler methodology. Confidence interval for the median survival time was calculated using the method by Brookmeyer and Crowley.

Cross-References: Figure 14.2.2.1, Table 14.2.4, Listing 16.2.6.2 PROGRAMMERS NOTES:

Only include if CR or PR responses are found in the database.

Life Table estimates are calculated using Kapian-Meier methodology, Confidence interval for the median duration time is calculated using the method by Brookineyer and Crowley.

Lipdate timepoint prior to last event per available data.

Present at every even numbered cycle for Part A dose level at 0.15, 8.3, 0.6, 1.2 mg/kg except Part A 1.6 mg/kg.



DIRECTORY/FILE.SAS

FINAL – ddmmmyy:hh:mm

NBF-006-001 Phase 1/1b


Table 14.2.2.2 Life Table Summary of Duration of Overall Response (Dose Expansion Part B) Efficacy Evaluable (N=n)

| | | NBF-006 Dose Exp | oansion (mg/kg) (Par | t B) |
|---|---|---|---|---|
| Duration of Overall Response | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | xx | xx | xx | xx |
| Number of Events | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Censored [1] | xx (xx.x%) | xx (xx.x%) | ×× (××.×%) | xx (xx.x%) |
| Duration of Overall Response [1][3] | | | | |
| 75% Progression-free | xxx days | xxx days | xxx days | xxx days |
| Median | xxx days | xxx days | xxx days | xxx days |
| Lower 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days |
| Upper 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days |
| 25% Progression-free | xxx days | xxx days | xxx days | xxx days |
| Last Observation | xxx days | xxx days | xxx days | xxx days |
| Duration of Overall CR [2][3] | | | | |
| 75% Progression-free | xxx days | xxx days | xxx days | xxx days |
| Median | xxx days | xxx days | xxx days | xxx days |
| Lower 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days |
| Upper 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days |
| 25% Progression-free | xxx days | xxx days | xxx days | xxx days |
| Last Observation | xxx days | xxx days | xxx days | xxx days |
| Progression-Free Rate | | | | |
| Baseline | 100.0% | 100.0% | 100.0% | 100.0% |
| 1 cycle (42 days) | xx.x % | xx.x % | xxx % | xx.x % |
| 2 cycles (84 days) | xx.x % | xx.x % | xx.x % | xx.x % |
| 3 cycles (126 days) | xx.x % | xx.x % | xx.x % | xx.x % |
| 4 cycles (168 days) | xx.x % | xx.x % | xx.x % | xx.x % |
| 5 cycles (210 days) | xx.x % | xx.x % | xx.x % | xx.x % |
| | | ••••• | | |
| Last Event (xxx days) | xx.x % | xx_x % | xx.x % | xx.x % |

<sup>[1]</sup> Duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Only

38

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan Final Version 2.0, March 14, 2023



patients with a confirmed CR or PR are included in the analysis. Symptomatic deterioration is not considered PD. For a patient without evidence of disease progression, duration of overall response will be censored at the date of last evaluable tumor assessment.

[2] Duration of overall complete response is measured from the time measurement interia are first met for CR until the first date that recurrent disease is objectively documented. Only patients with a confirmed CR are included in the analysis. Symptomatic deterioration is not considered PD. For a patient without evidence of disease progression, duration of overall CR will be censored at the date of last evaluable turnor assessment.

[3] Life Table estimates are calculated using Kaplan-Meler methodology. Confidence interval for the median survival time was calculated using the method by Brookmeyer and Crowley.

Cross-References: Figure 14.2.2.2 Table 14.2.4. Listing 16.2.6.2 PROGRAMMERS NOTES:

Only include if CR or PR responses are found in the database.

Life Table estimates are calculated using Kapian-Meier methodology, Confidence interval for the median duration time is calculated using the method by Brookineyer and Crowley.

Lipdate timepoint prior to last event per available data,

Present Part A and Part B output separately, adjust title for Part B accordingly.

Present at every cycle for Part 8 at 0.6, 1.2, 1.6 mg/kg including the 1.6 mg/kg from Part A.



Figure 84.2.2.1: Duration of Overall Response (Kaplan-Meler) (Dose Escalation Part A) Efficacy Evaluable (N=n)



## O O O Censored Patients

For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg.

Duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Only patients with a confirmed CR or PR (SAP section S.4.1) are included in the analysis. Symptomatic deterioration is not considered PD. For a patient without evidence of disease. progression, duration of overall response will be consored at the date of last evaluable tumor assessment. Cross-References: Table 14.2.2.1, Table 14.2.4, Listing 16.2.6.2 PROGRAMMER'S NOTES:

Kaplan-Meier curves are generated using log-rank test. Draw horizontal reference line representing 50% level (median).

Update timepoint prior to last event per available data.

Present for Part A at dose level at 0.15, 0.3, 0.6, 1.2 mg/kg except Part A 1.6 mg/kg, and overall.

Use different colors or patterns and legend to indicate 0.15, 0.3, 0.6, 1.2 mg/kg and Overall.

# <Use the above as template repeat for>

| N8F-006-001 | Statistical Analysis Plan | Final Version 2.0, March 14, 2023 |
|---|---|---|
| Copyright© 2016 by Therades Oncology®, Princeton NJ | Server and the server | |



### Figure 94.2.2.2: Duration of Overall Response (Kaplan-Meier) (Dose Expansion Part B) Efficacy Evaluable (N=r)

For Part B at 0.6, 1.2, 1.6 mg/kg including the 1.6 mg/kg from Part A. Cross-References: Table 14.2.2, Table 14.2.4, Listing 16.2.6.2 PROGRAMMER'S NOTES:

Add 1.6 mg/kg for Dose Expansion (Part 8), Present Part A and Part B output separately, adjust title for Part B accordingly. Present for Part B at 0.6, 1.2, 1.6 mg/kg including the 1.6 mg/kg from Part A.

Use different colors or patterns and legend to indicate 0.6, 1.2, 1.6 mg/kg and Overall.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 41




Figure 164.2,2.3: Duration of Overall Complete Response (Kaplan-Meier) (Dose Escalation Part A) Efficacy Évaluable (N=n)



# O O O Censored Patients

# For Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg.

Duration of overall complete response is measured from the time measurement criteria are first met for CR until the first date that recurrent or progressive disease is objectively documented. Only confirmed CR is included. Symptomatic deterioration is not considered PD. For a patient without evidence of disease progression, duration of overall complete response will be consored on the date of last evaluable turnor assessment.

Cross-References: Table 14.2.2.1, Table 14.2.4, Listing 16.2.6.2
PROGRAMMERS NOTES:

Kaplan-Meier curves are generated using log-rank test. Draw horizontal reference line representing 50% level (inedian).

Update timepoint prior to last event per available data.

Present for Part Alat dose level at 0.15, 0.3, 0.6, 1.2 mg/kg except Part All.6 mg/kg, and overall. Use different colors or patterns and legend to indicate 0.15, 0.3, 0.6, 1,2 mg/kg and Overall.

# <Use the above as template repeat for>

| N8F-006-001 | Statistical Analysis Plan | Final Version 2.0, March 14, 2023 |
|---|---|---|
| Copyright© 2016 by Theradex Oncology®, Princeton NJ<br>All rights reserved | 42 | Confidential - Entire Page |



### Figure 114.2.2.4: Duration of Overall Complete Response (Kaplan-Meler) (Dose Expansion Part B) Efficacy Evaluable (N=n)

For Part B at 0.6, 1.2, 1.6 mg/kg including the 1.6 mg/kg from Part A.

Cross-References: Table 14.2.2.2, Table 14.2.4, Listing 16.2.6.2

PROCRAMMERS NOTES:

Add 1.6 mg/kg for Dese Expansion (Part B), Present Part A and Part B output separately, adjust title for Part B accordingly.

Present for Part B at 0.6, 1.2, 1.6 mg/kg including the 1.6 mg/kg from Part A.

Use different colors or patterns and legend to indicate 0.6, 1.2, 1.6 mg/kg and Overall.

NBF-006-001 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 43




Figure 124.2.2.5: Duration of Treatment per Dose Level with Patient's Response Overtime (Swimmer Plot) (Dose Escalation Part A)

Efficacy Evaluable (N=n)



Crass-References: Appendix Listing 16.2.6.2

PROGRAMMER'S NOTES:

The X-axis displays individual patient's tumor response overtime,

The Y-axis displays the individual patients that received the study drug.

Present patient 10 on the left.

Figure 134,2,2.6: Duration of Treatment per Expansion Cohort with Patient's Response Overtine (Swimmer Plot) (Dose Expansion Part B)

Efficacy Evaluable (N=n)

Cross-References: Appendix Listing 16.2.6.2

PROGRAMMER'S NOTES:

The X-axis displays individual patient's tumor response overtime,

The Y-axis displays the individual patients that received the study drug.

Present patient ID on the left.

NBF-006-001 Copyright© 2016 by Therades Occology®, Princeton NJ All rights reserved

Statistical Analysis Plan




DIRECTORY/FILE.SAS

FINAL – ddmmmyy:hh:mm Page 1 of x

Table 14.2.3.1

Life Table Analysis of Duration of Overall Response: Confidence Intervals for Point Estimates (Dose Escalation Part A)

Efficacy Evaluable (N=n)

| NBF-006 Dose | Number at | Cumulative | Progression-Free | 95% Confidenc | e Interval [2] |
|---|---|---|---|---|---|
| Timepoint | Risk | Events [1] | Rate | Lower | Upper |
| 0.15 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 6 cycles (252 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 8 cycles (336 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| | | | | ***** | |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 0.3 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 6 cycles (252 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 8 cycles (336 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| | <del></del> | | | | |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 0.6 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 6 cycles (252 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 8 cycles (336 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Onward | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan


ts reserved 45 Confidential – Entire Page



| 6 cycles (252 days) | nnn | non | xx.x46 | xx.x% | xx_x96 |
|-----------------------|----------|----------|--------|--------|--------|
| 8 cycles (336 days) | nnn | מחרו | XX.X% | XX.X96 | XX,X96 |
| 1404 | | . Colore | | 94444 | , |
| Last Event (xxx days) | non | nnn | **.×% | xx.x96 | XX.X96 |
| Overall | | | | | |
| Baseline | mm | mnn | 100.0% | xx.x96 | xx.x% |
| 2 cycles (84 days) | nnn | mnn | xx.x% | xx.x96 | XX.X96 |
| 4 cycles (168 days) | nnn | rinn | xx,x%- | xx.x96 | xx.x% |
| 6 cycles (252 days) | mm | rinn | жжж% | xx.x96 | xxx% |
| 8 cycles (336 days) | nan | מחרו | xx.x46 | xx.x56 | xx,x56 |
| 1000 | ******** | F-91944 | | 164616 | (man) |
| Last Event (xxx days) | nnn | rinn | ×x.x% | xx.x% | xx.x% |

<sup>[1]</sup> Duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Only patients with a confirmed CR or PR (SAP section 5.4.1) are included in the analysis. Symptomatic deterioration is not considered PD: For a patient without evidence of disease progression, duration of overall response will be censored at the date of last evaluable tumor assessment.

#### PROGRAMMER'S NOTES:

Life Table estimates are calculated using Kaplan-Meier methodology. Confidence interval for a point estimate on the survival distribution is calculated using the method by Kabifleisch and Prentice.

Present at every even numbered cycle for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg except Part A 1.6 mg/kg.

46

<sup>[2]</sup> Life Table estimates are calculated using Kaplan-Meier methodology. Confidence interval for a point estimate on the survival distribution is calculated using the method by Kalbfielsch and Prentice.

Cross-Reference: Table 14.2.4, Listing 16.2.6.2



DIRECTORY/FILE.SAS FINAL – ddmmmyy;hh;mm Page 1 of x

Table 14.2.3.2
Life Table Analysis of Duration of Overall Response: Confidence Intervals for Point Estimates (Dose Expansion Part B)
Efficacy Evaluable (N=n)

| NBF-006 Dose | Number at | Cumulative | Progression-Free | 95% Confidenc | e Interval [2] |
|---|---|---|---|---|---|
| Timepoint | Risk | Events [1] | Rate | Lower | Upper |
| 0.6 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 1 cycle (42 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 3 cycles (126 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 5 cycles (210 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 1.2 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 1 cycle (42 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 3 cycles (126 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 5 cycles (210 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 1.6 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 1 cycle (42 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 3 cycles (126 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 5 cycles (210 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Last Event (xxx days) | nnn | nnn | <br>xx.x% | <br>xx.x% | <br>xx.x% |
| Last Everit (AAA days) | 11111 | 111111 | 2010/4 | 20.070 | 00.079 |
| Overall | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 1 cycle (42 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 47 Final Version 2.0, March 14, 2023



| 2 cycles (84 days) | nnn | mon | ×x.x% | xx.x96 | XX.X96 |
|---|---|---|---|---|---|
| 3 cycles (126 days) | nnn | 1700 | xx.x% | XX.X96 | XX.X96 |
| 4 cycles (168 days) | ann | cinn | xx.xH | xx.x56 | xx.x56 |
| 5 cycles (210 days) | non | nnn | ×x.×% | xx.x96 | xx.x96 |
| Carrier Control of the Control of th | ****** | | | | ****** |
| Last Event (xxx days) | nnn | mnn | ×x.×16 | xx.x56 | xx.x96 |

[1] Duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Only patients with a confirmed CR or PR (SAP section 5.4.1) are included in the analysis. Symptomatic deterioration is not considered PD. For a patient without evidence of disease progression, duration of overall response will be censored at the date of last evaluable turnor assessment.

[2] Life Table estimates are calculated using Kaplan-Meier methodology. Confidence interval for a point estimate on the survival distribution is calculated using the method by Kalbifelsch and Prentice.

Cross-Reference: Table 14.2.4, Listing 16.2.6.2

#### PROGRAMMER'S NOTES;

Life Table estimates are calculated using Kaplan-Meier methodology, Confidence interval for a point estimate on the survival distribution is calculated using the method by Kabifleisch and Prentice.

Present Part A and Part B output separately, adjust title for Part B accordingly,

Present at every cycle for Part 8 at 0.6, 1.2, 1.6 mg/kg including the 1.6 mg/kg from Part A.



NBF-006-001 Phase 1/1b DIRECTORY/FILE-SAS FINAL - ddmmmyy;th;mm

# Table 14:2.4 Patient Listing for Duration of Overall Response Efficacy Evaluable (N=n)

| | | | | Date of | Date of | Date of | Date of | Date of | Date of | Duration of | Duration of |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | Study | NBF-006 | Date of | First CR | | | First uPR | Progression | Censoring | Overall Response | Overall CR |
| /Age/Sex Part Dose(mg/kg) First Dose | First Dose | [1] | m m m | | | | | (day) [2] | [3] | | |
| сс-рррр<br>жк/х | × | XXX | ddmmmyyyy | xxxx | | | | | | iox | XXX |
| cc-pppp | × | XXX | ddmmmyyyy | | | XXXXX | | | | xxx | XXX |
| сс-рррр<br>кк∕х | × | XXX | ddmmrnyyyy | | XXX | | | | | XXX | XXX |
| сс-рррр<br>жух | × | XXX | ddmmmyyyy | | | | xxxx | XXXX | | XXX | XXX |
| cc-pppp<br>xx/x | × | XXX | ddmmmyyyy | XXXX | | | | | | xxx | XXX |
| ccc-pppp | х | XXX | ddmmrryyyy | | | | | | XXXXXXX | xxx | XXX |

- [1] CR = Complete Response, PR = Partial Response, uCR = Unconfirmed Complete Response, uPR = Unconfirmed Partial Response
- (2) Duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Symptomatic deterioration is not considered PD. For a patient without evidence of disease progression, duration of overall response will be censored.
- (3) Duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented. Only patients with a confirmed CR are included in the analysis. For a patient without evidence of disease progression, duration of overall CR will be censored. Cross-Reference. Case Report Forms: Cycle Response Assessment (RS).

### PROGRAMMER'S NOTES:

Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number.

Data used in the SAS Life Table procedure.

NBF-006-001 Statistical Analysis Plan Copyright© 2016 by Therades Occology®, Princeton NJ All rights reserved 49




DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b

#### FINAL - ddmmmyy;hh;mm Page 1 of x

#### Table 14.2.5.1 Life Table Summary of Duration of Stable Disease (Dose Escalation Part A) Efficacy Evaluable (N=n)

| | | NBF-006 Dos | e Level (rng/kg) for | Escalation (Part A) | |
|---|---|---|---|---|---|
| Duration of Stable Disease | 0.15 | 0.3 | 0.6 | 1,2 | Overall |
| Number of Patients | xx | xx | xx | xx | xx |
| Number of Events | xx (xx.x46) | AN (NOLAH) | xx (xx.x96) | xx (xx,x96) | xx (xx.x95) |
| Number of Censored [1] | xx (xx.x36) | xx (xx_x16) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Duration of Stable Disease [1][2] | | | | | |
| 75% Progression-free | xxx days | xxx days | xxx days | xxx days | xxx days |
| Median | xxx days | xxx days | xxx days | xxx days | xxx days |
| Lower 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days | xxx days |
| Upper 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days | xxx days |
| 25% Progression-free | xxx days | xxx days | xxx days | xxx days | xxx days |
| Last Observation | xxx days | xxx days | xxx days | xxx days | xxx days |
| Progression-Free Rate | | | | | |
| 2 cycles (84 days) | xx,x % | xx.x % | 300.00 Hb | xx.x % | xx.x 95 |
| 4 cycles (168 days) | xx.x % | xx.x: % | XX.X % | XX.X % | XXLX 96 |
| 6 cycles (252 days) | xx,x % | XX.X 96 | xx_x % | xx,x % | 30CX 96 |
| 8 cycles (336 days) | xx.x % | ккж % | xx.x % | ××.× % | xx.x % |
| Last Event (xxx days) | xx.x % | XX.X: % | xx.x % | XX,X % | XX.X 96. |

[1] Stable Disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started. Only patients with a SD are included in the analysis. Follow-up measurements for SD must meet the SD criteria at least 5 weeks after study entry. Symptomatic deterioration is not considered PD, For a patient without evidence of disease progression, duration of stable disease will be consored at the date of last evaluable turnor assessment.

[2] Life Table estimates are calculated using Kaplan-Meier methodology. Confidence interval for the median survival time was calculated using the method by Brookmeyer and Crowley. Cross-References: Figure 14.2.5.1, Listing 16.2.6.2

PROGRAMMERS NOTES:

Life Table estimates are calculated using Kaplan-Meier methodology, Confidence interval for the median duration time is calculated using the method by Brookmeyer and Crowley.

Update timepoint prior to last event per available data.

Present at every even numbered cycle for Part A dose level at 0.15, 0.3, 0.6, 1,2 mg/kg except Part A 1.6 mg/kg.

Statistical Analysis Plan Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved 50.




FINAL - ddmmmyy;hh;mm Page 1 of x

# Table 14.2.5.2 Life Table Summary of Duration of Stable Disease (Dose Expansion Part B) Efficacy Evaluation (Non)

| | emacy | NPE ONE Date Sur | pansion (mg/kg) (Pan | 01 |
|---|---|---|---|---|
| Duration of Stable Disease | 0.5 | | CONTRACTOR OF THE PARTY OF THE | The second secon |
| TO THE PARTY OF TH | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | XX | XX | XX. | XX |
| Number of Events | xx (xx.x%) | xx (xx,x96) | xx (xx,x96) | xx (xx.x36) |
| Number of Censured [1] | xx (xx.x%) | xx (xx.x46) | юс (жжж96) | xx (xx.x%) |
| Duration of Stable Disease [1][2] | | | | |
| 75% Progression-free | xxx days | xxx days | xxx days | xxx days |
| Median | xxx days | xxx days | xxx days | xxx days |
| Lower 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days |
| Upper 95% Confidence Limit | xxx days | xxx days | xxx days | xxx days |
| 25% Progression-free | xxx days | xxx days | .xxx days | xxx days |
| Last Observation | xxx days | xxx days | xxx days | xxx days |
| Progression-Free Rate | | | | |
| 1 cycle (42 days) | xx.x % | XX.X % | XX.X-16 | xx.x % |
| 2 cycles (84 days) | xx.x % | xx,x % | XX.X 16 | ××,× % |
| 3 cycles (126 days) | **.* % | xx.x % | JOKUK 96 | xx.x % |
| 4 cycles (168 days) | xx.x % | xx.x % | XXLX 16 | xx.x % |
| 5 cycles (210 days) | xx.x % | xx.x % | xx.x 96 | xx.x % |
| | ***** | ***** | ****** | 60000 |
| Last Event (xxx days) | **.× % | xx.x 96 | AXX.X 16 | **.* % |

[1] Stable Disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started. Only patients with a SD are included in the analysis. Follow-up measurements for SD must meet the SD criteria at least 5 weeks after study entry. Symptomatic deterioration is not considered PD. For a patient without evidence of disease progression, duration of stable disease will be consored at the date of last evaluable turnor assessment.

[2] Life Table estimates are calculated using Kaplan-Meier methodology. Confidence interval for the median survival time was calculated using the method by Brookmeyer and Crowley.

Cross-References: Figure 14.2.5.2, Listing 16.2.6.2

PROGRAMMER'S NOTES:

Life Table estimates are calculated using Kaplan-Meier methodology. Confidence interval for the median duration time is calculated using the method by Brookmeyer and Crowley.

Update timepoint prior to last event per available data,

Present at every cycle for Part 8 at 0.6, 1.2, 1.6 mg/kg including the 1.6 mg/kg from Part A.

NBF-005-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan




Figure 144.2.5.1: Duration of Stable Disease (Kaplan-Meier) (Dose Escalation Part A) Efficacy Evaluable (N=n) NBF-006-001 Phase 1/1b Phase I Study



#### O O O Censored Patients

For Part A dose level at 0.75, 0.3, 0.6, 1.2 mg/kg.

Stable Disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started. Only patients with a SD are included in the analysis. Follow-up measurements for SD must meet the SD criteria at least 5 weeks after study entry. For a patient without evidence of disease progression, duration of stable disease will be censored at the date of last evaluable tumor assessment. Cross-References: Table 14.2.5.1, Listing 16.2.6.2

#### PROGRAMMER'S NOTES:

Kaplan-Meier curves are generated using log-rank test. Draw horizontal reference line representing 50% level (median). Update timepoint prior to last event per available data.

Present Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg except Part A 1.6 mg/kg, and overall.

Figure 154.2.5.2: Duration of Stable Disease (Kaplan-Meier) (Dose Expansion Part B) Efficacy Evaluable (N=n)

For Part B at 0.6, 1.2, 1.6 mg/kg including the 1.6 mg/kg from Part A.

Cross-References: Table 14.2.5.2, Listing 16.2.6.2

#### PROGRAMMER'S NOTES:

Present Part A and Part B output separately, adjust title for Part B accordingly Present for Part B at 0.6, 1.2, 1.6 mg/kg including the 1.6 mg/kg from Part A.

Use different colors or patterns and legend to indicate 0.6, 1.2, 1.6 mg/kg and Overall.

Statistical Analysis Plan Final Version 2.0, March 14, 2023 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved 52 Confidential - Entire Page



DIRECTORY/FILE.SAS FINAL – ddmmmyy.hh:mm Page 1 of x

Table 14.2.6.1

Life Table Analysis of Duration of Stable Disease: Confidence Intervals for Point Estimates (Dose Escalation Part A)

Efficacy Evaluable (N=n)

| NBF-006 Dose | Number at | Cumulative | Progression-Free | 95% Confidenc | e Interval [2] |
|---|---|---|---|---|---|
| Timepoint | Risk | Events [1] | Rate | Lower | Upper |
| 0.15 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 6 cycles (252 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 8 cycles (336 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 0.3 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 6 cycles (252 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 8 cycles (336 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| | | | | ***** | |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 0.6 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 6 cycles (252 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 8 cycles (336 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 1.2 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 6 cycles (252 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 53 Final Version 2.0, March 14, 2023



| 8 cycles (336 days) | nnn | non | xx.x46 | xx.x56 | xx.x96 |
|-----------------------|--------|------|--------|--------|--------|
| | ****** | | ****** | | ***** |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x56 |
| Overall | | | | | |
| Baseline | nnn | חחכו | 100.0% | xx.x46 | xx.x% |
| 2 cycles (84 days) | nnn | rinn | xx.x% | xx.x96 | xx.x% |
| 4 cycles (168 days) | nnn | מחרו | xx.x% | XX.X56 | XX.X96 |
| 6 cycles (252 days) | nnn | mnn | xx,x16 | xx.x56 | xx.x% |
| 8 cycles (336 days) | nnn | rinn | ××.κ% | ×x.x96 | xx.x% |
| | nnn | | ***** | ***** | ****** |
| Last Event (xxx days) | nnn | mnn | xx.x96 | xx,x56 | xx,x96 |

<sup>[1]</sup> Stable Disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started. Only patients with a SD are included in the analysis, Follow-up measurements for SD must meet the SD criteria at least 5 weeks after study entry. For a patient without evidence of disease progression, duration of stable disease will be censored.

# PROGRAMMER'S NOTES;

<sup>[2]</sup> Life Table estimates are calculated using Kaplan-Meier methodology, Confidence interval for a point estimate on the survival distribution is calculated using the method by Kalbfielsch and Prentice. Cross-Reference: Table 14.2.7, Listing 16.2.6.2

Life Table estimates are calculated using Kaplan-Meier methodology, Confidence interval for a point estimate on the survival distribution is calculated using the method by Kalofleisch and Prentice.

Present at every even numbered cycle for Part A dose level at 0.15, 0.3, 0.6, 1.2 mg/kg except Part A 1.6 mg/kg and overall.



DIRECTORY/FILE.SAS FINAL – ddmmmyy:hh:mm


Table 14.2.6.2

Life Table Analysis of Duration of Stable Disease: Confidence Intervals for Point Estimates (Dose Expansion Part B)

Efficacy Evaluable (N=n)

| NBF-006 Dose | Number at | Cumulative | Progression-Free | 95% Confidenc | e Interval [2] |
|---|---|---|---|---|---|
| Timepoint | Risk | Events [1] | Rate | Lower | Upper |
| 0.6 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 1 cycle (42 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 3 cycles (126 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 5 cycles (210 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 1.2 mg/kg | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 1 cycle (42 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 3 cycles (126 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 5 cycles (210 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Last Event (xxx days) | nnn | nnn | <br>xx.x% | <br>xx.x% | <br>xx.x% |
| 1.6malka | | | | | |
| 1.6mg/kg<br>Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |
| 1 cycle (42 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 2 cycles (84 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 3 cycles (126 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 4 cycles (168 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| 5 cycles (210 days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Last Event (xxx days) | nnn | nnn | xx.x% | xx.x% | xx.x% |
| Overall | | | | | |
| Baseline | nnn | nnn | 100.0% | xx.x% | xx.x% |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan
55




| 1 cycle (42 days) | nnn | mnn | xx.x96 | xx.x96 | XX.X96 |
|-----------------------|-----|--------|--------|--------|---------|
| 2 cycles (84 days) | nnn | 1700 | xx.x% | XX.X96 | XX.X96 |
| 3 cycles (126 days) | ann | cinn | жж.ж% | xx.x56 | xx.x56 |
| 4 cycles (168 days) | enn | mnn | ××.×% | xx.x96 | XX.X96 |
| 5 cycles (210 days) | nnn | non | xx.x% | xx.x56 | xx.x96 |
| 4464 | | Feiner | - | +++++ | pinner. |
| Last Event (xxx days) | nnn | mnn | xx,x% | xx.x% | xx,x% |

[1] Stable Disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started. Only patients with a SD are included in the analysis. Follow-up measurements for SD must meet the SD criteria at least 5 weeks after study entry. For a patient without evidence of disease progression, duration of stable disease will be censored.

Life Table estimates are calculated using Kaplan-Meier methodology. Confidence interval for a point estimate on the survival distribution is calculated using the method by Kalbfleisch and Prentice.

Present Part A and Part B output separately. Present at every cycle for Part B at 0.6, 1.2, 1.6 mg/kg including the 1.6 mg/kg from Part A

<sup>[2]</sup> Life Table estimates are calculated using Kaplan-Meier methodology. Confidence interval for a point estimate on the survival distribution is calculated using the method by Kalbfeisch and Prentice. Cross-Reference: Table 14-2-7, Listing 16-2-6-2 PROGRAMMERS NOTES:



#### DIRECTORY/FILE.SAS


#### Table 14.2.7 Patient Listing of Duration of Stable Disease Efficacy Evaluable (Nen)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006<br>Dose (mg/kg) | Date of<br>First Dose | Date of<br>First CR [1] | Date of<br>First PR [1] | Date of<br>Progression | Date of<br>Censoring | Duration of<br>SD (day)(1)[2] |
|---|---|---|---|---|---|---|---|---|
| ccc-pppp<br>/xx/x | ж. | XX | ddmmmyyyy | ddmmmyyyy | | ddmmmyyyy | | XXX |
| еес-рррр<br>/ю/х | × | XX | ddmmmyyyy | | ddmmmyyyy | | ddmmmyyyy | XXX |
| сес-рррр<br>/ю/х | × | XX | ddmmmyyyy | | ddmmmyyyy | ddmmmyyyy | | XXX |
| ccr-pppp<br>/xx/x | <b>.</b> × | XX | ddmmmyyyy | | ddmmmyyyy | | ddmmmyyyy | XXX |

Sort "Patient" in ascending order using "pppp", and then "ccc" portion of patient number. Data used in the SAS Life Table procedure.


<sup>[1]</sup> CR- complete response, PR- partial response, SD- stable disease
[2] Stable Disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started. Only patients with a SD are included in the analysis. Follow-up measurements for SD must meet the SD criteria at least 5 weeks after study entry. For a patient without evidence of disease progression, duration of stable disease will be consored.

Cross-Reference: Case Report Forms: Cycle Response Assessment (RS) PROGRAMMER'S NOTES:



14.3.1 Display of Adverse Events



# Table 14.3.1.1 Coverall Summary of Treatment-Emergent Adverse Events (Dose Escalation Part A) Safety Evaluable (N=n)

| | N8F-006 D | ase Level (mg | /kg) for Escala | gion (Part A) | NBF-006 Dose Expansion (mg/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment-Emergent Adverse Event [1][2] | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | nnn | nnn | DIPIT | nnn | nnn | nno | nnn |
| Patients | | | | | | | | |
| With Any TEAEs | mn(xx,x46) | mn(xx,x%) | nn(xx,x96) | nn(xx.x%) | mm(xxxx94) | nn(xx.x%) | rin(xx.x%) | пиросж46 |
| With Orug Related TEAEs [3] | nn(xx.x46) | rin(xx,x%) | ne(xx,x%) | nn(xx.x16) | rin(xxxx96) | nn(xx,x%) | nn(xx,x%) | nn(xx.x16 |
| With Severity Grade 3, 4, or 5 | mm(xxxx16) | rin(xx,x%) | nn(xx.x96) | nn(xx.x46) | nn(xxxx96) | nn(xx,x96) | rin(xx,x%) | пп(хх,х% |
| With Severity Grade 3, 4, or 5 Drug Related TEAEs [3] | nn(xx.x46) | mn(xx,x%) | nn(xx,x96) | nn(xx.x36) | rin(xx.x94) | nn(xx,x%) | nn(xx.x96) | ппросхн |
| With Any Serious TEAEs | nn(xxxx46) | mn(xx.x96) | rm(xx.x96) | nn(xx.x%) | mm(xxxx96) | nn(xx.x96) | nn(xx,x96) | mpxx46 |
| With Any Serious, Drug Related TEAEs [3] | mn(xxxx/H) | nn(xx.x%) | rin(xx.x96) | nn(xx.x%) | nn(xx.x%) | nn(xx,x96) | nn(xx,x%) | nntxxx46 |
| Who Discontinued Treatment Due to TEAEs | nn(xxxx16) | mn(xx,x94) | rm(xx,x%) | nn(xx.x46) | rin(xx.x96) | nn(xx.x94) | nn(xx,x%) | ппросен |
| Who Died Due to Any TEAEs | mm(xxxxx46) | nn(xx.x96) | nn(xx,x96) | nn(xx.x36) | mm(xxxx96) | nn(xx.x96) | nn(xx.x96) | mpocx® |
| Who Experienced DLT [4] | nr16xx_x36) | nn(xx,x%) | nn(xx,x56) | nn(xxxx16) | nn(xxx96) | nn(xx,x96) | nn(xx.x96) | nntxxxx86 |

<sup>[1]</sup> Number of Patients is used as denominator to calculate percentages.

PROGRAMMER'S NOTES:

Sort in descending order using "Overall" frequency column.

Excludes events with incomplete information for grade or drug relationship. Add footnote if required: See Listing 16.2.7.4 for excluded events,

Present Part A and Part B output separately, adjust title for Part B accordingly.

NBF-006-001 Copyright© 2016 by Therades Occology®, Princeton NJ All rights reserved

Statistical Analysis Plan


<sup>[2]</sup> Treatment-Emergent Adverse Events (TEAEs) are defined as adverse events that occurred on and after the first dose date up to 30 days post last dose date. Patients with multiple TEAEs were counted once within a summary category; system organ class, preferred term, maximum grade, or relationship to treatment. Patients with events in more than one category were counted once within each category.

<sup>[2]</sup> Number of Patients is used as denominator to calculate percentages.

<sup>[3]</sup> Drug Related include relationship as Definite or Probable or Possible.

<sup>[4]</sup> DLT: Dose-limiting taxicity

Cross-References: Listing 16.2.7.1, 16.2.7.4



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b


#### Table 14,3,1,2 Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Dose Escalation Part A) Safety Evaluable (N=n)

| MedDRA System Organ Class | NBF-00 | 6 Dase Level (m | g/kg) for Escalat | ion (Part A) | NBF-006 Dose Expansion (mg/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|---|
| MedDRA Preferred Term [1] | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | onn | nnn | nnn | non | nnn. | non | nnn |
| Patients with Any TEAE [2][3] | nn(xx.x96) | nn(xxx46) | nn(xxxx96) | nn(xx.x%) | nn(xx.x90) | nn(xx.x96) | nn(xxx%) | nn(xx,x96) |
| MedDRA System Organ Class | nn(xx,x96) | nn(xxx%) | nn(xx_x96): | nn(xx.x%) | rm(xx.x95) | rint(xx,x%) | nn(xx.x%) | nn(xx,x96) |
| MedDRA Preferred Term | mm(xx,x96) | nn(xxx%) | mm(xxxxx96) | rm(xx.x56) | mm(xxxx94) | rint(xx,x56) | пп(хх.х;Ні) | nn(xx.x94) |
| MedDRA Preferred Term | mm(xx,x%) | nn(xx.x%) | mm(xxxx96) | rint(xx,x96) | mn(xx,x96) | ryrr(xx.x46) | nn(xx.xH) | nn(xx.x%) |
| MedDRA Preferred Term | mm(xx,x96) | nn(xxxH) | mm(xx,x96) | rin(xx,x96) | rm(xx.x96) | rint(xx.x96) | пп(хж.ж%) | nn(xx,x96) |
| MedDRA Preferred Term | nn(xx.x96) | nn(xxx4) | mm(xx.x96) | rm(xx.x56) | mn(xx,x96) | rm(xx.x56) | rin(xx.xH) | nn(xx.x96) |
| MedDRA System Organ Class | mm(xx.x96) | nn(xxxH) | mm(xx_x96) | nn(xx.x96) | rm(xx.x96) | rin(xx.x%) | nn(xxxx%) | nn(xx.x96) |
| MedDRA Preferred Term | mm(xx.x96) | nn(xxx4i) | mm(xxx.x96) | rin(xx.x96) | mm(xx.x94) | nn(xx.x56) | пп(хх.жн) | nn(xx.x94) |
| MedDRA Preferred Term | nn(xx.x96) | nn(xx.x%) | mm(xxxx96) | nn(xx.x%) | mn(xxx,x96) | nn(xx.x96) | nn(xxx%) | nn(xx,x96) |
| MedDRA Preferred Term | mm(xx.x%) | nn(xx.x%) | mm(xx.x%) | rin(xx.x96) | rm(xx,x94) | rin(xx.x96) | nn(xx.x%) | nn(xx.x96) |

<sup>[1]</sup> MedDRA version 21.1

Sort System Organ Class and then Preferred term in descending order using "Overall" frequency column.

Excludes events with incomplete information for grade or drug relationship. Add footnote if required: See Listing 16.2.7.4 for excluded events. Medical writer will determine the appropriate percentage cut-off point e.g., 5% or 10 % in CSR.

Present Part A and Part B output separately, adjust title for Part B accordingly.

NBF-006-001 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 60


<sup>[2]</sup> Number of Patients used as denominator to calculate percentages.

<sup>[3]</sup> Treatment-Emergent Adverse Event (TEAEs) are defined as adverse events that occurred on and after the first dose date up to 30 days post last dose date. Patients with multiple TEAEs were only counted once within a summary category; system organ class, preferred term. Patients with events in more than one category were counted once within each category. Cross-References; Usting 16.2.7.1, 16.2.7.4 PROGRAMMERS NOTES:



#### DIRECTORY/FILE.SAS

FINAL - ddmmmyy:hh:mm Page 1 of x

Table 14.3.1.3 Summary of Treatment-Emergent Adverse Events by System Organ Class (Dose Escalation Part A)
Safety Evaluable (N=n)

| | | Drug-Related[4] An | ıv | Drug-Related |
|---|---|---|---|---|
| MedDRA System Organ Class [1][2] | All TEAE | Grade [5] | Grade>= 3 [5] | >=Grade 3 [4][5] |
| Number of Patients | nnn | nnn | nnn | nnn |
| Number of Patients with Any TEAE [3] | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Blood and lymphatic system disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Cardiac disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Ear and labyrinth disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Eye disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Gastrointestinal disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| General disorders and administration site conditions | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| nfections and infestations | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| nvestigations | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Metabolism and nutrition disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Musculoskeletal and connective tissue<br>disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Neoplasms benign, malignant and unspecified<br>incl cysts and polyps) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Nervous system disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Psychiatric disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Renal and urinary disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Reproductive system and breast disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Respiratory, thoracic and mediastinal disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Skin and subcutaneous tissue disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| Vascular disorders | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |

Statistical Analysis Plan

61

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved Final Version 2.0, March 14, 2023

<sup>[1]</sup> MedDRA version 21.1 [2] Number of Patients used as denominator to calculate percentages.



[3] Treatment-Emergent Adverse Events (TEAEs) are defined as adverse events that occurred on and after the first dose date up to 30 days post last dose date. Patients with multiple TEAEs were only counted once within a summary category; system organ class, preferred term, maximum grade, or relationship to treatment. Patients with events in more than one category were counted once within each category.

[4] Orug Related include relationship as Definite or Probable or Possible.

[5] Grade: 1=Mild, 2=Moderate, 3=Severe, 4=Life threatening, 5= Death

Cross-References: Listing 16.2.7.1, 16.2.7.4 PROGRAMMERS NOTES:

Sort System Organ Class in descending order using "All TEAF" frequency column. Excludes events with incomplete information for grade or drug relationship. Add footnote if required: See Listing 16.2.7.4 for excluded events.

## Repeat for

<0.3 mg/kg>

anwards

<Overall for Dose Escalation>

Present Part A and Part B output separately, adjust title for Part B accordingly.



DIRECTORY/FILE.SAS


Table 14.3.1.4 Summary of Drug-Related, Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Dose Escalation Part A) Safety Evaluable (N=n)

| NBF-00 | 6 Dase Level (m | g/kg) for Escalat | ion (Part A) | NBF-006 Dose Expansion (mg/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|
| 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| nnn | nnn | nnn | nnn | non | 19971 | non | nnn |
| nn(xx.x%) | nn(xxx%) | nn(xxxx%) | ne(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xxx46) | nn(xx,x96 |
| nn(xx.x96)<br>nn(xx,x96) | nn(xxx%)<br>nn(xxx%) | nn(xx.x%)<br>nn(xx.x%) | nn(xx.x%)<br>nn(xx.x%) | nn(xx.x96)<br>nn(xx,x96) | nn(xx.x%)<br>nn(xx.x%) | nn(xxxXII) | nn(xx.x% |
| mm(xx,x96) | nn(xxx%)<br>nn(xxx%) | mm(xx=x96) | rm(xx.x%) | mn(xx.x94) | rm(xx,x96) | (Hx.xx)nn | nn(xx.x%<br>nn(xx.x%<br>nn(xx.x% |
| nn(xx.x96) | nn(xx.x%) | mn(xxxx96) | nn(xx.x96) | mn(xx.x94) | nn(xx.x96) | rin(ax.x%) | nn(xx.x96 |
| nn(xx.x96)<br>nn(xx.x96) | nn(xx.x%)<br>nn(xx.x%) | mm(xx.x96) | nn(xx.x96)<br>nn(xx.x96) | mn(xx,x96)<br>mn(xx,x96) | nn(xx.x%)<br>nn(xx.x%) | nn(xx.x%) | nn(xx.x96<br>nn(xx.x96<br>nn(xx.x96 |
| | 0.15 nn(xx.x%) | 0.15 0.3 nnn nnn nn(xx.x%) nn(xx.x%) nn(xx.x%) | 0.15 0.3 criwards nnn nnn nn(xx,x%) nn(xx,x%) nn(xx,x%) | nnn | 0.15 0.3 onwards Overall 0.6 nnn nnn nnn nnn nnn nnn nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) nn(xx,x%) | 0.15 0.3 onwards Overall 0.6 1.2 | 0.15 0.3 criwards Overall 0.6 1.2 1.6 |

Sort System Organ Class and then Preferred term in descending order using "Overall" frequency column.

Excludes events with incomplete information for grade or drug relationship. Add footnote if required: See Listing 16.2.7.4 for excluded events. Present Part A and Part 8 output separately, adjust title for Part 8 accordingly.

NBF-006-001 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 63


<sup>[2]</sup> Number of Patients used as denominator to calculate percentages.

<sup>[3]</sup> Treatment-Emergent Adverse Events (TEAEs) are defined as adverse events that occurred on and after the first dose date up to 30 days post last dose date. Patients with multiple TEAEs were counted once within a summary category; system organ class, preferred term, or relationship to therapy. Patients with events in more than one category were counted once within each category.

<sup>[4]</sup> Drug Related include relationship as Definite or Probable or Possible.

Cross-References: Listing 16.2.7.1, 16.2.7.4
PROGRAMMERS NOTES:



DIRECTORY/FILE.SAS

FINAL - ddmmmyychhomm. Page 1 of x

Table 14.3.1.5 Summary of Grade 3 or Greater, Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Dose Escalation Part A) Safety Evaluable (N=n)

| MedDRA System Organ Class<br>MedDRA Preferred Term [1][2] | NBF-006 Dose Level (ing/kg) for Escalation (Part A) | | | | NBF-006 Dose Expansion (mg/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|---|
| | 0.15 | 0.3 | orwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | mner | nnn | nnn | nnn | nnn | nnn | nnn |
| Number of Patients with Any Grade 3 or Greater TEAE [3][4] | nn(xx,x%) | nn(xx,x%) | nn(xx,x%) | nn(xx,x%) | rin(xx,x%) | nn(xx.x56) | nn(xx,x%) | nn(xx.x% |
| MedDRA System Organ Class | nn(xx,x96) | nn(xx.x%) | mm(xx.x96) | rin(xx,x%) | mn(xx,x96) | nn(xx,x56) | nn(xx.x46) | nn(xx.x96 |
| MedDRA Preferred Term | mm(xx,x96) | nn(xxxH) | mm(xx,x96) | rin(xx.x%) | rm(xx.x96) | ryrr(xx,x96) | пп(жжжіі) | nn(xx.x96 |
| MedDRA Preferred Term | mm(xx,x96) | nn(xxx%) | mm(xxxx96) | rm(xx.x96) | mm(xxxx94) | rint(xx,x96) | nn(xx,xH) | nn(xx.x96 |
| MedDRA Preferred Term | nn(xx,x%) | nn(xx,x46) | rin(xx.x96) | rim(xx,x%) | mn(xx,x%) | rm(xx.x46) | nn(xx,x%) | nn(xx.x% |
| MedDRA Preferred Term | nn(xx.x%) | nn(xxxH) | mm(xx_x96) | nn(xx.x96) | mn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x96 |
| MedDRA System Organ Class | nn(xx.x%) | mn(xx,x96) | mm(xxxx96) | nn(xx.x%) | /m(xxxx96) | rin(xx.x96) | nn(xxx%) | nn(xx.x96 |
| MedDRA Preferred Term | mm(xx.x%) | nn(xxxHi) | mm(xx.x96) | rm(xx.x96) | rrr(xx.x96) | rin(xx.x96) | пп(хх.х%) | nn(xx.x96 |
| MedDRA Preferred Term | nn(xx,x94) | nn(xx.x%) | rin(xxxx96) | rin(xx.x56) | nn(xx.x94) | rim(xx.x56) | nn(xx.x%) | nn(xx.x96 |
| MedDRA Preferred Term | mm(xx.x96) | mn(xx,x46) | rin(xx.x96) | nntkk.x96) | rin(xx, x96) | nnexx.x960 | nn(xx,x46) | nn(xx.x% |

<sup>[1]</sup> MedDRA version 21.1

Cross-References: Listing 16.2.7.1, 16.2.7.4
PROGRAMMERS NOTES:

Sort System Organic lass and then Preferred term in descending order using "Overall" frequency column. Excludes events with incomplete information for grade or drug relationship. Add footnote if required: See Listing 16.2.7.4 for excluded events. Medical writer will determine the appropriate percentage cut-off point e.g., 5% or 10 % in CSR.

Present Part A and Part B output separately, adjust title for Part B accordingly.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 64


<sup>[2]</sup> Number of Patients used as denominator to calculate percentages.

<sup>[3]</sup> Treatment-Emergent Adverse Events (TEAEs) are defined as adverse events that occurred on and after the first dose date up to 30 days post last dose date. Patients with multiple TEAEs were counted once within a summary category; system organiclass, preferred term, or maximum grade. Patients with events in more than one category were counted once within each category,

<sup>[4]</sup> Grade: 3=Severe, 4=Life threatening, 5=Fatal


DIRECTORY/FILE.SAS


### Table 14,3,1,6 Summary of Grade 3 or Greater, Drug-Related, TEAE by System Organ Class and Preferred Term (Dose Escalation Part A) Safety Evaluable (N=n)

| MedDRA System Organ Class | NBF-00 | 6 Dase Level (m | g/kg) for Escalat | ion (Part A) | NB | F-006 Dose Exp. | ansion (mg/kg) ( | Part B) |
|---|---|---|---|---|---|---|---|---|
| MedDRA Preferred Term [1][2] | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | onn | nnn | nnn | non | nnn. | non | nnn |
| Number of Patients with Any Drug-<br>Related Grade >=3 TEAE [3][4][5] | nn(xx.x96) | nn(xxx%) | nn(xxxx96) | ne(xx.x%) | nn(xx.x%) | nn(xx.x56) | nn(xxx4) | nn(xx,x96 |
| MedDRA System Organ Class<br>MedDRA Preferred Term | nn(xx,x%)<br>nn(xx,x%) | nn(xx.x%)<br>nn(xx.x%) | nn(xx.x%)<br>nn(xx.x%) | rm(xx.x96)<br>rm(xx.x96) | nn(xx,x%)<br>nn(xx,x%) | nn(xx.x%)<br>nn(xx.x%) | nn(xx.xH)<br>nn(xx.xH) | nn(xx.x96<br>nn(xx.x96 |
| MedDRA Preferred Term<br>MedDRA Preferred Term<br>MedDRA Preferred Term | nn(xx,x%)<br>nn(xx,x%)<br>nn(xx,x%) | nn(xx.x%)<br>nn(xx.x%) | nn(xx.x%)<br>nn(xx.x%)<br>nn(xx.x%) | nn(xx.x%)<br>nn(xx.x%)<br>nn(xx.x%) | mn(xx.x94)<br>mn(xx.x94)<br>mn(xx.x96) | nn(xx,x96)<br>nn(xx,x96)<br>nn(xx,x96) | nn(xx,x%)<br>nn(xx,x%) | nn(xx.x%<br>nn(xx.x%<br>nn(xx.x% |
| MedDRA System Organ Class<br>MedDRA Preferred Term<br>MedDRA Preferred Term<br>MedDRA Preferred Term | nn(xx.x96)<br>nn(xx.x96)<br>nn(xx.x96)<br>nn(xx.x96) | nn(xx.x%)<br>nn(xx.x%)<br>nn(xx.x%) | nn(xxx96)<br>nn(xxx96)<br>nn(xxx96)<br>nn(xxx96) | nn(xx.x%)<br>nn(xx.x%)<br>nn(xx.x%)<br>nn(xx.x%) | nn(xx.x%)<br>nn(xx.x%)<br>nn(xx.x%) | nn(xx.x96)<br>nn(xx.x96)<br>nn(xx.x96)<br>nn(xx.x96) | nn(xxx%)<br>nn(xxx%)<br>nn(xxx%) | nn(xx.x96<br>nn(xx.x96<br>nn(xx.x96 |

#### PROGRAMMER'S NOTES:

Sort System Organic lass and then Preferred term in descending order using "Overall" frequency column. Excludes events with incomplete information for grade or drug relationship. Add footnote if required: See Listing 16.2.7.4 for excluded events. Medical writer will determine the appropriate percentage cut-off point e.g., 5% or 10 % in CSR.

Present Part A and Part B output separately, adjust title for Part B accordingly.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 65


<sup>[2]</sup> Number of Patients used as denominator to calculate percentages.

<sup>[3]</sup> Treatment-Emergent Adverse Events (TEAEs) are defined as adverse events that occurred on and after the first dose date up to 30 days post last dose date. Patients with multiple TEAEs were counted once within a summary category; system organ class, preferred term, maximum grade, or relationship to therapy. Patients with events in more than one category were counted once within each category.

<sup>[4]</sup> Grade: 3=Severe, 4=Life threatening, 5=Fatal.

<sup>[5]</sup> Drug Related include relationship as Definite or Probable or Possible,

Cross-References: Listing 16.2.7.1, 16.2.7.4



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b


### Table 14.3.1.7 Summary of TEAE by Maximum Severity Grade, System Organ Class and Preferred Term (Dose Escalation Part A) Safety Evaluable (N=n)

| MedDRA System Organ Class<br>MedDRA Preferred Term | NBF-00 | 6 Dose Level (m) | g/kg) for Escalat | ion (Part A) | NBF-006 Dose Expansion (rng/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|---|
| Maximum Severity Grade [1][2] | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | mnn | min | nnn | nnn | nnn | nnn | nnn |
| Patients with Any TEAE [3] | m(xx.x96) | mn(xx.x%) | nn(xx.x96) | nn(xx,x96) | nn(xx.x96) | nn(xx.x%) | nn(xx.x56) | пп(жжжі6) |
| MedDRA System Organ Class | mn(xxxx96) | nn(xxxx9li) | mn(xx.x96) | nn(xxxx96) | rm(xx.x96) | nn(xx.x96) | nn(xxxx56) | nn(xx.x% |
| MedDRA Preferred Term | mm(xx.x96) | rm(xx.x96) | mm(xx,x95) | rin(xx,x96) | mn(xx.x94) | mn(xx.x%) | nn(xx.x%) | пп(хосж% |
| < Grade 3 | mn(xx.x94) | mn(xx,x96) | mm(xx,x96) | mm(xxxx96) | rm(xx.x94) | mn(xxxx96) | nn(xx.x/6) | rintocx16 |
| Grade 1 | mn(xx,x96) | mn(xxxx9li) | nn(xx,x95) | nn(xxx96) | nn(xx.x96) | nn(xxxx46) | nn(xx.x96) | nn(xx.x% |
| Grade 2 | nn(xx,x96) | nn(xx_x%) | rin(xx,x96) | nn(xx,x96) | nn(xx,x96) | nn(xx.x%) | nn(xx,x96) | nnoxxii |
| Grade 3 | mn(xx.x96) | mn(xxxx96) | rrrr(xxx.x95) | mm(xxxx96) | rm(xx.x96) | mn(xx.x%) | nn(xx.x66) | nntocx46 |
| Grade 4 | mm(xx, x96) | nn(xxx94) | mm(xxx.x96) | rin(xxxx96) | mn(xx.x96) | nn(xxxx46) | rin(xx,x96) | nn(xx.x% |
| Grade 5 | mn(xx,x96) | nn(xx.x%) | mn(xx.x95) | mm(xx,x96) | nn(xx,x96) | mn(xx.x96) | nn(xx.x96) | nntxxxX |
| >= Grade 3 | mn(xx,x96) | mn(xxxx96) | rtrs(xx,x95) | mm(xxxx96) | rm(xx.x96) | nn(xxxH) | nn(xx,x96) | nnfxx.x% |

<sup>[1]</sup> MedDRA version 21,1

Cross-References: Listing 16.2.7,1, 16.2.7,4
PROGRAMMERS NOTES:

Sort System Organ Class and then Preferred term in descending order using "Overall" frequency column.

Excludes events with incomplete information for grade or drug relationship, Add footmate if required: See Listing 16.2.7.4 for excluded events.

Present Part A and Part B output separately, adjust title for Part B accordingly.

NBF-006-001 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 66


<sup>[2]</sup> Number of Patients used as denominator to calculate percentages.

<sup>[3]</sup> Treatment-Emergent Adverse Event (TEAEs) are defined as adverse events that occurred on and after the first dose date up to 30 days post last dose date. Patients with multiple TEAEs were only counted once within a summary category; system organiclass, preferred term or maximum grade. Patients with events in more than one category were counted once within each category.



DIRECTORY/FILE.SAS


NBF-006-001 Phase 1/1b Table 14.3.1.8

# Summary of Drug-Related, TEAE by Maximum Severity Crade, System Organ Class and Preferred Term (Dose Escalation Part A) Safety Evaluable (N=n)

| MedDRA System Organ Class<br>MedDRA Preferred Term | NBF-006 | Dose Level (m) | g/kg) for Escalat | ion (Part A) | NBF-006 Dose Expansion (mg/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|---|
| Maximum Severity Grade [1][2] | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | nnn | inin | מתיו | nnn | nnn | nnn | nnn |
| Patients with Any Drug-Related TEAE[3][4] | nn(xxxx96) | nn(xx.x%) | nn(xx.x46) | nn(xx.x46) | nn(xx.x%) | nn(xx,x%) | mm(xx.x56) | пп(хосх% |
| MedDRA System Organ Class | mm(xxx.x96) | nn(xxxx96) | mm(xxxx16) | nn(xx.x46) | mm(xxxx96) | nn(xx,x%) | mn(xx.x%) | nn(xxxX |
| MedDRA Preferred Term | rm(xxxx96) | mm(xxx,x96) | mm(xxxxxHb) | mn(xxx46) | mm(xx,x96) | nn(xx.x%) | nn(xx,x%) | nn(xxxXi |
| < Grade 3 | nn(xx.x%) | nn(xxxx94) | mm(xxxxx46) | nrt(xxxx46) | mn(xx_x%) | nn(xx.x%) | mm(xx.x%) | nn(xxxx¥ |
| Grade 1 | nn(xx.x96) | nn(xxxx96) | mm(boxxx96) | nn(xxx%) | mm(xx_x96) | nn(xxxx96) | mn(xx.x90) | nn(xx.x% |
| Grade 2 | nn(xx.x%) | mm(xx,x%) | mn(xx.x;16) | nnpocx46) | nn(xx,x96) | nn(xx,x%) | nn(xx,x%) | nntxxx4 |
| Grade 3 | rin(xxx.x96) | nn(xxxx96) | mn(xxxxx16) | mm(xxx,x46) | rm(xx.x%) | nn(xxx96) | mm(xx.x%) | nn(xx.xH |
| Grade 4 | nn(xxx.x96) | nn(xxxx96) | mn(xx.x36) | nn(xx.x%) | nn(xx_x%) | nn(xxxx96) | mn(xx.x96) | nn(xx.x% |
| Grade 5 | nn(xx_x%) | rintxx.x96) | nn(xx.xx10) | nn(xxxx16) | (dex.xx)(nn | nn(xx,x%) | mn(xx,x%) | nnboux# |
| >= Grade 3 | rim(xxx.x96) | mm(xxxx96) | nm(xxxxx46) | nn(xxxx46) | mn(xx_x%) | nn(xx.x96) | mn(xx.x96) | nn(xx.xX |

<sup>[1]</sup> MedDRA version 21,1

# PROGRAMMER'S NOTES:

Surf System Organ Class and then Preferred term in descending order using "Overall" frequency column.

Excludes events with incomplete information for grade or drug relationship. Add footnote if required: See Listing 16.2.7.4 for excluded events. Present Part A and Part 8 output separately, adjust title for Part 8 accordingly.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 67


<sup>[2]</sup> Number of Patients used as denominator to calculate percentages.

<sup>[3]</sup> Treatment-Emergent Adverse Event (TEAEs) are defined as adverse events that occurred on and after the first dose date up to 30 days post last dose date. Patients with multiple TEAEs were only counted once within a summary category: system organ class, preferred term, maximum grade or relationship to therapy. Patients with events in more than one category were counted once within each category.

<sup>[4]</sup> Drug Related include relationship as Definite or Probable or Possible. Cross-References: Listing 16.2.7.1, 16.2.7.4



DIRECTORY/FILE.SAS


Table 14.3.1.9

# Summary of Serious Adverse Events by System Organ Class and Preferred Term (Dose Escalation Part A) Safety Evaluable (N=n)

| MedDRA System Organ Class | NBF-00 | 6 Dose Level (in | g/kg) for Escalat | ion (Part A) | NB | F-006 Dose Expi | ansion (mg/kg) ( | Part B) |
|---|---|---|---|---|---|---|---|---|
| MedDRA Preferred Term [1][2] | 0.15 | 0.3 | orwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | mner | nnn | nnn | rinn | mm | nnn | nnn |
| Number of Patients with Any Serious<br>Adverse Event | nn(xx,x%) | nn(xx,x%) | nn(xx,x%) | nn(xx,x%) | rin(xx,x%) | nn(xx.x56) | nn(xx,x%) | nn(xx.x% |
| MedDRA System Organ Class | nn(xx,x96) | nn(xx,x%) | nn(xx.x%) | nn(xx,x%) | nn(xx,x96) | nn(xx.x56) | nn(xx.x%) | nn(xx.x96 |
| MedDRA Preferred Term | nn(xx,x96) | nn(xxxH) | mm(xx_x96) | rin(xx,x96) | rm(xx,x96) | rint(xx.x96) | пп(хжжіі) | nn(xx,x% |
| MedDRA Preferred Term | rm(xx,x96) | mn(xxx%) | mm(xx_x96) | rm(xx.x96) | mn(xxxx94) | rint(xx,x56) | (iffx.xx)nn | nn(xx.x96 |
| MedDRA Preferred Term | nn(xx,x%) | nn(xx,x16) | rin(xx.x96) | nn(xx,x%) | mn(xx,x%) | rm(xx.x46) | nn(xx,x%) | nn(xx.x% |
| MedDRA Preferred Term | nn(xx.x%) | nn(xxxH) | mm(xx_x96) | nn(xx.x96) | mn(xx.x96) | nn(xx.x%) | nn(xxxXII) | nn¢xx.x% |
| MedDRA System Organ Class | nn(xx.x%) | mn(xx,x96) | mm(xxxx96) | nn(xx.x%) | 717(xxx,x96) | rin(xx.x96) | nn(xxx%) | nn(xx.x96 |
| MedDRA Preferred Term | mm(xx,x%) | nn(xx.x%) | mm(xx.x96) | rm(xxxx96) | 7177(xx,x96) | rin(xx.x96) | пп(хх.х%) | nn(xx.x96 |
| MedDRA Preferred Term | mm(xx,x94) | nn(xx.x%) | mm(xxxxx96) | rin(xx.x56) | mn(xx.x94) | rim(xx.x56) | nn(xx.x%) | nn(xx.x96 |
| MedDRA Preferred Term | mm(xx, x96) | nn(xxx36) | rin(xx,x96) | ne(xx.x%) | rrn(xx,x96) | nin(xx.x96) | nn(xx,x46) | nn(xx.x9) |

<sup>[1]</sup> MedDRA version 21.1

Cross-References: Listing 16.2.7.1, 16.2.7.4

## PROGRAMMER'S NOTES:

Use Serious Code > 1. Serious: 1=Not serious, 2=Results in Death, 3=Life threatening, 4=Requires or Prolongs Hospitalization, 5=Persist or Significant Disability/Incapacity, 6=Congenital Anomaly or Birth Defect, 7=Other Medically Important Serious Event.

Sort System Organ Class and then Preferred term in descending order based on "Overall" column frequency.

Present Part A and Part B output separately, adjust title for Part B accordingly.

NBF-006-001 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 68


<sup>[2]</sup> Number of Patients used as denominator to calculate percentages.



#### DIRECTORY/FILE.SAS


### Table 14.3.1.10 Summary of Death On-Study or within 30 Days Post Last Dose (Dose Escalation Part A) Safety Evaluable (N=n)

| | NBF-006 Das | se Level (mg/kg) | for Escalation ( | Part A) | NBF-006 Dos | se Expansion (it | g/kg) (Part E) | |
|---|---|---|---|---|---|---|---|---|
| Primary Cause of Death(1) | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | novi | nnn | nnn | nnn | nnn. | non | nnn | nnn |
| All Death | | | | | | | | |
| Primary Cause | mn(xxx,x46). | rin(xx.x96) | nn(xx,xH) | mm(xxxx46) | mm(xxx.x96) | пп(юсжні) | nn(xx.xH) | nnčkx.x%) |
| Primary Cause | mm(xx.x%) | nn(xx.x96) | nn(xx.x94) | nn(xxx%) | mm(xxxx94) | mm(xxxx46) | mm(xx.x%) | rm(xx,x%) |
| Primary Cause | nn(xx.x%) | nn(xx.x94) | nn(xxx46) | nn(xx.x9b) | nn(xxx94) | nn(xxx46) | mn(xx.x%) | ппфкк.ж90) |
| Death within 30 days of Last Dose | | | | | | | | |
| Primary Cause | nn(xx.x%) | nn(xx,x94) | mn(xx_x?4) | nn(xx.x9b) | mm(xxxx94) | nn(xxxx46) | nn(xx.x%) | rinoxx.x96) |
| Primary Cause | nn(xx.x16) | nn(xx.x96) | nn(xx,x96) | nn(xxx%) | nn(xxxx96) | nn(xxxx16) | nn(xx,x%) | nn(xx.x%) |
| Primary Cause | mm(xxxx46) | mm(xx.x96) | nn(xxxxHs) | nn(xxxx%) | mm(xxx.x94) | mm(xxxx46) | nn(xx.x%) | rintkx.x96) |

<sup>[1]</sup> Number of Patients used as denominator to calculate percentages. Cross-References: Listing 16.2.7.4

PROGRAMMER'S NOTES:

Present Part A and Part B output separately, adjust title for Part B accordingly.



| 14.3.2 Listings of Death, O | Other Serious and | Significant Adve | rse Events |
|---|---|---|---|
|---|---|---|---|



#### DIRECTORY/FILE.SAS FINAL - ddmmmyychhimm Page 1 of x

# Table 14.3.2.1 Patient Listing of Treatment-Errergent Adverse Events Leading to Death Safety Evaluable (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006<br>Dose (mg/kg) | MedDRA<br>Preferred Term | Day [1] | Grade<br>[2] | Duration<br>(day) [3] | Drug<br>Related[4] | Outcome<br>[5] |
|---|---|---|---|---|---|---|---|---|
| ecc-pppp/xx/x | × | 33. | XXX | × | xx | .KX | Possible. | × |
| | | | XXX | × | XX | XX | Possible | × |
| | | | XXX | × | xx | XX | Related | × |
| ccc-pppp/xx/x | × | XX | XXX | × | жx | XX<br>XX | Possible | × |
| | | | NXX | × | ×× | XX | Possible | × |
| | | | XXX | × | ×× | XX. | Possible | × |
| ccc-ppppp/xx/x | × | XX | XXX | × | xx | XX<br>XX<br>XX | Related | × |
| | | | XXX | × | xx | 303 | Possible | × |

## MedDRA version 21.1

- [1] Day is relative to the first dose date.

- [1] Grade: 1=Mild, 2=Moderate, 3=Severe, 4=Life threatening, 5=Fatal.
  [3] Duration of adverse event is calculated in days from Onset Date to Resolution Date.
  [4] Drug Related include relationship as Definite or Probable or Possible.
  [5] Outcome: 1=Recovered/Resolved, 2=Recovered/Resolved with sequelae, 3=Recovering/Resolving, 4=Not Recovered /Not Resolved, 5=Fatal, 6=Unknown

Cross-References: Listing 16.2.7.1, 16.2.7.4
PROGRAMMER'S NOTES:

Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 71




DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b

# Table 14,3,2,2 Patient Listing of Serious Adverse Events Safety Evaluable (N=n)

FINAL - ddmmmyythhtmm


| Patient<br>/Age/Sex | Study<br>Part | NBF-006<br>Dose (mg/kg) | MedDRA<br>Preferred Term | (1) | Grade<br>[2] | Duration<br>(day) [3] | Orug<br>Related[4] | Outcome<br>[5] |
|---|---|---|---|---|---|---|---|---|
| ccc-pppp/xx/x | × | xx | XXX | × | xx | XX | Possible | × |
| STATE OF THE STATE | | | XXX | × | xx | XX | Possible | × |
| | | | XXX<br>XXX | × | XX | XX | Related | × |
| ccc-pppp/xx/x | * | 100 | XXX | × | xx | XX | Possible | × |
| | | | 300X | × | жx | 300 | Possible | × |
| | | | XXX | × | XX | XX | Possible | × |
| ccc-pppp/xx/x | × | sx: | XXX | × | ×× | XX. | Related | × |
| | | | XXX | × | xx | .KK | Possible | × |

# MedDRA version 21.1

- [1] Day is relative to the first dose date.
- [2] Grade: 1=Mild. 2=Moderate, 3=Severe, 4=Life threatening, 5=Fatal.
- [3] Duration of adverse event is calculated in days from Onset Date to Resolution Date.
  [4] Drug Related include relationship as Definite or Probable or Possible.
- [5] Outcome: 1=Recovered/Resolved, 2=Recovered/Resolved with sequelae, 3=Recovering/Resolving, 4=Not Recovered /Not Resolved, 5=Fatal, 6=Unknown

Cross-References: Listing 16.2.7.1, 16.2.7.3, 16.2.7.4
PROGRAMMER'S NOTES:

Sort "Patient" in ascending order using "pppp", and then "cor" portion of patient number.



# Table 14.3.2.3 Patient Listing of Treatment-Emergent Adverse Events Leading to Drug Withdrawn Safety Evaluable (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006<br>Dose (mg/kg) | MedDRA<br>Preferred Term | Day<br>[1] | Grade<br>[2] | Duration<br>(Days) [3] | Drug<br>Related[4] | Outcome<br>[5] |
|---|---|---|---|---|---|---|---|---|
| ccc-pppp | × | xx | MedORA PT | × | ж | × | Possible | x |
| | | xx | MedDRA PT | * | ************************************** | XX | Related | × |
| ccc-pppp | × | άx | MedDRA PT | × | xx | × | Unrelated | × |
| | | XX | MedORA PT | × | - XX | XX<br>XX | Possible | X |
| | | xx<br>xx | MedDRA PT | * | XX<br>XX | XX | Related | × |
| ссс-рррр<br>/юс/х | x | xx | MedORA PT | × | xx | xx | Possible | x |
| 1000 | | xx | MedORA PT | × | XX | 206 | Related | × |

#### MedDRA version 21.1

- [1] Day is relative to the first dose date.
- [2] Grade: 1=Mild, 2=Moderate, 3=Severe, 4=Life threatening, 5=Fatal.

- [3] Duration of adverse event is calculated in days from Onset Date to Resolution Date.
  [4] Drug Related include relationship as Definite or Probable or Possible.
  [5] Outcome: 1=Recovered/Resolved, 2=Recovered/Resolved with sequelae, 3=Recovering/Resolving, 4=Not Recovered /Not Resolved, 5=Fatal, 6=Unknown, Cross-References: Listing 16.2.7.1, 16.2.7.2.3, 16.2.7.4

  PROGRAMMERS NOTES:

Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number,



# Table 14,3.2,4 Patient Listing of Dose Limiting Toxicities DLT Evaluable (N=n)

| Patient/<br>Age/Sex | Study<br>Part | NBF-006<br>Dose (mg/kg) | MedDRA<br>Preferred Term | Day<br>[1] | Grade<br>[2] | Duration<br>(Days) [3] | Drug<br>Related[4] | Outcome<br>[5] |
|---|---|---|---|---|---|---|---|---|
| ccc-pppp/<br>xx/x | x | xx | MedDRA PT | × | xx | ×× | Possible | × |
| | | | MedDRA PT | × | XX | XX | Related | × |
| ссс-рррр/<br>хм/х | × | xx | MedDRA PT | × | XX | xx | Unrelated | к |
| | | | MedDRA PT | × | XX | xx | Possible | × |
| | | | MedDRA PT | × | xx<br>xx | 300 | Related | × |
| ccc-pppp/<br>xx/x | × | xx | MedDRA PT | × | xx | xx | Possible: | × |

## MedDRA version 21.1

- DLT- Dose Limiting Taxicity
- [1] Day is relative to the first dose date.

- [1] Grade: 1=Mild, 2=Moderate, 3=Severe, 4=Life threatening, 5=Fatal.
  [2] Grade: 1=Mild, 2=Moderate, 3=Severe, 4=Life threatening, 5=Fatal.
  [3] Duration of Adverse Event calculated in days from the Onset Date to the Resolution Date.
  [4] Drug Related include relationship as Definite or Probable or Possible.
  [5] Outcome: 1=Fatal, 2= Not Recovered/Not Resolved, 3= Recovered/Resolved, 4= Recovered/Resolved with sequelae, 5=Recovering/Resolving, 6=Unknown Cross-References; Listing 16.2.7.1, 16.2.7.4

  PROGRAMMIER'S NOTES:

Sort "Patient" in ascending order using "pppp", and then "coc" portion of patient number.



# 14.3.3 Adverse Events of Special Interest

Statistical Analysis Plan



# Table 14.3.3.1 Summary of Dose Limiting Toxicities by System Organ Class and Preferred Term During Cycle One DLT Evaluable (N=n)

| | NBF-006 D | ose Level (mg/kg) for | Escalation (Part A) | | |
|---|---|---|---|---|---|
| 0.15 | 0.3 | 0.6 | 1,2 | 1.6 | Overall |
| nnn | nnn. | nnn | ann | | nnn |
| mn(xxxxXb) | mn(xxxx16) | nn(xx.x46) | mn(xxxx96) | nn(xx,x46) | nn(xx.x36) |
| mn(xxx,x16) | nn(xxxx)hn | mm(xxxx46) | rin(xxxxHs) | nn(xx,x16) | nn(xx,x%) |
| mn(xxxx46) | nn(xxxx96) | nn(xxx46) | mn(xxxx46) | mm(xx.x96) | nn(xx.x16) |
| mm(xxxx46) | mm(xxxxx94) | mm(xxx.x46) | mm(xxxxxHe) | rsr(xx.x46) | nn(xx.x%) |
| nn(xx.x%) | mm(xxxx96) | mm(xxxx36) | nn(xxxx%) | nn(xx.x46) | nn(xxx%) |
| nn(xxxx16) | mm(xxxxx46) | mm(xxx.x46) | mn(xxxxx46) | mr(xx.x%) | nn(xx.x16) |
| nn(xx.x46) | rin(societi) | mm(xxxx96) | nn(xx.xHi) | nn(xx.x16) | nn(xx.x%) |
| nn(xx,x%) | nn(xxx%) | nn(xxxx16) | mm(xxxxx16) | nn(xxxx16) | nn(xx.x%) |
| mm(xxxx46) | rint(xxxx94) | mm(xxx.x46) | mn(xxxxx4e) | rvn(xxx.x46) | mm(xx.x46) |
| nn(xx.x%) | mm(xxxxx9b) | nn(xxxx96) | nn(xxxxiii) | nm(xxxx96) | nn(xx.x46) |
| | nn(xx,x%) | 0.15 0.3 nnn nnn nn(xxx%) | 0.15 0.3 0.6 nnn nnn nnn nn(xx,****) nn(xx,***) nn(xx,****) nn(xx,***) nn(xx,****) nn(xx,***) nn(xx,****) nn(xx,****) nn(xx,***) nn(xx,****) nn(xx,****) nn(xx,****) nn(xx,****) nn(xx,****) | nnn nnn nnn nnn nn(pocxHb) nn(pocxHb) nn(pocxHb) nn(pocxHb) nn(pocxHb) nn(pocxHb) nn(pocxHb) nn(pocxHb) | 0.15 0.3 0.6 1.2 1.6 nnn nnn nnn nnn nnn nnfocxib nnfocxib nnfocxib nnfocxib nnfocxib nnfocxib nnfocxib nnfocxib nnfocxib nnfocxib |

DLT= Dose Limiting Toxicity
[1] MedDRA version 21.1

Sort System Organ Class and then Preferred term in descending order using "Overall" frequency column. Excludes events with incomplete information for grade or drug relationship. Add footnote if required: See Listing 16,2.7.4 for excluded events.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 76


<sup>[2]</sup> Number of Patients used as denominator to calculate percentages.

<sup>[3]</sup> Only those DLTs occurring during Cycle 1 will be used to make decisions regarding dose escalation and tolerability. Cross-References: Table 14.3.2.4, Listing 16.2.7.1, 16.2.7.4 FROGRAMMERS NOTES;



#### DIRECTORY/FILE.SAS


NBF-006-001 Phase 1/1b Table 14,3.3.2

## Summary of Infusion-Related Reaction by Maximum Severity Gradie, System Organ Class and Preferred Term (Dose Escalation Part A) Safety Evaluable (N=n)

| MedDRA System Organ Class<br>MedDRA Preferred Term | NBF-00 | Dose Level (m) | g/kg) for Escalat | ion (Part A) | NBF-006 Dose Expansion (rng/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|---|
| Maximum Severity Grade [1](2) | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | nnn | nnn | non | nnn | nnn | nnn | nnn |
| Patients with Any TEAE [3] | mm(xx,x96) | nn(xx,x%) | nn(xx.x96) | nr(xx.x96) | nn(xx.x%) | nn(xxxx96) | nn(xx.x96) | mm(xxx,x96) |
| MedDRA System Organ Class | mn(xx.x96) | nn(xxx96) | nn(xx.x94) | nn(xx.x%) | nn(xx.x%) | пп(хосжіі) | nn(xx.x%) | nnpocx96 |
| MedDRA Preferred Term | rim(xx,x96) | rim(xxi.x%) | rin(xx,x95) | rin(xx.x96) | nn(xx,x%) | mn(xxxxx/46) | nn(xx.x46) | nn(xxxx96) |
| < Grade 3 | mn(xx.x94) | mm(xxx.x96) | mn(xx,x95) | mm(xx.x96) | mn(xx.x%) | mn(xxxxxYi) | nn(xxx96) | rintxx.x% |
| Grade 1 | nn(xx.x96) | .mm(xxLx96) | nn(xx.x95) | nn(xx.x96) | mn(xx.x96) | nn(xxxx46) | rin(xxxx96) | mm(xxx.x96) |
| Grade 2 | nn(xx,x94) | nn(xx_x%) | nn(xxxx96) | nn(xx.x96) | nn(xx,x%) | mn(xxxx96) | nn(xx,x36) | nn(xx,x%) |
| Grade 3 | mn(xx.x96) | mm(xxxx96) | rm(xx.x95) | mm(xx.x96) | nn(xx,x46) | nn(xxxx46) | nn(xxx96) | rin(xxxx94) |
| Grade 4 | mm(xx,x96) | nn(xxxx96) | nn(xx.x96). | nn(xx.x96) | mn(xx.x46) | nn(xxxx46) | rin(xxxx96) | nn(xx.x96) |
| Grade 5 | nn(xx,x96) | nn(xx_x96) | nn(xx.x96) | rin(xx,x96) | nn(xx,x%). | mn(xxxx96) | nn(xx,x36) | nn(xx,x96) |
| >= Grade 3 | mm(xx,x96) | rm(xxxx96) | rm(xx.x94) | mm(xx, x96) | nn(xx.x%) | nn(xx.x96) | mm(xx,x96) | rim(xxx.x94) |

<sup>[1]</sup> MedDRA version 21,1

## PROGRAMMER'S NOTES:

Sort System Organ Class and then Preferred term in descending order using "Overall" frequency column.

Excludes events with incomplete information for grade or drug relationship, Add footnote if required: See Listing 16.2.7.4 for excluded events.

Present Part A and Part B output separately, adjust title for Part B accordingly.

NBF-006-001 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan


<sup>[2]</sup> Number of Patients used as denominator to calculate percentages.

<sup>[3]</sup> Infusion-related reaction (IAR) signs and symptoms include back pain, fever and/or shaking chills, flushing and/or itching, alterations in heart rate and blood pressure, dyspriea or chest discomfort, skin rashes, or anaphylaxis (e.g., generalized urticaria, angioederna, wheezing, hypotension, tachycardia, etc.). Cross-References: Listing 16.2,7.1, 16.2.7.4



# 14.3.4 Abnormal Laboratory Value Listing

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan Final Version 2.0, March 14, 2023

78



#### Table 14,3,4 Patient Listing of Grade 3 and 4 Abnormal Laboratory Values During Treatment Safety Evaluable (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006<br>Dose (mg/kg) | Abnormal Laboratory<br>Test (unit) | Baseline<br>Grade [1] | Grade<br>Grade [1] | Day<br>[Z] | Lab<br>Result | Reference<br>Range Indicator |
|---|---|---|---|---|---|---|---|---|
| tec-pppp | × | ж | Test Name (xxx) | × | x | xx | × | High |
| | | xx · | Test Name (xxx) | × | × | 300 | ×× | Law |
| ecc-pppp<br>/xx/x | x | xx . | Test Name (xxx) | × | × | ×х | x | Low |
| | | XX | Test Name (xxx) | × | × | XX | XX | High |
| | | KX<br>KX | Test Name (xxx) | × | × | ×х | xx | High |
| ссс-рррр<br>/ю/х | X. | xx | Test Name (xxx) | × | × | жx | XX | Low |
| | | XX | Test Name (xxx) | 34. | × | XX | xx | Low |

<sup>[1]</sup> Grade: 3= Severe, 4= Life threatening, 5= Fatal.

[2] Day is relative to the first dose date.

Cross-References: Listing 162.8.1-16.2.8.3

PROGRAMMER'S NOTES:

Sort "Patient" in ascending order using "pppp", and then "ccc" and "ii" portions of patient number.

During Treatment is the period from first dose up to 30 days post last dose study drug.



14.3.5 Other Safety Data Summary Tables

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan

80




DIRECTORY/FILE.SAS

FINAL – ddmmmyy:hh:mm Page 1 of x

Table 14.3.5.1.1

Summary of NBF-006 Administration and Compliance for Cycle One (Dose Escalation Part A)

Safety Evaluable (N=n)

| | NRF-0 | 006 Dose Level (m | ng/kg) for Escalati | ion (Part A) |
|---|---|---|---|---|
| NBF-006 Administration | 0.15 | 0.3 | onwards | Overall |
| Number of Patients | nnn | nnn | nnn | nnn |
| Duration of Exposure [1] | | | | |
| N | nnn | nnn | nnn | nnn |
| Mean | XX.X | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx |
| Median | xx.x | xx.x | XX.X | xx.x |
| Minimum | XX | xx | xx | XX |
| Maximum | xx | xx | xx | xx |
| Total Actual Dose (mg) [2] | | | | |
| N | nnn | nnn | nnn | nnn |
| Mean | XX.X | xx.x | XX.X | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx |
| Median | XX.X | XX.X | XX.X | XX.X |
| Minimum | xx | xx | xx | xx |
| Maximum | xx | xx | xx | xx |
| Total Target Dose (mg/kg) [3] | | | | |
| N | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | XX.X | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx |
| Median | xx.x | xx.x | xx.x | xx.x |
| Minimum | xx | xx | xx | xx |
| Maximum | xx | xx | xx | xx |
| Compliance (%) [4][5] | | | | |
| >100% | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| 100% | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |
| <100% | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) | nn(xx.x%) |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved Statistical Analysis Plan 81 Final Version 2.0, March 14, 2023



Cycle one length = 6 weeks (42 days)

- Cycle one length = 6 weeks (42 days)

  [1] Duration of Exposure is the duration between the first dose and last dose of NBF-006 during the study.

  [2] Total Actual Dose is the sum of all NBF-006 administered over the entire course of the study.

  [3] Total Target Dose is the sum of intended NBF-006 doses during the duration of exposure, based on no modifications to dose or schedule.

  [4] Percent Compliance is the total actual NBF-006 dose divided by total target NBF-006 dose multiplied by 100% for each patient.

  [5] Number of patients used as denominator to calculate percentages.

  Cross-References: Listing 16.2.5.1

  PROGRAMMERS NOTES:

  Compliance categories may need to be modified based on the data.

Compliance categories may need to be modified based on the data.



DIRECTORY/FILE.SAS

FINAL – ddmmmyy:hh:mm Page 1 of x

Table 14.3.5.1.2

Summary of NBF-006 Administration and Compliance for All Treatment Cycles (Dose Escalation Part A)

Safety Evaluable (N=n)

| | N | NBF-006 Dose Leve | l (mg/kg) for Escalati | on (Part A) | NBF-00€ | Dose Expan | sion (mg/kg) | (Part B) |
|---|---|---|---|---|---|---|---|---|
| NBF-006 Administration | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Number of Cycles [1] | | | | | | | | |
| N | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean | XX.X | XX.X | XX.X | xx.x | XX.X | xx.x | xx.x | xx.x |
| Standard Deviation | X.XX | X.XX | x.xx | X.XX | x.xx | x.xx | x.xx | x.xx |
| Median | xx.x | XX.X | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x |
| Minimum | XX | XX | XX | XX | xx | xx | xx | xx |
| Maximum | xx | xx | xx | xx | XX | xx | xx | XX |
| Duration of Exposure [2] | | | | | | | | |
| N | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | X.XX | x.xx | X.XX | x.xx | X.XX | x.xx | X.XX |
| Median | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x |
| Minimum | xx | xx | xx | xx | xx | xx | xx | xx |
| Maximum | xx | xx | xx | xx | XX | xx | xx | XX |
| Total Actual Dose (mg) [3] | | | | | | | | |
| N | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | X.XX | x.xx | x.xx | x.xx | x.xx |
| Median | XX.X | XX.X | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x |
| Minimum | xx | xx | xx | xx | xx | xx | xx | xx |
| Maximum | xx | xx | xx | xx | xx | xx | xx | xx |
| Total Target Dose (mg) [4] | | | | | | | | |
| N | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan




| Median | XX.X | XXXX | XX_X | xx.x | XXX | XX.X | NK.X | XX.X |
|---|---|---|---|---|---|---|---|---|
| Minimum | XX | XX | XX | XX: | XX. | XX | XX | XX |
| Maximum | 300 | xx | ×× | NX. | xx | XX | XX | 300 |
| Compliance (%) [5] | | | | | | | | |
| >100% | mn(xxLx16) | rintpocx46) | nm(xx.x96) | mn(xx,x96) | nn(xxxx%) | rin(xx,x%) | nn(xx,x56) | mn(xxxxH) |
| 100% | mm(xxxx46) | mrt(xxx.x%) | ппфок.х.96) | mn(xx,x/6) | nn(xx.x%) | nn(xx.x%) | nm(xx,x56) | mm(xxx,x96) |
| <100% | mm(xxxx468 | mmbox.x460 | nni(xx,x96) | mm(xx,x96) | nntxxxx(N) | nn(xx,x96) | nnéxx.x56) | mn(xxxx96) |

Compliance categories may need to be modified based on the data.

Present Part A and Part B output separately, adjust title for Part B accordingly.

<sup>[1]</sup> Incomplete treatment cycles are included in counts.
[2] Duration of Exposure is the duration between the first dose and last dose of NBF-006 during the study.
[3] Total Dose is the sum of all NBF-006 administered over the entire course of the study.
[4] Total intended Dose is the sum of intended NBF-006 doses during the duration of exposure, based on no modifications to dose or schedule.
[5] Percent Compliance is the total NBF-006 doses divided by Total Intended NBF-006 dose multiplied by 100% for each patient.

Cross-References: Listing 16.2.5.1

PROGRAMMERS NOTES:



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b

FINAL - ddmmmyy;hh;mm Page 1 of x

### Table 14.3.5.1.3 Summary of NBF-006 Dose Delayed/Interrupted/Withdrawn (Dose Escalation Part A) Safety Evaluable (N=n)

| | NBF-006 | Dose Level (mg | g/log) for Escala | tion (Part A) | NBF-006 Do | se Expansion ( | mg/kg) (Part B) | Same |
|---|---|---|---|---|---|---|---|---|
| NBF-006 Administration | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | nna | nnn | nnn | nnn | nnn | onn | nan |
| Patients with Dose Delayed [1] | nn(xxx96) | nn(xxxx96) | nn(xxxx4h) | nn(xx.x96) | nn(xx.x46) | nn(xx.x46) | nn(xx.x96) | mn(xx.x%) |
| Yes | nn(xx,x%) | nn(xx.x96) | mm(back96) | nn(xx.x96) | nn(xx,x%) | nn(xxxx16) | nn(xx.x96) | nn(xx.x%) |
| Adverse Event | rim(xxxx96) | rnn(xx.x56) | mn(xxxxx4) | nn(xx.x94) | nn(xx.x%) | mm(xxxx26) | mn(xx.x95) | nn(xx,x%) |
| Non-compliance | mm(xxxx96)- | rin(xx.x56) | rm(xxxxx4b) | nn(xx.x9b) | nn(xx.x36) | mm(xx.x46). | nn(xx.x96) | mn(xx,x%) |
| Other | nn(xx,x96) | nn(xx,x56) | rin(xxxx96) | nn(xx.x%) | nn(xx,x%) | en(xxxx46) | mm(xx.x96) | inn(xx,x%) |
| No | nn(xx.x%) | nn(xx.x16) | mn(xxxXIII) | nn(xx,x96) | nn(xx,x%) | nn(xx.x46) | nn(xx.x%) | mn(xx,x96) |
| Patients with Dose Interrupted [1] | nn(xx,x96) | nn(xx,x56) | mm(xxxxx96) | nn(xx,x96) | nn(xx,x%) | nn(bocx(6) | nn(xx.x%) | nn(xx,x%) |
| Yes | nn(xx,x%) | nn(xx,x96) | mn(xxxx%) | nn(xx,x96) | nn(xx,x46) | nn(xx,x36) | nn(xx,x%) | mn(xx,x%) |
| Adverse Event | nn(xxx96) | nn(xx.x56) | nn(xxxxxi) | nn(xx.x96) | nn(xx,x%) | nn(xx_x16) | nn(xx.x95) | nn(xx,x%) |
| Non-compliance | nn(xx.x96) | nn(xx,x96) | rim(xxxxx96) | nn(xx.x96) | nn(xx,x/l6) | nn(xxxx16) | nn(xx.x96) | nn(xx.x%) |
| Other | rin(xx,x96) | nn(xx,x16) | mm(xxxxW) | nn(xx,x96) | nn(xx.x%) | nn(xx,x%) | nn(xx,x96) | nn(xx,x%) |
| No | nn(xx.x%) | rm(xx,x%) | nn(xxxx%) | nn(xx.x%) | nn(xx.x%) | пп(хэджіі) | nn(xx,x%) | mn(xx,x%) |
| Patients with Dose Skipped[1] | nn(xx,x96) | nm(xx.x46) | mn(xxxx%) | nn(xx,x96) | mm(xx,x%) | nn(xx,x36) | nn(xx,x96) | nn(xx.x%) |
| Yes | rirr(xx,x%) | rm(xx.x%) | mm(xxxx96) | nn(xx.x%) | mm(xx,x46) | nn(xxxx16) | rim(xx,x96) | mn(xx,x%) |
| Adverse Event | mm(xxxx96) | mm(xx.x96) | nn(xxxx94) | nn(xx.x96) | mn(xx.x96) | mm(xxxx46) | nn(xx.x%) | nn(xx.x%) |
| Non-compliance | nn(xx,x%) | rin(xx,x56) | mn(accade) | nn(xx,x%) | nn(xx.x%) | nn(xxxx36) | nn(xx,x%) | nn(xx,x%) |
| Other | mm(xxxx96) | nn(xx.x%) | mm(xxxx94) | nn(xx,x94) | nn(xx.x46) | mm(xxxxx16) | rim(xx,x96) | nn(xx,x%) |
| No | mn(xx.x96) | nn(xx.x96) | nn(xxxx%) | mn(xx.x96) | nn(xx,x%) | mm(xxx46) | nn(xx.x%) | nn(xx.x%) |
| Patients with NBF-006 Withdrawn Due to | | | | | | | | |
| Adverse Event | mm(xx,x96) | rm(xx.x96) | nn(xxxx94) | mn(xx.x96) | nn(xx,x%) | mm(xxxx46) | rm(xx.x96) | nn(xx.x%) |
| XXXXXX | nn(xxx96) | nn(xx,x96) | nn(xxxx9b) | nn(xx,x96) | nn(xx,x36) | nn(xxxx16) | nn(xx.x96) | nn(xx.x16) |
| XXXXX | rm(xxxx96) | rm(xx,x96) | rin(socx%) | nn(xx.x90) | nn(xx,x46) | пп(холонь) | nn(xx,x96) | nn(xx.x%) |

[1] Number of Patients used as denominator to calculate percentages. Cross-References: Listing 16.2.7.2.1-3.

PROGRAMMER'S NOTES:

Based on the CAF NBF-006 Exposure page and Adverse Events page.

Present Part A and Part 8 output separately, adjust title for Part B accordingly.

Present Dose Skipped after Cycle 3 only data is available.

Copyright© 2016 by Therades Oncology®, Princeton NJ

Statistical Analysis Plan


All rights reserved

85



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b


### Table 14.3.5.1.4 Summary of Concomitant Measures (Dose Escalation Part A) Safety Evaluable (N=n)

| WHO-DD ATC Class Category Level II | NBF-00 | 6 Dose Level (m | g/kg) for Escalat | ion (Part A) | NB | F-006 Dose Expi | ansion (mg/kg) ( | Part B) |
|---|---|---|---|---|---|---|---|---|
| WHO-DD Preferred Term [1][2] | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | nnn | ann | nan | nnn | nnn | nnn | onn |
| Number of Patients Taking | mn(xx.x%) | nn(xx,x16) | m(xx.x%) | nn(xx.x%) | rm(xxx96) | nn(xx.x%) | mn(xxxx46) | nn(xx.x96) |
| Concomitant Measures[3][4] | | | | | | | | |
| WHO-DD ATC Class Category Level II | mn(xx.x96) | nn(xx.x46) | 7777(xx_x96) | rin(xx.x96) | mm(xxxx95) | nn(xx.x%) | mn(xxxxH) | mn(xx.x96) |
| WHO-DD Preferred Term | rrrr(xx,x96) | nn(xx,x%) | mm(xxxx96) | rim(xxx.x96) | rm(xxxx96) | nn(xx.x%) | mn(xxxxX) | nn(xx.x96) |
| WHO-DD Preferred Term | mm(xxx.x96) | nn(xx.x%) | nn(xx.x44) | rin(xx.x96) | rim(xxxx90) | nn(xx.x96) | nn(xxxx46) | mn(xx.x96) |
| WHO-DD Preferred Term | nn(xx.x%) | mn(xx,x46) | nn(xxx9b) | nn(xx,x96) | nn(xxxx96) | nn(xx,x%) | rin(xxxx16) | rin(xx,x96) |
| WHO-DD Preferred Term | nn(xx.x%) | nn(xx.x46) | nn(xxxx46) | nn(xx.x96) | nn(xxx94) | nn(xx.x96) | nn(xxxxiii) | m(xx.x94) |
| WHO-DD ATC Class Category Level II | nn(xx,x96) | nn(xx,x%) | nn(xxxxiii) | nn(xx.x96) | nn(xxxx96) | nn(xx.x%) | nn(xx.x46) | nn(xx,x96) |
| WHO-DD Preferred Term | nn(xx,x%) | nn(xx,x%) | nn(xxxx4i) | nn(xx,x96) | rm(xxxx96) | mm(xxxx96) | mm(xxxxx46) | rin(xx.x94) |
| WHO-DD Preferred Term | nn(xx,x96) | nn(xx,x%) | nn(xx_xq6) | rin(xx.x96) | nn(xxxx96) | nn(xx,x96) | nn(xxxx46) | mn(xx,x96) |
| WHO-DD Preferred Term | nn(xx,x%) | nn(xx,x16) | nn(xx.xiii) | nn(xx,x%) | nn(xxx%) | nn(xx,x%) | nn(xxxx16) | nn(xx.x96) |

<sup>[1]</sup> World Health Organization Drug Dictionary (WHO-DD) version 2018

Include all "Therapeutic Class" categories found in the database.

Sort "Therapeutic Class" column in descending order based on "Overal" column frequency count.

Present Part A and Part B output separately, adjust title for Part B accordingly

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 86


<sup>[2]</sup> Number of Patients used as denominator to calculate percentages.

<sup>[3]</sup> Patients may be counted in more than one therapeutic class; patients are only counted once within a therapeutic class.

<sup>[4]</sup> Summarizes medications (except for study drug) taken on or after the date of the first study drug dose up to last dose+30 days. Cross-References: Listing 16.2.10.1, 16.2.10.2 PROGRAMMERS NOTES:



NBF-006-001 Phase 1/15 DIRECTORY/FILE.SAS FINAL - ddmmmyychhomm Page 1 of x

## Table 14,3.5.2.1 Summary of Change from Baseline during Treatment Period for Hematology Tests (Dose Escalation Part A) Safety Evaluable (N=n)

| Hematology Test | | | | | | Dose Level (mg. | rkg) for Esta | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timepaint | | 0.15 | | - | 0.3 | | | onward | | - | Overal | |
| Statistics | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Chang |
| Lab Parameter 1 | | | | | | | | | | | | |
| (unit) | | | | | | | | | | | | |
| Baseline | | | | | | | | | | | | |
| N | nnn | | | nnn | | | mon | | | mmn | | |
| Mean | XX.X | | | XXXX | | | XX.X | | | XX.X | | |
| Standard | A.XX | | | XXX | | | X.XX | | | XXX | | |
| Deviation | | | | | | | | | | | | |
| Mediair | XX.X | | | XX.X | | | XX.X | | | XX.X | | |
| Minimum | XX | | | XX | | | XX. | | | XX | | |
| Maximum | xx | | | XXX<br>XXX | | | XX | | | xx<br>xx | | |
| Timepoint | | | | | | | | | | | | |
| N | non | rinni | nnn | nnn | mon | eron | nnn | non | mm | nnn | non | non |
| Mean | XX.X | XX.X | XX.X | XXX | xx.x | 10LK | XX.X | xxx | xx.x | XX.X | xx.x | XX.X |
| Standard | 8.300 | XXX | X.XX | XXX | x.xx | KIKK | XXX | N.XX | x.xx | x.xx | XXX. | x.xx |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | | | 30K.K | | | 30X,X | | | XXX | XX.X | |
| Minimum | xx<br>xx | XX | XX. | XXX<br>XXX | XX | XX | XX<br>XX | XX | XX | xx<br>xx | ××. | XX<br>XX |
| | 1000 | XX | XX | . 600 | XX | XX | WW | XX | XX | KK. | XX | XX. |

Cross-Reference: Listing 16.2.8.1

PROGRAMMERS NOTES:
Hematology Tests: hemographin, hematocrit, platelets, RBC and WBC and differentials, combined other cells.
Protocol Study Event Schedule and windowing will be used.

Copyright© 2016 by Therades Oncology®, Princeton NJ

Statistical Analysis Plan 87


All rights reserved



NBF-006-001 Phase 1/15 DIRECTORY/FILE.SAS FINAL - ddmmmyychhomm

### Table 14.3.5.2.1 Summary of Change from Baseline during Treatment, Period for Hematology Tests (Dose Expansion Part B) Safety Evaluable (N=n)

| Hematology Test | | | | | NBF-6 | 006 Dose Expan | nsion (mg/k | g) (Part B) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timepaint | 13 months | 0.6 | POLICE LITTLE SERVICE | Narresy Little | 1.2 | Sayad - Sales | | 1.6 | 2010 | o security. | Overal | les conserve |
| Statistics | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Change |
| Lab Parameter 1 | | | | - 1100 | | | | | | | | |
| (unit) | | | | | | | | | | | | |
| Baseline | | | | | | | | | | | | |
| N | non | | | nnn | | | mon | | | mmn | | |
| Mean | XX,X | | | XXXX | | | XX.X | | | XX.X | | |
| Standard | X.XX | | | XXX | | | XXX. | | | XXX | | |
| Deviation | | | | | | | | | | | | |
| Mediair | XX.X | | | XX.X | | | xx.x | | | XX.X | | |
| Minimum | XX | | | XX | | | XX | | | XX | | |
| Maximum | xx | | | XXX<br>XXX | | | XX | | | xx<br>xx | | |
| Timepoint | | | | | | | | | | | | |
| N | non | mmin | nnn | nnn | more | oran | nno | non | mm | nnn | nnn | non |
| Mean | XX.X | XX.X | XXX | 30K.K | xx.x | XXII.X | XX.X | XXX | xx.x | XX.X | xx.x | XX.X |
| Standard | x.xx | X.XX | X.XX | XXX | x.xx | XXX | XXX | x.xx. | X.XX | x.xx | XXX. | x.xx |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | XXXX | XXXX | 30K.K | XX.X | 30C.X | XXXX | XXX | XXX | XXX | XX.X | XX.X |
| Minimum | XX. | XX | XX | 300 | XX | XX | XX | XX. | KK | XX. | *X | XX |
| Maximum | XX | XX | XX | XX | XX | XX | XX | XX | XX | xx<br>xx | XX | xx<br>xx |

Cross-Reference: Listing 16.2.8.1 PROGRAMMER'S NOTES:

Hematology Tests: hemographic, hematocrit, platelets, RBC and WBC and differentials, combined other cells. Protocol Study Event Schedule and windowing will be used. Present Part A and Part B output separately, adjust title for Part B accordingly.

88

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan Final Version 2.0, March 14, 2023




NBF-006-001 Phase 1/15 DIRECTORY/FILE.SAS FINAL - ddmmmyychhomm

## Table 14.3.5.2.2 Summary of Change from Baseline during Treatment Period for Blood Chemistry Tests (Dose Escalation Part A) Safety Evaluable (N=n)

| Chemistry Test | | | | | NBF-006 I | lose Level (mg | rkg) for Esta | elation (Par | (A) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timepaint | Barrier | 0.15 | economic en | Authory III | 0.3 | | | onward | 5 | o team in the | Overal | es constant |
| Statistics | Actual | Change | %Change | Actual | Change | 954Change | Actual | Change | %Change | Actual | Change | %Change |
| Lab Parameter 1 | | | | - 1100 | | | | | | | | |
| (unit) | | | | | | | | | | | | |
| Baseline | | | | | | | | | | | | |
| N | non | | | nnn | | | mon | | | mmn | | |
| Mean | XX.X | | | XXXX | | | XX.X | | | XX.X | | |
| Standard | x.xx | | | XXX | | | x.xx | | | XXX | | |
| Deviation | | | | | | | | | | | | |
| Mediair | XX.X | | | XX.X | | | XX.X | | | XX.X | | |
| Minimum | XX | | | 300 | | | XX | | | XX | | |
| Maximum | xx | | | XXX<br>XXX | | | XX | | | xx<br>xx | | |
| Timepoint | | | | | | | | | | | | |
| N | nnn | mmin | nnn | nnn | more | eron | nno | non | mnn | nnn | non | non |
| Mean | XXX | XX.X | XXX | XXXX | xx.x | 10E.K | XX.X | XXX | XX.X | XX.X | xx.x | XX.X |
| Standard | 8.30 | X.XX | X.XX | XXX | x.xx | XXX | XXX | XXX. | X.XX | x.xx | x.xx | x.xx |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | XXXX | XXX | 30K.K | xx.x | 30C.X | 30X.X | XXX | KX.X | XXX | XX.X | XX.X |
| Minimum | XX | XX | XX | 300 | XX | xxc | XX | XX. | KK | XX. | ××. | XX |
| Maximum | 308 | XX. | XX | XX | XX | 300 | XX | XX | XX | xx<br>xx | XX | xx<br>xx |

Cross-Reference: Listing 16.2.8.2 PROGRAMMERS NOTES:

Blood Chemistry Tests: BUN, Sodium, Chloride, Phosphatase, Bicarbonate, Uric Acid, Direct Billrubin, Total Billrubin, Alkaline Phosphatase, SGPT/ALT, SGOT/AST, GGT, Creatine, Potassium, Calcium, Magnesium, Creatine Kinase, Total Protein, Albumin, Glucose, Protocol Study Event Schedule and windowing will be used.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 89




NBF-006-001 Phase 1/15 DIRECTORY/FILE.SAS FINAL - ddmmmyychhomm Page 1 of x

### Table 14,3,5,2,2 Summary of Change from Baseline during Treatment Period for Blood Chemistry Tests (Dose Expansion Part 8) Safety Evaluable (N=n)

| Chemistry Test | | | | | NBF-6 | 006 Dose Expan | sion (mg/k | g) (Part B) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timepoint | Barrie | 0.6 | SANTEN SE | Network 150 | 1.2 | Sayar Salar | | 1.6 | 524.6% | uses in | Overal | la compania |
| Statistics | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Change |
| Lab Parameter 1 | | | | - 1100 | | | | | | | | |
| (unit) | | | | | | | | | | | | |
| Baseline | | | | | | | | | | | | |
| N | non | | | nnn | | | mon | | | mmn | | |
| Mean | XXX | | | XXXX | | | XXX | | | XX.X | | |
| Standard | x.xx | | | XXX | | | x.xx | | | XXX | | |
| Deviation | | | | | | | | | | | | |
| Mediair | XX.X | | | XX.X | | | XX.X | | | XX.X | | |
| Minimum | XX | | | XX | | | | | | XX | | |
| Maximum | xx | | | XX | | | XX<br>XX | | | XX<br>XX | | |
| Timepoint | | | | | | | | | | | | |
| N | non | mmin | nnn | nnn | mm | oran | nino: | non | mnn | nnn | nnn | non |
| Mean | XX.X | XX.X | XXX | XXLX | xx.x | 10LX | XX.X | XXX | xx.x | XX.X | xx.x | XX.X |
| Standard | 36.30X | XXX. | X.XX | XXX | x.xx | XXX | x;xx | x.xx. | x.xx | x.xx | x.xx | x.xx |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | XXX | XXXX | 30K.K | xx.x | 30C.X | XX.X | XXX | KX.X | XXX | XX.X | XX.X |
| Minimum | XX. | XX | XX | 300 | XX | xxc | XX | XX. | KK | XX. | ××. | XX |
| Maximum | XX | XX | XX | XX | XX | 300 | XX | XX | XX | xx<br>xx | XX | XX<br>XX |

Cross-Reference: Listing 16.2.8.2 PROGRAMMER'S NOTES;

Blood Chemistry Tests: BUN, Sodium, Chloride, Phosphutase, Bicarbonate, Uric Acid, Direct Billrubin, Total Billrubin, Alkaline Phosphatase, SGPT/ALT, SGOT/AST, GGT, Creatine, Potassium, Calcium, Magnesium, Creatine Kinase, Total Protein, Albumin, Glucose, Protocol Study Event Schedule and windowing will be used.

Present Part A and Part B output separately, adjust title for Part B accordingly.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 90




NBF-006-001 Phase 1/15 DIRECTORY/FILE.SAS FINAL - ddmmmyychhomm

# Table 14,3,5,2,3 Summary of Change from Baseline during Treatment Period for Urinalysis Tests (Dose Escalation Part A) Safety Evaluable (N=n)


| Urinalysis Test | | | | | NBF-006 D | lose Level (mg | /kg) for Esta | slation (Par | (A) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timepaint | 1 Store and | 0.15 | dougrames. | Network Co. | 0.3 | August 1 | 43.6 | onward | 5 | a general and | Overal | Learner La |
| Statistics | Actual | Change | %Change | Actual | Change | 954Change | Actual | Change | %Change | Actual | Change | %Change |
| Lab Parameter 1 | | | | | | | | | | | | |
| (unit) | | | | | | | | | | | | |
| Baseline | | | | | | | | | | | | |
| N | non | | | nnn | | | mon | | | mmn | | |
| Mean | XX.X | | | 30CX | | | XX.X | | | XX.X | | |
| Standard | x.xx | | | XXX | | | x.xx | | | XXX | | |
| Deviation | | | | | | | | | | | | |
| Mediair | XX.X | | | XX.X | | | XX.X | | | XX.X | | |
| Minimum | XX | | | 300 | | | XX | | | XX | | |
| Maximum | xx | | | XXX<br>XXX | | | XX | | | xx<br>xx | | |
| Timepoint | | | | | | | | | | | | |
| N | non | mmin | nnn | nnn | mon | oran | nno | non | mm | nnn | non | non |
| Mean | XX.X | XX.X | XXX | XXLX | xx.x | 10LX | XX.X | XXX | xx.x | XX.X | xx.x | XX.X |
| Standard | 8.88 | XXX. | X.XX | XXX | x.xx | XXX | XXX | XXX. | X.XX | x.xx | XXX. | x.xx |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | XXX | XXXX | 30K.K | xx.x | 30C.X | XXXX | XXX | KX.X | XXX | XX.X | XX.X |
| Minimum | XX | XX | XX | 300 | XX | XX | XX | XX. | KK | XX | *X | XX |
| Maximum | 308 | XX. | XX | XX | XX | 300 | XX | XX | XX | xx<br>xx | XX | XX<br>XX |

Cross-Reference: Listing 16.2.6.3

PROGRAMMERS NOTES:
Urinalysis Test: Specific gravity, pH, Glucose, Protein, Ketones Nitrite, and Leukocyte Esterase, and microscopic tests.
Protocol Study Event Schedule and windowing will be used.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan

91




NBF-006-001 Phase 1/15 DIRECTORY/FILE.SAS FINAL - ddmmmyychhomm

# Table 14,3,5,2,3 Summary of Change from Baseline during Treatment Period for Uninalysis Tests (Dose Expansion Part B) Safety Evaluable (N=n)


| Lirinalysis Test | | | | | NBF-6 | 006 Dose Expa | ision (mg/k | gl (Part B) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timepaint | Barrier | 0.6 | Santilla de | naracy III. | 1.2 | Sayad-G-Mari | | 1.6 | 2010 39 | outen in | Overal | les conserv |
| Statistics | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Chang |
| Lab Parameter 1 | | | | | | | | | | | | |
| (unit) | | | | | | | | | | | | |
| Baseline | | | | | | | | | | | | |
| N | nnn | | | nnn | | | nnn | | | nnn | | |
| Mean | XX.X | | | 300.00 | | | 30K.R | | | XX.X | | |
| Standard | x,xx | | | X,XX | | | x,xx | | | x.xx | | |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | | | 300.00 | | | 300.30 | | | XX.X | | |
| Minimum | XX | | | XX | | | XX | | | XX | | |
| Maximum | ×× | | | ж | | | жк | | | ж | | |
| Timepoint. | | | | | | | | | | | | |
| N | nnn | mm | nnn | nnn | TITAL | non: | mnn | nns | mmm | nnn | nnn | nnn |
| Mean | XX.X | XX.X | XXX | 30C.X | xx.x | 300,00 | XX.X | xx.x | KK.K | XX.X | xx.x | XX.X |
| Standard | XXX | X-XX | X.XX | XXX | x.xx | X_XX | XXX. | X.XX | XXX | x.xx | K.XX | XXX |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | XXX | NOCK. | 300.00 | XX.X | 3008 | XX.X | XXX | XX.X | XX.X | XX.X | KK.K |
| Minimum | XX<br>XX | XX | XX | XX<br>XX | XX | 3000 | XX | XX. | XX | XX | XX | XX |
| Maximum | жx | XX<br>XX | 300 | 206 | XX | XX | XX<br>XX | xx | KK | XX<br>XX | xx<br>xx | XX |
| Lab Parameter 2 | | | | | | | | | | | | |
| (unit) | | | | | | | | | | | | |
| Baseline | | | | | | | | | | | | |

Cross-Reference: Usting 16,2,8,3

PROGRAMMERS NOTES:

Limaysia Test: Specific gravity, pH, Glucose, Protein, Ketones, Nitrite, and Leukocyte Esterase, and microscopic tests, 
Protocol Study Event Schedule and windowing will be used.

Present Part A and Part B output separately, adjust title for Part B accordingly.

Copyright© 2016 by Therades Oncology®, Princeton NJ

Statistical Analysis Plan 92


All rights reserved



DIRECTORY/FILE.SAS

FINAL - ddmmrnyychhamm


Table 14.3.5.3.1

Summary of Shift from Baseline to Maximum CTCAE Grade during Treatment Period for Hematology Tests (Dose Escalation Part A) Safety Evaluable (N=n)

| Hematology Test | Baseline Severity Grade | | | | | |
|---|---|---|---|---|---|---|
| NBF-006 Dose<br>Maximum CTCAE Grade [1][2] | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Overall |
| Lab Parameter 1 (unit) | | | | | | |
| 0.15 mg/kg | | | | | | |
| Grade 0 | nn(xxxx36) | mn(xx,x96) | mm(xxxxXIII) | rm(xx.x96) | nn(xx,x36) | rin(xx,x96) |
| Grade 1 | nn(xxxx46) | mn(xx.x96) | mm(xxxx36) | nn(xx.x96) | nn(xx,x%) | rim(xx.x96) |
| Grade 2 | nn(xx.x96) | mn(xx.x96) | mm(xxxx46) | mn(xx.x94) | mm(xxxx46) | mn(xx,x94) |
| Grade 3 | nn(xxxx9i) | rm(xx,x96) | nn(sococits) | rin(xxxx96) | mn(xxxx96) | rin(xx.x96) |
| Grade 4 | nn(xxx%) | (69x,xx)nn | nn(xx.x%) | nn(xx,x96) | mm(xx,x%) | rm(xx.x%) |
| Overall | nn(xxxXII) | rm(xx.x96) | mn(xxxxX6) | rm(xx.x96) | nn(xx.x%) | nnn (100.0%) |
| 0.3 mg/kg | | | | | | |
| Grade 0 | nn(xxxx96) | 1111(XX,X96) | mm(xxxx46) | mn(xx,x96) | mn(xxxx46) | mn(xx.x96) |
| Grade 1 | nn(xx,x%) | nn(xx.x36) | nn(xxxx46) | rin(xx,x96) | mn(xxxx46) | nn(xx.x%) |
| Grade 2 | mm(xxxx26) | rtrr(xx_x96) | mm(xxxx46) | mn(xx.x94) | mn(xxxx)6) | rm(xx,x94) |
| Grade 3 | mn(xxxx96) | (1111(xx,x96) | nn(xx.x%) | mn(xx.x96) | mn(xxxx%) | rin(xx,x96) |
| Grade 4 | nn(xxxx96) | mn(xx.x96) | nn(xx_x36) | rin(xx.x%) | mn(xx,x%) | nn(xx.x%) |
| criwards | | | | | | |
| Overall | rtm(xxx,x96) | nn(xx.x96) | mn(xxx.x16) | mn(xx.x%) | mm(xxxx96) | mnn (100,0%) |

Lab Parameter 2 (unit)

Overall for All Dose Levels

[1] Number of patients with both a baseline evaluation and an on-study evaluation used as denominator to calculate percentages,

[2] Maximum CTCAE Grade was defined as the highest CTCAE Grade reported for a patient after first dose.

Cross-References: Listing 16.2.8.1
PROGRAMMER'S NOTES:

Grand total used as denominator to calculate percentages within each category.

Hematology Parameters: hemoglobin, hematocnit, platelets, RBC and WBC and differentials, combined other cells.

Only gradable parameters are included in the table.

Present Part A and Part B output separately, adjust title for Part B accordingly.

Statistical Analysis Plan Copyright© 2016 by Therades Oncology®, Princeton NJ


All rights reserved



DIRECTORY/FILE.SAS

FINAL - ddmmmyychbonm Page 1 of x

Table 14.3.5.3.2

Summary of Shift from Baseline to Maximum CTCAE Grade during Treatment Period for Blood Chemistry Tests (Dose Escalation Part A)
Safety Evaluable (N=n)

| Blood Chemistry Test | Baseline Severity Grade | | | | | |
|---|---|---|---|---|---|---|
| NBF-006 Dose<br>Maximum CTCAE Grade (1)(2) | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Overall |
| Lab Parameter1 (unit) | ======================================= | | | | | |
| 0.15 mg/kg | | | | | | |
| Grade 0 | rrrr(xxx,x96) | nn(xx.x96) | mn(xxxx96) | nn(xx.x%) | mm(xxxxxHb) | rim(xx.x%) |
| Grade 1 | rin(xxxx96) | rin(xx,x46) | mm(xxxxxHb) | nn(xx,x56) | nn(xxx.x16) | nn(xx.x96) |
| Grade 2 | mm(xxxxx96) | rm(xx.x%) | nn(xxxxXXX) | nr(xx.x%) | nn(xx,xx46) | mm(xxxx44) |
| Grade 3 | mm(xxx,x94) | mn(xx.x96) | mm(xxxxxHi) | mm(xx.x46) | mm(socacifé) | mm(xxx,x94) |
| Grade 4 | mn(xxxx96) | rvt(xx.x96) | mm(poc.x96) | nn(xx.x46) | mm(xxxx46) | rm(xx.x96) |
| Overall | mm(xx.x%) | nn(xx.x95) | nn(xxxiii) | nn(xx.x46) | nn(xxxXII) | rinn (100.0%) |
| 0.3 mg/kg | | | | | | |
| Grade 0 | mn(xx.x96) | nn(xx.x%) | nn(xx_x%) | nn(xx.x56) | mm(xxxx46) | rin(xx.x%) |
| Grade 1 | mm(xxx.x96) | rin(xx,x%) | 71n(xxxx16) | nn(xx,x96) | mn(xxxx46) | nn(xxxx96) |
| Grade 2 | mm(soc.x96) | rm(xx.x56) | mn(xxxxHi) | mm(xxx.x96) | mn(xxxx) | rrrr(xx.x96) |
| Grade 3 | mn(xxxx96) | nn(xx.x96) | mm(xx2x96) | nn(xx.x56) | mn(xxxx16) | rin(xxxx94) |
| Grade 4 | mn(xxx.x96) | nn(xx,x%) | nn(xx,x36) | nn(xx.x86) | mm(pocx46) | nn(xxxx96) |
| onwards | | | | | | |
| Overall | rin(xxxx96) | nn(xx.x%) | nn(xxxx96) | nn(xx.x46) | mm(xxxx46) | nnn (100,0%) |
| 77.2 | | | | | | |

Lab Parameter2 (unit)

Overall for All Dose Levels

Cross-References: Listing 16.2.8.2 PROGRAMMER'S NOTES:

Grand total used as denominator to calculate percentages within each category.

Blood Chemistry tests: BUN, Sodium, Chloride, Phosphatase, Bicarbonate, Uric Acid, Direct Billirubin, Total Billirubin, Alkaline Phosphatase, SGPT/ALT, SGOT/AST, GGT, Creatine, Potassium, Calcum, Magnesium, Creatine Kinase, Total Protein, Albumin, Glucose.

Only gradable parameters are included.

Present Part A and Part B output separately, adjust title for Part B accordingly.

| N8F-006-001 | Statistical Analysis Plan | Final Version 2.0, March 14, 2023 |
|---|---|---|
| Copyright© 2016 by Therudex Oncology®, Princeton NJ | Providence and Commence of the | |

<sup>[1]</sup> Number of patients with both a baseline evaluation and an on-study evaluation used as denominator to calculate percentages.

<sup>[2]</sup> Maximum CTCAE Grade was defined as the highest CTCAE Grade reported for a patient after first dose.



DIRECTORY/RLE.SAS

FINAL - ddmmmyychbanm


Table 14.3.5.3.3

Summary of Shift from Baseline to Maximum CTCAE Grade during Treatment Period for Urinalysis Tests (Dose Escalation Part A)
Safety Evaluable (Nint)

| Urinalysis Test | Baseline Severity Grade | | | | | |
|---|---|---|---|---|---|---|
| NBF-006 Dose<br>Maximum CTCAE Grade [1][2] | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Overall |
| ab Parameter1 (unit) | 7.0 | | | | | |
| 0.15 mg/kg | | | | | | |
| Grade 0 | nn(xx.xH <sub>b</sub> ) | nn(xx.x56) | mm(xxx.x46) | nn(xx.x96) | mn(xx,x46) | rtrr(xxx,x95) |
| Grade 1 | mm(xxx,x%) | nn(xx.x%) | mn(xxxx96) | (25.xx)rrr | тп(жжжіі) | rrrr(xxx.x96) |
| Grade 2 | nn(xxxx%) | nn(xx,x96) | mm(xxxxXH) | nn(xx.x96) | nn(xx,x96) | rin(xx,x96) |
| Grade 3 | nn(xxxxH <sub>b</sub> ) | nn(xx.x%) | mn(xxxx46) | nn(xx.x%) | mm(xx,x%) | rin(xx.x95) |
| Grade 4 | nn(xx,x%) | nn(xx.x%) | nn(xx.x%) | mn(xx,x96) | nn(xxx46) | mm(xx.x96) |
| Overall | nn(xxx%) | nr(xx.x%) | nn(xxxx%) | mr(xx.x96) | mm(xxx46) | ппп (100.0%) |
| 0.3 mg/kg | | | | | | |
| Grade 0 | mn(xxxx46) | nn(xx.x%) | nn(xxxx16) | mn(xx,x%) | mmbxxx46) | nn(xx.x%) |
| Grade 1 | mm(xxx,x46) | mm(xx.x96) | an(xxx46) | nn(xx,x94) | mm(xxxx96) | rrrr(xxx.x94) |
| Grade 2 | mn(xxxx46) | nn(xx.x96) | mm(xxxx44) | nn(xx.x96) | mm(xx,x96) | mn(xx,x96) |
| Grade 3 | mn(xx,x%) | nn(xx,x%) | 710(XXX46) | mn(xx,x96) | mn(xxxx46) | nn(xx.x%) |
| Grade 4 | nrr(socue#6) | nn(xx.x96) | mn(xx_x%) | mn(xx.x94) | mn(xxx%) | rrrr(xxx.x94) |
| onwards | | | | | | |
| Overall | nn(xx,xHi) | nn(xx,x%) | mn(xx.x%) | rin(xx.x96) | mn(xxxx66) | rinn (100.0%) |

Lab Parameter2 (unit)

Overall for All Dose Levels

Cross-References: Usting 16.2.8.3
PROGRAMMERS NOTES:

Grand total used as denominator to calculate percentages within each category.

Urinalysis Tests: Specific gravity, pH. Glucose, Protein, Ketones, Nitrite, and Leukocyte Esterase, and microscopic tests.

Only gradable parameters are included in the table.

Present Part A and Part B output separately, adjust title for Part B accordingly.

Statistical Analysis Plan Final Version 2.0, March 14, 2023 Copyright© 2016 by Therades Oncology®, Princeton NJ Confidential - Entire Page All rights reserved 95

<sup>[1]</sup> Number of patients with both a baseline evaluation and an on-study evaluation used as denominator to calculate percentages.

<sup>[2]</sup> Maximum CTCAE Grade was defined as the highest CTCAE Grade reported for a patient after first dose.



Table 14.3.5.4

Vital Signs at Baseline Including Weight and Height (Dose Escalation Part A)

Safety Evaluable (N=n)

| | NI | BF-006 Dose Le | evel (mg/kg) for Esca | alation (Part A) | NBF-006 Dose Expansion (mg/kg) (Part B) | | | |
|---|---|---|---|---|---|---|---|---|
| Vital Signs | 0.15 | 0.3 | onwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| Number of Patients | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Systolic Blood Pressure (mmHg) | | | | | | | | |
| N | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| Median | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x |
| Minimum | xx | xx | xx | xx | xx | xx | xx | xx |
| Maximum | XX | XX | xx | xx | XX | xx | XX | XX |
| Diastolic Blood Pressure (mmHg) | | | | | | | | |
| N | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| Median | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x |
| Minimum | xx | xx | xx | xx | xx | xx | xx | xx |
| Maximum | XX | XX | xx | xx | xx | xx | XX | XX |
| Pulse ( /min) | | | | | | | | |
| N | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| Median | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x |
| Minimum | xx | xx | xx | xx | xx | xx | xx | xx |
| Maximum | xx | xx | xx | xx | xx | xx | xx | XX |
| Temperature (°C) | | | | | | | | |
| N | nnn | nnn | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x |
| Standard Deviation | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| Median | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x | xx.x | xx.x |
| Minimum | xx | xx | xx | xx | xx | xx | xx | xx |
| Maximum | xx | xx | xx | xx | xx | xx | xx | xx |

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 96




| 201000000000000000000000000000000000000 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Respiration ( /min) | | | | | | | | |
| N | nnn | non | nnn | nnn | nnn | nnn | unu | nnn |
| Mean | XXX | NX.N | xx.x | XXX | XX.X | xx.x | XX.X | XX.X |
| Standard Deviation | x,xx | 8.88 | X.XX | x,xx | X.XX | x.xx | x.xx | X.XX |
| Median | XXX | xx,x | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| Minimum | XX: | XX. | XX | XX | KK | KK. | KK. | XX |
| Maximum | ×× | XX | xx | ×× | ×× | XX | XX | XX |
| Weight (kg) | | | | | | | | |
| N | nnn | nnn- | nnn | man | non | non | rien | nnn |
| Mean | XXX | xx,x | XX.X | XXX | xx.x | xx.x | xx,x | XX,X |
| Standard Deviation | x,xx | 30,300 | x.xx | x,xx | x.xx | x.xx | x.xx | X.XX |
| Median | xx.x | XX.X | xx.x | XX-X | XX.X | XX.X | XX.X | XX.X |
| Minimum | xx | xx | xx | xx | XX | XX | ×× | XX |
| Maximum | xx. | XX | xx | ×× | кx | KK | KK | ЖK |
| Height (cm) | | | | | | | | |
| N | nnn | ririn: | nnn | nnn | nnn | mm. | mm | mm |
| Меап | XX.X | MX.X | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Standard Deviation | x.xx | N.XX | x.xx | x.xx | x.xx | x.xx | x.xx | XXX |
| Median | xx.x | NX.X | xx.x | xx.x | xx.x | xx.x | xx.x | XX.X |
| Minimum | XX. | ×× | XX. | ×× | XX | XX | XX | XX |
| Maximum | xx. | xx | XX | xx | xx | ×× | xx | XX |
| BSA | | | | | | | | |
| N | nnn | nna | nnn | nnn | nnn | nnn | nnn | nnn |
| Mean | xx.x | xx.x | xx,x | xxx | xx.x | XX.X | XX.X. | XX.X |
| Standard Deviation | x.xx | ×.×× | x.xx | x.xx | x.xx | x,xx | x.xx | x.xx |
| Median | XXX | XXX | xx,x | XXX | XX.X | XX.X | XXX | XXX |
| Minimum | xx | ×× | xx | ×× | ×× | ×× | XX | XX |
| Maximum | xx | ×× | xx | ×× | ×× | XX | XX | KK |

Cross-Reference: Listing 16.2.9.1
PROGRAMMERS NOTES:
Present Part A and Part B output separately, adjust title for Part B accordingly.

NBF-006-001 Copyright© 2016 by Theradex Oscology®, Princeton N7 All rights reserved

Statistical Analysis Plan Final Version 2.0, March 14, 2023

97



NBF-006-001 Phase 1/1b DIRECTORY/FILE.SAS FINAL - ddmmmyythhtmm Page 1 of x

### Table 14.3.5.5.1 Summary of ECG Data and Change from Baseline by Visit (Dose Escalation Part A) Safety Evaluable (N=n)

| ECG Parameter | NBF-006 Dose Level (mg/kg) for Escalation (Part A) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timepoint | 0.15 | | | _ | 0.3 | | | onwards: | | | Overal | |
| Statistics | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | <b>WChange</b> |
| ECG Parameter 1 | | | | | | | | | O Section 1 | | | |
| (unit) | | | | | | | | | | | | |
| Baseline | | | | | | | | | | | | |
| N | nnn | | | nnn | | | nnn | | | nnn | | |
| Mean | XX.X | | | XX.X | | | XX.X | | | XX,X | | |
| Standard | x.xx | | | 10,000 | | | x.xx | | | x,xx | | |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | | | XX.X | | | xx,x | | | XXXX | | |
| Minimum | XX | | | 300 | | | XX. | | | XX | | |
| Maximum | XX | | | 306 | | | XX | | | xx | | |
| Timepoint | | | | | | | | | | | | |
| N | nnn | mm | mm | nnn: | nnn | nem | mmn | mnn | nnn | mm | non | nnn |
| Mean | XX.X | XXX | XXX | XX.X | XX.X | XXLX | XX.X | XX.X | XXX | XXX | XXX | XX.X |
| Standard | x.xx | x.xx | 30.000 | KXX | x.xx | x.xx | x.xx | x.xx | X.XX | x.xx | x.xx | X,XX |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | XXX | XXX | XXX | 8X.8 | XXX | XX.X | XXX | XXX | XX.X | XX.X | XXXX |
| Minimum | xx | XX | XX. | 300 | XX | XX | XX | XX | кx | жx | ×× | XX |
| Maximum | XX | XX. | XX | 301 | XX | XX | XX | XX. | <b>KK</b> | XX | ××. | XX |

«Repeat timepoint>

ECG Parameter 2 (unit)

QT=QT interval, QTcF= QT corrected by Fridericia's formula

Cross-Reference: Usting 16.2.9.3 PROGRAMMERS NOTES:

ECG parameters; heart rate, PR, QT, QTcF Protocol Study Event Schedule and windowing will be used.

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan

98




NBF-006-001 Phase 1/1b DIRECTORY/FILE.SAS FINAL - ddmmmyythhtmm Page 1 of x

### Table 14.3.5.5.2 Summary of ECG Data and Change from Baseline by Visit (Dose Expansion Part B)

Safety Evaluable (N=n) ECG Parameter NBF-006 Dose Expansion (mg/kg) (Part 8) Overall Timepoint 0.6 1.2 1.6 Statistics Actual Change %Change Actual Change %Change Change %Change Actual Change %Change ECG Parameter 1 (unit) Baseline nnn nnn ninn nnn Mean XX.X XX.X XX.X XXX Standard X,XX XXX X.XX XXX Deviation Median XX.X XX.X XXX.R XX.X Minimum xx XX XX XX Maximum XX xx XX XX Timepoint: nm mmm nnn nnn mmin mnn nnn mmn nnn nnn nhn nnn Mean XX.X. XXX XX.X XX.X XX.X XX.X XX.X XX.X KK.X. XX.X XX.X KK.K Standard x.xx X.XX X.XX XXX X.XX XXX X.XX X.XX X.XX XXX. X.XX X.XX Deviation Median XX.X XXX XXX XXX XX.X XXX XX,X XX.X KK,X XX.X xx.x XX.X Minimum XX Maximum xx ж XX xx KX ĸĸ хx XX ХX XX. xx XX.

<Repeat. timepoint>

ECG Parameter 2 (unit)

QT=QT interval, QTcF= QT corrected by Fridericia's formula

Cross-Reference: Usting 16.2.9.3

PROGRAMMERS NOTES:

ECG parameters: heart rate, FR, QT, QTcF

Protocol Study Event Schedule and windowing will be used.

Present Part A and Part B output separately, adjust title for Part B accordingly.

Statistical Analysis Plan Copyright© 2016 by Therades Oncology®, Princeton NJ


All rights reserved

99



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b


# Table 14,3,5,6,1 Summary of ECG Parameter QT and QTcF Data by Visit (Dose Escalation Part A) Safety Evaluable (N=n)

| Timepoint | NBF-00 | NBF-006 Dose Expansion (mg/kg) (Part B) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| ECG Parameter | 0.15 | 0.3 | anwards | Overall | 0.6 | 1.2 | 1.6 | Overall |
| lumber of Patients | nnn | nnn | rinn | nnn | rinn | nnn | nnn | nnn |
| Baseline | | | | | | | | |
| QT interval | mn(xx.x96) | nn(xx.x46) | (dPx_xx)nn | rm(xx.x96) | mm(xxxx95) | nn(xx.x56) | mn(xxxx46) | rin(xx.x96 |
| s450 msec | mm(xx,x96) | nn(xx,x%) | nn(xx.x46) | rm(xx,x96) | rim(xxxx94) | nn(xx.x%) | nn(xxxx4i) | nn(xx.x9 |
| >450 msec | mm(xx.x96) | nn(xx,x%) | (Africacions | nn(xx.x96) | rm(xxxx94) | nn(xx,x%) | nn(xx.x4b) | nn(xx.x9) |
| >480 msec | mn(xx.x96) | nn(xx,x%) | mn(xx,x%) | ran(xx.x96) | mm(xxxx96) | nn(xx.x%) | mn(xxxx16) | rin(xx.x9i |
| >500 msec | mm(xx.x96) | nn(xx,x%) | nn(xxxx96) | rm(xx.x96) | rm(xxxx96) | nn(xx.x%) | nn(xxxxX) | nn(xx.x9) |
| Increase > 30 | nn(xx.x%) | nn(xx,x%) | nn(xx.x%) | nn(xx.x96) | nn(xxx96) | nn(xx,x%) | nn(xxxxiii) | nn(xx,x96 |
| Increase > 60 | nn(xx.x96) | nn(xx.x46) | nn(xxxx46) | nm(xx.x96) | rin(xxx.x96) | nn(xx.x96) | mm(xxxxx46) | nn(xx.x9 |
| QTc Interval | | | | | | | | |
| s450 msec | nn(xx,x95) | nn(xx,xl6) | nn(xxxx96) | nn(xx.x96) | rin(xxxx96) | nn(xxx96) | mm(xxxxx46) | nn(xx.x9) |
| >450 to 480 msec | nn(xx,x96) | nn(xx.x%) | (dPx_xx)nn | mn(xx,x96) | nn(xxxx96) | nn(xx,x56) | nn(xxxxXii) | mn(xx.x90 |
| >480 to 500 msec | nn(xx,x%) | nn(xx,xi6) | mn(xx.x96) | nn(xx.x%) | nn(xxx96) | nn(xx,x%) | mm(xxxx96) | nn(xx.x% |
| >500 msec | nn(xx.x%) | nn(xx.x%) | mm(xx,x;Hi) | nm(xx,x%) | nn(xxx%) | nn(xx.x96) | пп(жжжі) | nn(xx.x9 |
| increase > 30 | nn(xx,x95) | nn(xx,xl6) | nn(xxx%) | nn(xx.x%) | nn(xxxx96) | nn(xx,x%) | nn(xxxx16) | nn(xx.x% |
| increase > 60 | nn(xx.x%) | nn(xx,x%) | mm(xx_x/6) | nm(xx,x%) | mn(xxxx46) | nn(xx,x%) | mm(xxxx/H) | mn(xx.x9) |

QT-QT interval, QTof-- QT corrected by Fridericia's formula

ECC parameters: heart rate, PR, QT, QTcF
Present Part A and Part B output separately, adjust title for Part B accordingly.

Statistical Analysis Plan

100

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved


<sup>111</sup> Number of Patients used as denominator to calculate percentages.
Cross-Reference: Listing 16.2.9.3
PROGRAMMERS NOTES:


DIRECTORY/FILE.SAS NBF-006-001 Phase 1/15

FINAL - ddmmmyythhtmm Page 1 of x

#### Table 14.3.5.7.1 Summary of Shift from Baseline to Maximum ECOG Score (Dose Escalation Part A) Safety Evaluable (N=n)

| NBF-006 Dose | | Baseline ECOG Perform | ance | |
|---|---|---|---|---|
| Maximum Score [1][2] | Scare 0 | Score 1 | Score 2 | Overall |
| 0.15 mg/kg | | | | |
| Score 0 | non (xx.x96) | nnm (xx.x96) | nnn (xxxxH) | nnn (xxxx96) |
| Score 1 | nnn (xx.x96) | mmm (xx.x96) | mm (xxxXH) | nnin (xxxx96) |
| Score 2 | ninn (xx,x96) | rinn (xx,x%) | nnn (xxxxib) | rinn (xxxx96) |
| Score 3 | nnn (xx,x96) | nnm (xx.x96) | mm (xxxxH) | nnn (xxxx96) |
| Score 4 | nnn (xx.x96) | rinn (xx.x96) | mm (xxx46) | nnin (xxxx94) |
| Score 5 | non (kx.x96) | nnn (xx.x96) | nnn (xxx%) | mmm (xxxx94) |
| Overall | nnn (xx.x96) | nnn (xx.x96) | mm (xxxx4) | nnn (xxxx%) |
| Onwards | | | | |
| Score 0 | nnn (xx,x96) | nnn (xx.x96) | nnn (xxxx96) | /mm (xxxx96) |
| Score 1 | nnn (xx.x96) | ninn (xx.x96) | mm (xxx%) | nnn (xxxx94) |
| Score 2 | nnn (kx.x96) | nnn (xx.x96) | non (xxxx96) | mmm (xxxx94) |
| Score 3 | nnn (xx,x96) | nnn (xx.x96) | nnn (xxxx%) | nnn (xxxx96) |
| Score 4 | nnn (xx.x96) | nnn (xx.x96) | nnn (xxxxH) | mm (xxxx9b) |
| Score 5 | nnn (xx.x96) | ninn (xx.x96) | non (xxx96) | nnn (xxxx96) |
| Overall | nnn (xx.x96) | nnn (xx.x%) | non (xxx4) | nnn (xxxx96) |
| Overall | | | | |
| Score 0 | mm (xx,x%) | nnn (xx.x96) | min (xxxx96) | nnn (xxxx96) |
| Score 1 | non (xx,x%) | nnn (xx.x96) | man (xx.x%) | mm (xxx.x%) |
| Score 2 | nnn (xx.x96) | nnn (xx.x96) | nrin (xxxx%) | nnn (xxxx96) |
| Score 3 | nnn (xx,x%) | nnn (xx,x96) | mm (xxxx96) | nnn (xx,x%) |
| Score 4 | nnn (xx.x%) | ninn (xx.x96) | nnn (xx.x%) | mm (xxxx96) |
| Score 5 | mmm (xxx.x96) | nnn (xx.x96) | mm (xxxx%) | mm (xxxx94) |

Cross-References: Listing 16.2.9.4 PROGRAMMERS NOTES:

Grand total used as denominator to calculate percentages within each category

Statistical Analysis Plan Final Version 2.0, March 14, 2023 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved Confidential - Entire Page 101

Overall for All Dose Levels

[1] Number of patients with both a baseline evaluation and an on-study evaluation used as denominator to calculate percentages.

<sup>[2]</sup> Maximum score are the highest ECOG for a patient after first dose.



NBF-006-001 Phase 1/15

DIRECTORY/FILE.SAS

FINAL - ddmmmyythhtmm Page 1 of x

Table 14.3.5.7.2 Summary of Shift from Baseline to Maximum ECOG Score (Dose Expansion Part B)

| NBF-006 Dose | | Baseline ECOG Performs | arce. | |
|---|---|---|---|---|
| Maximum Score [1][2] | Scare 0 | Score 1 | Score 2 | Overall |
| 0.15 mg/kg | | | | |
| Score 0 | nnn (xx.x96) | ninn (xx.x%) | nnn (accx96) | nnn (xxxx96) |
| Score 1 | nnn (xx.x96) | nnin (xx,x96) | nnn (xxxx4) | nnn (xxxx%) |
| Score 2 | mm (xx,x96)- | rinin (xx,x96) | mm (access) | nnn (xxxx96) |
| Score 3 | ninn (xx.x96) | rinn (xx.x%) | nnn (xxxxiii) | rinn (xxxx96) |
| Score 4 | nnm (xx.x96) | nnin (xx,x96) | mm (xxxx4) | mmm (xxxx96) |
| Score 5 | nnn (xx.x95) | rinn (xx.x96) | nnn (xxxx46) | nnn (xxxxx96) |
| Overall | nnn (xx.x96) | nnn (xx.x96) | nnin (xxxx96) | mm (xxxx94) |
| Onwards | | | | |
| Score 0 | nnn (xx.x96) | nnn (xx.x96) | mm (xxxx96) | nnn (xxxx94) |
| Score 1 | nnn (xx,x96) | nna (xx.x96) | nnn (xxxx96) | nnn (xxxx96) |
| Score 2 | nnn (xx.x96) | nnn (xx.x%) | mm (xxxx46) | nnn (xxxx94) |
| Score 3 | nnn (kx.x96) | nnn (xx.x96) | non (xxx96) | nnn (xxxx94) |
| Score 4 | nnn (xx,x96) | nnn (xx.x96) | nnn (xxxx%) | nnn (xxxx96) |
| Score 5 | nnn (xx.x96) | nnn (xx.x96) | mm (xxxx9b) | nnn (acce9i) |
| Overall | nnn (xx.x96) | mm (xx.x96) | nnn (xxx96) | nnn (xxx96) |
| Overall | | | | |
| Score 0 | nnn (xx.x96) | nnn (xx.x96) | nort (xxxx96) | mnn (xxxx96) |
| Score 1 | nnn (xx,x96) | nnn (xx.x96) | nnn (xxx96) | mnn (xxxxx4) |
| Score 2 | nnn (xx.x%) | nnn (xx.x96) | mm (xxx96) | mm (xxx96) |
| Score 3 | nnn (xx.x%) | nnn (xx.x96) | nm (xxx%) | nnn (xxxx94) |
| Score 4 | nnn (xx.x96) | nnn (xx,x96) | mm (xxxx96) | nnn (xxxx%) |
| Score 5 | nnn (xx.x%) | ninin (xx.x96) | mm (accade) | mm (xxxx%) |

## Overall for All Dose Levels

Grand total used as denominator to calculate percentages within each category.

Present Part A and Part B output separately, adjust title for Part B accordingly.

Statistical Analysis Plan Final Version 2.0, March 14, 2023 Copyright© 2016 by Therades Oncology®, Princeton NJ 102 Confidential - Entire Page All rights reserved

<sup>[1]</sup> Number of patients with both a baseline evaluation and an on-study evaluation used as denominator to calculate percentages.

<sup>[2]</sup> Maximum score are the highest ECOG for a patient after first dose.

Cross-References: Usting 16,2,9,4
PROGRAMMERS NOTES:



14.4 Biomarker Data Summary Tables

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan

103




NBF-006-001 Phase 1/1b DIRECTORY/FILE.SAS FINAL - ddmmmyychhomm Page 1 of x

# Table 14.4.1.1 Summary of Mean Change from Baseline in TNF-o Overtime (Dose Escalation Part A) Safety Evaluable (N=n)

| Timepoint | 13 marin | 0.15 | | | 0.3 | 4.00 | | onward | 5 | or a Sewart of Sewart | Overal | · January Commercial |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Statistics | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Chang |
| Baseline | | | | | | | | | | | | |
| N | nnn | | | nnn | | | nnn | | | nnn | | |
| Mean | XX.X | | | XX.X | | | XX.X | | | XX,X | | |
| Standard | x.xx | | | K.XX | | | x.xx | | | x.xx | | |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | | | AXCX | | | xx,x | | | XXXX | | |
| Minimum | XX. | | | 300 | | | XX | | | XX | | |
| Maximum | XX | | | XX | | | XX<br>XX | | | xx | | |
| Timepoint | | | | 300 | | | ××. | | | xx | | |
| N | nnn | nnn | min | non | nnn | ment | nnn | mnn | men | nnn | non | nnn |
| Mean | XX.X | XXX | XXX | XX.X | XX.X | XXC.X | XX.X | XXX | XXX | XXXX | XX.X | XXX |
| Standard | x.xx | x.xx | X.300 | K.XX | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | XXX | XXXX | XXX | XX.X | XXLX | XX.X | XXX | XXXX | XX.X | XXX | XX.X |
| Minimum | xx | XX | XX. | | XX | XX | XX | XX | кx | жx | ×× | XX |
| Maximum | XX | XX | XX | 30X<br>30X | XX | 300 | 300 | XX. | <b>KK</b> | XX | ××. | XX |

Cross-Reference: Figure 14.4.1.1, Listing 16.2.9.7
PROGRAMMERS NOTES:

NBF-006-001 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 104




NBF-006-001 Phase 1/15 DIRECTORY/FILE.SAS FINAL - ddmmmyychhomm Page 1 of x

#### Table 14.4.1.2 Summary of Mean Change from Baseline in TNF-a Overtime (Dose Expansion Part B) Safety Evaluable (N=n)

| | | | | | NBF-6 | 006 Dose Expa | nsion (mg/k | g) (Part B) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timepoint | Barrier | 0.6 | SAME TO SE | nuesesym on | 1.2 | Sand S. Was | | 1.6 | 52405 36 | u seemi in a | Overal | la conserva |
| Statistics | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Change | Actual | Change | %Change |
| Baseline | 10163 | | | | | | | | | | | |
| N | nnn | | | non | | | nnn | | | mm | | |
| Mean | MX.W | | | XXX | | | XX.X | | | XX.X | | |
| Standard | X,XX | | | XXX | | | X.XX | | | x.xx | | |
| Deviation | | | | | | | | | | | | |
| Median | - xx.x | | | 300.00 | | | 300.8 | | | XX.X | | |
| Minimum | xx | | | XX | | | XX | | | XX | | |
| Maximum | жx | | | ж. | | | жĸ | | | XX<br>XX | | |
| Timepoint | | | | xx | | | XX | | | XX | | |
| N | nnn | nnn | nnn | nnn | nrvn | non | nnn | nnn | nnn | nnn | nhn | nnn |
| Mean | 38.X | XXX | XXX | XXX | XX.X | XXX.X | XX.X | xx.x | XX.X | XX.X | xx.x | KK.K |
| Standard | x.xx | X.XX | XXX | XXX | x.xx | XXX | x.xx | X.XX | X.XX | XXX. | XXX | XXX. |
| Deviation | | | | | | | | | | | | |
| Median | XX.X | XXXX | XXXX | XXXX | xx.x | 300,8 | 300.8 | XXX | KK.X | XX.X | xx.x | XX.X |
| Minimum | XX | XX | XX. | XX | XX | 200 | XX | XX. | XX | XX | XX | XX |
| Maximum | ×× | XX | XX | XX | KK. | 300 | XX | XX | жx | XX. | XX<br>XX | XX |

Present Part A and Part B output separately, adjust title for Part B accordingly.

Present Part B only if data is available (cytokines to be collected if there are symptoms indicative of cytokine induction, e.g., IRRs). PROGRAMMERS NOTES:

Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 105




< Repeat for>

#### Table 14.4.2.1 Summary of Mean Change from Baseline in IL-1β Overtime (Dose Escalation Part A) Safety Evaluable (N=n)

Cross-Reference: Figure 14.4.2.1, Listing 16.2.9.7
PROGRAMMERS NOTES:

#### Table 14.4.2.2

Summary of Mean Change from Baseline in IL-1β Overtime (Dose Expansion Part B) Safety Evaluable (N=n)

Cytokines only collected in Part B at 1.6 mg/kg if cytokine induction was seen at 1.6 mg/kg in Part A, or if there are symptoms indicative of cytokine induction. Cross-References: Figure 14.4.2.2, Listing 16.2.9.7

PROGRAMMER'S NOTES:

Present Part B only if data is available (cytokines to be collected if there are symptoms indicative of cytokine induction, e.g., IRRs).

Table 14,4.3.1 Summary of Mean Change from Baseline in It-6 Overtime (Dose Escalation Part A) Safety Evaluable (N=n)

Cross-References; Figure 14.4.3.1, Listing 16.2.9.7 PROGRAMMER'S NOTES:

Table 14,4,3.2

Summary of Mean Change from Baseline in IL-6 Overtime (Dose Expansion Part B) Safety Evaluable (N=n)

Cytokines only collected in Part B at 1.6 mg/kg if cytokine induction was seen at 1.6 mg/kg in Part A, or if there are symptoms indicative of cytokine induction. Cross-Referencest Figure 14.4.3,2, Listing 16.2.9.7

PROGRAMMER'S NOTES:

Present Part 8 only if data is available (cytokines to be collected if there are symptoms indicative of cytokine induction, e.g., IRRs).

NBF-006-001 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan


106



#### Table 14.4.4.1

Summary of Mean Change from Baseline in IFN-y Overtime (Dose Escalation Part A) Safety Evaluable (N=n)

Cross-References: Figure 14.4.4.1. Listing 16.2.9.7

PROGRAMMER'S NOTES:

#### Table 14,4,4,2

Summary of Mean Change from Baseline in IFN-y Overtime (Dose Expansion Part B) Safety Evaluable (N=n)

Cytokines only collected in Part B at 1.6 mg/kg if cytokine induction was seen at 1.6 mg/kg in Part A, or if there are symptoms indicative of cytokine induction. Cross-References: Figure 14,4,4,2, Listing 16,2,9,7

PROGRAMMER'S NOTES:

Present Part B only if data is available (cytokines to be collected if there are symptoms indicative of cytokine induction, e.g., IRRs).

### Table 14.4.5.1

Surremary of Mean Change from Baseline in Complement-CH50 Overtime (Dose Escalation Part A) Safety Evaluable (N=n)

Cross-References: Figure 14.4.5.1, Listing 16.2.9.8 PROGRAMMERS NOTES:

#### Table 14.4.5.2

Summary of Mean Change from Baseline in Complement-CH50 Overtime (Dose Expansion Part B) Safety Evaluable (N=n)

Cross-References: Figure 14.4.5.2, Listing 16.2,9.8 PROGRAMMERS NOTES:

#### Table 14,4.6.1

Summary of Mean Change from Baseline in Complement-Bb Overtime (Dose Escalation Part A) Safety Evaluable (N=n)

Cross-References: Figure 14.4.6.1, Listing 16.2.9.8 PROGRAMMER'S NOTES:

Statistical Analysis Plan


Copyright© 2016 by Therades Oncology®, Princeton NJ

All rights reserved

107



#### Table 14.4.6.2

Summary of Mean Change from Baseline in Complement-Bb Overtime for Dose Expansion (Part B)

Safety Evaluable (N=n)

Cross-References: Figure 14.4.6.2, Listing 16.2.9.8

PROGRAMMER'S NOTES:

Table 14,4,7,1

Summary of Mean Change from Baseline in Complement-C3a Overtime (Dose Escalation Part A) Safety Evaluable (N=n)

Cross-References: Figure 14.4.7.1, Listing 16.2.9.8 PROGRAMMERS NOTES:

Table 14.4.7.2

Summary of Mean Change from Baseline in Complement-C3a Overtime (Dose Expansion Part B) Safety Evaluable (N=n)

Cross-References: Figure 14.4.7.2, Listing 16.2.9.8

PROGRAMMER'S NOTES

Table 14,4,8,1

Summary of Mean Change from Baseline in Complement-C5a Overtime (Dose Escalation Part A) Safety Evaluable (N=ri)

Cross-References: Figure 14.4.8.1, Listing 16.2.9.8 PROGRAMMER'S NOTES:

Table 14.4.8.2

Summary of Mean Change from Baseline in Complement-CSa Overtime (Dose Expansion Part B) Safety Evaluable (N=n)

Cross-References: Figure 14.4.8.2, Listing 16.2.9.8

PROGRAMMER'S NOTES:

NBF-006-001

Statistical Analysis Plan


Copyright© 2016 by Therades Oncology®, Princeton NJ

All rights reserved

108



Figure 164.4.1.1: Spaghetti Plot for individual Change from Baseline in TNF-o Overtime (Dose Escalation Part A)
Safety Evaluable (N=n)



Cross-References: Table 14.4.1.1, Listing 16.2.9.7
PROGRAMMERS NOTES:
Y-axis scale should always be -100 to 100 to avoid presenting extreme values.
Use line colors/ patterns to represent different dose levels.

#### Repeat for

Figure 174.4.1.2: Spagnetti Plot for Individual Change from Baseline in TNF-o Overtime (Dose Escalation Part B)

Cross-References: Table 14.4.1.2. Listing 16.2.9.7

NBF-006-001 Copyright© 2016 by Therades Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 109




#### PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Present Part Bionly if data is available (cytokines to be collected if there are symptoms indicative of cytokine induction, e.g., IRRs).

Figure 184.4.2.1: Spaghetti Plot for Individual Change from Baseline in IL-1β Overtime (Dose Escalation Part A)

#### Cross-References: Table 14.4.2.1, Listing 16.2.9.7

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Present Part Blonly if data is available (cytokines to be collected if there are symptoms indicative of cytokine induction, e.g., IRRs).

Figure 194.4.2.2; Spaghetti Plot for Individual Change from Baseline in IL-1β Overtime (Dose Escalation Part B)

#### Cross-References: Table 14.4.2.2, Listing 16.2.9.7

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Present Part Bionly if data is available (cytokines to be collected if there are symptoms indicative of cytokine induction, e.g., IRRs).

Figure 204.4.3.1; Spagnetti Plot for Individual Change from Baseline in IL-6 Overtime (Dose Escalation Part A)

### Cross-References: Table 14.4.3.1, Listing 16.2.9.7

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Present Part 8 only if data is available (cytokines to be collected if there are symptoms, indicative of cytokine induction, e.g., IRRs).

Figure 214.4.3.2: Spagnetti Plot for Individual Change from Baseline in IL-6 Overtime (Dose Escalation Part B)

#### Cross-References: Table 14.4.3.2. Listing 16.2.9.7

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Present Part 8 only if data is available (cytokines to be collected if there are symptoms indicative of cytokine induction, e.g., IRRs).

Copyright© 2016 by Theradex Oncology®, Princeton NJ

Statistical Analysis Plan


All rights reserved



Figure 224.4.4.1: Spagnetti Plot for Individual Change from Baseline in IFN-y Overtime (Dose Escalation Part A)

Cross-References: Table 14.4.4.1. Listing 16.2.9.7

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Present Part Blonty if data is available (cytokines to be collected if there are symptoms indicative of cytokine induction, e.g., IRRs).

Figure 234.4.4.2: Spagnetti Plot for Individual Change from Baseline in IFN-y Overtime (Dose Escalation Part B)

Cross-References: Table 14.4.4.2. Listing 16.2.9.7

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Present Part Biorily if data is available (cytokines to be collected if there are symptoms indicative of cytokine induction, e.g., (RRs),

Figure 244.4.5.1: Spaghetti Plot for Individual Change from Baseline in Complement-CH50 Overtime (Dose Escalation Part A)

Cross-References: Table 14.4.5.1, Listing 16.2.9.8

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Figure 254.4.5.2: Spaghetti Piot for Individual Change from Baseline in Complement-CH50 Overtime (Dose Escalation Part B)

Cross-References: Table 14.4.5.2, Listing 16.2.9.8

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Figure 264.4.6.1: Spaghetti Plot for Individual Change from Baseline in Complement-Bb Overtime (Dose Escalation Part A)

Cross-References: Table 14.4.6.1, Listing 16.2,9.8

Copyright© 2016 by Therades Oncology®, Princeton NJ

Statistical Analysis Plan


All rights reserved

111



PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Figure 274.4.6.2: Spaghetti Piot for Individual Change from Baseline in Complement-Bb Overtime (Dose Escalation Part B)

Cross-References: Table 14.4.6.2, Listing 16.2.9.8

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Figure 284.4.7.1: Spaghetti Piot for Individual Change from Baseline in Complement-C3a Overtime (Dose Escalation Part A)

Cross-References: Table 14.4.7.1, Listing 16.2.9.8

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Figure 294.4.7.2: Spaghetti Plot for Individual Change from Baseline in Complement-C3a Overtime (Dose Escalation Part B)

Cross-References: Table 14.4.7.2, Listing 16.2.9.8

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Figure 304.4.8.1: Spaghetti Plot for Individual Change from Baseline in Complement-C5a Overtime (Dose Escalation Part A)

Cross-References: Table 14.4.8.1, Listing 16.2.9.8

PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Figure 314.4.8.2: Spaghetti Plot for individual Change from Baseline in Complement-C5a Overtime (Dose Escalation Part 8)

Cross-References: Table 14.4.8.2, Listing 16.2.9.8

Copyright© 2016 by Therades Oncology®, Princeton NJ

Statistical Analysis Plan 112


All rights reserved



#### PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values. Use line colors/ patterns to represent different dose levels.

Figure 324.4.9.1: Spaghetti Piot for Individual Change from Baseline in GSTP1 mRNA Level Overtime (Dose Escalation Part A)

# Crass-References: Listing 16.2.9.14 PROGRAMMER'S NOTES:

Y-axis scale should always be -100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.

Figure 334.4.9.2: Spaghetti Plot for Individual Change from Baseline in GSTP1 mRNA Level Overtime (Dose Escalation Part 8)

Cross-References; Listing 16.2.9.14
PROGRAMMERS NOTES:
Y-axis scale should always be +100 to 100 to avoid presenting extreme values.

Use line colors/ patterns to represent different dose levels.



# 4.0 Index of Listing

| Listing 16.2.1.1 Patient Disposition | . 116 |
|---|---|
| Listing 16.2.2.1 Inclusion/Exclusion Criteria | . 117 |
| Listing 16.2.4.1 Demographics | . 118 |
| Listing 16.2.4.2.1 Disease Related Characteristics | . 119 |
| Listing 16.2.4.2.2 Baseline KRAS Mutation Assessment | . 120 |
| Listing 16.2.4.3 Medical History | . 121 |
| Listing 16.2.4.4 Prior Cancer Therapy | . 122 |
| Listing 16.2.4.5 Prior Medications | . 123 |
| Listing 16.2.4.6 Prior Cancer Radiation | . 124 |
| Listing 16.2.4.7 Prior Cancer Surgeries | . 125 |
| Listing 16.2.4.8 Pregnancy Test | . 126 |
| Listing 16.2.5.1 NBF-006 Administration | . 127 |
| Listing 16.2.6.1 Extent of Disease: Target and Non-Target Lesions | . 128 |
| Listing 16.2.6.2 Cycle Response Assessment | . 130 |
| Listing 16.2.7.1 Adverse Events | . 131 |
| Listing 16.2.7.2.1 Treatment-Emergent Adverse Events Leading to Dose<br>Interrupted | . 132 |
| Listing 16.2.7.2.2 Treatment-Emergent Adverse Events Leading to Dose Delayed | . 133 |
| Listing 16.2.7.2.3 Treatment-Emergent Adverse Events Leading to Drug Withdrawn | . 134 |
| Listing 16.2.7.3 Serious Adverse Events | . 135 |
| Listing 16.2.7.4 Patients with Incomplete Adverse Event Information Excluded from Summary Tables | . 136 |
| Listing 16.2.7.5 Death Summary | . 137 |
| Listing 16.2.8.1 Clinical Laboratory Tests - Hematology | . 138 |
| Listing 16.2.8.2 Clinical Laboratory Tests - Blood Chemistry | . 139 |
| Listing 16.2.8.3 Clinical Laboratory Tests - Urinalysis | . 140 |

All rights reserved



| Listing 16.2.9.1 Vital Signs | 141 |
|--------------------------------------------------------------------|-----|
| Listing 16.2.9.2 Physical Examination | 142 |
| Listing 16.2.9.3 Electrocardiogram | 143 |
| Listing 16.2.9.4 ECOG Performance Status | 145 |
| Listing 16.2.9.5 Infusion-Related Reactions | 146 |
| Listing 16.2.9.6 Pain Assessment | 147 |
| Listing 16.2.9.7 Immune Activation Markers - Cytokines Assessment | 148 |
| Listing 16.2.9.8 Immune Activation Markers – Complement Assessment | 149 |
| Listing 16.2.9.9 Anti-Drug Antibody (ADA) Assay | 150 |
| Listing 16.2.9.10 KRAS Mutation Assessment | 151 |
| Listing 16.2.9.11 GSTT1 Genotyping | 152 |
| Listing 16.2.9.12 Exploratory Tumor Biopsy | 153 |
| Listing 16.2.9.13 GSTP mRNA KD Sample | 154 |
| Listing 16.2.9.14 GST Family - GSTP1 mRNA Level | 155 |
| Listing 16.2.9.15 GST Family - GSTT1 mRNA Level | 156 |
| Listing 16.2.9.16 GST Family - MGST3 mRNA Level | 157 |
| Listing 16.2.9.17 GST Family – GSTM3 mRNA Level | 158 |
| Listing 16.2.9.18 Pharmacokinetics Data Collection | 159 |
| Listing 16.2.10.1 Concomitant Measures | 160 |
| Listing 16.2.10.2 Concomitant Measures - Palliative Radiotherapy | 161 |

All rights reserved



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b


Listing 16.2.1.1 Patient Disposition All Enrolled (N=n)

| | Study | NBF-006 Dose | Date of | Day | | ITT | Safety | Efficacy |
|---|---|---|---|---|---|---|---|---|
| Patient/Age/Sex | Part | (mg/kg) | Last Dose | [1] | Reason | [2] | Evaluable [3] | Evaluable [4] |
| ссс-роролог/к | × | XXX | ddmmmyyyy | XXX | Reason | Yes | Yes | Yes |
| ccc-pppp/xx/x | × | XXX | ddmmmyyyy | KKK | Reason | Yes | Yes | Yes |
| rcc-pppp/xx/x | × | XXX | ddmmmyyyy | XXX | Other: Specify | Yes | Yes | Yes |
| ccc-pppp/xx/x | × | XXX | ddmmmyyyy | xxx | Reason | Yes. | Yes | Yes |
| cc-pppp/xx/x | × | XXX | ddmmmyyyy | XXX | Reason | Yes | Yes | Yes |
| x/xx/qqqqq | × | XXX | ddmmmyyyy | XXX | Other: Specify | Yes | Yes | Yes |
| cc-pppp/xx/x | × | xxx | ddmmmyyyy | xxx | Reason | Yes | Yes | Yes |
| ccc-ppppp/xx/x | × | xxx | ddmmmyyyy | xxx | Reason | Yes | Yes | Yes |
| ccc-ppppp/xx/x | × | XXX | ddmmmyyyy | XXX | Other: Specify | Yes. | Yes | Yes |

<sup>[1]</sup> Day is relative to first dose date of NBF-006-001.

#### PROGRAMMER'S NOTES:

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "occ" portion of patient number.

NBF-006-001

Statistical Analysis Plan


All rights reserved

Copyright© 2016 by Theradex Oncology®, Princeton NI

116

<sup>[2]</sup> Intent-to-Treat (ITT) includes all participants who were enrolled (signed consent) into the study, irrespective of whether study medication was administrated or not, [3] Safety Evaluable include all patients who received any component of study treatment.

<sup>[4]</sup> Efficacy Evaluable include patients with measurable disease by RECIST 1.1 who had a baseline assessment and at least one post-baseline assessment. Cross-References: Case Report Form OFF-STUDY SUMMARY (OF)



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b


# Listing 16.2.2.1 Inclusion/Exclusion Criteria All Enrolled (N=n)

| | Study | NBF-006 Dose | | Protocol | | |
|---|---|---|---|---|---|---|
| Patient/Age/Sex | Part | (mg/kg) | Eligibility | Version Date | Category Not Met | Walver Number |
| ссс-рррр/ю/х | × | XXX | Yes | XX | | |
| есс-рррр/ж/х | × | XXX | Yes | XX<br>XX | | |
| ccc-pppp/xx/x | 8 | XXX | No | 100 | Inclusion x | |
| ccc-pppp/xx/x | × | XXX | Yes | XX<br>XX | | |
| ссс-рррр/ж/х | × | XXX | Yes | XX | | |
| ccc-pppp/xx/x | × | XXX | No, but waiver granted | XX | Exclusion x | XXXXXX |
| ccc-pppp/xx/x | × | XXX | Yes | XX<br>XX | | |
| ссс-рррр/ж/ж | × | XXX | Yes | XX | | |
| ссс-ррррллог/х | × | XXX | No | XX | Inclusion x | |
| ccc-ppppp/xx/x | × | XXX | Yes | XX | | |

Cross-References: Case Report Form INCLUSION/EXCLUSION CRITERIA (IE)
PROGRAMMERS NOTES:

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "ccc" portion of patient number.

Copyright© 2016 by Theradex Oncology®, Princeton NI

Statistical Analysis Plan


All rights reserved

117



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/To


Listing 16.2.4.1 Demographics Intent-to-Treat (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006 Dase<br>(mg/kg) | Birth<br>Date | | Ethnicity | Registration<br>Date | ICF<br>Date | ICF Signature<br>Date | Protocol<br>Amend # | | Withdraw Content<br>from Main Study | Withdraw Content<br>for Biopsies | Date |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ccc-papps/w/x | × | xxx | XXX | × | XXX | ddmmmyyyy | xxx | XXX | × | ddmmmyyyy | Yes | XXX | XXX |
| x/xx/qqqqqxxx/x | x | XXX | XXX | × | XXX | üdmmmyyyy | XXX | xxx | × | ddmmmyyyy | No | XXX | жж |
| x/xx/qqqqq-xxx | X | xxx | XXX | × | XXX | ddmmmyyyy | | | × | ddmmmyyyy | No | 3000 | 3000 |
| ссс-рарруххух | x | xxx | XXX | × | XXX | ddmmmyyyy | XXX | XXX | × | ddmmmyyyy | Yes | XXX | XXX |
| ссе-пррружж/х | x | XXX | XXX | × | XXX | ddmmmyyyy | XXX | xxx | × | ddmmmyyyy | No | XXX | XXX |
| x/xx/qqqqq-333 | × | XXX. | XXX | × | XXX | ddmmmyyyy | XXX | XXX | × | ddmmmyyyy | No | 2003 | XXX |

[1]Race; A-Asian, W-White, B-Black or African American, N-Native Hawalian or Pacific Islander, I- American Indian or Alaska native, NR-Not Reported, O-Other Cross-References: Case Report Form DEMOGRAPHICS (DM), Informed Consent (IC)

PROGRAMMER'S NOTES:

Data will be presented in mixed case for formatted variables and upper case only for uniformatted variables. Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number.

118




DIRECTORY/FILE.SAS NBF-006-001 Phase 1/Tb

# Listing 16.2.4.2.1 Disease Related Characteristics intent-to-Treat (N=n)

FINAL- ddmmmyychh:mm


| Patient<br>/Age/Sex | Study<br>Part | NBF-006 Dose<br>(mg/kg) | Primary Site<br>(Site Class) | Initial Diagnosis<br>Date | Day<br>[1] | Duration of<br>Disease (m) [2] | Histology<br>[3] | Disease<br>Stage | EGFR<br>Mutation | ALK/ROS1<br>Gene Fusion | KRAS Genotype<br>Mutated |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ες-ρορο/κυ/κ | × | XXX | Site (Class) | ddmmmyyy | XXXX | XXX.X | XXXX | XXXX | Yes, specify | Yes | Yes |
| cc-ppppp/xx/x | × | XXX | Site (Class) | ddmmmyyyy | XXXX | KKKKK | XXXX | XXXX | No | No | No |
| cc-ppppp/xx/x | × | XXX | Site (Class) | ddmmmyyyy | 8XXX | XXX.X | 30000 | XXXX | No | No | Unknown |
| сс-раррухх/х | × | XXX | Site (Class) | ddmmmyyyy | XXXX | XXXX | XXXX | XXXX | Yes, specify | Yes | Yes |
| сс-рррружж/х | × | XXX | Site (Class) | ddmmmyyyy | XXXX | XXXX | Other | XXXX | No | Unknown | No |
| cc-ppppp/xx/x | × | xxx. | Site (Class) | ddmmmyyyy | XXXX | xxx.x | XXXX | XXXX | Unknown | No | No |

[1] Days to first dose date.

[2] Duration of Disease+ (Date ICF signed - Initial Diagnosis Date) in month

[3] ICO- version xxx

Cross-References: Case Report Form DEMOGRAPHICS (DM)

PROGRAMMER'S NOTES:

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "cor" portion of patient number.

Statistical Analysis Plan


Copyright© 2016 by Theradex Oncology®, Princeton NI

All rights reserved

119



DIRECTORY/FILE.SAS FINAL- ddmmmyychh:mm NBF-006-001 Phase 1/Tb Page 1 of x

# Listing 16,2.4.2.2 Baseline KRAS Mutation Assessment Intent-to-Freat (N=n)

| Patient | Study | NBF-006<br>Dose | Assessment | Genomic<br>Turnor<br>Profile | Date of | Archived Tissue | Sample | Fresh<br>Sample | Sample | Biopsy | If nat, | KRAS<br>Mutation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (reg/kg) | Completed? | | Analysis | Sample<br>Obtained? | Date | Required | Date | Performed? | Reason | |
| εςς-<br>αρορ/xx/x | × | xxx | | Yes | ddrnmmyyyy | Yes | ddrnmmyyyy | Yes | ddmmmyyyy | Yes | | XXXX |
| ccc-<br>pppp/xx/x | × | XXX | | Yes | ddminimyyyy | Yes | dd:mmmyyyy | Yes | ddmmmyyyy | Yes | | жжж |
| | | | Yes | Yes | ddmmmyyyy | Ves . | ddmmmyyyy | Yes | ddmmmyyyy | Yes | | XXXXXX |
| cc-<br>pppp/xx/x | × | xxx | Yes | Yes | ddmmmyyyy | Yes | ddrnmmyyyy | No | | | | XXXXX |
| | | | Yes | Yes | ddmmmyyyy | Yes | ddmmmyyyy | No | | | | XXXXXX |
| ccc-<br>apap/xx/x | × | xxx | No | No | 9333 | Yes | ddmmmyyyy | Yes | ddmmmyyyy | Yes | | |
| cc-<br>pppp/xx/x | X | XXX | Yes | Yes | ddmmmyyyy | Ves | ddmmmyyyy | Yes | ddmmmyyyy | Yes | | XXXXX |
| CASH CANA | | | Yes | Yes | ddmmmyyyy | Yes | ddrnmmyyyy | Yes | ddmininyyyy | Yes | | 300000 |
| | | | Yes | Yes | ddmmmyyyy | Yes | ddmmmyyyy | Yes | ddmmmyyyy | Yes | | XXXXXX |
| ccc-<br>pppp/xx/x | × | XXX | Yes | Yes | ddmmmyyyy | Yes | ddmmmyyyy | Yes. | ddmmmyyyy | No | XXXXXX | 300000 |

Cross-References: Case Report Form KRAS MUTATION ASSESSMENT (TM5)
PROGRAMMER'S NOTES:
Sort "Patient" in ascending order using "papp", and then "ccc" portion of patient number.

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NT All rights reserved

Statistical Analysis Plan 120




DIRECTORY/FILE.SAS NBF-006-001 Phase 1/To


Listing 16.2.4.3 Medical History Intent-to-Treat (N=n)

| Patient | Study | NBF-006 Dose | Start | Study | Condition<br>(Preferred Term) | | | Related to | Therapy |
|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Date | Day [1] | (System Organ Class) [2] | Ongoing | Grade | Study Disease | Given |
| ecc-pppp<br>/xx/x | × | KXX | ddmrnmyyyy | -XX | Condition<br>(MedDRA Preferred Term)<br>(MedDRA System Organ Class) | No | Mild | No | Np |
| | | | | | Condition<br>(MedDRA Preferred Term)<br>(MedDRA System Organ Class) | No | Moderate | No | Yes |
| xxxx<br>fxx/x | × | XXX | ddmirenyyyy | -xx | Condition<br>(MedDRA Preferred Term)<br>(MedDRA System Organ Class) | Yes | Mild | No | No |

<sup>[1]</sup> Day is relative to the first dose date of NBF-006 or ongoing.

Grade: 1=Mild, 2=Moderate, 3=Severe, Unknown, and Not Applicable.

Data will be presented in mixed case for formatted variables and upper case only for uniformatted variables. Sort "Patient" in ascending order using "papp", and then "ccc" portion of patient number.

NBF-006-001

Statistical Analysis Plan


All rights reserved

Copyright© 2016 by Theradex Oncology®, Princeton NI

121

<sup>(2)</sup> MedDRA version 21.1

Cross-References: Case Report Form MEDICAL HISTORY (MH)
PROGRAMMER'S NOTES:



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b

FINAL- ddmmmyychbcmm Page 1 of x

#### Listing 16.2.4.4 Prior Cancer Therapy Intent-to-Treat (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006 Dase<br>(mg/kg) | Regimen<br>Number | Agent/Treatment | Therapy<br>Type | Start<br>Date | Stop<br>Date | Stop<br>Day [1] | Reason | Best<br>Response |
|---|---|---|---|---|---|---|---|---|---|---|
| ccc-ppppp/xx/x | × | XXX | × | Prior Therapy Name | Type | ddmmmyyyy | ddmmmyyyy | -xx | XXX | Response |
| cc-pppp/xx/x | * | KKK | × | Prior Therapy Name | Type | ddmmmyyyy | dammmyyyy | -xx | 3000 | Response |
| - FREE | | | × | Prior Therapy Name | Type | ddrnmmyyyy | ddmmmyyyy | -xx | 300X | Response |
| cc-ppppp/xx/x | × | XXX | × | Prior Therapy Name | Type | ddmmmyyyy | ddmmrryyyy | -xx | XXX | Response |
| Series Series | | | × | Prior Therapy Name | Type | ddmmmyyyy | 0.0000000000000000000000000000000000000 | | | A COMMITTEE STATE |
| cc-pppp/xx/x | × | XXX | × | NO PRIOR THERAPY | | | | | | |
| сс-раррухх/х | × | XXX | × | Prior Therapy Name | Type | ddmmmyyyy | ddmmmyyyy | -xx | XXX | Response |
| Section Section 1 | | | × | Prior Therapy Name | Type | ddmmmyyyy | ddmmmyyyy | -xx | 3000 | Response |
| | | | × | Prior Therapy Name | Type | ddmmmyyyy | ddmmrryyyy | -xx | 300X | Response |
| сс-раррухх/х | × | XXX | * | Prior Therapy Name | Type | ddmmmyyyy | ddmmmyyyy | -xx | 3000 | Response |

[1] Stop day is relative to the first dose date of NBF-006 or ongoing. Cross-References: Case Report Form PRIOR CANCER THERAPY (PT) PROGRAMMERS NOTES:

PROCHAMMERS NOTES:

Prior Therapy Type includes: Chemotherapy, Hormonal Therapy, Immunotherapy, and Other.

Best Response includes: Complete Response, Partial Response, Statue Disease, Progressive Disease, Unknown, and Not Applicable.

When "No Prior Therapy" is indicated, enter "NO PRIOR THERAPY" in the "Agent/Treatment" column.

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "popp", and then "coc" portion of patient number.

Sort "Start Date" in ascending order within "Patient".

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan

122




DIRECTORY/FILE.SAS NBF-006-001 Phase 1/To


Listing 16.2.4.5 Prior Medications Intent-to-Treat (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006 Dose<br>(mg/kg) | Agent/Treatment | Start<br>Date | Stop<br>Date | Stop<br>Day [1] | Time | Dose | Unit | Route | Other |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ccc-ppppp/xx/x | × | xxx | Prior Therapy Name | ddmmmyyyy | ddmmmyyy | -000 | hhomm | 500X | 2000 | xxx | |
| есе-раррухх/х | * | XXX | Prior Therapy Name | ddmmmyyyy | ddmmmyyyy | *XX | bhanm. | XXX | 300X | XXX | |
| | | | Prior Therapy Name | ddmmmyyyy | ddmmmyyyy | -XX | hhomm | XXX | X000 | 300X | |
| cc-ppppy/xx/x | × | xxx | Prior Therapy Name | ddmmmyyyy | ddmmmyyyy | -3000 | hhamm | 500,X | 2000 | XXX | |
| | | | Prior Therapy Name | ddmmmyyyy | ddmmmyyyy | -XX | bhamm. | XXX | 3000 | Other | XXX |
| сс-равру/хх/х | × | xxx | NO PRIOR THERAPY | | | | | | | | |
| ссс-рарруххух | × | xxx | Prior Therapy Name | ddmm/nyyyy | ddmmmyyyy | -800 | hhamm | 300X | 2000 | XXX. | |
| | | | Prior Therapy Name | ddmmmyyyy | ddmmmyyyy | -90% | bhamm | xxx | 3000 | 3000 | |
| | | | Prior Therapy Name | ddmmmyyyy | ddmmmyyyy | -XX | hhamm | XXX | 2000 | 3000 | |
| ссе-раррухх/х | × | xxx | Prior Therapy Name | ddmmmyyyy | ddmmmyyyy | -XX | hhamm | 50CX | 2000 | XXX | |

[1] Stop day is relative to the first dose date of NBF-006 or ongoing,

Cross-References: Case Report Form PRIOR MEDICATIONS (PM)

PROGRAMMER'S NOTES:
Prior Therapy Type includes: Chemotherapy, Hormonal Therapy, Immunotherapy, and Other.

Best Response includes: Complete Response, Partial Response, Stable Disease, Progressive Disease, Unknown, and Not Applicable.

When "No Prior Therapy" is indicated, enter "NO PRIOR THERAPY" in the 'Agent/Treatment' column.

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "popps", and then "coc" portion of patient number.

Sort "Start Date" in ascending order within "Patient",

Copyright© 2016 by Theradex Oncology®, Princeton NI

Statistical Analysis Plan


All rights reserved

123



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b

FINAL- ddmmmiyythh;mm Page 1 of x

#### Listing 16.2.4.6 Prior Cancer Radiation Intent-to-Treat (N=n)

| | Study | NBF-006 Dose | | Start | Stop | Stop | Best |
|---|---|---|---|---|---|---|---|
| Patient/Age/Sex | Part | (mg/kg) | Site | Date | Date | Day [1] | Response |
| есс-арара/жу/х | × | xxx | NO PRIOR RADIATION | | | | |
| ccc-ppgp/xx/x | × | XXX | Reported Site | ddmmmyyyy | ddmmrryyyy | -xx | XXX |
| ccc-pppp/xx/x | × | XXX | Reported Site | ddmmmyyyy | ddmmrryyyy | -830 | XXX |
| εεε-αμαρ/χι/χ | × | XXX | Reported Site | ddmmmyyyy | ddmmrryyyy | *XX | XXX |
| ccc-popp/xx/x | × | XXX | Reported Site | ddmmmyyyy | ddmmrryyyy | -xx | XXX |
| ссс-рарар/ж/х | × | XXX | Reported Site | ddmmmyyyy | ddmmrryyyy | -836 | XXX |
| ссс-рара/хх/х | × | XXX | Reported Site | ddmmmyyyy | ddmmrryyyy | -xx | XXX |
| ccc-poop/xx/x | × | XXX | Reported Site | ddmmmyyyy | ddmmrryyyy | -xx | XXX |

[1] Stop day is relative to the first dose of NBF-006 or orgoing. Cross-References: Case Report Form PRIOR CANCER RADIATION (PR) ROGRAMMER'S NOTES:

When "No Prior Radiation" is indicated, enter "NO PRIOR RADIATION" in the "Site" column.

Best Response includes: Complete Response, Partial Response, Stable Disease, Progressive Disease, Unknown, and Not Applicable
Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Papent" in ascending order using "pppp", and then "ccc" portion of patient number.

Sort "Start Date" in ascending order within "Patient".

Statistical Analysis Plan


All rights reserved

Copyright© 2016 by Theradex Oncology®, Princeton NI

124



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b


Listing 16.2.4.7 Prior Cancer Surgeries Intent-to-Treat (N=n)

| Patient/Age/Sex | Study<br>Part | NBF-006 Dose<br>(mg/kg) | Procedure<br>(including ste) | Procedure<br>Date | Study Day<br>[1] | Findings (Pathology/Cytology) |
|---|---|---|---|---|---|---|
| The state of the s | | | *************************************** | | 717/02/1 | |
| ccc-ppppp/xx/x | - 14 | XXX | Procedure and Site | ddmmmyyyy | -xx | Description of Findings |
| | | | Procedure and Site | ddmmmyyyy | *XX | Description of Findings |
| есс-рррр/ж/х | - X | XXX | Procedure and Site | ddmmmyyyy | -xx | Description of Findings |
| | | | Procedure and Site | ddmmmyyyy | -xx | Description of Findings |
| | | | Procedure and Site | ddmmmyyyy | -XX | Description of Findings |
| сес-рррр/ж/х | × . | XXX | Procedure and Site | ddmmmyyyy | ·xx | Description of Findings |
| 200 44 (400) | | | Procedure and Site | ddmmmyyyy | -xx | Description of Findings |
| | | | Procedure and Site | ddmmmyyyy | -xx | Description of Findings |
| εεε-ρρημ/χν/χ | × | XXX | Procedure and Site | ddmmmyyyy | -xx | Description of Findings |
| Sec. Colonial Sec. | | | Procedure and Site | ddmmmyyyy | -xx | Description of Findings |

[1] Day is relative to the first dose date of NBF-006. Cross-References: Case Report Form PRIOR CANCER SURGERIES (SG)

### PROGRAMMER'S NOTES:

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

125

Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number. Sort "Procedure Date" in ascending order within "Patient".

Statistical Analysis Plan Copyright© 2016 by Theradex Oncology®, Princeton NI

All rights reserved




DIRECTORY/FILE.SAS NBF-006-001 Phase 1/To


Listing 16.2.4.8 Pregnancy Test Intent-to-Treat (N=n)

| Patient/Age/Sex | Study | NBF-006 Dose | | | Study Day | | | |
|---|---|---|---|---|---|---|---|---|
| | Part | (rrg/kg) | Visit | Date | [1] | Method | Result | Reason Not Done |
| ccc-pppp/xx/x | × | XXX | XXX | ddmmmyyyy | -xx | Urine | Negative | |
| | | | 300X | ddmmmyyyy | -XX<br>XX | Serum | Negative | |
| | | | 2000 | ddmmmyyyy | XX | Serum | Negative | |
| ccc-pppp/xx/x | × | XXX | 2000 | ddmmmyyyy | -xx | Serum | Negative | |
| | | | 300X | ddmmmyyyy | XX | Urine | Negative | |
| | | | XXX | ddmmmyyyy | 300 | Urine | Negative | |
| ccc-pppp/xx/x | × | XXX | XXX | ddmmmyyyy | -xx | Urine | Negative | |
| 131101 | | | XXXX | NOT PERFORMED. | | | | Post-Menopausal |
| | | | XXX | ddmmrryyyy | *** | Urine | Negative | |

<sup>[1]</sup> Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Form PRECNANCY (RP)
PROGRAMMER'S NOTES:

If Pregnancy Test is not performed, enter "NOT PERFORMED" in the "Sample Date" column.

Data will be presented in mixed case for formatted variables and upper case only for uniformatted variables.

Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number.

Statistical Analysis Plan


All rights reserved

Copyright© 2016 by Theradex Oncology®, Princeton NI

126



NBF-006-001 Phase 1/1b

#### DIRECTORY/FILE.SAS

FINAL- ddmmmyychhoron Page 1 of x

#### Listing 16.2.5.1 NBF-006 Administration Safety Evaluable (N=n)

| Patient<br>/Age/Sex | Study<br>Part | Visit | Start<br>Date | Day<br>[1] | Start<br>Time | Stop<br>Time | Dose Level<br>(mg/kg) | | Total infused<br>Dose (mg) | Infusion<br>Rate | Dose<br>Delay[2] | Reason | Dose<br>Interrupted[3] | Reason | AE<br># |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ccc-pppp | × | XX | ddmmmyyyy | XX | hhaman | hhamm | xxx | × | DOOK | XXX | Yes | XXX | No | | |
| | | | ddmmmyyyy | XX | hh:mm | hhamm | 300K | × | 3000 | XXX | No | XXX | No | | |
| /xx/x | | | ddmmmyyyy | XX | hh:mm | hhamm | XXX | × | pox | KXX. | No | | Ves | xxx | XX |
| | | XX: | ddmmmyyyy | XX. | hhann | hhamm | 300X | × | 300X | XXX | No | | No | | |
| | | | ddmmmyyyy | XX | hhimm | hhamm | XXX | × | 3000 | | No | | No | | |
| | | | ddmmmyyyy | XX. | hhamm | hhamin | XXX | × | DOOK | хжк | Yes | XXX | No | | |
| ссс-роро | × | xx | ddmmmyyyy | XX | hhamm | hhamm | XXX | | 3000 | XXX | No | | No | | |
| /xx/x | | | ddmmmyyyy | XX | hh;mm | hhomm | 100X | × | 3000 | XXX | No | | No | | |
| | | 300 | ddmmmyyyy | XX | hh:mm | hhamm | 3000 | × | 3000 | XXX | No | | Yes | XXX | XX |

[1] Day is relative to first dose date of NBF-006. [2] Dose is not administrated on protocol scheduled timepoint.

[3] The infusion is temporarily interrupted and then resumed when symptoms are resolved. Cross-Reference: Case Report Form NBF-006 ADMINISTRATION (EX) PROGRAMMERS NOTES:

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "ccc" portion of patient number.

Sort "Start Date" in ascending order within "Patient", specify other,

There are 3 infusion rates, each subject may have 3 rows for 3 infusion rates.

The infusion will be implemented as a stepwise infusion:

- (1) 0.5 mL/min for 10 minutes.
- (2) then 1.5 mi/min for 10 minutes, and
- (3) finally 6 mL/min for the remaining volume

Statistical Analysis Plan


Copyright© 2016 by Theradex Oncology®, Princeton NI

All rights reserved

127



NBF-006-001 Phase 1/1b DIRECTORY/FILE.SAS FINAL- ddmmmyy;hh;mm

#### Listing 16.2.6.1 Extent of Disease: Target and Non-Target Lesions Efficacy Evaluable (Nan)

| Patient | Study | y NBF-006 Dose | | Date of | Day | Lesion | Lesian | Organ | | Previous RT | Progression |
|---|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Procedure | [1] | Туре | Number | (Other, specify) | Procedure | to Lesion | Since RT |
| ссс-рррр | × | 30KX | Screening | ddmmmyyyy | -XX | Target | x | Other: Specify | X-Ray | | |
| xx/x | | | | | | Target | × | Reported Organi | Other: Specify | Yes | Yes |
| | | | | | | Target | × | Reported Organ | PET/CT | | |
| | | | | | | Non-Target | × | Reported Organ | Other: Specify | | |
| | | | XXX | ddmmmyyyy | XX. | Target | × | Reported Organ | X-Ray | | |
| | | | | | | Target | × | Reported Organ | Other: Specify | | |
| | | | | | | Target | × | Reported Organ | CT Scan | | |
| | | | | | | Non-Target | × | Reported Organ | Other: Specify | | |
| | | | | | | Non-Target | × | Reported Organ | CT Scan | | |
| | | | | | | Non-Target | × | Reported Organ | X-Ray | | |
| ccc-pppp | | жж | XXX | ddmmmyyyy | хх | Target | × | Reported Organ | CT Scan | | |

[1] Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Forms TARGET LESIONS ASSESSMENT (TR1, TR2), NON-TARGET LESIONS ASSESSMENT (TR3, TR4), NEW LESIONS (TR5)

PAGGRAMMER'S NOTES:
When "No Target Lesions at Pretreatment", enter "NO TARGET LESIONS' in the "Lesion Type" column.

When "No Non-Target Lesions at Pretreatment", enter "NO NON-TARGET LESIONS' in the 'Lesion Type' column.

Data is presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "popp", and then "ccc" portions of patient number. Sort "Date" in ascending order within "Patient".

Sort "Lesion Type" in descending order within "Date". Sort "Lesion Number" in ascending order within "Lesion Type".

NBF-006-001 Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan 128




NBF-006-001 Phase 1/1b DIRECTORY/FILE.SAS FINAL- ddmmmyythbmm Page 1 of x

#### Listing 16.2.6.1 Extent of Disease: Target and Non-Target Lesions Efficacy Evaluable (N=n)

| Patient<br>/Age/Sex | | NBF-006 Dose<br>(mg/kg) | Visit | Date of<br>Procedure | | Lesion<br>Type | Lesion<br>Number | Anatomical Location | Lesion Assessable/<br>Non-Target Lesion Evaluation | RECIST<br>Measure (mm) | Total<br>Sum (mm) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ccc-pppp | x | xxx | Streening | ddrimmyyyy | -300 | Target | x | Reported Location | Yes | xx<br>xx | |
| /xxx/x | | | VI 1800 P. C. 1800 | | | Target | | Reported Location | Yes | XX | |
| | | | | | | Target. | x | Reported Location | Yes | xx | 3000 |
| | | | | | | Non-Target | × | Reported Location | | | |
| | | | | | | Non-Target | x | Reported Location | | | |
| | | | KKK: | ddmmmyyyy | XX. | Target | × | Reported Location | Yes | XX | |
| | | | | | | Target | x<br>x<br>x | Reported Location | Yes | XX | |
| | | | | | | Target | x | Reported Location | Yes | xx<br>xx | XXX |
| | | | | | | Non-Target | × | Reported Location | | | |
| | | | | | | Non-Target | x | Reported Location | | | |
| | | | | | | NewLesion | × | Reported Location | | | |
| ccc-pppp | | xxx | XXX | ddmmmyyyy | хх | Target | × | Reported Location | Yes | xx | |

[1] Day is relative to the first dose date of NBF-006.

(1) Day's rearise to the first observation of North Construction (TR3, TR4), NEW LESIONS ASSESSMENT (TR3, TR4), NEW LESIONS (TR5) PROGRAMMER'S NOTES:

When "No Target Lesions at Pretreatment", enter "NO TARGET LESIONS' in the "Lesion Type" column.

When "No Non-Target Lesions at Pretreatment", enter "NO NON-TARGET LESIONS' in the "Lesion Type" column.

Data is presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "popp", and then "ccc" portions of patient number. Sort "Date" in ascending order within "Patient".

Sort "Lesion Type" in descending order within "Date".

Sort "Lesion Number" in ascending order within "Lesion Type",

Copyright© 2016 by Theradex Oncology®, Princeton NI

Statistical Analysis Plan 129


All rights reserved



NBF-006-001 Phase 1/Tb

#### DIRECTORY/FILE.SAS


#### Listing 16.2.6.2 Cycle Response Assessment Efficacy Evaluable (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-806 Dose<br>(mg/kg) | Visit | Date of<br>Procedure | 1000 | Target Lesion<br>Response | Non-Target<br>Lesion<br>Response | New<br>Lesions | Symptomatic<br>Deterioration | Deterioration<br>Date | Overall<br>Response<br>for this Cycle |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ссс-рарр | x | XXX | XXX | ddammyyyy | XX | Stable Disease | NON-CR/NON-PD | No | | | Stable Disease |
| | | | XXX | ddmmmyyyy | XX. | Stable Disease | NON-CR/NON-PD | No | | | Stable Disease |
| | | | XXX | ddmmmyyyy | XX | Complete Response | Complete Response | No | | | Complete Response |
| | | | XXX | ddmmmyyyy | XX | Complete Response | Complete Response | No | | | Complete Response |
| сс-рррр | × | XXX | XXX | ddmmmyyyy | XX | Stable Disease | NON-CR/NON-PD | No | | | Stable Disease |
| | | | XXX | ddmmmyyyy | XX | Stable Disease | NON-CRANON-PO | No | Yes | ddmmmyyyy | Stable Disease |
| | | | XXX | ddmmmyyyy | XX | Complete Response | Complete Response | No | | | Complete Response |
| | | | XXX | ddmmmyyyy | XX. | Complete Response | Complete Response | No | | | Complete Response |
| сс-рррр | X | XXX | XXX | ddmmmyyyy | XX | Stable Disease | NON-CR/NON-PD | No | | | Stable Disease |
| xx/x | | | XXX | ddmmmyyyy | XX | Stable Disease | NON-CR/NON-PD | No | | | Stable Disease |
| | | | XXX | ddmmmyyy | xx | Progression | Progression | No | | | Progression |

<sup>[1]</sup> Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Form CYCLE RESPONSE ASSESSMENT (RS)
PROGRAMMER'S NOTES:

Data is presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "popp", and then "ccc" portions of patient number.

130




DIRECTORY/FILE.SAS NBF-006-001 Phase 1/1b

Listing 16.2.7.1 Adverse Events Safety Evaluable (N=n) FINAL- ddmmmyythbmm Page 1 of x

| | Carch (90) | World Industry | Adverse Event | naned | Onset | V. 2000 | | .00 | 004 | 1470-2 | TeXVI A L | A74.3 m | Aftern | late Cause |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>/Age/Sex | Study<br>Part | NBF-006<br>Dose (rng/kg) | (MedDRA Preferred Term)<br>(MedDRA System Organ Class) | DLT<br>[1] | Resolved<br>Dates | Day<br>[2] | Grade | Ser<br>[3] | Drug<br>Related | | Therapy<br>Given | Out<br>[5] | Primary<br>Disease | Comment |
| ccc-pppp<br>/xx/x | x | XXX | ADVERSE EVENT<br>(MedDRA Preferred Term)<br>(MedDRA System Organ Class) | | ddmmmyyyy<br>ddmmmyyyy | ж | Mid | × | probably | 1 | Yes | * | | |
| | | | ADVERSE EVENT<br>(MedDRA Preferred Term)<br>(MedDRA System Organ Class) | | ddmmmyyyy<br>engoing | ж | Mid | × | Unlikely | 3 | Yes | × | Yes | XXXXXX |
| ccc-pppp<br>/xx/x | × | xxx | ADVERSE EVENT<br>(MedDRA Preferred Term)<br>(MedDRA System Organ Class) | Yes | ddmmmyyyy | ж | Severe | | Unrelated | 2 | No | × | Yes | NXXXXX |

### MedDRA version 21.1

- [1] DLT= Dose Limiting Taxicity
- [Z] Day is relative to the first dose date of NBF-006.
- [3] Ser-Serious: 1=Not Serious, 2=Results in Death, 3=Life Threatening, 4=Requires or Prolongs Hospitalization, 5=Persistent or Significant Disability/Incapacity, 6=Congenital Anomaly or Birth Defect, 7=Other Medically Important Serious Eyent.
- [4] Act-Action Taken: 1-Dose NOT Changed, 2-Dose Interrupted, 3- Dose Delayed, 4- Drug Withdrawn.
- [5] Out-Outcome: 1-Recovered/Resolved, 2-Recovered/Resolved with sequelae, 3-Recovering/Resolving, 4-Not Recovered/Not Resolved, 5-Fatal, 6-Unknown,
- **DLT= Dose Limiting Toxicity**
- Cross-References: Case Report Form ADVERSE EVENTS (AE)

#### PROGRAMMER'S NOTES:

- Grade: 1-Mild, 2-Moderate, 3-Severe, 4-Life threatening, 5-Fatal, Use maximum grade for summary. Data will be presented in mixed case for formatted variables and upper case only for unformatted variables. Sort "Patient" in ascending order using "pppp", and then "ccc" portion of patient number. Sort "Onset Date" in ascending order within "Patient".

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan 131




NBF-006-001 Phase 1/1b DIRECTORY/FILE.SAS FINAL- ddmmmyychh:mm Page 1 of x

### Listing 16.2.7.2.1

#### Treatment-Emergent Adverse Events Leading to Dose Interrupted Safety Evaluable (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006<br>Dase(mg/kg) | Adverse Event<br>(MedDRA Preferred Term) | Day<br>[1] | Last Dose<br>to Onset[2] | Treatment<br>Duration [3] | Duration of TEAE (day) | Grade | Senous<br>[5] | Drug<br>Related |
|---|---|---|---|---|---|---|---|---|---|---|
| ecc-pppp | × | xxx | Adverse Event<br>(MedDRA Preferred Term) | XX | xxx | XXX | xxx | Mild | Na | Possible |
| ecc-pppp | × | xxx | Adverse Event<br>(MedDRA Preferred Term) | XX | XXX | XXX | 2003. | Severe | Yes | Unrelated |

[1] Day is relative to the first dose date of NBF-006.

[2] Last Dose to Onset is calculated in days.

[3] Treatment Duration is calculated from first dose to discontinuation of study drug.

[4] Duration of adverse event is calculated in days from Onset Date to Resolution Date.
[5] Ser-Serious:1=Not Serious, 2=Results in Death, 3=Life Threatening, 4=Requires or Prolongs Hospitalization, 5=Persistent or Significant Disability/Incapacity, 6=Congenital Anomaly or Birth Defect, 7=Other Medically Important Serious Event.

Cross-References: Case Report Form ADVERSE EVENTS (AE)
PROGRAMMER'S NOTES;

Sort "Patient" in ascending order using "pppp", and then "ccc" portion of patient number.

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan


132



NBF-006-001 Phase 1/1b DIRECTORY/FILE.SAS FINAL- ddmmmyychh:mm Page 1 of x

## Listing 16.2.7.2.2

#### Treatment-Emergent Adverse Events Leading to Dose Delayed Safety Evaluable (N=n)

| Patient<br>/Age/Sex | Study<br>Parl | NBF-006<br>Dase(mg/kg) | Adverse Event<br>(MedDRA Preferred Term) | Day<br>[1] | Last Dose<br>to Onset[2] | Treatment<br>Duration [3] | Duration of TEAE (day) | Grade | Serious<br>[5] | Drug<br>Related |
|---|---|---|---|---|---|---|---|---|---|---|
| ccc-pppp | × | xxx | Adverse Event<br>(MedDRA Preferred Term) | XX | XXX | жж | xxx | Mild | No | Possible |
| ccc-pppp<br>/xx/x | × | xxx | Adverse Event<br>(MedDRA Preferred Term) | XX | XXX | жж | 3000 | Severe | Yes | Unrelated |

[1] Day is relative to the first dose date of NBF-006.

[2] Last Dose to Onset is calculated in days.

[3] Treatment Duration is calculated from first dose to discontinuation of study drug.

[4] Duration of adverse event is calculated in days from Onset Date to Resolution Date.
[5] Ser-Serious:1=Not Serious, 2=Results in Death, 3=Life Threatening, 4=Requires or Prolongs Hospitalization, 5=Persistent or Significant Disability/incapacity, 6=Congenital Anomaly or Birth Defect, 7=Other Medically Important Serious Event.

Cross-References: Case Report Form ADVERSE EVENTS (AE)
PROGRAMMER'S NOTES;

Sort "Patient" in ascending order using "pppp", and then "ccc" portion of patient number.

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan




NBF-006-001 Phase 1/1b DIRECTORY/FILE.SAS FINAL- ddmmmyychh:mm Page 1 of x

### Listing 16.2.7.2.3

#### Treatment-Emergent Adverse Events Leading to Drug Withdrawn Safety Evaluable (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006<br>Dose(mg/kg) | Adverse Event<br>(MedDRA Preferred Term) | Day<br>[1] | Last Dose<br>to Onset[2] | Treatment<br>Duration [3] | Duration of TEAE (day) | Grade | Senous<br>[5] | Drug<br>Related |
|---|---|---|---|---|---|---|---|---|---|---|
| ссс-рррр<br>/хж/х | × | xxx | Adverse Event<br>(MedDRA Preferred Term) | XX | XXX | жж | xxx | Mild | Na | Possible |
| ccc-pppp | × | xxx | Adverse Event<br>(MedDRA Preferred Term) | XX | XXX | жж | 2003. | Severe | Yes | Unrelated |

[1] Day is relative to the first dose date of NBF-006.

[2] Last Dose to Onset is calculated in days.

[3] Treatment Duration is calculated from first dose to discontinuation of study drug.

[4] Duration of adverse event is calculated in days from Onset Date to Resolution Date.
[5] Ser-Serious:1=Not Serious, 2=Results in Death, 3=Life Threatening, 4=Requires or Prolongs Hospitalization, 5=Persistent or Significant Disability/Incapacity, 6=Congenital Anomaly or Birth Defect, 7=Other Medically Important Serious Event.

Cross-References: Case Report Form ADVERSE EVENTS (AE)
PROGRAMMER'S NOTES;

Sort "Patient" in ascending order using "pppp", and then "ccc" portion of patient number.

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan


134



NBF-006-001 Phase 1/Tb

#### DIRECTORY/FILE.SAS


Listing 16.2.7.3 Serious Adverse Events Safety Evaluable (N=n)

| | | NBF-006 SAE | | | Onset | Hospitalized | THE STATE OF | -0.0 | | 1-5-5 | 1 1 2 2 1 1 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>/Age/Sex | 100000 | Dase<br>(rig/kg) | | Previously<br>Reported | | <br>Admission<br>Discharge<br>Date | Drate Met SAE<br>Criteria | Rechallenge | Study Drug<br>Administrated? | Off-Treatment<br>Prior to SAE? | Patient<br>Withdrawn |
| cc-pppp | × | жж | SAE<br>(PT) | No | ddrammyyyy<br>ddrammyyyy | ddmmmyyyy | ddmmmyyyy | Yes | Yes | × | Yes |
| cc-pppp | × | XXX | SAE<br>(PT) | Yes | ddrnmmyyyy<br>ddrnmmyyyy | ddmmmyyyy | ddmmmyyyy | NA | No | x | No |

[1] MedDRA version 21.1

[2] Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Form SERIOUS ADVERSE EVENTS (SAE)

### PROGRAMMER'S NOTES:

Data will be presented in inixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number.

Sort "Onset Date" in ascending order within "Patient".

Statistical Analysis Plan 135


Copyright© 2016 by Theradex Oncology®, Princeton NT All rights reserved



DIRECTORY/FILE.SAS NBF-006-001 Phase 1/To

#### FINAL- ddmmmyychhomm Page 1 of x

#### Listing 16.2.7.4

#### Patients with Incomplete Adverse Event Information Excluded from Summary Tables Safety Evaluable (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006<br>Dose(mg/kg) | Adverse Event | Oriset | | Grade | Ser<br>[4] | Drug<br>Related | Act<br>[5] | Therapy<br>Given | Out<br>[6] | Alternate Cause | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | (MedDRA Preferred Term) DLT<br>(MedDRA System Organ [2]<br>Class) [1] | Resolved<br>Dates | Day<br>[3] | | | | | | | Primary<br>Disease | Comment |
| ccc-pppp<br>/xx/x | x | XXX | ADVERSE EVENT<br>(MedDRA Preferred Term)<br>(MedDRA System Organ<br>Class) | ddmmmyyyy<br>ddmmmyyyy | xx<br>xx | Mild | X | probably | 1 | Yes | × | | |
| | | | ADVERSE EVENT<br>(MedDRA Preferred Term)<br>(MedDRA System Organ<br>Class) | ddmmmyyyy<br>ongoing | xx | Mild | x | Unlikely | 3 2 | Yes | × | Yes | XXXXXX |
| ссс-рррр<br>/хж/х | х | XX | ADVERSE EVENT Yes<br>(MedDRA Preferred Term)<br>(MedDRA System Organ<br>Class) | ddmmmyyyy<br>ddmmmyyyy | xx<br>xx | Severe | | Unrelated | 1 | No | × | Yes | 3000000 |

<sup>[1]</sup> MedDRA version 21.1

#### Cross-References: Case Report Form ADVERSE EVENTS (AE)

#### PROGRAMMER'S NOTES:

Grade: 1-Mild, 2-Moderate, 3-Severe, 4-Life threatening, 5-Fatal, Use maximum grade for summary Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "ccc" portion of patient number.

Sort "Onset Date" in ascending order within "Patient".

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan


136

<sup>[2]</sup> DLT= Dose Limiting Toxicity

<sup>[3]</sup> Day is relative to the first dose date of NBF-006.

<sup>[4]</sup> Ser-Serious; 1-Not Serious, 2-Results in Death, 3-Life Threatening, 4-Requires or Prolongs Hospitalization, 5-Persistent or Significant Disability/Incapacity, 6-Congenital Anomaly or Birth Defect, 7=Other Medically Important Serious Event.

<sup>[5]</sup> Act=Action Taken: 1=Dose NOT Changed, 2=Dose Interrupted, 3= Dose Delayed, 4= Drug Withdrawn.

<sup>[6]</sup> Out-Outcome: 1-Recovered/Resolved, 2-Recovered/Resolved with sequelae, 3-Recovering/Resolving, 4-Not Recovered/Not Resolved, 5-Fatal, 6-Unknown.



Listing 16.2.7.5 Death Summary Safety Evaluable (N=n)

| Patient | Study | NBF-006 Dose | Date of | Primary | Date of | Date of | Date off- | Treatment | First Dose | Last Dose | Off-Study |
|---|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Death | Cause | First Dose | Last Dose | Study | Duration (Day) [1] | to Death (Day) | to Death (Day) | to Death (Day |
| ccc-pppp<br>/xx/x | × | xxx | ddmmmyyyy | XXXXX | ddmiriryyyy | ddmininyyyy | ddmmrryyyy | xx | xx | xx | кх |
| ccc-pppp | × | XXX | ddmininyyyy | XXXXXX | ddminiryyyy | ddmmmyyyy | ddmmrryyyy | XX | xx | xx | KK |

[1] Treatment duration is calculated from the first dose date to discontinuation date of study drug in days.

Cross-References: Case Report Form Case Report Forms DEATH SUMMARY (DS), NBF-006 ADMINISTRATION (EX) and OFF-STUDY SUMMARY (OF)
PROGRAMMER'S NOTES:

Sort "Patient" in ascending order using "poop", and then "cot" portion of patient number,



## Listing 16.2.8.1 Clinical Laboratory Tests - Hematology Safety Evaluable (N=n)

FINAL- ddmmmyychh:mm


| Patient | Study | NBF-006 Dose | | Sample | Sample | Day | Late | Laboratory T | est 1 (unit) (Z) | Laboratory 1 | fest 2 (unit) [2] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Date | Time | [II] | Code | Results | Normal Range | Results | Normal Range |
| ce-pppp | × | XXX | xx | ddmmmyyyy | hhonm | *XX | XXXX | XXXHG1 | XX.X.+ XX,X | xxx H G1 | XX.X - XX.X |
| xx/x | | | XX | ddmmmyyyy | hhamm | XX | XXXX | XX.X | XX.X - XX.X | XXX | XX,X - XX,X |
| | | | XX | ddrnmmyyyy | bbanm | XX | XXXX | xx.x | XXX - XXX | 30000 | XXXX - XXXX |
| ссс-рррр | x | XXX | xx | ddmmmyyyy | hhomm. | ×XX | XXXX | XXX | XX.X = XX.X | XXX | XXXX = XXXX |
| AxxX | | | XX | ddrnmmyyyy | hhomm | XX. | XXXX | XXXLG1 | XX.X = XX.X | XXX L G1 | XXX - XXX |
| 22.26 | | | XX | ddrnmmyyyy | hhanm | 300 | XXXX | XX.X | XX.X - XXX | 30000 | MXXX = XXXX |
| | | | xx | ddmmmyyyy | hhomm | XX | XXXX | XX.X | XX.X + XX.X | XXX | XXX - XXX |

<sup>[1]</sup> Day is relative to the first dose date of NBF-006.

(2) Reported Result: H = High (Above Normal Range), L = Low (Below Normal Range); Calculated CTCAE version 5 Grade 1 to 4. Cross-References: Case Report Form HEMATOLOGY (HM)

136

PROGRAMMER'S NOTES:

Onwards page as required.

Include following Hernatology Tests: Hernoglobin, Hernatocrit, Platelets, WBC, and WBC differential.

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "papp", and then "ccc" portion of patient number. Sort "Date" in ascending order within "Patient".

Remove footnote 'Calculated CTCAE version 5 Grade 1 to 4 if not needed.

Statistical Analysis Plan

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved




DIRECTORY/FILE.SAS FINAL- ddmmmyychbcmm Page 1 of x NBF-006-001 Phase 1/1b

#### Listing 16.2.8.2 Clinical Laboratory Tests - Blood Chemistry Safety Evaluable (N=n)

| Patient Study | NBF-006 Dose | | Sample | Sample | Diny | Lab | Laboratory 1 | est 1(unit) [2] | Laboratory 7 | Test 2 (unit) [2] |
|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex Part | (rrg/kg) | Visit | Date | Time | [1] | Code | Results. | Normal Range | Results | Normal Range |
| ссс-рарр х | xxx | XX | ddmmmyyyy | hhamm | -XX | XXXX. | XXX H G1 | NXX-XXX | xx.x H G1 | XX,X + XX,X |
| ov/x | | ЖX | ddmmmyyyy | Hhammi | KK | XXXX | 30K.X | XXX × XX.X | xx.x | XX,X = XX,X |
| | | XX. | ddmmmyyyy | hhomm | XX | XXXX | XXX | XX.X - XX.X | XX,X | XX.X - XX.X |
| | | XX. | ddmmmyyyy | Hhamm | +9000 | XXXX | XX.X | MX.X - XX.X | XX.X | $KX_{*}X + 300_{*}X$ |
| ccc-pppp x | XXX | XX- | ddrimmyyyy | hhammi | KK | XXXX | xx.x L G1 | XX.X × XX.X. | xx.x l, G1 | xx.x - xx.x |
| odx | | XX | ddmmmyyyy | hinamin | XX | XXXX | XXX | XXX - XXX | XX.X | XX.X - XX.X |
| | | ×× | ddmmmyyyy | hismin | XX | XXXX | XX.X | XX.X + XX.X | XX.X | XX,X = 300.X |

[1] Day is relative to the first dose date of NBF-006.

[2] Reported Result: H = High (Above Normal Range), L = Low (Below Normal Range); Calculated CTCAE version 5 Grade 1 to 4. Cross-References: Case Report Form BLOOD BIOCHEMISTRY (BC) PROGRAMMERS NOTES:

Coagulation collected only Pre-Study, revise footnote [1].

Orwards page as required,

Include following Blood Chemistry Tests: BUN, sodium, potassium, calcium, total bilirubin, total protein, ALT, AST, ALP, albumin, creatinine, and glucose.

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables. Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number. Sort "Date" in ascending order within "Patient". Remove footnote 'Calculated CTCAE version 5 Grade 1 to 4 if not needed.

Copyright© 2016 by Theradex Oncology®, Princeton NI

Statistical Analysis Plan


All rights reserved

139



DIRECTORY/FILE.SAS FINAL- ddmmmyychh:mm NBF-006-001 Phase 1/To Page 1 of x

## Listing 16.2.8.3 Clinical Laboratory Tests - Urinalysis Safety Evaluable (N=n)

| Patient Stu | dy | NBF-006 Dose | | Sample | Sample | Day. | Lab | Laboratory 7 | Test 1[2] | Laboratory 7 | Test 2[2] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex Part | rt | (mg/kg) | Visit | Date | Time | [1] | Cade | Results | Normal Range | Results | Normai Range |
| сес-рарр к | | xxx | жx | ddrammyyyy | Hhammi | 9XX | XXX | xxx H G1 | XXX×XXX | xx.x H G1 | xx.x - xx.x |
| hours. | | | XX. | ddmmmyyyy | hhomm | XX | XXX | XX,X | XX.X - XX.X | XX,X | XX.X - XX.X |
| | | | NX. | ddmmmyyyy | Hhamm | XX | 3000 | XX.X | AX.X - XX.X | XX.X | XX,X + 306,X |
| | | | XX- | ddrnmmyyyy | hhammi | HOE | XXX | 30K.X | XX.X × XX.X | XX.X | XX.X - XX.X |
| ссс-рррр к | | XXX. | XX. | ddmmmyyyy | hinarem | XX | XXX | XXXX L G1 | XXX - XXX | xx.x L G1 | XX.X - XX.X |
| /xx/x | | | XX | ddmmmyyyy | hhamm | KK | XXX | XX.X | XX.X - XX.X | XX.X | KX,X + 906_K |
| | | | XX | ddmmmyyyy | hiticimin | XX. | 3006 | XX.X | XX.X - XX.X | xx.x | XX.X · XX.X |
| | | | XX. | ddmmmyyyy | hhamm | XX | XXX | XXX | XXX - XXX | XX.X | XX.X - XX.X |

[1] Day is relative to the first dose date of NBF-006.

[2] Reported Result: H = High (Above Normal Range), L = Low (Below Normal Range); Calculated CTCAS version 5 Grade 1 to 4.

140

Cross-References: Case Report Form URINALYSIS (US)
PROGRAMMER'S NOTES:

Onwards page as required.

Include following Urinalysis Tests: Specific gravity, pH, Glucose, Protein, Ketones, Nitrite, and Leukocyte Esterase, and microscopic tests.

Data will be presented in mixed case for formatted variables and upper case only for uniformatted variables.

Sort "Patient" in ascending order using "oppp", and then "cot" portion of patient number. Sort "Date" in ascending order within "Patient". Remove footnote 'Calculated CTCAE version 5 Grade 1 to 4 if not needed.

Statistical Analysis Plan Copyright© 2016 by Theradex Oncology®, Princeton NI

Final Version 2.0, March 14, 2023 Confidential - Entire Page




Listing 16.2.9.1 Vital Signs Safety Evaluable (N=n)

| Age/Sex<br>cc-pppp | Part | Dose(mg/kg) | Visit | - | | Day | | Time | DIDDOM FIES | aut maint in the | Temperature | Heart Rate | Respiratory |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| or-mon | | | | Date | Time | [1] | Start | Stop | Systolic | Diastolic | (°C) | (/min) | (/min) |
| cc-bbbb | X | XXX | KX. | ddmmmyyyy | hhomm | xx | hhamm | bhomm | xxx | XX. | xx,x | XXX | XX |
| cx/x | | | | | | | | | XXX | ××. | xx.x | XXXX | XX |
| | | | | | | | | | XXX | XX. | XX.X | SOCK | xx |
| | | | | | | | | | xxx | XX | XX,X | XXX | xx<br>xx<br>xx |
| | | | KK: | ddmmmyyyy | hhomon | XX. | beamin | hhamm | XXX | ×× | xx.x | XXX | XX |
| | | | | | | | | | XXX | XX | xx.x | XXXX | XX |
| | | | | | | | | | xxx | XX | xx.x | XXX | XX |
| | | | | | | | | | XXX | XX | xx.x | XXX | XX |
| cc-pppp | × | XXX | XX | ddmmmyyyy | hhamm | XX | hhamm | hhomm | XXX | XX. | xx.x | XXX | XX<br>XX<br>XX<br>XX |
| ov/x | | | | | | | | | SOC | XX. | XX.X | мжж | XX |
| | | | | | | | | | 8308 | xx | xx.x | XXXX | xx |

[1] Day is relative to the first dose date of NBF-006,

Cross-References: Case Report Form VITAL SIGNS (VS. VS1)
PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column.

Add records for "Other unscheduled timepoints" within a day if necessary.

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "papp", and then "cot" portion of patient number.

Sort "Date Performed" in ascending order within "Patient", Sort "Time" in ascending order within "Date".

Present infusion Time only data is available or can be derived.

Statistical Analysis Plan Copyright© 2016 by Theradex Oncology®, Princeton NI


All rights reserved

141




Listing 16.2,9.2 Physical Examination Safety Evaluable (N=n)

| Patient<br>(Acade or | Study | NBF-006 Do | | Examination | Day | Any Clinically |
|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Date | [1] | Significant Findings |
| ccc-pppp/xx/x | × | XXX | Screening | ddmmmyyyy | -xx | No |
| | | | 300 | ddmininyyyy | XX | No |
| | | | XX | ddmmmyyyy | -XX<br>XX | No<br>No |
| | | | XX | ddmmmyyyy | 300 | No |
| cc-pppp/xx/x | × | XXX | Screening | ddmmmyyyy | *XX | No<br>Na<br>No |
| | | | XX | ddmmmyyyy | 308 | No |
| | | | XX. | ddmmmyyyy | 300 | No<br>Yes |
| | | | 300 | ddmmmyyyy | XX | |
| εεε-ρρρη/κν/κ | × | XXX | Screening | ddmmmyyyy | *XX | No<br>No |
| | | | XX | ddmmmyyyy | XX | No |
| | | | 300 | ddmmmyyyy | XX | No |
| | | | XX | ddmmmyyyy | 204 | No |

[1] Day is relative to the first dose date of NBF-006. Cross-References: Case Report Form PHYSICAL EXAMINATION (PE)

#### PROGRAMMER'S NOTES:

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "ccc" portion of patient number.

Statistical Analysis Plan

142


Copyright© 2016 by Theradex Oncology®, Princeton NT All rights reserved




Listing 16.2.9.3 Electrocardiogram Safety Evaluable (N=n)

| Patient | Study | NBF-006 Dose | | Visit | Day | Planned | | Infusion 1 | Time | Heart | PR | QT. | QTcF |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Date | [1] | Timepoint | Time | Start | End | Rate (bpm) | (rrs) | (ms) | (ms) |
| ccc-pppp/xx/x | × | xxx | Screening | ddmmmyyyy | -900 | xxx | Manin | Hecmm | hhamm | 300 | хх.х | XXX | xx.x |
| | | | | | | XXX | hhamm | hhomm | hhomm | xx | XX.X | XX.X | XX.X |
| | | | | | | xxx | hhanm- | hhamm | hhomm | 30X | XX,X | XX.X | XX.X |
| | | | XXX | ddmmmyyyy | xx | XXX | bhanm | hhamm | hhamm | xx | XX.X | XXX | XX.X |
| | | | xxx. | ddmmmyyyy | XX. | XXX | thann | hhamm | hhanm | xx | XX.X | XXX | XX.X |
| сес-пррр/хх/х | × | xxx | Screening | ddmmmyyyy | -900 | XXX. | Mann | rincimi | hhamm | xx | XX.X | XXX | xx.x |
| | | | | | | XXX | thanm | hhamm | hhamm | XX | XX.X | XXX | XX.X |
| | | | | | | xxx | hhanm | fythamm: | hhamm | 304 | XX.X | XX.X | XX.X |
| | | | XXX | ddmmmyyyy | xx | XXX | Manm | hhamm | hhomm | xx | XX.X | XXX | XX.X |
| | | | XXX. | ddmmmyyyy | XX | XXX | tharm | hhamm | hhomm | XX | XX.X | XXX | XX.X |

QT=QT interval, QTcF= QT corrected by Fridericia's formula

[1] Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Form ELECTROCARD/OGRAM (EG, EG1, EG2, EG3, EG4)

PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time column.

Add records for "Other unscheduled timepoints" within a day if necessary.

Data will be presented in mixed case for formatted variables and upper case only for uniformatted variables.

Sort "Patient" in ascending order using "popp", and then "cct" portion of patient number.

Sort "Date Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

Present Visit only if data are available.

Present Infusion Time only data is available or can be derived.

Copyright© 2016 by Theradex Oncology®, Princeton NI

All rights reserved

Statistical Analysis Plan 143





#### Listing 16.2.9.3 Electrocardiogram Safety Evaluable (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006<br>Dose(mg/kg) | Visit | Date | Day<br>[1] | Planned<br>Timepoint | Time | Clinical<br>Interpretation | Clinical<br>Significance | Conclusion | Collection<br>Status |
|---|---|---|---|---|---|---|---|---|---|---|---|
| сс-раррухх/х | × | xxx | Screening | ddrnmmyyyy | -XX | ddmmmyyyy | bhamm | ddmmmyyyy | XXX | XXX | XXX |
| | | | | | | ddmmmyyyy | hitomin | ddmmmyyyy | XXX | XXX | XXX |
| | | | | | | ddmmmyyyy | bhamm: | ddmmmyyyy | XXX | 3000 | XXX |
| | | | XXX | ddmmmyyyy | XX | ddmmmyyyy | bisamm | ddmmmyyyy | XXX | 300X | XXX |
| | | | xxx | ddimminyyyy | жx | ddmmmyyyy | hhanm | ddmmmyyyy | KKK | 300K | xxx |
| сс-рарружих | x | XXX | Screening | ddmmmyyyy | -XX | ddmmmyyyy | hhamm | ddmmmyyyy | XXX | XXX | XXX |
| | | | - 2 | 3 | | ddmmmyyyy | hhannn | ddmmmyyyy | XXX | 3000 | XXX |
| | | | | | | ddrnmmyyyy | hhamm | ddmmmyyyy | XXX | XXX | XXX |
| | | | XXX | ddmmmyyyy | XX | ddmmmyyyy | hhamm | ddmmmyyyy | XXX | 3000 | XXX |
| | | | XXX | ddmmmyyyy | XX | ddmmmyyyy | hhannn | ddmmmyyyy | XXX | 300X | XXX |

<sup>[1]</sup> Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Forms SCREENING ELECTROCARDIOGRAM (EG, EG1, EG2, EG3, EG4)
PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column. Add records for "Other unscheduled timepoints" within a day if necessary.

Data will be presented in mixed case for formatted variables and upper case only for uniformatted variables.

Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number.

Sort "Date Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

Remove "Collection Status" if not populated.

All rights reserved

Statistical Analysis Plan Copyright© 2016 by Theradex Oncology®, Princeton NI

144





# Listing 16.2,9.4 ECOG Performance Status Safety Evaluable (N=n)

| Patient | Study | NBF-006 Dose | | Date | Day | |
|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Assessed | [1] | ECOG Performance Status |
| ссс-рорр | × | XXX | Screening | ddmmmyyyy | -XX | 0 Fully active, able to carry on all pre-disease activities without restriction. |
| /xx/x | | | XXX | ddmmmyyyy | ж | 1 Restricted in physically strenuous activity but ambulatory and able to carry work of a light or sedentary<br>nature, e.g., light housework, office work. |
| | | | XXX | ddmmmyyyy | ж | 2 Ambulatory and capable of all self-care but unable to carry out work activities. Up and about more than<br>50% of waking hours. |
| | | | XXX | ddmmmyyyy | XX. | 3 Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. |
| | | | XXX | ddrmmmyyyy | XX | 4 Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. |
| | | | xxx | ddmmmyyyy | x | 5 Dead. |
| ссс-рара | X | XXX | Screening | ddmmmyyyy | -XX | 0 Fully active, able to carry on all pre-disease activities without restriction, |
| /xx/x | | | xxx | ddmmmyyyy | x | 1 Restricted in physically strenuous activity but ambulatory and able to carry work of a light or sedentary nature, e.g., light housework, office work. |
| | | | xxx | ddimmmyyyy | ж | 2 Ambulatory and capable of all self-care but unable to carry out work activities. Up and about more than<br>50% of waking hours. |
| | | | XXX | ddmmmyyyy | 300 | 3 Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. |

[1] Day is relative to the first dose date of NBF-006, Cross-References: Case Report Form PERFORMANCE STATUS (ES) PROGRAMMER'S NOTES:

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables. Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number. Sort "Date Performed" in ascending order within "Patient".

Statistical Analysis Plan


All rights reserved

Copyright© 2016 by Theradex Oncology®, Princeton NI

145



DIRECTORY/FILE.SAS FINAL- ddmmmyythh:mm NBF-006-001 Phase 1/To Page 1 of x

Listing 16.2,9.5 Infusion-Related Reactions

| Patient | Study | NBF-006 | Adverse Event<br>(MedDRA Preferred Term) | DLT | Onset<br>Resolved | Day | | Ser | Drug | Act | Therapy | Infusion ' | Time |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | Dose (mg/kg) | (MedDRA System Organ Class) | [1] | Date/Time | [2] | Grade | [3] | Related | [4] | Given | Start | Stop |
| ссс-рррр<br>/хж/х | * | XXX | ADVERSE EVENT<br>(MedDRA Preferred Term)<br>(MedDRA System Organ Class) | | XX XXX/XXXX<br>XX XXX/XXXX | XX | Mild | × | probably | 1 | Yes | bharnay | bhonm |
| | | | ADVERSE EVENT<br>(MedDRA Preferred Term)<br>(MedDRA System Organ Class) | | xxxx/xxxx<br>xxxx/xxxx | xx | Mild | × | Unlikely | 3 | Yes | hhomm | hhanin |
| /xx/x | × | XXX | ADVERSE EVENT<br>(MedDRA Preferred Term)<br>(MedDRA System Organ Class) | Yes | xxxxx/xxxx<br>xx xxx/xxxx | XX. | Severe | | Unrelated | 2 | No | bbann | hinanim |

### MedDRA version 21.1

[1] DLT= Dose Limiting Taxicity

[2] Day is relative to the first dose date of NBF-006.

[3] Ser-Serious: 1=Not Serious, 2=Results in Death, 3=Life Threatening, 4=Requires or Prolongs Hospitalization, 5=Persistent or Significant Disability/Incapacity, 6=Congenital Anomaly or Birth Defect, 7=Other Medically Important Serious Eyent.

[4] Act-Action Taken: 1-Dose NOT Changed, 2-Dose Interrupted, 3- Dose Delayed, 4- Drug Withdrawn.

DLT= Dose Limiting Toxicity

Influsion-related reactions includes back pain, fever and/or shaking chills, flushing and/or itching, alterations in heart rate and blood pressure, dyspnea or chest discomfort, skin rashes, or anaphylaxis (e.g. generalized urticaria, angloedema, wheezing hypotens ion, tachycardia, etc.)
Cross-References: Case Report Form ADVERSE EVENTS (AE)

#### PROGRAMMER'S NOTES:

Grade: 1-Mild, 2-Moderate, 3-Severe, 4-Life threatening, 5-Fatai. Use maximum grade for summary. Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "ccc" portion of patient number.

Sort "Onset Date" in ascending order within "Patient".

Influsion-related reactions includes back pain, fever and/or shaking chills, flushing and/or litching, alterations in heart rate and blood pressure, dyspries or chest discomfort, skin rashes, or anaphylaxis (e.g. generalized urticaria, angioedema, wheezing, hypotension, tachycardia, etc.)

Present infusion Time only data is available or can be derived.

Copyright© 2016 by Theradex Oncology®, Princeton NI

Statistical Analysis Plan


All rights reserved

146



FINAL- ddmmmyychnomm Page 1 of x

#### Listing 16,2,9.6 Pain Assessment Safety Evaluable (N=n)

| Patient<br>/Age/Sex | Study | Dose<br>(mg/kg) | Visit | Visit<br>Date | Infusion Start<br>/Stop Time | MedDRA<br>Preferred Term | Date<br>Collected | Day<br>[1] | Time<br>Callected | Pain<br>Rate[2] | Grade<br>[3] | Where | Duration<br>(unit) | Drug<br>Relationship | Trigger |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| - | | | | | | | | | | | 1977/19 | | | | |
| есс-рррр | × | XXX | XXX | XXX | hhamm | MedDRA PT | ddrnmmyyyy | xx | hhanm | XXX | × | XXX | KK.X | Unrelated | XXXXX |
| /xx/x | | | | | /hhamm | | | | | | | | | | |
| | | | | | hhamm | MedDRA PT | ddrnmmyyyy | XX | hhamm | NXX | × | XXX | XX.X | Linlikely | XXXXXX |
| | | | | | Principini | | | | | | | | | | |
| ссс-рррр | × | 3000 | 3000 | XXX | hitemin | MedDRA PT | ddmmmyyyy | XX | Trhimm | XXX | | XXX | NX.N | Possible | XXXXX |
| /xx/x | | | | | 7hhamm | MedDRA PT | ddmmmyyyy | XX | hhamm | XXX | | XXX | XX.X | | |

Pain rate scale of 0-10, 0 is no pain, 10 is the worst pain.

[1] Day is relative to the first dose date of NBF-006.

[2] Pain scale 0-10

[3] Grade: 1-Mild; 2-Moderate, 3-Severe, 4-Life threatening, 5-Fatal,

Cross-References: Case Report Form Pain Assessment (PA)

PROGRAMMER'S NOTES:

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables. Sort "Patient" in ascending order using "oppp", and then "occ" portion of patient number.

Sort "Date Performed" in ascending order within "Patient".

Influsion-related reactions includes back pain, fever and/or shaking chills, flushing and/or itching, alterations in heart rate and blood pressure, dyspines or chest discomfort, skin

rashes, or anaphylaxis (e.g. generalized urticaria, angioedema, wheezing, hypotension, tachycardia, etc.)

Present Visit/Visit Date only if data are available. Present pain rate only if data is available.

Added 3 columns MedDRA PT, Grade, Drug Relationship, but they are not on CRF Pain Assessment page, present only if they can be populated

Copyright© 2016 by Theradex Oncology®, Princeton NI

Statistical Analysis Plan 147


All rights reserved



NBF-006-001 Phase 1/To

DIRECTORY/FILE.SAS


#### Listing 16.2.9.7 Immune Activation Markers - Cytokines Assessment Intent-to-Treat (N=n)

| Patient | Study | N8F-006 | | Sample | Day | Scheduled | | | TNF-a | | L+1β | | 11.46 | | IFN-y |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | Dose(ing/kg) | Visit | Date | 111 | Timepoint | Time | Actual | 16Change | Actual | %Change | Actual | %Change | Actual | 16Change |
| εεε-ρρρργούχ | × | XXX | Screening | XXX | ×x. | XXX | hhomm | XXX | xx.x | XXX | XXX | XX.X | xx.x | XXX | xx.x |
| | | | | | | XXX | hhamm | XXX | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | | | | XXX | Monte | xx.x | xx.x | xx.x | xx,x | жж.ж | xx,x | XX.X | xx.x |
| ccc-pppp/xx/x | × | XXX | Screening | XXX | XX | XXX | hhamm | XXX | xx.x | XXX | XX.X | XX.X | xx.x | XX.X | xx.x |
| | | | | | | XXX | himmin | xx.x | xx.x | xx.x | xx,x | XX.X | xx.x | XXX | xx,x |
| | | | | | | XXX | hitamin | XX.X | xx.x | XXX | xx.x | xx,x | XX,X | XXX | xx.x |

Cytokines only collected in Part B at 1.6 mg/kg if cytokine induction was seen at 1.6 mg/kg in Part A, or if there are symptoms indicative of cytokine induction. [1] Day is relative to the first dose date of NBF-006,

[2] Change = Change from baseline. Baseline is defined as the last value prior to first dose of study drug.

Cross-References: Case Report Form IMMUNE ACTIVATION MARKERS - CYTOKINES ASSESSMENT (TM4)

PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time column.

Add records for "Other unscheduled timepoints" within a day if necessary.

Data will be presented in inixed case for formatted variables and upper case only for unformatted variables. Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number.

Sort "Date Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

Copyright© 2016 by Theradex Oncology®, Princeton NI

Statistical Analysis Plan


All rights reserved

148



DIRECTORY/FILE.SAS FINAL- ddmmmyychh:mm NBF-006-001 Phase 1/To Page 1 of x

#### Listing 16.2.9.8 Immune Activation Markers - Complement Assessment Intent-to-Treat (N=n)

| Patient | Study | NBF-006 | | Sample | Day | Scheduled | | / | CH50 | a | Bb | S-111 1 | C3a | Na | C5a |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | Dose(mg/kg) | Visit | Date | [1] | Timepoint | Time | Actual | 16Change | Actual | WChange | Actual | 6Otange | Actual | %Change |
| εεε-ρρρρ/κκ/χ | × | XXX | XXX | XXX | XXXXXX | xx | hhomm | XX.X | XX.X | XXX | xx.x | XX.X | XXX | XXX | xx.x |
| | | | | | | XX | hhamm | xx.x | XXX | XXX.X | XX.X | XX.X | XXX | XXX | XX.X |
| | | | | | | xx | hhamm | xx.x | XX.X | XX.X | xx.x | xx,x | xx.x | xx.x | xx.x |
| ccc-ppppp/xx/x | × | XXX. | XXX | XXX | XXXXXX | xx | hhamm | xx.x | XXX | XXX | xx.x | xx.x | XXXX | XX.X | XX.X. |
| | | | | | | XX. | hhomm | xx.x | XXX | XXX | xx,x | XX,X | 30K.X | XX,X | xx.x |
| | | | | | | xx | hhamm | XX.X | XXXX | XXX | XX.X | XX,X | NOCK,N | XX.X | XXX |

<sup>[1]</sup> Day is relative to the first dose date of NBF-006.

PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column.

Add records for "Other unscheduled timepoints" within a day if necessary.

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number.

Sort "Date Performed" in ascending order within "Patient", Sort "Time" in ascending order within "Date".

Statistical Analysis Plan


All rights reserved

Copyright© 2016 by Theradex Oncology®, Princeton NI

149

<sup>[2]</sup> Change = Change from baseline. Baseline is defined as the last value prior to first dose of study drug, Cross-References: Case Report Form IMMUNE ACTIVATION MARKERS - COMPLEMENT (TM)




#### Listing 16.2.9.9 Ariti-Drug Antibody (ADA) Assay intent-to-Treat (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006 Dose<br>(mg/kg) | Visit | Test | Sample<br>Date | Day<br>[1] | Scheduled<br>Timepoint | Time | Result | Titer |
|---|---|---|---|---|---|---|---|---|---|---|
| εεε-ρορο/κκ/κ | × | XXX | XXX | Screening | didminimyyyy | xx | xx | nhonm | Negative | |
| 77777 | × | XXX | XXX | Confirmatory | N/A | | | | | |
| | * | XXX | KKK | Titration | N/A | | | | | |
| сс-ррррухж/х | × | XXX | KKK | Screening | ddmmmyyyy | ×× | XX<br>XX | hhonm | Positive | |
| | × | XXX | XXX | Confirmatory | ddmmmyyyy | XX | XX | hhomm | Positive | |
| | × | XXX | XXX | Titration | ddmmmyyyy | XX | xx | thhomm | Positive | XXXX |
| | × | XXX | KKK. | XXX | ddmmmyyyy | xx | XX | htomm | Positive | |
| | × | XXX | XXX | Confirmatory | didimmmyyyy | XX | xx | thomm | Negative | |
| | × | XXX | XXX | Titration | N/A | | | | 8514 | |

<sup>[1]</sup> Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Form ANTI-DRUG ANTIBODY (ADA) ASSAY (TM1, TM2)
PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column. Add records for "Other unacheduled timepoints" within a day if necessary.

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "popp", and then "cor" portion of patient number.

Sort "Date Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

If Screening result is positive, the same sample will be tested again as a confirmatory assay. Assume that if only tier 1 done on sample, then would next result be blank or

Copyright© 2016 by Theradex Oncology®, Princeton NI

Statistical Analysis Plan


All rights reserved

150



# Listing 16.2.9.10 KRAS Mutation Assessment intent-to-Treat (N=n)

FINAL- ddmmmyychh:mm


| Patient | Study | NBF-006 Dose | | Assessment | Genomic Tumor | Date of | Day | | Archival Tissue | | Fresh | | If Yes, Biopsy | KRAS Mutation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Completed | Profile at Screen | Analysis | [1] | Result | Sample | Date | Sample | Date | Performed | Туре |
| εεε-ρρρογωνία | x | XXX | xxx | Ves | Yes | ddmmmyyyy | -XX | XXX | Yes | XXX | Yes | жх | Yes | XXX |
| ccc-pppp/xx/x | × | XXX | XXX | Yes | Yes | ddminimyyyy | ×XX | XXX | Yes | XXX | Yes | XXX | Yes | XXX |
| ccc-ppppp/xx/x | × | XXX | XXX | Yes | Yes | ddmmmyyyy | *XX | XXX | Yes | XXX | Yes | XXX | Yes | XXX |
| ссс-раррухх/х | x | KXX | XXX | Yes | Yes | ddmmmyyyy | -XX | XXX | Yes | XXX | Yes | XXX | Yes . | XXX |
| ccc-ppppp/xx/x | × | XXX | XXX | No | No | NOTDONE | *XX | XXX | No | | No | | No, xxx | |
| ccc-ppppp/xx/x | x | XXX | XXX | Yes | Yes | ddmmmyyyy | -XX | XXX | Yes | XXX | Yes | XXX | Yes | 300X |
| x/xx/aggg-pox | x | XXX | XXX | Yes | Yes | ddmmmyyyy | -xx | XXX | Yes | XXX | Yes | XXX | Yes | Other, specify |

[1] Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Form KRAS MUTATION ASSESSMENT (TM8)

#### PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column.

Data will be presented in mixed case for formatted variables and upper case only for uniformatted variables.

Sort "Patient" in ascending order using "pppp", and then "cor" portion of patient number.

Present Visit only if it is applicable.

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan 151





Listing 16.2.9.11 GSTT1 Genotyping Intent-to-Treat (N=n)

| Patient | Study | NBF-006 Dose | | Whole Blood | Date | Day | Time | | 1100 ton 1000 a |
|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Collected | Callected | [1] | Collected | Test | Result |
| εεε-ραρολούχ | ĸ | xxx | 3000 | Yes | ddmmmyyyy | -xx | hhamm | GSTT1 Ct Value | XX.XX |
| ccc-ppppp/xx/x | × | XXX | XXX | Yes | ddmmmyyyy | -XX | hh:mm | RNASE Ct Value | XX.XX |
| ccc-ppppp/xx/x | × | xxx | XXX | Yes | ddminmyyyy | *XX | hhamm | GSTT1 Genotype | GSTT1 Positive |
| ссс-раррухол/х | × | xxx | XXX | Yes | ddmmmyyyy | -xx | hhamas | GSTT1 Ct Value | Undetermined |
| ccc-ppppp/xx/x | × | XXX | XXX. | Yes | ddmmmyyyy | -830 | hhamm | RNASE CL Value | KX,XX |
| ccr-ppppp/xx/x | × | XXX | XXX | Yes | ddmmmyyyy | -XX | hhamm | GSTT1 Genotype | GSTT1 Positive |
| ссс-раррухомх | × | XXX | 3000 | No | | | | | |

GSTT1 - Glutathione S-Transferase theta class

[1] Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Form GSTT1 GENOTYPING (BS)

PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time column.

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "cor" portion of patient number.

Sort "Date Performed" in ascending order within "Patient", Sort "Time" in ascending order within "Date".

Present Visit only if it is applicable. Present result if data collected.

NBF-006-001

Copyright© 2016 by Theradex Oncology®, Princeton NJ All rights reserved

Statistical Analysis Plan 152 Final Version 2.0, March 14, 2023




# Listing 16.2.9.12 Exploratory Tumor Biopsy Intent-to-Treat (N=n)

| Patient<br>/Age/Sex | Study<br>Part | NBF-006 Dose<br>(mg/kg) | Visit | Date<br>Collected | Day<br>[1] | Reason<br>Not Collected | Time | Turner Biopsy<br>Location |
|---|---|---|---|---|---|---|---|---|
| ACRES CYCATULAS | | | | (A. M.) (C.) (C.) (C.) (C.) | | | | 79200 |
| εεε-ρρρρ/κκ/κ | × | XXX | XXX | ddmmmyyyy | -XX | | bhamm | XXX |
| ccc-pppp/xx/x | × | XXX | XXX | ddmmmyyyy | -XX | | tehornen | XXX |
| ccc-ppppp/xx/x | × | 3000 | XXX | ddrnmmyyyy | -KX | | bhamm | xxx |
| ссс-раррухол/х | × | 3000 | XXX | ddmmmyyyy | -XX | | hinamin | XXX |
| ccc-ppppp/xx/x | × | 3000 | XXX | ddmmmyyyy | *XX | | thomen | xxx |
| ccc-ppppp/xx/x | × | 3000 | XXX | ddrnmmyyyy | -KX | | hhamm | XXX |
| ccc-ppppp/xx/x | × | 2000 | XXX | NOT DONE | | XXXXXX | | |

[1] Day is relative to the first dose date of NBF-006. Cross-References; Case Report Form EXPLORATORY TLIMOR BIOPY (PR1, PR2)

#### PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column.

Data will be presented in mixed case for formatted variables and upper case only for uniformatted variables.

Sort "Patient" in ascending order using "pppp", and then "cor" portion of patient number.

Sort "Date Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

Present Visit only if it is applicable.

Statistical Analysis Plan


All rights reserved

Copyright© 2016 by Theradex Oncology®, Princeton NI

153




#### Listing 16.2.9.13 GSTP mRNA KD Sample Intent-to-Treat (N=n)

| Patient | Study | NBF-006 Dose | | Schedule | Sample | Day | | | |
|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Timepoint | Date | [1] | Time | Result | Unit |
| ссс-рарр/хж/х | × | XXX | XXX | XXX | ddmmmyyyy | -xx | hhanm | XXXXX | XXXX |
| ccc-ppppp/xx/x | ×. | XXXX | KKK | XXX | ddmmmyyyy | *XX | hhanm | XXXXX | XXXX |
| ccc-ppppp/xx/x | × | XXX | KKK. | 3000. | ddmmmyyyy | -XX | hhanm | XXXXX | XXXX |
| ссс-рарру/хх/х | x | XXX | XXX | XXX | ddmmmyyyy | -XX | hhimm | XXXXX | 30000 |
| ccc-ppppp/xx/x | ×. | XXX | KKK | XXX | ddmmmyyyy | *XX | Hhanim | XXXXX | 30000 |
| ccr-ppppp/xx/x | × | XXX | KKK. | XXX | ddmmmyyyy | -XX | hhanm | XXXXX | 33000 |
| ссс-рарру/хог/х | × | XXX | XXX | XXX | ddmmmyyyy | -xx | hhanm. | XXXXX | XXXX |

[1] Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Form GSTP MRNA KD SAMPLE (TM6, TM7)

#### PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column.

Add records for "Other unscheduled timepoints" within a day if necessary,

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "cor" portion of patient number.

Sort "Date Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

Present Visit only if it is applicable. Present result if data collected.

For any of the PBMC read-outs (GST mRNA levels), there will be some time points that fall due to insufficient sample. So for unit we may have to indicate ND and then footnote that sample insufficient for analysis.

Statistical Analysis Plan

154


Copyright© 2016 by Theradex Oncology®, Princeton NI

All rights reserved




#### Listing 16.2.9.14 GST Family - GSTP1 mRNA Level intent-to-Treat (N=n)

| Patient | Study | NBF-006 Dose | | Schedule | Sample | Day | | GSTP1 | |
|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (rng/kg) | Visit | Timepoint | Date | [1] | Time | mRNA Level | Unit |
| ccc-pppp/xx/x | × | XXX | XXX | XXX | ddmmmyyyy | -xx | bhamm | KXXXXX | XXX |
| ccc-ppppp/xx/x | × | XXX | XXX | XXX | ddmmrryyyy | -500 | tehomen | MANAGE | XXX |
| ccc-ppppp/xx/x | × | XXX | XXX | 2003 | ddmmmyyyy | HXX | tihamm | XXXXXX | XXX |
| ссс-раррухол/х | × | XXX | XXX | 3006 | ddmmmyyyy | -xx | hhamm | XXXXXX | XXX |
| ccc-ppppp/xx/x | × | XXX | SXX | XXX | ddmmrryyyy | -8X | teleponen | MACHOR | XXX |
| ccr-ppppp/xx/x | × | XXX | XXX | 3004 | ddmmmyyyy | -XX. | bhamm | 8XXXX | XXX |
| εεε-ραρρλούχ | × | XXX | XXX | XXX | ddmmmyyyy | -xx | hinsonon | KKKKK | XXX |

[1] Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Form GSTP MRNA KD SAMPLE (TM6, TM7)

#### PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column.

Add records for "Other unscheduled timepoints" within a day if necessary,

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "cor" portion of patient number.

Sort "Date Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

Present Visit only if it is applicable. Data will be from outside vendor.

For any of the PBMC read-outs (GST inRNA levels), there will be some time points that fall due to insufficient sample. So for unit we may have to indicate ND and then footnote that sample insufficient for analysis.

Statistical Analysis Plan


Copyright© 2016 by Theradex Oncology®, Princeton NI

All rights reserved

155



DIRECTORY/FILE.SAS FINAL- ddmmmyychhomm NBF-006-001 Phase 1/To

#### Listing 16.2.9.15 GST Family - GSTT1 mRNA Level Intent-to-Treat (N=n)


| Patient | Study | NBF-006 Dose | | Schedule | Sample | Day | | GSTT1 | |
|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Timepoint | Date | [1] | Time | mRNA Level | Unit |
| ссс-рара/хог/х | × | XXX | XXX | XXX | ddmmmyyyy | -xx | hfonor | XXXXXX | XXX |
| ccc-ppppp/xx/x | × | XXX | 3000 | KKK | ddmmmyyyy | -500 | hhomm | 300000 | XXX |
| ccc-pppp/xx/x | × | XXX | 3006 | XXX | ddmmmyyyy | HXX | hhemm | XXXXXX | XXX. |
| ссс-раррухол/х | × | XXX | XXX | XXX | ddmmmyyyy | -xx | hhamm | 300000 | XXX |
| ссс-рррру/хж/х | × | XXX | 3000 | KKK | ddmmmyyyy | -8X | hhomm | 3000000 | XXX |
| ccc-ppppp/xx/x | × | XXX | 3000 | XXX | ddmmmyyyy | -XX. | hhanm | XXXXXX | XXX |
| εεε-ραρφλούχ | × | XXX | XXX | XXX | ddmmmyyyy | -xx | hhomm | XXXXXX | XXX |

GSTT1 - Glutathione S-Transferase theta class

[1] Day is relative to the first dose date of NBF-006.

Cross-References:

#### PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time column.

Add records for "Other unscheduled timepoints" within a day if necessary.

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "popp", and then "cor" portion of patient number.

Sort "Date Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

Present Visit only If it is applicable. Data will be from outside vendor.

For any of the PBMC read-outs (GST mRNA levels), there will be some time points that fail due to insufficient sample. So for unit we may have to indicate ND and then footnote that sample insufficient for analysis.

Statistical Analysis Plan 156


Copyright© 2016 by Theradex Oncology®, Princeton NI

All rights reserved



#### Listing 16.2.9.16 GST Family - MGST3 mRNA Level Intent-to-Treat (N=n)

FINAL- ddmmmyychhamm


| Patient | Study | NBF-006 Dose | | Schedule | Sample | Day | | MGST3 | |
|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Timepoint | Date | [1] | Time | mRNA Level | Unit |
| ccc-pppp/xx/x | × | XXX | XXX | XXX | ddmmmyyyy | -xx | bhamm | XXXXXX | XXX |
| ccc-ppppp/xx/x | × | XXX | NXX | XXX | ddmmmyyyy | 1900 | hhamm | 300000 | XXX |
| ccc-ppppp/xx/x | × | XXX | XXX | XXX | ddmmmyyyy | -306 | hhamm | XXXXX | XXX |
| ссс-раррухол/х | × | XXX | XXX | XXX | ddmmmyyyy | -XX | hitenton | XXXXXX | XXX |
| ссс-рррру/хж/х | × | XXX | NOOK. | XXX | ddmmmyyyy | -900 | hinamin | XXXXXX | XXX |
| ccr-ppppp/xx/x | × | XXX | XXX | XXX | ddmmmyyyy | -XX | hhamm | XXXXX | XXX |
| εεε-ραρφλούχ | × | XXX | XXX | XXX | ddmmmyyyy | -xx | hinamin | XXXXXX | XXX |

[1] Day is relative to the first dose date of NBF-006.

Cross-References:

#### PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column.

Add records for "Other unscheduled timepoints" within a day if necessary,

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "cor" portion of patient number.

Sort "Date-Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

Present Visit only if it is applicable. Data will be from outside vendor.

For any of the PBMC read-outs (GST inRNA levels), there will be some time points that fail due to insufficient sample. So for unit we may have to indicate ND and then footnote that sample insufficient for analysis.

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan 157





#### Listing 16.2.9.17 GST Family - GST M3 mRNA Level Intent-to-Treat (N=n)

| Patient | Study | NBF-006 Dose | | Schedule | Sample | Day | | GSTM3 | |
|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (rng/kg) | Visit | Timepoint | Date | [1] | Time | mRNA Level | Unit |
| ccc-pppp/xx/x | × | XXX | XXX | XXX | ddmmmyyyy | -xx | Mann | XXXXXX | XXX |
| ccc-ppppp/xx/x | × | XXX | NXX | XXX | ddmmmyyyy | -90% | hhamm | XXXXXX | XXX |
| ccc-ppppp/xx/x | × | XXX | XXX | XXX | ddmmmyyyy | -306 | hhamm | X0000X | XXX |
| ссс-раррухол/х | × | XXX | XXX | XXX | ddmmmyyyy | →kX | hitemm | XXXXXX | XXX |
| ccc-ppppp/xx/x | × | XXX | NOOK. | JOICK | ddmmmyyyy | -900 | hinamin | XXXXXX | XXX |
| ccr-ppppp/xx/x | × | XXX | XXX | жж | ddmmmyyyy | -XX | hhamm | XXXXX | XXX |
| ccc-pgpp/xx/x | × | XXX | XXX | XXX | ddmmmyyyy | -900 | hinamin | XXXXX | XXX |

[1] Day is relative to the first dose date of NBF-006.

Cross-References:

#### PROGRAMMER'S NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column.

Add records for "Other unscheduled timepoints" within a day if necessary,

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "pppp", and then "cor" portion of patient number.

Soft "Date Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

Present Visit only if it is applicable. Data will be from outside vendor.

For any of the PBMC read-outs (GST inRNA levels), there will be some time points that fall due to insufficient sample. So for unit we may have to indicate ND and then footnote that sample insufficient for analysis.

Statistical Analysis Plan


Copyright© 2016 by Theradex Oncology®, Princeton NI

All rights reserved

158



DIRECTORY/FILE.SAS FINAL- ddmmmyychh:mm NBF-006-001 Phase 1/To Page 1 of x

#### Listing 16.2.9.18 Pharmacokinetics Data Collection Safety Evaluable (N=n)

| Patient | Study | NBF-006 Dose | | Planned | Date | Day | Time | SIRNA | Infusion T | Ime |
|---|---|---|---|---|---|---|---|---|---|---|
| /Age/Sex | Part | (mg/kg) | Visit | Timepoint | Collected | [1] | Collected | (rig/mL) | Start | Stop |
| ccc-pppp/xx/x | × | XXX | XXX | xxx | didminimyyyy | ·xx | hisanm | XXX | hhanm | htemm |
| сес-рарружжи | * | XXX | XXX | XXX | ddmmmyyyy | -xx | hhanm | 3000 | hhomm | hhamm |
| ccc-ppppp/xx/x | * | XXX | XXX | XXX | didmmmyyyy | +XX | htsmm | 3006 | hhamm | hhanm |
| ccc-ppppp/xx/x | × | XXX | XXX | XXX. | didirenmyyyy | *8X | hbanm | XXX | hhanin | hlomm |
| εεε-μαρφ/χχ/χ | × | XXX | XXX | XXX. | ddmmmyyyy | -8× | hforem | XXX | hhomm | hhemm |
| ccc-ppppp/xx/x | * | XXX | NXX | XXX | didminimyyyy | +xx | hhanm | XXX | hhanm | hhanm |
| есе-пррружух | х. | XXX | XXX | XXX | NOT DONE | | | | | |

(1) Day is relative to the first dose date of NBF-006.

Cross-References: Case Report Form PHARMACOKINETICS (PK, PKT), PHARMACOKINETICS DATA COLLECTION (PK1-2)
PROGRAMMERS NOTES:

When "Not done" is indicated, enter "NOT DONE" in the Time' column.

Add records for "Other unscheduled timepoints" within a day if necessary.

Data will be presented in mixed case for formatted variables and upper case only for unformatted variables.

Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number.

Sort "Date Performed" in ascending order within "Patient". Sort "Time" in ascending order within "Date".

Present Visit only if it is applicable. Present result if data collected.

Present Infusion Time only data is available or can be derived.

Statistical Analysis Plan


All rights reserved

Copyright© 2016 by Theradex Oncology®, Princeton NI

159




#### Listing 16.2.10.1 Concomitant Measures Safety Evaluable (N=n)

| Patient<br>/Age/Sex | | NBF-006 Dose<br>(mg/kg) | Start Date<br>Stop Date | Start Day<br>Stop Day<br>[1] | Drug Name or Treatment<br>(WHO-DD Preferred Term)<br>(WHO-DD ATC Class Category Level II) [2] | Dose | Unit | Route | Reason<br>For Use | AE<br>Number |
|---|---|---|---|---|---|---|---|---|---|---|
| ссс-рррр<br>/хж/х | × | xxx | ddmmrnyyyy<br>Ongoing | -90X<br>-XX | Concomitant Measure<br>(WHO-DD Preferred Term)<br>(WHO-DD ATC Class Category Level II) | XXX | XXX | Route | Reason | ×× |
| | | жж | ddmmrryyyy<br>ddmmrryyyy | xx<br>xx | Concomitant Measure<br>(WHO-DD Preferred Term)<br>(WHO-DD ATC Class Category Level II) | XXX | XXX | Route | Reason | XX |
| ccc-pppp<br>/xx/x | x | XXX | ddmmmyyyy<br>Ongoing | -xx<br>xx | Concomitant Measure<br>(WHO-DD Preferred Term)<br>(WHO-DD ATC Class Category Level II) | жх | 2000 | Other: specify | Reason | XX |

[1] Day is relative to the first dose date of NBF-006.
[2] WHO-DDE version 2018
Cross-References: Case Report Form CONCOMITANT MEASURES (CM)
PROGRAMMERS NOTES:

When "None" is indicated, enter "NO CONCOMITANT MEASURES" in the 'Drug Name or Treatment' column. Data will be presented in mixed case for formatted variables and upper case only for unformatted variables. Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number.

Sort "Start Date" in ascending order within "Patient".

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan 160




DIRECTORY/FILE.SAS FINAL- ddmmmyychh:mm NBF-006-001 Phase 1/1b Page 1 of x

# Listing 16.2,10.2 Concomitant Measures - Palliative Radiotherapy Safety Evaluable (N=n)

| Patient<br>/Age/Sex | 121111111 | / NBF-006 Dose<br>(mg/kg) | Start Date<br>Stop Date | Start Day<br>Stop Day<br>[1] | Drug Name or Treatment<br>(WHO-DD Preferred Term)<br>(WHO-DD ATC Class Category Level II) [2] | Dose | Unt | Route | Reason<br>For Use | On<br>Target<br>Lesion |
|---|---|---|---|---|---|---|---|---|---|---|
| сес-рррв<br>/хж/х | х | xxx | ddmmreyyyy<br>Ongoing | -90X<br>+80X | Concomitant Measure<br>(WHO-DD Preferred Term)<br>(WHO-DD ATC Class Category Level II) | XXX | XXX | Route | Reason | No |
| | | xxx | ddmmmyyyy<br>ddmmmyyyy | xx<br>xx | Concomitant Measure<br>(WHO-DD Preferred Term)<br>(WHO-DD ATC Class Category Level II) | XXX | XXX | Route | Reason | No. |
| ccc-pppp<br>/xx/x | × | XXXX | ddrammyyyy<br>Ongoing | -xx<br>xx | Concomitant Measure<br>(WHO-DD Preferred:Term)<br>(WHO-DD ATC Class Category Level II) | XXX | xxx | Other: specify | Reason | Yes |

Palliative radiotherapy is allowed as medically indicated after completion of the first treatment cycle, and after discussion with medical monitor.
[1] Day is relative to the first dose date of NBP-006.

Cross-References: Case Report Form CONCOMITANT MEASURES (CM)
PROGRAMMERS NOTES:

When "None" is indicated, enter "NO CONCOMITANT MEASURES" in the 'Drug Name or Treatment' column.

Data will be presented in mixed case for formatted variables and upper case only for uniformatted variables.

Sort "Patient" in ascending order using "popp", and then "ccc" portion of patient number,

Sort "Start Date" in ascending order within "Patient".

May removed some columns if data is not available.

Copyright© 2016 by Theradex Oncology®, Princeton NI All rights reserved

Statistical Analysis Plan 161


# Nitto NBF-006-001\_TLF Plan Part A & B Final 2.0\_clean\_14Mar2023

Final Audit Report 2023-03-21

Created: 2023-03-16

By: Zachary Albaugh (ZAlbaugh@theradex.com)

Status: Signed

Transaction ID: CBJCHBCAABAAKOujWJ7v6JNMvGU0l6sxgHxLGq5zPyzQ

# "Nitto NBF-006-001\_TLF Plan Part A & B Final 2.0\_clean\_14Mar 2023" History

- Document created by Zachary Albaugh (ZAlbaugh@theradex.com) 2023-03-16 - 2:23:11 PM GMT- IP address: 65.126.24.19
- Document emailed to Dailan Danforth (DDanforth@theradex.com) for signature 2023-03-16 - 2:25:33 PM GMT
- Document emailed to Judy DeChamplain (jdechamplain@theradex.com) for signature 2023-03-16 - 2:25:33 PM GMT
- Document emailed to Jose Mejias (jmejias@theradex.com) for signature 2023-03-16 - 2:25:33 PM GMT
- Document emailed to Zachary Albaugh (ZAlbaugh@theradex.com) for signature 2023-03-16 - 2:25:33 PM GMT
- Document emailed to Joachim Gullbo (jgullbo@theradex.com) for signature 2023-03-16-2:25:33 PM GMT
- Document emailed to sonya.zabludoff@nitto.com for signature
- Zachary Albaugh (ZAlbaugh@theradex.com) authenticated with Adobe Acrobat Sign. 2023-03-16 - 2:25:52 PM GMT
- Document e-signed by Zachary Albaugh (ZAlbaugh@theradex.com)
  Signing reason: approval
  Signature Date: 2023-03-16 2:25:52 PM GMT Time Source; server- IP address: 65:128:24.19



Email viewed by Dailan Danforth (DDanforth@theradex.com) 2023-03-16 - 2:28:15 PM GMT-IP address: 104.47.56.254

Dailan Danforth (DDanforth@theradex.com) authenticated with Adobe Acrobat Sign. 2023-03-18 - 2:29:05 PM GMT

6 Document e-signed by Dailan Danforth (DDanforth@theradex.com)

Signing reason: author

Signature Date: 2023-03-16 - 2:29:05 PM GMT - Time Source: server- IP address: 24.2:241.195

Email viewed by Judy DeChamplain (jdechamplain@theradex.com) 2023-03-16 - 3:03:11 PM GMT- IP address: 104.47.56.254

Judy DeChamplain (jdechamplain@theradex.com) authenticated with Adobe Acrobat Sign. 2023-03-16 - 3:03:36 PM GMT

Document e-signed by Judy DeChamplain (jdechamplain@theradex.com)

Signing reason: approval

Signature Date: 2023-03-16 - 3:03:36 PM GMT - Time Source: server- IP address: 72.94.90.100

Email viewed by Joachim Gullbo (jgullbo@theradex.com) 2023-03-17 - 12:53:57 PM GMT- IP address: 104.47.56.254

Joachim Gullbo (jgullbo@theradex.com) authenticated with Adobe Acrobat Sign. 2023-03-17 - 12:54:20 PM GMT

Document e-signed by Joachim Gullbo (jgullbo@theradex.com)

Signing reason: approval

Signature Date: 2023-03-17 - 12:54:20 PM GMT - Time Source: server- IP address: 73:255,180:248

Email viewed by sonya.zabludoff@nitto.com 2023-03-20 - 7:13:05 PM GMT-IP address: 104.47.23.190

Signer sonya.zabludoff@nitto.com entered name at signing as Sonya Zabludoff 2023-03-20 - 7:13:48 PM GMT- IP address: 138.226.67.6

Sonya Zabludoff (sonya.zabludoff@nitto.com) authenticated with Adobe Acrobat Sign. 2023-03-20 - 7:13:50 PM GMT

Sonya Zabludoff (sonya.zabludoff@nitto.com)

Signing reason: approval

Signature Data: 2023-03-20 - 7:13:50 PM GMT - Time Source; server- IP address: 136:226.67.6

Jose Mejias (jmejias@theradex.com) authenticated with Adobe Acrobat Sign, 2023-03-21 - 12:58:05 PM GMT

Document e-signed by Jose Mejias (jmejias@theradex.com) Signing reason approval



Signature Date: 2023-03-21 - 12:58:05 PM GMT - Time Source: server- IP address: 73:226:136:254

Agreement completed.

2023-03-21 - 12:58:05 PM GMT

Names and email addresses are entered into the Acrobat Sign service by Acrobat Sign users and are unverified unless otherwise noted.